

# STATISTICAL ANALYSIS PLAN

SEP361-308

AN 8-WEEK, OPEN-LABEL STUDY EVALUATING THE EFFECTIVENESS, SAFETY AND TOLERABILITY OF SEP-363856 IN SUBJECTS WITH SCHIZOPHRENIA SWITCHED FROM TYPICAL OR ATYPICAL ANTIPSYCHOTIC AGENTS

PHASE: PHASE III

AUTHOR: PPD

VERSION NUMBER AND DATE: FINAL VERSION 1.0, 06MAY20244

Author: PPD Version Number: 1.0 Version Date: 06MAY2024

# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan Version 1.0 (Date 07MAY2024) for Protocol SEP361-308.

| | Name | Signature | Date | |
|---|---|---|---|---|
| Author: | PPD | DocuSigned | May 8, 2024<br>PPD | |
| Position: | PPD Biostatistics | PPD | | ove this document<br>2024 7:23:21 AM PD |
| Company: | Sumitomo Pharma America, Inc | c | D9B74E6EBF126E878D21636D | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.









### **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| Stable Draft | 30MAY2023 | PPD | Not applicable – First Version |
| Version 1.0 | 07MAY2024 | PPD | Change in the enrolled subjects definition. Change in sample size. Addition of AEs leading to dose increase and decrease analyses. Addition of Treatment-related AEs by PT analysis. Addition of haloperidol equivalent doses for lumateperone. |


# **TABLE OF CONTENTS**

| 1. Introduction 12 | | | |
|---|---|---|---|
| 2. Study Objectives and Endpoints 12 | | | |
| 2.1. Study Objectives | | | 12 |
| 2.1.1. Primary Objective | | | 12 |
| <ul><li>2.1.2. Secondary Objective</li><li>2.1.3. Other Objectives</li></ul> | | | 12<br>13 |
| 2.2. Study Endpoints | | | 14 |
| 2.2.1. Primary Endpoint | | | 14 |
| 2.2.2. Secondary Endpoint | | | 14 |
| 2.2.3. Other Endpoints | | | 14 |
| 3. Study Design 15 | | | |
| 3.1. General Description | | | 15 |
| 3.2. Method of Assigning Subjects to Treatment Group | s | | 16 |
| 3.3. Blinding | | | 16 |
| 3.4. Determination of Sample Size | | | 16 |
| 3.5. Changes in the Conduct of the Study | | | 17 |
| 3.6. Schedule of Events | | | 17 |
| Document: PPD | | _ | |
| Author: PPD | Version Number:<br>Version Date: | 1.0<br>06MAY2024 | |



| 3.7. | Changes to Analysis from Protocol | | | 17 |
|---|---|---|---|---|
| 4. P | anned Analyses 18 | | | |
| 4.1. | Data and Safety Monitoring Board | | | 18 |
| 4.2. | Interim Analysis | | | 18 |
| 4.3. | Final Analysis | | | 18 |
| 5. A | nalysis Populations 18 | | | |
| 5.1. | Safety [SAF] Population | | | 19 |
| 5.2. | Per Protocol [PP] Population | | | 19 |
| 5.3. | Effectiveness [EFF] Population | | | 19 |
| 6. G | eneral Considerations 19 | | | |
| 6.1. | Reference Start Date and Study Day | | | 19 |
| 6.2. | Baseline | | | 20 |
| 6.3. | Derived Timepoints | | | 23 |
| 6.4. | Retests, Unscheduled Visits, and Early Termination Dat | ta | | 26 |
| 6.5. | Windowing Conventions | | | 26 |
| 6.6. | Statistical Tests | | | 27 |
| 6.7. | Common Calculations | | | 27 |
| 6.8. | Software Version | | | 27 |
| Doc | ıment: PPD | | | |
| Auth | or: PPU | Version Number: Version Date: | 1.0<br>06MAY2024 | |



| 7. Statistical Considerations 27 | | |
|---|---|---|
| 7.1. Adjustments for Covariates and Factors to be Inclu | ded in Analyses | |
| 7.2. Multicenter Studies | | |
| 7.3. Missing Data | | |
| 7.4. Multiple Comparisons/ Multiplicity | | |
| 7.5. Examination of Subgroups 7.5.1. Derivation of Subgroups | | |
| 8. Output Presentations32 | | |
| 9. Disposition and Withdrawals 32 | | |
| 9.1. Derivations | | |
| 10. Important Protocol Deviations 34 | | |
| 11. Demographic and Other Baseline Characteristics | 34 | |
| 11.1. Derivations | | |
| 12. Medical History 38 | | |
| 13. Medications 38 | | |
| 14. Study Medication Exposure 39 | | |
| 14.1. Derivations | | |
| 15. Study Medication Compliance 40 | | |
| 15.1. Derivations | | |
| 16. Effectiveness Outcomes 41 | | |
| Document: PPD | | |
| Author: PPD | Version Number:<br>Version Date: | 1.0<br>06MAY2024 |



# Sumitomo Pharma

| 16.1. | PANSS | | | | 41 |
|---|---|---|---|---|---|
| 16.1.1. | PANSS Total Score | | | | 44 |
| 16.1.2. | Proportion of Subjects Wh | no Achieve a Response | | | 44 |
| 16.1.3. | PANSS Subscale Scores | | | | 45 |
| 16.1.4. | PANSS Marder Factor Sco | res | | | 46 |
| 16.1.5. | PANSS UPSM factor score | s and the UPSM total fa | actor score | | 46 |
| 16.2. | Clinical Global Impression-S | everity | | | 48 |
| 16.3. | Brief Negative Symptom Sca | ale (BNSS) Total Score a | and Subscale Scores | | 48 |
| 16.4. | 12-Item Short Form Survey | (SF-12) | | | 49 |
| 16.5. | PSP total score and individu | al domain scores | | | 49 |
| 16.6. | Medication Satisfaction Que | estionnaire (MSQ) | | | 51 |
| 16.7. | Clinical Global Impressions | - Improvement Scale ( | CGI-I) | | 51 |
| 16.8. | Healthcare Resource Utiliza | tion | | | 52 |
| 16.9. | Nicotine Use | | | | 52 |
| 16.10. | Missing Data Method | | | | 53 |
| 17. Safet | y Outcomes 53 | | | | |
| 17.1. | Discontinuation due to Clini | cal Reasons | | | 54 |
| 17.2. | Discontinuation due to Any | Reasons | | | 54 |
| 17.3. | Adverse Events and Pre-trea | atment Events | | | 54 |
| | All AEs | Additional Events | | | 57 |
| 17.3.1. | | | | | 57 |
| 17.3 | | medication | | | 57 |
| Docume | | | | | 3, |
| Author: | ראח | | Version Number: | 1.0 | |
| Author. | FFD | | Version Date: | 06MAY2024 | |



# Sumitomo Pharma

| 17.3.2. | AEs Leading to Discontinuation from Study | | | 58 |
|---|---|---|---|---|
| 17.3.3. | AEs Leading to Study Medication Withdrawal | | | 58 |
| 17.3.4. | AEs Leading to Study Medication Interruption, stu | ldy dose increase and reduced | | 58 |
| 17.3.5. | Serious Adverse Events | | | 58 |
| 17.3.6. | Adverse Events Leading to Death | | | 59 |
| 17.3.7. | Adverse Events of Potential Drug Abuse and Depe | endence | | 59 |
| 17.3.8. | Extrapyramidal Adverse Events | | | 59 |
| 17.3.9. | Adverse Events by Subgroups | | | 59 |
| 17.3.10 | . Psychiatric Adverse Events Leading to Discontinua | ation from Study (PAEDCs) | | 59 |
| 17.4. | Laboratory Evaluations | | | 60 |
| 17.4.1. | Laboratory Specific Derivations | | | 61 |
| 17.4.2. | Laboratory Reference Ranges | | | 61 |
| 17.5. | ECG Evaluations | | | 62 |
| 17.5.1. | QTc Interval Prolongation Criteria | | | 63 |
| 17.5.2. | ECG Potentially Clinically Significant Criteria | | | 64 |
| 17.6. | Vital Signs | | | 64 |
| 17.6.1. | Vital Sign Specific Derivations | | | 65 |
| 17.6.2. | Vital Sign Potentially Clinically Significant Criteria | | | 66 |
| 17.7. | Physical Examination | | | 66 |
| 17.8. | Other Safety Assessments | | | 67 |
| 17.8.1. | Columbia Suicide Severity Rating Scale (C-SSRS) | | | 67 |
| 17.8.2. | Abnormal Involuntary Movement Scale (AIMS) | | | 70 |
| 17.8.3. | Barnes Akathisia Rating Scale (BARS) | | | 70 |
| 17.8.4. | Simpson-Angus Scale (SAS) | | | 71 |
| 17.8.5. | Pittsburgh Sleep Quality Index | | | 72 |
| 17.9. | Subgroup Analysis of Safety Variable(s) | | | 72 |
| 18. Pharn | nacokinetic Analysis 72 | | | |
| Documei | nt: PPD | | _ | |
| 200dillo | | | | |
| Author: | טאא | Version Number:<br>Version Date: | 1.0<br>06MAY2024 | |



| 19. Data Not Sumn | narized or Presented 73 | | |
|---|---|---|---|
| 20. References | 73 | | |
| APPENDIX 1. | <b>Programming Conventions for Outputs</b> 75 | | |
| IQVIA Output Conv | entions | | 75 |
| Dates & Times | | | 70 |
| Spelling Format | | | 76 |
| Presentation of Tre | eatment Groups | | 76 |
| Listings | | | 77 |
| APPENDIX 2. | Partial Date Conventions 78 | | |
| Algorithm for Adve | rse Events | | 78 |
| Algorithm for Prior | / Concomitant / Post-Treatment Medications | | 80 |
| Partial Date Imputa | ation Rules for Initial Onset of Schizophrenia | | 82 |
| Partial Date Imputa | ation Rules for Current Onset of Acute Exacerbation | | 82 |
| Partial Date Imputa | ation Rules for First Hospitalization | | 82 |
| Partial Date Imputa | ation Rules for First Anti-psychotic Drug Therapy | | 83 |
| Partial Date Imputa | ation Rules for Onset of Initial Behavioral Disturbance | | 83 |
| Rules for Assigning | DOSEON/DOSEA | | 84 |
| APPENDIX 3. | Uncorrelated PANSS Score Matrix (UPSM) 85 | | |
| APPENDIX 4. | Internationally Agreed Order for System Organ Class 87 | | |
| Document: | PPD | | |
| Author: | Version Number:<br>Version Date: | 1.0<br>06MAY2024 | |

96



Statistical Analysis Plan

APPENDIX 5. Adverse Events of Potential Drug Abuse and Dependence 88

**APPENDIX 6.** Extrapyramidal Adverse Events 92

APPENDIX 7. Predefined Potentially Clinically Significant (PCS) Criteria in SI Units 96

Standard PCS Criteria for Laboratory Parameters – SI Units

APPENDIX 8. PSQI Scoring Sheet 98

APPENDIX 9. Classification of Patient Type from UPSM Factor Scores 101

APPENDIX 10. Marder PANSS Negative Symptoms (MPNS) Heterogeneity Index Method 131

APPENDIX 11. Schedule of Events 133




### 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of safety, effectiveness and pharmacokinetic (PK) data for Protocol SEP361-308. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 5.00, dated 06NOV2023.

A Pre-Lock Data Review (PLDR) and Important Protocol Deviation (IPD) Review Plan will be written to describe the process and the outputs to be delivered during the IPD/BDR meetings.

The scope of this SAP does not include calculation and statistical analysis of PK parameters of SEP-363856; individual SEP-363856 PK parameters will be determined using population PK approach and results will not be reported in the clinical study report (CSR).

### 2. STUDY OBJECTIVES AND ENDPOINTS

### 2.1. STUDY OBJECTIVES

#### 2.1.1. PRIMARY OBJECTIVE

The primary objective is to evaluate the safety and effectiveness of switching clinically stable outpatients with schizophrenia from a typical antipsychotic to SEP-363856 over a period of 8 weeks as assessed by the percentage of subjects who discontinue from the study due to an adverse event or lack of efficacy

#### 2.1.2. SECONDARY OBJECTIVE

The secondary objective is to evaluate the safety and effectiveness of switching clinically stable outpatients with schizophrenia from a typical or atypical antipsychotic to SEP-363856 over a period of 8 weeks as assessed by the percentage of subjects who discontinue for any reason (ie, all causes of discontinuation)

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | טאא | Version Number: | 1.0 |
| | | Version Date: | 06MAY2024 |



#### 2.1.3. OTHER OBJECTIVES

- To evaluate the tolerability and safety of switching clinically stable outpatients with schizophrenia from a typical or atypical antipsychotic to SEP-363856 over a period of 8 weeks using:
  - o Adverse event reports
  - o Clinical laboratory tests
  - o Vital sign measurements
  - o 12-lead electrocardiograms (ECG)
  - o Columbia Suicide Severity Rating Scale (C-SSRS)
  - o Barnes Akathisia Rating Scale (BARS)
  - o Abnormal Involuntary Movement Scale (AIMS)
  - o Simpson-Angus Scale (SAS)
- To evaluate the effectiveness of SEP-363856 using:
  - o Positive and Negative Syndrome Scale (PANSS)
  - o Clinical Global Impression-Severity (CGI-S) scale
  - o Clinical Global Impression-Improvement (CGI-I) scale
  - o Brief Negative Symptom Scale (BNSS)
- To evaluate the effects of SEP-363856 on health-related quality of life as measured by the Short Form Health Survey (SF-12)
- To evaluate the effects of SEP-363856 on functional capacity as measured by the Personal and Social Performance Scale (PSP)
- To evaluate medication satisfaction as measured by the Medication Satisfaction Questionnaire (MSQ)
- To evaluate sleep as measured by the Pittsburg Sleep Quality Index (PSQI)
- To evaluate the impact of SEP-363856 on healthcare resource utilization (HCRU)




### 2.2. STUDY ENDPOINTS

#### 2.2.1. PRIMARY ENDPOINT

Percentage of subjects who discontinue for clinical reasons (ie, discontinued due to an adverse event [AE] or lack of efficacy)

#### 2.2.2. SECONDARY ENDPOINT

Percentage of subjects who discontinue for any reason (ie, all causes for discontinuation)

#### 2.2.3. OTHER ENDPOINTS

- The incidence of overall AEs, serious adverse events [SAE]s, and AEs leading to discontinuation
- Observed values and changes from Baseline in clinical laboratory tests (hematology, chemistry and urinalysis)
- Observed values and changes from Baseline in vital signs (including body weight, body mass index [BMI], waist circumference, temperature, blood pressure [supine and standing], heart rate [supine and standing] and respiratory rate)
- Observed values and changes from Baseline in 12-lead ECG parameters
- Frequency of subjects with suicidal ideation and suicidal behavior based on the C-SSRS
- Changes from Baseline in BARS, AIMS and SAS scores
- Changes from Baseline to Week 8 in:
  - o PANSS total score and subscale scores (positive, negative, and general psychopathology)
  - o PANSS Marder Factor (five-factor) scores (positive, disorganized, negative, hostility, and depression/anxiety), and Uncorrelated PANSS Score Matrix (UPSM)

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | PPD | Version Number: | 1.0 |

- o CGI-S score
- BNSS total score
- o SF-12 scores
- o PSP total score
- o MSQ score
- PSQI global score
- CGI-I score at Week 8
- HCRU (including numbers of physician office visits, emergency room [ER] visits and hospitalizations, length of hospital stays, employment status and average number of hours caregiver(s) spends helping subjects per week.)
- Nicotine use at baseline and Week 8 (end of treatment [EOT]/early termination [ET])

### 3. STUDY DESIGN

### 3.1. GENERAL DESCRIPTION

This is an 8-week, outpatient, multicenter, open-label, single-group, flexible-dose study designed to evaluate the safety and tolerability, as well as effectiveness of switching clinically stable adult subjects with schizophrenia from a typical or atypical antipsychotic to SEP-363856. This study is projected to enroll approximately 120 subjects into a single treatment group (SEP-363856). Over the 8-week treatment period, subjects will receive flexibly dosed SEP-363856 (50 to 100 mg/day) and the investigator will have the discretion to discontinue each subject's pre-switch antipsychotic treatment by the end of Week 2, 3, 4, 5, or 6.

Once the pre-switch antipsychotic has been fully discontinued, subjects will continue to receive SEP-363856 flexible 50 to 100 mg/day until study endpoint, at the end of Week 8. Study medication will be taken at the same time each evening at bedtime and can be taken with or without food.

The study will consist of three periods: Screening/Washout (up to 21 days), Treatment (8 weeks) and a Follow-up visit (7 ± 2 days after the last dose of study medication for those subjects who discontinue prior to the Week 8 visit or who complete the study but do not enroll in the open-label extension study SEP361-309). If necessary, subjects may return to the clinic at any time for an unscheduled visit.

A study schematic is presented in Figure 1.

| Document: | PPD |
|-----------|-----|

Figure 1: Study schematic



### 3.2. METHOD OF ASSIGNING SUBJECTS TO TREATMENT GROUPS

This is an open label study. There is no randomization planned in this study. All subjects will receive flexible dosing with SEP-363856 (50 to 100 mg/day).

### 3.3. BLINDING

This is an open-label study. All subjects will receive flexible dosing with SEP-363856 (50 to 100 mg/day).

### 3.4. DETERMINATION OF SAMPLE SIZE





The sample size was determined by the width of the 95% confidence interval for the proportion of subjects who may discontinue due to clinical reasons by Week 8 to ensure the precision of the estimate of the true discontinuation rate due to clinical reasons. Assuming, 1) 15% of SEP-363856 treated subjects will experience discontinuation due to clinical reasons by Week 8, and 2) 6.4% as the half width (the distance between the upper/lower limits to the point estimate) of the 95% confidence interval (ie, [8.6%, 21.4%]), approximately 120 subjects was planned for enrollment. Due to higher than predicted rates for enrollment, retention, and completers in study 308, the SMPA team decided to revisit the assumption of 15% SEP-363856 treated subjects discontinuation rate due to clinical reasons by Week 8. Using the proportion from the data at time of revisiting, the discontinuation rate due to clinical reasons by Week 8 was approximately 7.2%. With 7.2% as the assumption, 100 subjects would provide a half width of 5.1% half width and was deemed to be sufficient. 101 subjects were enrolled.

### 3.5. Changes in the Conduct of the Study

The first subject was screened on 19DEC2022 under protocol Version 3.00 (dated 12OCT2022). Additional protocol versions and amendments are listed below.

Protocol version 1.00 (24-Aug-2022)

Protocol version 2.00 (22-Sep-2022); Substantial Amendment 1.00 (22-Sep-2022)

Protocol version 3.00 (12-Oct-2022); Substantial Amendment 2.00 (12-Oct-2022)

Protocol version 4.00 (28-Mar-2023); Substantial Amendment 3.00 (28-Mar-2023)

Protocol version 5.00 (06-Nov-2023); Substantial Amendment 4.00 (06-Nov-2023)

### 3.6. SCHEDULE OF EVENTS

Schedule of events can be found in Section 1, Table 2 of the Clinical Study Protocol (CSP). These tables are also included in APPENDIX 11 of the SAP.

### 3.7. CHANGES TO ANALYSIS FROM PROTOCOL

There are no changes to analysis from the protocol.

| Document: | PPD |
|-----------|-----|



### 4. PLANNED ANALYSES

The following analyses will be performed for this study:

Final Analysis

### 4.1. DATA AND SAFETY MONITORING BOARD

There is no DSMB planned for this study.

### 4.2. INTERIM ANALYSIS

There is no interim analysis planned for this study.

### 4.3. FINAL ANALYSIS

All final, planned analyses specified in this SAP will be performed by IQVIA following Sunovion authorization of this SAP, Sunovion authorization of Analysis Populations, Database Lock

Some minor modifications may be necessary to the planned design of tables, figures, and listings to accommodate data collected during the actual study conduct.

### 5. ANALYSIS POPULATIONS

Agreement and authorization of subjects included/excluded from each analysis population will be conducted prior to database lock.

Enrolled subjects in 361-308 will include all subjects who signed the informed consent form (ICF) of study 361-308 and did not screen fail.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | טיי | Version Number: | 1.0 |



# 5.1. SAFETY [SAF] POPULATION

The safety population will consist of all subjects who are enrolled and receive study medication (SEP-363856). All safety and tolerability assessments will be performed using the safety population.

# 5.2. PER PROTOCOL [PP] POPULATION

The per protocol (PP) population will consist of all EFF population subjects who satisfy the following conditions:

- Have 7 days or more overall exposure to study medication
- Have no important protocol deviations that can potentially impact the integrity of the effectiveness endpoint analysis

Selected effectiveness endpoints will be analyzed using the PP population. Subjects will be analyzed according to the treatment to which they receive.

# **5.3.** EFFECTIVENESS [EFF] POPULATION

The effectiveness population will consist of all subjects who are enrolled, have received at least one dose of study medication, and have a Baseline and at least one post-Baseline effectiveness measurement in PANSS or CGI-S. Subjects will be included in the population regardless of any protocol deviation. The effectiveness population will be the primary population for the effectiveness analyses.

### 6. GENERAL CONSIDERATIONS

Study medication refers to SEP-363856 unless otherwise specified.

# 6.1. REFERENCE START DATE AND STUDY DAY

Study Day will be calculated from the reference start date and will be used to show the start/stop day of assessments and events.

| Document: | PPD |
|-----------|-----|



Reference start date is defined as the date of the first dose of study medication (Day 1 is the Study Day of the first dose of study medication).

• If the date of assessment or event is prior to the reference start date, then:

Study Day = (date of assessment or event - reference start date).

If the date of assessment or event is on or after the reference start date, then:

Study Day = (date of assessment or event - reference start date) + 1.

In the situation where the assessment or event date is partial or missing, Study Day and any corresponding durations will appear missing in the listings. Partial assessment or event dates will however be presented as is in the listings.

### 6.2. BASELINE

Unless otherwise specified, Baseline is defined as the last non-missing measurement taken prior to the first dose of study medication (including unscheduled assessments).

Whenever available, the time information should be accounted for in the derivation of Baseline values. In the case where time is not available and the date of the last non-missing measurement and the date of the first dose of study medication coincide, that measurement will be considered the Baseline.

Baseline will be derived for the following outcome measures:

- PANSS: total score, subscale scores, Marder factor scores, uncorrelated PANSS score matrix (UPSM) factor scores and total factor score, and individual item scores. For a given subject, the Baseline values for all PANSS summary and individual item scores should come from the same assessment (i.e., have the same visit number and assessment start date/time) and it should be the last assessment prior to first dose where PANSS total score is available (i.e., not set to missing). In the rare event where no PANSS total score is available before first dose due to partially completed assessments, the assessment prior to first dose with most PANSS item scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.
- CGI-S score.
- BNSS: total score, subscale scores, and individual item scores. For a given subject, the Baseline values for all BNSS summary and individual item scores should come from the same assessment and it should be the last assessment prior to first dose where BNSS total score is available. In the

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראט | Version Number: | 1.0 |



rare event where no BNSS total score is available before first dose due to partially completed assessments, the assessment prior to first dose with most BNSS item scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.

- SF-12 Score.
- PSP: total score, individual domain scores, and the derived binary variables. For a given subject, the Baseline values for all PSP data should come from the same assessment and it should be the last assessment prior to first dose where PSP total score is available. In the rare event where no PSP total score is available before first dose due to partially completed assessments, the assessment prior to first dose with most PSP individual domain scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.
- MSQ score.
- C-SSRS: Suicidal ideation categories 1-5 (yes/no) and suicidal behavior categories 6-10 (yes/no); C-SSRS composite endpoints: any suicidal ideation (yes/no), any suicidal behavior (yes/no), any suicidality (yes/no); the suicidal ideation score (0-5). See Section 17.8.1 for the definition of a C-SSRS Baseline.
- SAS: mean score and individual item scores. For a given subject, the Baseline values for all SAS summary and individual item scores should come from the same assessment and it should be the last assessment prior to first dose where SAS mean score is available. In the rare event where no SAS mean score is available before first dose due to partially completed assessments, the assessment prior to first dose with most SAS item scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.
- BARS: total score and individual item scores. For a given subject, the Baseline values for all BARS summary and individual item scores should
  come from the same assessment and it should be the last assessment prior to first dose where BARS total score is available. In the rare event
  where no BARS total score is available before first dose due to partially completed assessments, the assessment prior to first dose with most
  BARS item scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.
- AIMS: total score and individual item scores. For a given subject, the Baseline values for all AIMS summary and individual item scores should
  come from the same assessment and it should be the last assessment prior to first dose where AIMS total score is available. In the rare event
  where no AIMS total score is available before first dose due to partially completed assessments, the assessment prior to first dose with most
  AIMS item scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.
- PSQI: global score, component scores, and individual item scores. For a given subject, the Baseline values for all PSQI summary and individual item scores should come from the same assessment and it should be the last assessment prior to first dose where PSQI global score is available.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ארט | Version Number: | 1.0 |



In the rare event where no PSQI global score is available before first dose due to partially completed assessments, the assessment prior to first dose with most PSQI item scores available should be taken as the Baseline assessment for all raw and derived scores as applicable.

- Clinical laboratory parameters (blood chemistry, hematology, urinalysis, HOMA-IR (if collected)). For a given subject, the Baseline values for the clinical laboratory parameters do not have to all come from the same assessment; the only exception is: the Baseline flag for the counts of leukocytes and its differential should be applied to records from the same assessment and it should be the last assessment prior to first dose where counts of leukocytes and its differential are reported. Baseline flag does not need to be derived for RBC morphology findings, WBC morphology findings, and urinalysis microscopic examination findings (excluding urine erythrocytes and leukocytes).
- Urine drug screening: For a given subject, the Baseline values for all urine drug screening parameters should come from the same assessment and it should be the last assessment prior to first dose where a urine drug screening test was administered.
- Vital sign parameters (supine and standing systolic blood pressure [SBP], supine and standing diastolic blood pressure [DBP], supine and standing pulse rate, respiratory rate, oral temperature), height, weight, BMI, and waist circumference. For a given subject, the Baseline values for all vital sign parameters, height, weight, BMI, and waist circumference do not have to come from the same assessment; the only exceptions are: (1) the Baseline flag for weight and BMI should be applied to records from the same assessment and it should be the last assessment prior to first dose where weight is available, (2) the Baseline flag for supine SBP and DBP, standing SBP and DBP, and the derived corresponding orthostatic endpoints (i.e., standing SBP supine SBP; standing DBP supine DBP) should be applied to records from the same assessment and it should be the last assessment prior to first dose where all four BP measures are available, (3) the Baseline flag for supine and standing pulse rate and the derived corresponding orthostatic endpoint (i.e., standing pulse rate supine pulse rate) should be applied to records from the same assessment and it should be the last assessment prior to first dose where both pulse rate measures are available.
- ECG parameters: For a given subject, the Baseline values for all ECG parameters do not have to come from the same assessment. Baseline flag does not need to be derived for ECG parameters in the category of "FINDINGS".
- Nicotine use data: Baseline of this outcome measure should be taken strictly from the assessment given at Visit 1 without regard to its temporal relationship to the first dose of study medication.
- Healthcare resource utilization data: Baseline of this outcome measure should be taken strictly from the assessment given at Visit 2 without regard to its temporal relationship to the first dose of study medication.

The Baseline flag may be derived for additional outcome measures based on the needs during analyses.

| Document: | PPD |
|-----------|-----|



### 6.3. DERIVED TIMEPOINTS

The last non-missing post-Baseline (i.e., post-first dose) measurement collected during the study up to and including the Visit 10 (EOT/ET) measurement will be carried forward and defined as the last observation carried forward (LOCF) endpoint. Both scheduled and unscheduled assessments as well as the early termination assessments that are collected during this period will contribute to the derivation of the LOCF endpoint. However, unscheduled measurements taken after the Visit 10 (EOT/ET) measurement will not be used in the derivation.

The LOCF endpoint will be derived for the following outcome measures:

- PANSS: total score, subscale scores, Marder factor scores, UPSM factor scores and total factor score, individual item scores, and derived binary variables for PANSS response. For a given subject, the LOCF values for all PANSS summary and individual item scores and derived binary variables should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where PANSS total score is available. In the rare event where no PANSS total score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- CGI-S score.
- BNSS: total score, subscale scores, and individual item scores. For a given subject, the LOCF values for all BNSS summary and individual item scores should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where BNSS total score is available. In the rare event where no BNSS total score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- SF-12.
- PSP: total score, individual domain scores, and the derived binary variables. For a given subject, the LOCF values for all PSP data should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where PSP total score is available. In the rare event where no PSP total score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- MSQ score.
- C-SSRS suicidal ideation score (0-5).

| Document: | PPD |
|-----------|-----|



- SAS: mean score and individual item scores. For a given subject, the LOCF values for all SAS summary and individual item scores should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where SAS mean score is available. In the rare event where no SAS mean score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- BARS: total score and individual item scores. For a given subject, the LOCF values for all BARS summary and individual item scores should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where BARS total score is available. In the rare event where no BARS total score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- AIMS: total score and individual item scores. For a given subject, the LOCF values for all AIMS summary and individual item scores should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where AIMS total score is available. In the rare event where no AIMS total score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- PSQI: global score, component scores, and individual item scores. For a given subject, the LOCF values for all PSQI summary and individual item scores should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where PSQI global score is available. In the rare event where no PSQI global score is available after first dose due to partially completed assessments, the last post-Baseline assessment up to and including Visit 10 should be taken as the LOCF assessment for all raw and derived scores as applicable.
- CGI-I.
- Clinical laboratory parameters (blood chemistry, hematology, urinalysis, HOMA-IR (if collected). For a given subject, the LOCF values for the clinical laboratory parameters do not have to all come from the same assessment; the only exception is: the LOCF flag for the counts of leukocytes and its differential should be applied to records from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where counts of leukocytes and its differential are reported. LOCF endpoint does not need to be derived for RBC morphology findings, WBC morphology findings, and urinalysis microscopic examination findings (excluding urine erythrocytes and leukocytes).
- Urine drug screening: For a given subject, the LOCF values for all urine drug screening parameters should come from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where a urine drug screening test was administered.
- Vital sign parameters (supine and standing SBP, supine and standing DBP, supine and standing pulse rate, respiratory rate, oral temperature), weight, BMI, and waist circumference. For a given subject, the LOCF values for all vital sign parameters, height, weight, BMI, and waist circumference do not have to come from the same assessment; the only exceptions are: (1) the LOCF flag for weight and BMI should be applied

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | PPU | Version Number: | 1.0 |



to records from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where weight is available (2) the LOCF flag for supine SBP and DBP, standing SBP and DBP, and the derived corresponding orthostatic endpoints (i.e., standing SBP – supine SBP; standing DBP – supine DBP) should be applied to records from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where all four BP measures are available, (3) the LOCF flag for supine and standing pulse rate and the derived corresponding orthostatic endpoint (i.e., standing pulse rate – supine pulse rate) should be applied to records from the same assessment and it should be the last post-Baseline assessment up to and including Visit 10 where both pulse rate measures are available.

- ECG parameters: For a given subject, the LOCF values for all ECG parameters do not have to come from the same assessment. LOCF endpoint does not need to be derived for ECG parameters in the category of "FINDING".
- Nicotine use data: LOCF of this outcome measure should come from the same assessment and it should be the last assessment post first dose up to and including Visit 10 where any data are reported.
- Healthcare resource utilization data: LOCF of this outcome measure should come from the same assessment and it should be the last assessment post first dose up to and including Visit 11 where any data are reported.

The study visits will be mapped to analysis visits for table summaries and statistical analyses where applicable (Table 1).

Table 1: Mapping of study visits to analysis visits.

| Study Visit | : | Analysis Visit Number | Analysis Visit | |
|---|---|---|---|---|
| Visit 1 | | 1 | Screening/Visit 1 | |
| Visit 2 | | 2 | Pre-switch Baseline/ | √isit 2 |
| Visit 3 | | 3 | Week 1/Visit 3 | |
| Visit 4 | | 4 | Week 2/Visit 4 | |
| Visit 5 | | 5 | Week 3/Visit 5 | |
| Visit 6 | | 6 | Week 4/Visit 6 | |
| Visit 7 | | 7 | Week 5/Visit 7 | |
| Visit 8 | | 8 | Week 6/Visit 8 | |
| Document: | PPD | | | |
| Author: | ארט | | ersion Number:<br>ersion Date: | 1.0<br>06MAY2024 |



| Study Visit | Analysis Visit Number | Analysis Visit |
|---|---|---|
| Visit 9 | 9 | Week 7/Visit9 |
| Visit 10 (if representing true EOT visit). For ET visit mapping see Section 6.4. | 10 | Week 8/Visit 10 |
| Visit 11 | 11 | Week 9/Follow-up/Visit 11 |

Original study visit collected on the case report forms (CRFs) will be displayed in the listings.

## 6.4. RETESTS, UNSCHEDULED VISITS, AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the planned visits where assessment is intended to be given will be presented, as well as the derived Baseline value and the LOCF value.

Unscheduled measurements will not be included in by-visit summaries as a separate time point. Unscheduled measurements collected prior to the first dose of study medication will contribute to the derivation of the Baseline value. Unscheduled measurements collected post Baseline will contribute to the derivation of the LOCF value, the potential clinically significant (PCS) value, and the best/worst case value where required (e.g., shift table).

In the case of a retest, the assessment recorded under the planned visit will be used for by-visit summaries, and the assessment(s) recorded under unscheduled visit(s) will be presented in listings only.

As per protocol, study Visit 10 can be a Week 8/End of Treatment (EOT) visit or an Early Termination (ET) visit. If a subject terminates early, his/her measurements taken at the ET visit will be mapped to the next planned visit (after the last scheduled visit the subject attended) during which that assessment was expected to be performed as specified by the Schedule of Assessments table in the protocol. This applies to both safety and effectiveness data.

Listings will include scheduled, unscheduled, retest and early discontinuation data with original dates and visits displayed.

### **6.5.** WINDOWING CONVENTIONS

| No visit windowin | ng will be performed during the analysis for this study. Data will be analyzed according to t | he sch <u>edu</u> le outlined in the CSP. |
|---|---|---|
| Document: | PPD | |

Author: Version Number: 1.0 Version Date: 06MAY2024



### 6.6. STATISTICAL TESTS

The default significance level will be 5%; confidence intervals (CIs) will be 95%. All CIs will be two-sided, unless otherwise specified in the description of the analyses or the outputs.

### 6.7. COMMON CALCULATIONS

For quantitative measurements, change from Baseline will be calculated as:

Test Value at Visit X - Baseline Value

For PANSS total score, percentage change from Baseline will be calculated as:

(Test Value at Visit X - Baseline Value) × 100 / (Baseline Value - 30)

For other quantitative measurements, percentage change from Baseline will be calculated as:

• (Test Value at Visit X - Baseline Value) × 100 / Baseline Value

# **6.8. SOFTWARE VERSION**

All analyses will be conducted using SAS version 9.4 or later.

### 7. STATISTICAL CONSIDERATIONS

# 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

No statistical comparison will be conducted, so no adjustments for covariates and factors are to be considered.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראח | Version Number: | 1.0 |



### 7.2. MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple centers in the US.

Center pooling will not be implemented in analyses for this study.

### 7.3. MISSING DATA

Individual missing items in any scale will not be imputed in any analysis. When calculating a total score, subscale score, or any summary scores based on more than one item, if one or more items are missing at a visit, then the associated summary score will be set to missing. For additional details, see the individual scale description sections.

- Handling of missing effectiveness data, if any, is described in Sections 16.10.
- Handling of missing safety data, if any, is described in Sections 17.3 and 17.8.
- See APPENDIX 2 for details of handling incomplete/missing dates.

# 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

No statistical comparison will be conducted, so no multiplicity adjustment will be performed.

### 7.5. EXAMINATION OF SUBGROUPS

Subgroup analyses will be conducted for subjects as stated in Section 16.1 for PANSS, Section 16.2 for CGI-S, and Section 17.3.9 for Adverse Events.

The following subgroups will be assessed. The subgroup haloperidol (hal) equivalent doses will be based on appendix III of the protocol. For lumateperone, 5.5 mg is equivalent to 1 mg of haloperidol (Leucht-2020).

Sex:



- o Female
- o Male
- Age group:
  - o ≤40 years
  - o >40 years
- Race (in 3 categories):
  - o White (White)
  - o Black (Black or African American)
  - o Other (All other races combined)
- BMI (kg/m²) categories:
  - o Underweight: <18.5 kg/m<sup>2</sup>
  - o Normal: ≥18.5 to <25.0 kg/m²</p>
  - o Overweight: ≥25.0 to <30.0 kg/m²
  - o Obese: ≥30.0 kg/m<sup>2</sup>
- Baseline patient type based on UPSM factor scores at Baseline (Hopkins S., Ogirala, Loebel, & Koblan, 2020) (only used in the subgroup analysis of PANSS total score):
  - o Type 1: Prominently Disorganized
  - o Type 2: Prominently Negative
  - o Type 3: Prominently Hostile
  - o Type 4: Prominently Positive
  - o Type 5: Prominently Affective

Subjects will be classified into one of 5 patient types based on their PANSS UPSM factor scores at Baseline. See APPENDIX 9 for details of how the classification will be made.

• Primary Reason for Switch:

| Document: | PPD |
|-----------|-----|

- Sumitomo Pharma
  - Side Effect
  - Lack of Efficacy
  - Duration of Switch:
    - 2 weeks
    - 3 weeks
    - 4 weeks
    - 5 weeks
    - 6 weeks
  - Type of Pre-switch Antipsychotic
    - Partial Agonist
    - Strong M1/H1 Antagonist
    - Strong D2/3 Antagonist
    - Sedating
    - Non-sedating
  - Pre-switch AP Dose Level
    - <= 6 mg HAL equivalent
    - o > 6 mg HAL equivalent
  - Metabolic Status
    - Metabolic Syndrome
    - No Metabolic Syndrome

PPD Document: PPU Author: Version Number: 1.0 Version Date: 06MAY2024



- Reason for Clinical Discontinuation
  - Adverse Event
  - Lack of Efficacy

#### 7.5.1. DERIVATION OF SUBGROUPS

#### Metabolic Status

If a male subject meets at least 3 out of 5 of the characteristics listed below, the subject is considered metabolically impaired at Baseline.

- 1. Baseline waist circumference ≥ 102 cm
- 2. Baseline fasting triglycerides ≥ 150 mg/dL (1.7 mmol/L) or use of drug treatment for elevated triglycerides at Baseline
- 3. Baseline fasting HDL < 40 mg/dL (1.0 mmol/L) or use of drug treatment for reduced HDL at Baseline
- 4. (Baseline supine systolic blood pressure ≥ 130 mmHg and/or Baseline supine diastolic blood pressure ≥ 85 mmHg) or use of anti-hypertensive medications at Baseline
- 5. Baseline fasting glucose ≥ 100 mg/dL or use of antidiabetic medications at Baseline

If a female subject meets at least 3 out of 5 of the characteristics listed below, the subject is considered metabolically impaired at Baseline.

- 1. Baseline waist circumference ≥ 88 cm.
- 2. Baseline fasting triglycerides ≥ 150 mg/dL (1.7 mmol/L) or use of drug treatment for elevated triglycerides at Baseline
- 3. Baseline fasting HDL < 50 mg/dL (1.3 mmol/L) or use of drug treatment for reduced HDL at Baseline
- 4. (Baseline supine systolic blood pressure ≥ 130 mmHg and/or Baseline supine diastolic blood pressure ≥ 85 mmHg) or use of anti-hypertensive medications at Baseline
- 5. Baseline fasting glucose ≥ 100 mg/dL or use of antidiabetic medications at Baseline

| Document: | PPD |
|-----------|-----|



#### 8. OUTPUT PRESENTATIONS

APPENDIX 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA.

#### 9. DISPOSITION AND WITHDRAWALS

Unless otherwise specified, the disposition summary tables will include the columns: SEP-363856 50 to 100 mg/day.

All subjects who were enrolled will be accounted for in this study.

The number and percentage of subjects who were screened, screen failed, enrolled in study SEP361-308, enrolled but did not receive study medication, received at least one dose of study medication, and completed or discontinued from the treatment period (including reasons for discontinuation) will be presented. In addition, the number and percentage of subjects who rolled over to the open-label extension study (SEP361-309) will be presented.

With respect to the above, the following definitions apply:

- Screened Subjects: Any subject who signed the study specific informed consent.
- Screen Failures: Any subject who signed the study specific informed consent but either failed to meet study requirements during screening or met study requirements at screening but was not dosed.

Subjects who were screened more than once will be counted only once in the disposition summary based on the outcome of the last screening. If a subject failed multiple screenings, they will only be counted once as a screen failure. If a subject is dosed after multiple screenings, they will only be counted once as an enrolled subject.

Discontinuation by visit will be summarized for the enrolled subjects.

The number and percentage of enrolled subjects will also be summarized by Site.

Lastly, the number and percentage of enrolled subjects included in and excluded from each analysis population will be summarized, along with the reason for exclusion.

| Document: | PPD |
|-----------|-----|



#### COVID-19 related analysis updates:

The number of subjects who failed screening due to COVID-19 related reasons, who discontinued early due to COVID-19 related reasons, and who completed the treatment period but did not roll over to the open-label extension study due to COVID-19 related reasons will be summarized in the disposition table.

Subjects affected by COVID-19 related study disruptions will be provided in data listings. These subjects will be identified as:

- Subjects who failed screening due to COVID-19.
- Subjects who were enrolled but discontinued from the treatment period due to COVID-19.
- Subjects who completed the treatment period but did not roll over to the open-label extension study (SEP361-309) due to COVID-19.
- Subjects who experienced a pre-treatment event / adverse event related to COVID-19.
- Subjects who had any protocol deviations related to COVID-19.
- Subjects who had any investigator comments related to COVID-19.

A subject may be identified in one or more categories listed above.

### 9.1. DERIVATIONS

• Time to discontinuation of the treatment in days.

For the purpose of this analysis, a subject's last dose date will be derived as follows:

- o If a subject's observed last dose date is before or on the date of Study Day 56, the derived last dose date will be set to the observed last dose date.
- If a subject's observed last dose date is after the date of Study Day 56, the derived last dose date will be set to the date of Study Day 56.

Time to discontinuation (days) = Derived last dose date - First dose date + 1.

The event of interest is the discontinuation of treatment. Subjects who completed the treatment will be censored on the derived last dose date.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ררט | Version Number: | 1.0 |



### 10. IMPORTANT PROTOCOL DEVIATIONS

Important protocol deviations (IPDs) will be identified and documented based on data listings and the protocol deviations log; the data will be presented separately.

Unless otherwise specified, the IPD summary tables will include the following columns: SEP-363856 50 to 100mg/day.

The IPD categories may include, but may not be limited to:

- Did not satisfy inclusion and/or exclusion criteria.
- Received prohibited medication.
- Overall compliance rate <75% or >125%.

IPDs will be identified and presented in a data listing. The number and percentage of subjects within each IPD category will be summarized for the SAF population.

A dedicated listing will present protocol deviations related to COVID-19.

### 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Unless otherwise specified, the demographic and Baseline characteristics summary tables will include the column: SEP-363856 50 to 100 mg/day.

Demographic data and other Baseline characteristics will be presented for the SAF population, EFF population, and PP population. The data will be presented by the treatment group.

No statistical testing will be carried out for demographic or other Baseline characteristics.

The following demographic and other Baseline characteristics will be reported for this study.

Age (years) - calculated relative to date of informed consent; as a continuous variable

Age (years) categories:

0 <18 years</p>

| Document: | PPD |
|-----------|-----|

1.0

06MAY2024

PPU

Author:

### Statistical Analysis Plan

| | 0 | ≥18 to ≤40 years<br>>40 to ≤65 years<br>>65 years |
|---|---|---|
| • | Age (years) categories for ClinicalTrials.gov (CTR.GOV): | |
| • | o<br>o<br>Age (years) o | ≤18 years >18 to <65 years ≥65 years categories for European Union Drug Regulating Authorities Clinical Trials Database (EudraCT): |
| | 0 0 | <12 years ≥12 to <18 years ≥18 to <65 years ≥65 years |
| • | Sex: | |
| • | o o | Female<br>Male |
| | 0 0 0 | American Indian or Alaska Native Asian Black or African American Native Hawaiian or Other Pacific Islander White Multiracial Other |
| • | Ethnicity: | |
| Docu | o<br>o<br>ment: | Hispanic or Latino Not Hispanic or Latino PD |

Version Number:

Version Date:

- Country:
- United States
- Baseline Height (cm), as a continuous variable
- Baseline Weight (kg), as a continuous variable
- Baseline BMI (kg/m²), as a continuous variable
- Baseline BMI (kg/m²) category:
  - Underweight: <18.5 kg/m²</li>
  - o Normal: ≥18.5 to <25.0 kg/m<sup>2</sup>
  - o Overweight: ≥25.0 to <30.0 kg/m<sup>2</sup>
  - o Obese: ≥30.0 kg/m²
- Baseline Waist Circumference (cm), as a continuous variable
- Baseline PANSS Total Score, as a continuous variable
- Baseline PANSS Total Score categories:
  - < Overall median Baseline value</li>
  - ≥ Overall median Baseline value
- Baseline PANSS Subscale Scores, as continuous variables
- Baseline PANSS Subscale Score categories:
  - < Overall median Baseline value</li>
  - ≥ Overall median Baseline value
- Baseline PANSS Positive vs Negative Subscale Score categories:

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | טיי | Version Number: | 1.0 |


### Statistical Analysis Plan

- Positive Subscale Score < Negative Subscale Score</li>
- o Positive Subscale Score ≥ Negative Subscale Score
- Patient type based on Baseline UPSM factor scores:
  - o Type 1: Prominently Disorganized
  - o Type 2: Prominently Negative
  - o Type 3: Prominently Hostile
  - o Type 4: Prominently Positive
  - o Type 5: Prominently Affective
- Baseline CGI-S Score, as a continuous variable
- Baseline CGI-S Score categories:
  - o <4
  - o ≥4 to ≤5
  - o >5
- Prior Antipsychotic Drug Administration
  - o 1
  - o 2
- Number of subjects who agreed to tokenization
- DSM-5 schizophrenia subtype diagnosis:
  - o 295.90 Schizophrenia
  - o 293.89 Schizophrenia with Catatonia
- Any other current psychiatric disorders:
  - o Yes
  - o No

Diagnosis and DSM-5 code for any other current psychiatric disorders will be summarized in a separate table. These other current psychiatric disorders will be coded using Medical Dictionary for Regulatory Activities (MedDRA) central coding dictionary, Version 22.0 or higher, and presented by System Organ Class (SOC) and Preferred Term (PT).

| Document: | PPD |
|-----------|-----|



### 11.1. DERIVATIONS

BMI expressed in kg/m<sup>2</sup>:

Weight (kg)/ height (m)2.

## 12. MEDICAL HISTORY

Unless otherwise specified, the medical and surgical history summary tables will include the column: SEP-363856 50 to 100 mg/day.

Medical and surgical history information, including both past and concomitant medical conditions and major surgical history, as collected on the "Medical History" CRF form, will be coded using MedDRA, Version 22.0 or higher, and presented by SOC and PT for the SAF population by the actual treatment group. Data will be sorted by SOC based on the internationally agreed order (APPENDIX 4) and by PT in decreasing frequency.

### 13. MEDICATIONS

Unless otherwise specified, the medications summary tables will include the following columns: SEP-363856 50 to 100 mg/day.

Medications will be coded to Anatomical Therapeutic Chemical (ATC) Levels and Preferred Names according to World Health Organization Drug (WHODRUG) dictionary, Version 01MAR2019 or later.

Whenever available, the time information should be accounted for in the derivation of prior, concomitant, and post-treatment medications. See APPENDIX 2 for the handling of partial dates for medications. In the case where it is not possible to define a medication as prior, concomitant, or post treatment, the medication will be classified by the worst case; i.e., concomitant.

- Prior medications are medications which stopped prior to the first dose of study medication.
- Concomitant medications are medications which started at the same time of or after the first dose of study medication and at the same time of or before the last dose of study medication; or started prior to and ended at the same time of or after the first dose of study medication; or started at the same time of or prior to the last dose of study medication and marked as ongoing.
- Post-treatment medications are medications which started after the last dose of study medication.

| Document: | PPD |
|-----------|-----|



Prior and concomitant medication use will be summarized by ATC Level 3 and Preferred Base Name for the SAF population by the actual treatment group. Medications will be sorted by ATC Level 3 alphabetically and by Preferred Base Name in decreasing frequency in the "SEP-363856 50 to 100 mg/day" column. Similar summary for primary and secondary prior antipsychotic drug administration will also be presented separately.

Descriptive statistics of primary prior antipsychotic drug dosage at each visit will be presented. The number of subjects who complete the down tapering will also be presented by week.

Prior, concomitant, and post-treatment medications will be provided in data listings.

Psychotropic and/or Sedating Medications taken by subjects prior to each visit as collected on the "Timing of last dose of Psychotropic and/or Sedating Medications" CRF form will be summarized by ATC Level 3 and Preferred Base Name for the SAF population by the actual treatment group and visit.

## 14. STUDY MEDICATION EXPOSURE

Unless otherwise specified, the study medication exposure summary tables will include the column: SEP-363856 50 to 100 mg/day.

Exposure to study medication data will be summarized for the SAF population by the actual treatment group.

Duration of exposure (in days) will be summarized both as a continuous variable for the treatment period and categorically:

- Number and percentage of subjects with exposure  $\geq 1$ ,  $\geq 7$ ,  $\geq 14$ ,  $\geq 21$ ,  $\geq 28$ ,  $\geq 35$ ,  $\geq 42$ ,  $\geq 49$ , and  $\geq 56$  days
- Number and percentage of subjects with exposure for 1 6, 7 13, 14 20, 21 27, 28 34, 35 41, 42 48, 49 55 and ≥ 56 days

Total person-years of exposure will be calculated for all subjects.

Mean daily dose and modal daily dose will be calculated for the treatment period and summarized.

The dose adjustment decision at each visit will be summarized in a shift table.

Lastly, the number of days that a subject received the 50 mg/day dose level, the 75 mg/day dose level and 100 mg/day dose level will be summarized for the SAF population both as a continuous variable and categorically:

Number and percentage of subjects with exposure to a particular dose level for 1 - 6, 7 - 13, 14 - 20, 21 - 27, 28 - 34, 35 - 41, 42 - 48, 49 - 55 and
 ≥ 56 days

| Document: | PPD |
|-----------|-----|

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



### 14.1. DERIVATIONS

- Duration of exposure (days) = date of last dose of study drug date of first dose of study drug + 1. Interruptions in exposure (i.e., missed doses) and dose changes (if any) are not considered in the calculation of overall exposure.
- Total person-years of exposure is the sum of all durations of exposure in days / 365.25.
- Mean daily dose (mg/day):

 $\frac{\sum \mathsf{Dose} \; \mathsf{per} \; \mathsf{tablet} \; \mathsf{for} \; \mathsf{Visit} \; j \; * \; (\mathsf{\#} \; \mathsf{Tablets} \; \mathsf{Dispensed} \; \mathsf{for} \; \mathsf{Visit} \; j \; - \; \mathsf{\#} \; \mathsf{Tablets} \; \mathsf{Returned} \; \mathsf{for} \; \mathsf{Visit} \; j \; - \; \mathsf{\#} \; \mathsf{Tablets} \; \mathsf{Lost} \; \mathsf{for} \; \mathsf{Visit} \; j)}{\mathsf{Duration} \; \mathsf{of} \; \mathsf{Exposure}}$ 

If the number of tablets dispensed, returned, and/or lost as collected on the "Study Treatment Administration as Collected / Drug Accountability Log" CRF form is missing for one or more visits, the mean daily dose will be calculated based on visits with complete drug accountability data available. That is, the numerator of the formula above will only include visits with the number of tablets dispensed, returned, and lost available, and the denominator should be adjusted to exclude dosing periods covered by visits excluded from the calculation (i.e., Duration of Exposure – dosing periods [sum of (EXENDTC – EXSTDTC+1)] covered by visits with missing or incomplete accountability data). If the dose level of a visit is unknown, that visit should be excluded from the calculation as well in both the numerator and the denominator.

- Modal daily dose will be determined as the daily dose that is taken for the most time (in terms of number of days) among all doses taken. A subject's modal daily dose may fall in one of the categories below:
  - o SEP-363856 50 mg/day
  - o SEP-363856 75 mg/day
  - o SEP-363856 100 mg/day
  - o Tie between xx and yy (i.e. the subject was on xx mg/day and yy mg/day for the same amount of time) (if needed)

# 15. STUDY MEDICATION COMPLIANCE

Unless otherwise specified, the study medication compliance summary tables will include the column SEP-363856 50 to 100 mg/day.

Compliance to study medication will be presented for the SAF population, by the actual treatment group.

| Document: | PPD |
|-----------|-----|



Percent compliance will be calculated overall for the treatment period. Non-compliance is defined as less than 75% or more than 125% non-missing compliance for the treatment period. Subjects with missing compliance will not be classified as non-compliant. Compliance will be summarized both as a continuous variable and categorically (i.e., number and percentage of subjects with compliance < 75%, 75% - 125%, > 125%, and missing).

## 15.1. DERIVATIONS

Overall Compliance (%) to study medication in percentage will be calculated as follows:

$$\frac{\sum (\text{\# Tablets Dispensed for Visit }j - \text{\# Tablets Returned for Visit }j - \text{\# Tablets Lost for Visit }j)}{\text{\# Tablets should be taken per day} \times \text{Duration of Exposure}} \times 100\%$$

If the number of tablets dispensed, returned, and/or lost as collected on the "Study Treatment Administration / Drug Accountability Log" CRF form is missing for one or more visits, the overall compliance will be calculated based on visits with complete drug accountability data available. That is, the numerator of the formula above will only include visits with the number of tablets dispensed, returned, and lost available, and the denominator should be adjusted to exclude dosing periods covered by visits excluded from the calculation (i.e., change "Duration of Exposure" to be Duration of Exposure – dosing periods [sum of (EXENDTC – EXSTDTC+1)] covered by visits with missing or incomplete accountability data).

### 16. EFFECTIVENESS OUTCOMES

Unless otherwise specified, the effectiveness analysis and summary tables will include the columns: SEP-363856 50 to 100 mg/day.

All analyses of the effectiveness variables will be based on the EFF population and, for selected variables/analyses, the PP population by the actual treatment group.

Descriptive statistics presented for effectiveness outcomes include sample size, mean, standard deviation, minimum, median, maximum, and a 95% confidence interval. Confidence intervals will be based on means and standard deviations estimated without adjustment for any center or baseline effects.

## **16.1. PANSS**

The PANSS (Positive and Negative Syndrome Scale) is an interview-based measure of the severity of psychopathology in adults with psychotic disorders and comprises 30 items and 3 subscales. The positive subscale assesses hallucinations, delusions, and related

| Document: | PPD |
|-----------|-----|



symptoms (7 items); the negative subscale assesses emotional withdrawal, lack of motivation, and related symptoms (7 items); and the general psychopathology subscale assesses other symptoms such as anxiety, somatic concern, and disorientation (16 items). An anchored Likert scale from 1 to 7 (1 = absent, 7 = extreme, with values of 2 and above indicating the presence of progressively more severe symptoms) is used to score each item.

Individual items are summed to derive the following scores:

Total score = sum of all 30 items. Total score ranges from 30 to 210.

Subscale scores = sum of items within each of the following subscales:

- Positive subscale: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. The subscale score ranges from 7 to 49.
- Negative subscale: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. This subscale score ranges from 7 to 49.
- General psychopathology subscale: somatic concern, anxiety, guilt feelings, tensions, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, active social avoidance. This subscale score ranges from 16 to 112.

Marder factor scores = sum of items within each of the following factors (Marder, Davis, Chouinard. 1997):

- Negative symptoms: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of spontaneity and flow of conversation, motor retardation, active social avoidance. This Marder factor score ranges from 7 to 49.
- Positive symptoms: delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution, stereotyped thinking, somatic concern, unusual thought content, lack of judgment and insight. This Marder factor score ranges from 8 to 56.

| Document: | PPD |
|-----------|-----|



- Disorganized thought: conceptual disorganization, difficulty in abstract thinking, mannerisms and posturing, poor attention, disturbance of volition, preoccupation, disorientation. This Marder factor score ranges from 7 to 49.
- Uncontrolled hostility/excitement: excitement, hostility, uncooperativeness, poor impulse control. This Marder factor score ranges from 4 to 28.
- Anxiety/depression: anxiety, guilt feelings, tension, depression. This Marder factor score ranges from 4 to 28.

UPSM (Uncorrelated PANSS Score Matrix) factor scores = PANSS item scores of each subject at each visit transformed using the UPSM to obtain scores of 7 transformed PANSS factors (Hopkins et al. 2018):

- POS: Positive
- DIS: Disorganized
- NAA: Negative apathy/avolition
- NDE: Negative deficit of expression
- HOS: Hostility
- ANX: Anxiety
- DEP: Depression

The transformation will be done as follows:

- [Transformed PANSS Factor Data] $_{(N\times7)} = [PANSS Data]_{(N\times30)} * [UPSM]_{(30\times7)}$
- where

[Transformed PANSS Factor Data] $_{(N\times7)}$  is the transformed matrix with N sets of scores for the 7 transformed PANSS factors.

| Document: | PPD |
|-----------|-----|

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



[PANSS Data] $_{(N\times30)}$  is a matrix with N PANSS assessments and 30 columns containing the scores of 30 PANSS items ordered in the same way as shown in UPSM.

[UPSM] $_{(30\times7)}$  is a matrix with 30 rows (one for each PANSS item) and 7 columns (one for each of the 7 transformed PANSS factors). This matrix is presented in <u>APPENDIX 3</u>.

UPSM total factor score = sum of the 7 UPSM factor scores.

PANSS is assessed at these study visits: Visit 1, Visit 2, Visit 3, Visit 4, Visit 6, Visit 8 and Visit 10.

#### 16.1.1. PANSS TOTAL SCORE

PANSS is assessed at these study visits: Visit 1, Visit 2, Visit 3, Visit 4, Visit 6, Visit 8, and Visit 10. The Baseline PANSS total score will be derived as described in Section 6.2. The change from Baseline in PANSS total score at Week 8, as well as at the other post-Baseline time points, will be derived as described in Section 6.7.

The observed PANSS total score and the change from Baseline values will also be summarized descriptively by treatment group and visit.

The observed PANSS total score and the change from Baseline values will also be summarized descriptively by treatment group and visit for each subgroup listed in Section 7.5.

#### 16.1.2. Proportion of Subjects Who Achieve a Response

PANSS response is defined as a 20% or greater improvement (i.e. decrease) in PANSS total score from Baseline.

The percent change in PANSS total score from Baseline will be calculated by:

PANSS total score at a visit or the Week 8 LOCF endpoint - PANSS total score at Baseline × 1009

PANSS total score at Baseline - 30

For each subject, the responder indicator will be set to 1 if the percent change is negative and the magnitude is equal to or greater than 20%. The indicator will be set to 0 if the percentage is negative but the magnitude is less than 20% or the percentage is non-negative. The

| Document: | PPD |
|-----------|-----|



indicator will be set to missing if the percentage is missing.

In addition, PANSS response defined by two more stringent thresholds will be assessed; that is, having a 30% or greater and 50% or greater improvement in PANSS total score from Baseline.

PANSS response at all three thresholds will be derived for all post-Baseline time points.

The number and percentage of subjects who achieve a PANSS response will also be summarized descriptively by treatment group and visit.

The proportion of subjects achieving a given percentage change threshold in PANSS total score from Baseline at the LOCF endpoint will be calculated for each treatment group. This calculation will be performed at multiple thresholds, starting from -100% and increases at 5% increments or until all subjects are accounted for in all treatment groups, with 5% increments.

#### 16.1.3. PANSS SUBSCALE SCORES

Individual items from the PANSS scale are summed to derive the following subscale scores:

- Positive subscale: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility. This subscale score ranges from 7 to 49.
- Negative subscale: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. This subscale score ranges from 7 to 49.
- General psychopathology subscale: somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, active social avoidance. This subscale score ranges from 16 to 112.

PANSS is assessed at these study visits: Visit 1, Visit 2, Visit 3, Visit 4, Visit 6, Visit 8, and Visit 10. The Baseline PANSS subscale scores will be derived as described in Section 6.2. The change from Baseline in PANSS subscale scores at each post-Baseline time point will be derived as described in Section 6.7.

The observed values of PANSS subscale scores at Baseline and each scheduled post-Baseline visit will be summarized descriptively. The Baseline PANSS subscale scores will be derived as described in Section 6.2.

The change from Baseline in PANSS subscale scores will be summarized for each scheduled post-Baseline visit. The change from Baseline in PANSS

| Document: | PPD |
|-----------|-----|



subscale scores will be derived as described in Section 6.7.

#### 16.1.4. PANSS MARDER FACTOR SCORES

Individual items from the PANSS scale are summed to derive the following Marder factors (Marder, Davis, & Chouinard, 1997;58:538–46):

- Negative symptoms: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of spontaneity and flow of conversation, motor retardation, and active social avoidance. This Marder factor score ranges from 7 to 49.
- Positive symptoms: delusions, hallucinatory behavior, grandiosity, suspiciousness/persecution, stereotyped thinking, somatic concern, unusual thought content, and lack of judgment and insight. This Marder factor score ranges from 8 to 56.
- Disorganized thought: conceptual disorganization, difficulty in abstract thinking, mannerisms and posturing, poor attention, disturbance of volition, preoccupation, and disorientation. This Marder factor score ranges from 7 to 49.
- Uncontrolled hostility/excitement: excitement, hostility, uncooperativeness, and poor impulse control. This Marder factor score ranges from 4 to 28.
- Anxiety/depression: anxiety, guilt feelings, tension, and depression. This Marder factor score ranges from 4 to 28.

PANSS is assessed at these study visits: Visit 1, Visit 2, Visit 3, Visit 4, Visit 5, Visit 6, Visit 7, Visit 8, and Visit 10. The Baseline PANSS Marder factor scores will be derived as described in Section 6.2. The change from Baseline in PANSS Marder factor scores at each post-Baseline time point will be derived as described in Section 6.7.

The observed values of PANSS Marder factor scores at Baseline and each scheduled post-Baseline visit will be summarized descriptively. The Baseline PANSS Marder factor scores will be derived as described in Section 6.2.

The change from Baseline in PANSS Marder factor scores will be summarized for each scheduled post-Baseline visit. The change from Baseline in PANSS Marder factor scores will be derived as described in Section 6.7.

#### 16.1.5. PANSS UPSM FACTOR SCORES AND THE UPSM TOTAL FACTOR SCORE

The PANSS item scores of each subject at each visit will be transformed using the UPSM, to obtain the scores of 7 transformed PANSS factors (Hopkins S., Ogirala, Loebel, & Koblan, 2018;44(3):593-602):

POS: Positive

| Document: | PPD |
|-----------|-----|



### Statistical Analysis Plan

DIS: Disorganized

NAA: Negative apathy/avolition

NDE: Negative deficit of expression

HOS: Hostility

ANX: Anxiety

DEP: Depression

The transformation will be done as follows:

[Transformed PANSS Factor Data]<sub>(N×7)</sub> = [PANSS Data]<sub>(N×30)</sub> \* [UPSM]<sub>(30×7)</sub>

#### where

- o [Transformed PANSS Factor Data] $_{(N\times7)}$  is the transformed matrix with N sets of scores for the 7 transformed PANSS factors.
- o  $[PANSS Data]_{(N\times30)}$  is a matrix with N PANSS assessments and 30 columns containing the scores of 30 PANSS items ordered in the same way as shown in UPSM.
- [UPSM] $_{(30\times7)}$  is a matrix with 30 rows (one for each PANSS item) and 7 columns (one for each of the 7 transformed PANSS factors). This matrix is presented in APPENDIX 3.

Lastly, the UPSM total factor score will be calculated as the sum of the 7 UPSM factor scores.

PANSS is assessed at these study visits: Visit 1, Visit 2, Visit 3, Visit 4, Visit 5, Visit 6, Visit 7, Visit 8, and Visit 10. The Baseline PANSS UPSM factor scores and UPSM total factor score will be derived as described in Section 6.2. The change from Baseline in PANSS UPSM factor scores and UPSM total factor score at each post-Baseline time point will be derived as described in Section 6.7.

The observed values of PANSS UPSM factor scores at Baseline and each scheduled post-Baseline visit will be summarized descriptively. The Baseline PANSS UPSM factor scores will be derived as described in Section 6.2.

The change from Baseline in PANSS UPSM factor scores will be summarized for each scheduled post-Baseline visit. The change from Baseline in PANSS UPSM factor scores will be derived as described in Section 6.7.

The observed values of PANSS UPSM total factor score at Baseline and each scheduled post-Baseline visit will be summarized descriptively. The Baseline PANSS UPSM total factor score will be derived as described in Section 6.2.

| Document: | PPD |
|-----------|-----|

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



The change from Baseline in PANSS UPSM total factor score will be summarized for each scheduled post-Baseline visit. The change from Baseline in PANSS UPSM total factor score will be derived as described in Section 6.7.

# 16.2. CLINICAL GLOBAL IMPRESSION-SEVERITY

The CGI-S (Clinical Global Impression-Severity) is a clinician-rated assessment of the subject's current illness state on a 7-point scale, where a higher score is associated with greater illness severity. The CGI-S score takes one of the following values: 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill patients).

CGI-S is assessed at these study visits: Visit 1, Visit 2, Visit 3, Visit 4, Visit 6, Visit 8, and Visit 10. The Baseline CGI-S score will be derived as described in Section 6.2. The change from Baseline in CGI-S score at Week 8, as well as at the other post-Baseline time points, will be derived as described in Section 6.7.

The observed CGI-S score and the change from Baseline values will also be summarized descriptively by treatment group and visit.

The observed CGI-S score and the change from Baseline values will also be summarized descriptively by treatment group and visit for each subgroup.

# 16.3. BRIEF NEGATIVE SYMPTOM SCALE (BNSS) TOTAL SCORE AND SUBSCALE SCORES

The BNSS (Brief Negative Symptom Scale) is a rating scale that measures the current level of severity of negative symptoms in schizophrenia and schizoaffective disorder. The measure is comprised of 13 individual items organized into 6 subscales: blunted affect (items 9, 10, 11), alogia (items 12, 13), avolition (items 7, 8), anhedonia (items 1, 2, 3), asociality (items 5, 6), and distress (item 4). Each of the items are scored on a Likert-type 7-point scale from 0-6, where values of 0 indicates the symptom is absent and a value of 6 means the symptom is a severe form. The subscale scores are calculated by summing the individual items within each scale. The 13 items are also summed to provide a total score which ranges from 0 to 78.

BNSS is assessed at these study visits: Visit 2, Visit 6, Visit 10.

The observed values of BNSS total score and BNSS subscale scores at Baseline and each scheduled post-Baseline visit will be summarized descriptively. The Baseline BNSS total score and BNSS subscale scores will be derived as described In Section 6.2.

The change from Baseline in BNSS total score and BNSS subscale scores will be summarized for each scheduled post-Baseline visit. The change from Baseline in BNSS total score and BNSS subscale scores will be derived as described in Section 6.7.

| Document: | PPD |
|-----------|-----|



# 16.4. 12-ITEM SHORT FORM SURVEY (SF-12)

The SF-12 is a 12-item self-reported questionnaire that is a subset of the SF-36 Health Survey. The survey captures physical and mental health. There are 8 subscales including: Physical functioning, Role-physical, Bodily pain, General health, Vitality, Social Functioning, Role emotional, and Mental health. The responses are reported on a 3- or 5-point Likert scale, depending on the question. The SF-12 uses 2-items each to estimate scores for 4 of the 8 health concepts (physical functioning, role-physical, role-emotional, and mental health). Score for the remaining 4 healthy concepts (bodily pain, general health, vitality, and social functioning) are estimated using 1 item each. Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12) are computed using the scores of 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The norm-based subdomain scores are the scores normed to the US population to have a mean of 50 and standard deviation of 10.

The observed values of the SF-12 for each subdomain (both raw and norm-based) such as general health, physical functioning, role physical, bodily pain, vitality, role emotional, mental health, social functioning, and both PCS and MCS composite scores and health utility index score at Baseline and each scheduled post-Baseline visit will be summarized descriptively.

The change from Baseline will be summarized for each scheduled post-Baseline visit.

### 16.5. PSP TOTAL SCORE AND INDIVIDUAL DOMAIN SCORES

The PSP (Personal and Social Performance Scale) is a 100-point single-item rating scale of personal and social functioning. The 100-point rating scale is subdivided into 10 equal intervals (or 10-point categories). The rating is based on the assessment of a patient's functioning in four areas: 1) socially useful activities, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behaviors. Each area is evaluated using the degree of severity: Absent, Mild, Manifest, Marked, Severe and Very Severe. For the purpose of analysis, the following numerical values will be assigned to the degrees of severity:





A PSP total score (range 1 to 100) is assigned by the rater based on the subject's functioning in the four areas.

Higher PSP total scores indicate better functioning. Scores of 1-30 indicate functioning so poor that intensive support or supervision is needed; scores of 31-70 indicate varying degrees of difficulty; and scores of 71-100 reflect only mild difficulties.

PSP is assessed at these study visits: Visit 2 and Visit 10. The Baseline PSP total score will be derived as described in Section 6.2. The change from Baseline in PSP total score at each post-Baseline time point will be derived as described in Section 6.7.

In addition, the following binary outcomes based on PSP total score will be derived:

- PSP total score ≥71 at Baseline and each scheduled visit (Week 8/Visit 10)
- Improvement of ≥1 PSP 10-point category from Baseline to each scheduled visit (Week 8/Visit 10)

For each subject, the indicator for each of the binary outcomes described above will be set to Y if the subject satisfied the condition, and N if the subject failed to satisfy the condition. The indicator will be set to missing if the data necessary for the derivation is missing (e.g., the PSP total score is missing at a particular time point).

The observed PSP total score and individual domain scores and the change from Baseline values will also be summarized descriptively by treatment group and visit.

The number and percentage of subjects satisfying each binary outcome listed below at Week 8/Visit 10 will be summarized descriptively by treatment group and visit.

- PSP total score ≥71 at Baseline and each scheduled visit (Week 8/Visit 10)
- Improvement of ≥1 PSP 10-point category from Baseline to each scheduled visit (Week 8/Visit 10)

In addition, the number and percentage of subjects that fall in each of the following PSP categories will be summarized descriptively by treatment group and visit:

- o Total score 100-71 (mild to no impairment).
- Total score 70-51 (moderate impairment)
- o Total score 50-31 (marked impairment)
- o Total score 30-1 (severe impairment)

| Document: | PPD |
|-----------|-----|



# 16.6. MEDICATION SATISFACTION QUESTIONNAIRE (MSQ)

The MSQ is a single-item, patient-rated, rater administered questionnaire that requires the subject to use a 7-point, Likert-type scale to rate how satisfied they are with their current antipsychotic medication. The subject will be asked the following question: "Overall, how satisfied are you with your current antipsychotic medication".

Subjects will select 1 of 7 potential responses based on their level of satisfaction from extremely dissatisfied (1) to extremely satisfied (7) as follows:

- (1) Extremely dissatisfied
- (2) Very dissatisfied
- (3) Somewhat dissatisfied
- (4) Neither dissatisfied nor satisfied
- (5) Somewhat satisfied
- (6) Very satisfied
- (7) Extremely satisfied

MSQ is assessed at these study visits: Visit 2 and Visit 10. The Baseline MSQ score will be derived as described in Section 6.2. The change from Baseline in MSQ score at each post-Baseline time point will be derived as described in Section 6.7.

The analysis of MSQ data will be limited to subjects who were being treated with an antipsychotic medication at the time of screening or had been treated with antipsychotic medications within 30 days prior to the Screening visit.

The observed MSQ score and the change from Baseline values will also be summarized descriptively by treatment group and visit. In addition, the frequency distribution of the MSQ score will be summarized descriptively by treatment group and visit.

# 16.7. CLINICAL GLOBAL IMPRESSIONS — IMPROVEMENT SCALE (CGI-I)

The CGI-I scale is a standard 7-point scale (Guy-1976) that requires the clinician to assess how much the subject's overall symptoms have improved or worsened relative to a baseline state.

The observed CGI-S score and the change from Baseline values will also be summarized descriptively by treatment group and visit.

| Document: | PPD |
|-----------|-----|

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



The observed CGI-S score and the change from Baseline values will also be summarized descriptively by treatment group and visit for each subgroup.

# 16.8. HEALTHCARE RESOURCE UTILIZATION

Healthcare resource utilization is assessed at these study visits: Visit 2 and Visit 10.

The number of physician's office visits, ER visits, and hospitalizations (for any reason and those related to schizophrenia) per month at Baseline and at Week 8/Visit 10, as well as the average length of hospital stays (for any reason and those related to schizophrenia) at Baseline and at Week 8/Visit 10, will be summarized. The frequency and percentage of subjects receiving unpaid care at Baseline and at Week 8/Visit 10, along with the average number of hours a caregiver spends per week helping the subject, will also be summarized.

The change in the number of physician's office visits, ER visits, and hospitalizations, the average length of hospital stays, and the average number of hours a caregiver spends per week helping the subject from Baseline at Week 8/Visit 10 will be summarized.

Shift from Baseline to Week 8/Visit 10 in whether the subjects receive unpaid care will also be summarized.

# 16.9. NICOTINE USE

Nicotine use is assessed at these study visits: Visit 1 and Visit 10. Nicotine use data will be summarized descriptively by treatment group and visit.

For each nicotine type, the amount being used at Week 8/Visit 10 and LOCF in comparison with the amount being used at Baseline will be classified as "increased", "decreased", or "unchanged" for every subject, based on the reported amount used in a given period. If a subject quit using a particular type of nicotine since Baseline, the amount used for that nicotine type will be classified as "decreased". If a subject newly started or restarted using a particular type of nicotine since Baseline, the amount used for that nicotine type will be classified as "increased".

Then for subjects whose changes in amount for all nicotine types between Baseline and each scheduled post-Baseline visit (Week 8/Visit 10 and LOCF) are not in opposite directions, a subject's overall nicotine consumption at each scheduled post-Baseline visit in comparison with Baseline will be classified as "increased", "decreased", or "unchanged" based on the following:

- If the change in amount for each nicotine type is either "increased" or "unchanged", the subject's overall consumption will be classified as "increased".
- If the change in amount for each nicotine type is either "decreased" or "unchanged", the subject's overall consumption will be classified as "decreased".

| Document: | PPD |
|-----------|-----|



• If the change in amount for all nicotine types is "unchanged", the subject's overall consumption will be classified as "unchanged".

The number and percentage of subjects in each overall consumption amount change category will be summarized by treatment group.

In addition, for subjects who reported using "Cigarettes" at either Baseline or each scheduled post-Baseline visit (Week 8/Visit 10 and LOCF) or at both time points, the number of cigarettes used per day will be derived for both time points. The following conversion will be applied if necessary:

- Amount: 1 Pack = 20 Cigarettes.
- Time period: 1 Week = 7 Days; 1 Month = 30 Days.

The amount of cigarette used per day and the change from Baseline values will be summarized by treatment group and visit.

# 16.10. MISSING DATA METHOD

Any individual missing item in any scale will not be imputed.

For derived scores that depend on more than one individual item (e.g., PANSS total score, PANSS subscale scores, PANSS Marder factor scores, PANSS UPSM factor scores and UPSM total factor score, BNSS total score, BNSS subscale scores, MADRS total score), if one or more items are missing at a visit, the derived score will be set to missing. The corresponding change from Baseline value at a given post-Baseline time point will be set to missing if the Baseline derived score is missing or if the derived score at that time point is missing.

For PANSS response, any subject with a missing PANSS total score at Baseline or at any post-Baseline time point will have their PANSS response set to missing for that time point.

For PSP binary variables based on the PSP total score, if the PSP total score is missing at Baseline or at any post-Baseline time point, the affected binary variable will be set to missing.

# 17. SAFETY OUTCOMES

Unless otherwise specified, the safety analysis and summary tables will include the column SEP-363856 50 to 100 mg/day All analyses of the safety outcomes will be based on the SAF Population, by treatment group.

| Document: | PPD |
|-----------|-----|



### 17.1. DISCONTINUATION DUE TO CLINICAL REASONS

Discontinuation for clinical reasons is defined as reasons due to AE or lack of efficacy. AE will follow the definition as in section 17.3.

The percentage of subjects who discontinued for clinical reasons will be calculated by a proportion consisting of the number of subjects who experience a discontinuation event due to clinical reasons as the numerator divided by the number of subjects in the safety population as the denominator multiplied by 100 along with a corresponding 95% confidence interval (CI).

The number and percentage of subjects, who discontinued early from the open-label treatment period (including both clinical reasons, ie, discontinued due to an AE or lack of efficacy (primary endpoint) and any reason for discontinuation (secondary endpoint)) will be presented.

The time-to-discontinuation for clinical reasons will be summarized descriptively, (eg, n, median, 25th percentile, 75th percentile, minimum and maximum, and 95% CI on median, where possible).

Time to discontinuation for clinical reasons since first dose of study medication will be plotted using Kaplan-Meier curves for the safety population by treatment group. Probability of remaining on treatment at Day 56, median time to discontinuation, and their 95% confidence intervals will be estimated using the Kaplan-Meier method for the safety population by treatment group.

# 17.2. DISCONTINUATION DUE TO ANY REASONS

The percentage of subjects who discontinued for any reason (ie, all cause discontinuation). The percentage will be calculated similarly as that of the primary endpoint along with a corresponding 95% CI.

Kaplan-Meier analysis as in section 17.1 will be performed for time to discontinuation for any reasons.

## 17.3. ADVERSE EVENTS AND PRE-TREATMENT EVENTS

Adverse events (AEs) and pre-treatment events will be coded using MedDRA central coding dictionary, Version 22.0 or higher.

Any COVID-19 related Adverse Events and pre-treatment events will be identified using a pre-defined search:

| Document: | PPD |
|-----------|-----|

| Lower Level<br>Term | Lower Level<br>Term Code | Preferred<br>Term | Preferred<br>Term Code | Search Criteria for COVID-19<br>Related Adverse Events or<br>Pre-treatment Events |
|---|---|---|---|---|
| Coronavirus test positive | 1007025 | Coronavirus test positive | 10070255 | Preferred Term Code = 10070255 or 10053983 |
| Coronavirus infection | 10051905 | Corona virus infection | 10053983 | |

AEs are defined as untoward medical occurrences that started at the same time of or after the first dose of study drug. Untoward medical occurrences that started prior to the first dose of study drug are pre-treatment events.

Whenever available, the time information should be accounted for in the derivation of AEs vs. pre-treatment events. In the case where time is not available, untoward medical occurrences that started on or after the day of the first dose of study drug will be considered AEs; those that started before the day of the first dose of study drug will be considered pre-treatment events.

See APPENDIX 2 for handling of partial dates for AEs. In the case where it is unclear whether an untoward medical occurrence is an AE or a pretreatment event, the algorithm uses a conservative approach where the untoward medical occurrence is classified by the worst case; i.e., AE.

AEs (including serious adverse events (SAEs)) are collected into the clinical database until the last study visit. For subjects who do not roll over to study 361-309, the last study visit will be Visit 11 (the follow-up visit) which per protocol should occur 7 (± 2) days after the last dose of study drug. For subjects continuing into study 361-309, the last 361-308 study visit will be Visit 10 (the end of treatment visit). If an AE (or a pre-treatment event) started in 361-308 and was ongoing at rollover, this adverse event (pre-treatment event) will be marked Ongoing in the 361-308 database. It will also be re-entered into the 361-309 database and its outcome will be monitored and updated in the 361-309 database.

Overall summary of the incidence of all AEs, AEs related to COVID-19, study medication-related AEs, severe AEs, serious AEs, AEs leading to discontinuation from study, AEs leading to study medication withdrawal, AEs leading to study medication interruption, and AEs leading to death will be provided by treatment group. This overall incidence summary will also be separately presented for the following subgroups: country, sex, age group, number of prior hospitalizations for treatment of schizophrenia, duration of schizophrenia, and BMI category.

Listings will be provided for all AEs, AEs related to COVID-19, study medication-related AEs, severe AEs, serious AEs, AEs leading to discontinuation from the study, AEs leading to study medication withdrawal, AEs leading to study medication interruption, AEs leading to death, AEs of potential drug abuse and dependence and extrapyramidal AEs. A listing of the pre-treatment events will also be presented. When complete event start date and complete event end date are available, duration of AEs/pre-treatment events will be calculated as: event end date – event start date + 1. Duration will be presented in data listings.

| Document: | PPD |
|-----------|-----|



PROTOCOL SEP361-308 

For all summaries, each subject will be counted only once within each category (e.g., an AE type, a severity level, a relationship category, a SOC, a high level term (HLT), and a PT). If not otherwise specified, all summaries will present the number and percentage of subjects as well as the number of events. For summaries by SOC and PT, AEs will be sorted by SOC based on the internationally agreed order (see APPENDIX 4) and then by PT in decreasing frequency in the "SEP-363856 50 to 100 mg/day" column. For summaries by SOC, HLT, and PT, AEs will be sorted by SOC based on the internationally agreed order and then by HLT and PT in decreasing frequency in the "SEP-363856 50 to 100 mg/day" column.

COVID-19 related pre-treatment events related pre-treatment events and AEs will be displayed similarly as any other pre-treatment events and AEs.

| Document: | PPD |
|-----------|-----|



#### 17.3.1. ALL AES

All AEs will be summarized by PT, by SOC and PT, as well as by SOC, HLT, and PT. The summary by SOC and PT will also be presented for the following subgroups: sex, age group and BMI category.

Summary tables (by SOC and PT) will be generated for those AEs starting after the last dose of study drug and those AEs starting more than 1 day after the last dose of study drug.

AEs reported by ≥ 2.0% (without rounding) of subjects in any treatment group will be summarized by SOC and PT.

Non-serious AEs reported by > 5.0% (without rounding) of subjects will be summarized by SOC and PT.

The summary by SOC and PT will be broken down further by maximum severity and by strongest relationship to study medication. These summaries are described in the sections below.

#### **17.3.2. SEVERITY**

Severity is classed as mild/moderate/severe (increasing severity). AEs with a missing severity will be classified as severe.

If a subject reported an AE more than once within the same SOC/ PT with different severity levels, the subject will be assigned to a severity level for that SOC/ PT based on the worst case severity (i.e., maximum severity). Event counts will not be included in this summary.

In a separate table, severe AEs will be summarized by SOC and PT.

#### 17.3.3. RELATIONSHIP TO STUDY MEDICATION

Relationship to study medication, as indicated by the Investigator, is classed as "not related" ("probable" ("definite" (increasing strength of relationship). A "related" AE is defined as an AE with a relationship to study medication as "possible", "probable" or "definite". AEs with a missing relationship to study medication will be regarded as related to the study medication. For this summary, AEs will be presented in 2 categories, related and not related.

If a subject reported an AE more than once within the same SOC/ PT in different relationship categories, the subject will be assigned to a category for that SOC/ PT based on the worst case relationship (i.e., strongest relationship). Event counts will not be included in this summary.

In separate tables, study medication-related AEs will be summarized by SOC and PT and summarized by PT.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראח | Version Number: | 1.0 |



#### 17.3.4. AES LEADING TO DISCONTINUATION FROM STUDY

AEs leading to discontinuation from the study are those AEs with "Caused Study Discontinuation" = "Yes" on the "Adverse Events" CRF form.

AEs leading to discontinuation from the study will be summarized by SOC and PT.

#### 17.3.5. AES LEADING TO STUDY MEDICATION WITHDRAWAL

AEs leading to permanent withdrawal from the study medication are those AEs with "Action Taken with Study Treatment" = "Drug Withdrawn" on the "Adverse Events" CRF form.

AEs leading to study medication withdrawal will be summarized by SOC and PT.

#### 17.3.6. AES LEADING TO STUDY MEDICATION INTERRUPTION, STUDY DOSE INCREASE AND REDUCED

AEs leading to study medication interruption, study dose increase, study dose reduce are those AEs with "Action Taken with Study Treatment" = "Drug Interrupted", "Action Taken with Study Treatment" = "Dose Increased", "Action Taken with Study Treatment" = "Dose Reduced" respectivelyon the "Adverse Events" CRF form.

AEs leading to study medication interruption will be summarized by SOC and PT.

#### 17.3.7. SERIOUS ADVERSE EVENTS

SAEs are those AEs recorded as "Serious" on the "Adverse Events" CRF form.

SAEs will be summarized by SOC and PT. The summary will also be presented for the following subgroups: country, sex, age group, number of prior hospitalizations for treatment of schizophrenia, duration of schizophrenia, and BMI category.

In a separate table, SAEs starting within 7 days, after the last dose of study drug will be summarized by SOC and PT as well.




#### 17.3.8. Adverse Events Leading to Death

AEs leading to death are those AEs with "Outcome" = "Fatal" on the "Adverse Events" CRF form.

AEs leading to death will be summarized by SOC and PT.

#### 17.3.9. Adverse Events of Potential Drug Abuse and Dependence

AEs associated with potential drug abuse and dependence will be identified as described in APPENDIX 5.

These AEs will be summarized by PT only.

#### 17.3.10. EXTRAPYRAMIDAL ADVERSE EVENTS

Extrapyramidal AEs will be identified by MedDRA SMQ 20000095 Extrapyramidal syndrome as described in APPENDIX 6.

These AEs will be summarized by PT only.

#### 17.3.11. ADVERSE EVENTS BY SUBGROUPS

The subgroup factors of interest for AE summaries include: country, sex, age group, number of prior hospitalizations for treatment of schizophrenia, duration of schizophrenia, and BMI category (see Section 7.5). AE by subgroup summaries are described in the individual sections above.

# 17.3.12. PSYCHIATRIC ADVERSE EVENTS LEADING TO DISCONTINUATION FROM STUDY (PAEDCS)

Additional information is collected for the non-serious psychiatric AEs that led to discontinuation from the study as well as for all serious psychiatric AEs within the study. The information is recorded in separate trackers and not part of the CRF. This information will be presented in separate data listings only.

| Document: | PPD |
|-----------|-----|



### 17.4. LABORATORY EVALUATIONS

Results from the central laboratory to be reported for this study include Hematology, Chemistry (including lipid panel and thyroid panel), Urinalysis, Urine drug screening, Rapid Urine Drug Screening, Serology panel, Serum pregnancy (β-HcG) (in female subjects only), Urine pregnancy (in female subjects only), Rapid Urine Pregnancy Test (in female subjects only), Follicle stimulating hormone (FSH) (in female subjects with suspected menopause).

Serum and urine pregnancy results in female subjects, FSH level in female subjects, serology panel in subjects, and any unexpected lab parameters not specified in protocol Section 22 (APPENDIX IV. CLINICAL LABORATORY TESTS) will only be listed. Laboratory parameters prespecified in protocol Section 22 under the categories of "HEMATOLOGY", "BLOOD CHEMISTRIES" (plus HOMA-IR if collected), "URINALYSIS", and "URINE DRUG SCREENING" will be summarized in tables as well as presented in listings.

Listing presentations will use both standard international (SI) Units and conventional units (CV). Table summaries will also be provided using both SI units and conventional units.

Quantitative laboratory measurements reported as "< X", i.e., below the lower limit of quantification (BLQ), or "> X", i.e., above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but they will be presented as recorded, i.e., as "< X" or "> X" in the listings.

The following summaries will be provided:

- By-visit summary of observed values and change from Baseline values for quantitative measurements in hematology, chemistry, and urinalysis.
   Serum prolactin results will be summarized overall and separately by sex. Glucose, insulin and lipid panel results (total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides) will be summarized by fasting status: fasting only and overall (fasting, non-fasting, or fasting status unknown combined). Change from Baseline for glucose, insulinand lipid panel results will only be calculated if post-Baseline fasting status is matching Baseline fasting status.
- By-visit summary of the number and percentage of subjects in each outcome category for qualitative measurements in urinalysis (as applicable) and for urine drug screening results. Urine drug screening results will be reported as "Positive"/ "Negative".
- Shift in laboratory results (chemistry, hematology, urinalysis) from Baseline to Week 8/Visit 10 and LOCF Endpoint according to the reference range criteria. The existing reference range indicators provided by the central laboratory will be mapped as needed to categories of "Normal" (within the reference range) / "Abnormal" (outside the reference range) for urinalysis non-pH results, and to categories of "Low" (below the reference range) / "Normal" (within the reference range) / "High" (above the reference range) for chemistry and hematology results as well as urinalysis pH results.

| Document: | PPD |
|-----------|-----|



• Number and percentage of subjects with at least one potentially clinically significant (PCS) laboratory value (see APPENDIX 7) post Baseline. The period of evaluation includes the follow-up period, including unscheduled visits. Subjects will be counted in a particular PCS category if they met that PCS criteria at least once post Baseline, regardless of their Baseline value.

All laboratory data will be provided in data listings, with the values outside the reference ranges flagged. In addition, separate listings will be provided to present the laboratory data that met the PCS criteria.

Boxplots will be created to present Baseline and Week 8/Visit 10 values by treatment group for lipid parameters (total cholesterol, LDL, HDL, and triglycerides), glucose, insulinby fasting status: fasting only and overall (fasting, non-fasting, or fasting status unknown combined). In addition, boxplots will be created to present Baseline and Week 8/Visit 10 prolactin values by treatment group by sex: Overall, males, females. Lastly, the values of HbA1c will be presented for Baseline and Week 8/Visit 10 by treatment group in boxplots as well. Each of these boxplots will be repeated to present the change from Baseline values.

#### 17.4.1. LABORATORY SPECIFIC DERIVATIONS

No applicable derivations.

#### 17.4.2. LABORATORY REFERENCE RANGES

Laboratory reference range indicators will be provided by the laboratory vendor and used in statistical analyses. Only if a reference range indicator is missing in the data transfer will it be derived in the analysis step as described below.

- Quantitative laboratory measurements (that are not urinalysis erythrocytes or urinalysis leukocytes) will be compared with the relevant laboratory reference ranges in <u>original</u> units and categorized as:
  - o Low: Below the lower limit of the laboratory reference range.
  - o Normal: Within the laboratory reference range (upper and lower limit included).
  - o High: Above the upper limit of the laboratory reference range.
- For laboratory parameters with categorical outcomes as well as urinalysis erythrocytes and urinalysis leukocytes, if the result is within the reference range, the indicator is "NORMAL"; if the result is not within range, the indicator is "ABNORMAL".

| Document: | PPD |
|-----------|-----|



# 17.5. ECG EVALUATIONS

Data from the centrally over-read ECG (Electrocardiogram) results will be included in the reporting of this study.

The following ECG parameters will be reported for this study:

- PR Interval (msec)
- RR Interval (msec)
- QRS Duration (msec)
- QRS Axis (deg)
- QT Interval (msec)
- QTcF Interval (msec) (Fridericia's Correction of QT interval)
- QTcB Interval (msec) (Bazett's Correction of QT interval)
- Heart Rate (bpm)
- Overall assessment of ECG as determined by the central over-read:
  - o Normal
  - o Abnormal, Insignificant
  - o Abnormal, Potentially Significant
  - o Abnormal, Significant
  - o Exclusion Alert (only given for the Screening visit). In table summaries, the category of "Exclusion Alert" will be combined into the category of "Abnormal, Significant".
  - o Not Evaluable
- ECG findings

| Document: | PPD |
|-----------|-----|



ECG findings will only be listed. Other ECG data will be summarized in tables as well as presented in listings.

The following summaries will be provided:

- By-visit summary of observed values and change from Baseline values for quantitative measurements.
- By-visit summary of ECG overall assessment results as determined by the central over-read ("Normal", "Abnormal, Insignificant", "Abnormal, Potentially Significant", "Abnormal, Significant", "Not Evaluable").
- Shift in ECG overall assessment as determined by the central over-read from Baseline to Week 8/Visit 10, and LOCF endpoint.
- Number and percentage of subjects who met each of the QTc interval prolongation criteria (see Section 17.5.1). The period of evaluation includes both the treatment period and the follow-up period, including unscheduled visits.
- Number and percentage of subjects with at least one PCS ECG value (see Section 17.5.2) post Baseline. The period of evaluation includes both the treatment period and the follow-up period, including unscheduled visits. Subjects will be counted in a particular PCS category if they met that PCS criteria at least once post Baseline, regardless of their Baseline value.

All ECG parameters, overall assessment as determined by the central over-read, and findings will be provided in a data listing. In addition, separate listings will be generated to present the QTc interval data of subjects who met at least one QTc prolongation criterion and the ECG data that met the PCS criteria.

### 17.5.1. QTc Interval Prolongation Criteria

QTc interval prolongation will be identified in accordance with the following predefined criteria (same criteria apply to both QTcF and QTcB):

- > 450 msec at any post-Baseline time point (including unscheduled visits) not present at Baseline
- > 480 msec at any post-Baseline time point (including unscheduled visits) not present at Baseline
- > 500 msec at any post-Baseline time point (including unscheduled visits) not present at Baseline
- ≥ 30 msec increase from Baseline for at least one post-Baseline measurement (including unscheduled visits) and < 60 msec increase from Baseline for all post-Baseline measurements (including unscheduled visits)

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראט | Version Number: | 1.0 |



• ≥ 60 msec increase from Baseline for at least one post-Baseline measurement (including unscheduled visits)

#### 17.5.2. ECG POTENTIALLY CLINICALLY SIGNIFICANT CRITERIA

Potentially clinically significant ECG measurements will be identified in accordance with the following predefined PCS criteria:

Table 3: Predefined ECG PCS criteria.

| ECG Parameter | PCS Low | PCS High |
|------------------------|---------|----------|
| Heart Rate (beats/min) | | ≥ 100 |
| PR Interval (msec) | | ≥ 210 |
| QRS Interval (msec) | | ≥ 120 |

# 17.6. VITAL SIGNS

The following vital sign measurements will be reported for this study:

- Supine and Standing Systolic Blood Pressure (mmHg)
- Supine and Standing Diastolic Blood Pressure (mmHg)
- Supine and Standing Pulse Rate (bpm)
- Respiratory Rate (breaths/min)
- Temperature (°C)
- Height (cm)
- Weight (kg)





### Statistical Analysis Plan

- BMI (kg/m²)
- Waist Circumference (cm)

Height will be summarized as part of the Baseline characteristics only.

The following summaries will be provided:

- By-visit summary with 95% CI of the mean of observed values and change from Baseline values for vital sign measurements, including Week 9/Follow-up/Visit 11.
- Number and percentage of subjects with at least one PCS vital sign value (see Section 17.6.2) post Baseline. The period of evaluation includes both the treatment period and the follow-up period, including unscheduled visits. Subjects will be counted in a particular PCS category if they met that PCS criteria at least once post Baseline, regardless of their Baseline value.
- Number and percentage of subjects with orthostatic hypotension and/or orthostatic tachycardia (see Section 17.6.1). The data will be summarized for Baseline and the overall post-Baseline period (which covers both the treatment period and the follow-up period, including unscheduled visits), as well as by visit, including Week 9/Follow-up/Visit 11.
- By-visit summary of BMI category (see Section 7.5) and shift in BMI category from Baseline to each post-Baseline time point.
- By-visit summary with 95% CI of the mean of observed values and change from Baseline values for vital signs measurements by BMI category (see Section 7.5).

All vital signs data will be provided in a data listing. In addition, a separate listing will be generated to present the vital signs data that met the PCS criteria. All occurrences of orthostatic hypotension and orthostatic tachycardia will also be presented in a listing.

Boxplots will be created to present weight data by time point and treatment group. The boxplots will be repeated to present the change from Baseline values.

#### 17.6.1. VITAL SIGN SPECIFIC DERIVATIONS

BMI expressed in kg/m<sup>2</sup> = Weight (kg)/ height (m)<sup>2</sup>.

| Document: | PPD |
|-----------|-----|



The height collected at Visit 1 will be used to derive BMI where needed throughout the study.

- Orthostatic hypotension is defined as a decrease of ≥ 20 mmHg in systolic blood pressure or ≥ 10 mmHg in diastolic blood pressure after a subject has been standing for at least 2 to 4 minutes, compared to the systolic blood pressure and diastolic blood pressure measured in the supine position, respectively.
- Orthostatic tachycardia is defined as a heart rate increase of ≥ 20 bpm after a subject has been standing for at least 2 to 4 minutes compared to the heart rate measured in the supine position, and a heart rate of > 100 bpm after the subject has been standing for at least 2 to 4 minutes.

#### 17.6.2. VITAL SIGN POTENTIALLY CLINICALLY SIGNIFICANT CRITERIA

Potentially clinically significant vital sign measurements will be identified in accordance with the following predefined PCS criteria:

Table 5: Predefined vital sign PCS criteria.

| Vital Sign Parameter | PCS Low | PCS High |
|---|---|---|
| Systolic Blood Pressure (Supine, Standing) (mmHg) | Value ≤ 90 and ≥ 20 decrease from Baseline | Value ≥ 180 and ≥ 20 increase from Baseline |
| Diastolic Blood Pressure (Supine, Standing) (mmHg) | Value ≤ 50 and ≥ 15 decrease from Baseline | Value ≥ 105 and ≥ 15 increase from Baseline |
| Pulse Rate (Supine, Standing) (beats/min) | Value ≤ 50 and ≥ 15 decrease from Baseline | Value ≥ 120 and ≥ 15 increase from Baseline |
| Weight (kg) | ≥ 7% decrease from Baseline | ≥ 7% increase from Baseline |
| Temperature (°C) | NA | Value ≥ 38.3°C and ≥ 0.8°C increase from Baseline |

# 17.7. PHYSICAL EXAMINATION

As all physical and neurological findings will be recorded as medical history or AEs, no specific analysis of physical and neurological




examination will be performed.

### 17.8. OTHER SAFETY ASSESSMENTS

### 17.8.1. COLUMBIA SUICIDE SEVERITY RATING SCALE (C-SSRS)

The C-SSRS is a tool designed to systematically assess and track suicidal behavior and suicidal ideation for lifetime, one month prior to the screening visit for suicidal ideation and 6 months prior to the screening visit for suicidal behavior, and throughout the study. The strength of this suicide classification system is in its ability to comprehensively identify suicidal events while limiting the over-identification of suicidal behavior. The C-SSRS Baseline/Screening Version is used at the screening visit and the C-SSRS Since Last Visit Version is used from Visit 2 and onward. Subjects with Type 4 (active suicidal ideation with some intent to act, without specific plan) or Type 5 (active suicidal ideation with specific plan and intent) suicidal ideation during the study will be discontinued from the study and referred to a mental health professional.

C-SSRS includes two main sections: Suicidal Ideation and Suicidal Behavior.

The following outcomes are C-SSRS categories and have binary responses (yes/no). The categories are re-ordered from the scale to facilitate the definitions of the C-SSRS endpoints, and to provide clarity in the presentation of the results.

- Suicidal ideation is measured by 5 categories, representing 5 subtypes of suicidal ideation with increasing severity:
  - o Category 1: Wish to be Dead
  - o Category 2: Non-specific Active Suicidal Thoughts
  - o Category 3: Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act
  - o Category 4: Active Suicidal Ideation with Some Intent to Act, without Specific Plan
  - o Category 5: Active Suicidal Ideation with Specific Plan and Intent
- Suicidal behavior is measured by 5 categories, representing 5 subtypes of suicidal behavior:
  - o Category 6: Preparatory Acts or Behavior
  - o Category 7: Aborted Attempt
  - o Category 8: Interrupted Attempt
  - o Category 9: Actual Attempt (non-fatal)
  - o Category 10: Completed Suicide

| Document: | PPD |
|-----------|-----|



The 10 categories above are not mutually exclusive. Subjects will be counted in each category for which they have an event.

Self-injurious behavior without suicidal intent is a non-suicide-related C-SSRS outcome, and also has a binary response (yes/no).

For the purpose of C-SSRS analysis, "Baseline" and the overall "post-Baseline" periods are defined as follows.

| Time point | Study Visit | C-SSRS Version | Derivation Rule |
|---|---|---|---|
| Baseline | Visit 1 | Baseline/Screening – Past 1<br>Month for Suicidal Ideation /<br>Past 6 Months for Suicidal<br>Behavior | Most severe outcome |
| | Visit 2* | Since Last Visit | |
| Post-<br>Baseline | All post-Baseline visits up<br>to and including Visit 10<br>(the follow-up visit),<br>including unscheduled<br>visits | Since Last Visit | Most severe outcome |

<sup>\*</sup> Note: The Visit 2 C-SSRS assessment must be administered prior to the first dose of study medication in order to be used in the C-SSRS Baseline derivation.

The following C-SSRS composite endpoints will be derived for each time point of interest (i.e., Baseline, overall post-Baseline, and each scheduled visit including Week 9/Follow-up/Visit 11) as follows:

- Any suicidal ideation: A "yes" answer to any one of the 5 suicidal ideation questions on C-SSRS (Categories 1-5).
- Any suicidal behavior: A "yes" answer to any one of the 5 suicidal behavior questions on the C-SSRS (Categories 6-10).
- Any suicidality: A "yes" answer to any one of the 10 suicidal ideation and behavior questions on the C-SSRS (Categories 1-10).

For each subject, the suicidal ideation score at each time point of interest (i.e., Baseline, overall post-Baseline, the LOCF endpoint, and each scheduled visit including Week 9/Follow-up/Visit 11) is defined as the maximum suicidal ideation category (1-5) present for the time point of interest. If no ideation is present a score of 0 is assigned.

The number and percentage of subjects with any suicidality, any suicidal ideation and subtypes of ideation, any suicidal behavior and subtype of

| Document: | PPD |
|-----------|-----|



behavior, and any non-suicidal self-injurious behavior will be presented for:

- Baseline (as defined above)
- The overall post-Baseline period (as defined above)
- Each scheduled visit: Screening/Visit 1 (lifetime; past 1 month for ideation/past 6 months for behavior), Pre-switch Baseline/Visit 2, Week1/Visit 3, Week2/Visit 4, Week 3/Visit 5, Week 4/Visit 6, Week 5/Visit 7, Week 6/Visit 8, Week 7/Visit 9, Week 8/Visit 10 and Week 9/Follow-up/Visit 11.

Shift in suicidal ideation score from Baseline to the overall post-Baseline period, to each of the scheduled visits (Week1/Visit 3, Week2/Visit 4, Week 3/Visit 5, Week 4/Visit 6, Week 5/Visit 7, Week 6/Visit 8, Week 7/Visit 9, Week 8/Visit 10 and Week 9/Follow-up/Visit 11), and to the LOCF endpoint will be presented.

Intensity of ideation for the most severe ideation subtype is measured in terms of frequency, duration, controllability, deterrents, and reasons for ideation. Each is measured with responses ranging from 1 to 5 for frequency and duration, and from 0 to 5 for controllability, deterrents, and reasons for ideation. The ideation intensity total score is the sum of responses to the five items and can range from 2 to 25 for subjects with endorsed suicidal ideation. For subjects with endorsed suicidal ideation, if one or more of these five items are missing at an assessment, the total score will be set to missing. If a subject did not endorse any suicidal ideation, a score of 0 for the ideation intensity total score will be given.

Actual lethality associated with actual attempts is rated on a 6-point scale from 0 = 'No physical damage or very minor physical damage' to 5 = 'Death'. Potential lethality of actual attempts (if actual lethality = 0) is rated on a 3-point scale from 0 = 'Behavior not likely to result in injury' to 2 = 'Behavior likely to result in death despite available medical care'.

Responses to each C-SSRS question will be listed. The ideation intensity total score and the actual lethality and potential lethality of actual attempts will only be presented in data listings.




### 17.8.2. ABNORMAL INVOLUNTARY MOVEMENT SCALE (AIMS)

The AIMS is a clinician-rated assessment of abnormal movements consisting of unobtrusive observation of the subject at rest (with shoes removed) and several questions or instructions directed toward the subject. It contains seven items related to: facial, lip, jaw, and tongue movements (items 1 - 4), upper and lower extremity movements (items 5 - 6), and trunk movements (item 7). Three other items assess the subject at a global level (items 8 - 10), and two items assess dental status (items 11 - 12).

The (non-global) AIMS total score is the sum of items 1 through 7. (Items 8 through 12 are not used in AIMS total score calculation.) The possible range for AIMS total score is 0 to 28. Higher values of the AIMS total score indicate increased severity in abnormal movement. If one or more of the 7 items contributing to AIMS total score calculation are missing at a visit, the total score will be set to missing for that visit.

AIMS total score at each visit is classified as 'abnormal' if: either at least two items (out of items 1 - 7) have a response of 'Mild' or higher (i.e., item score  $\geq 2$ ); or at least one item (out of items 1 - 7) has a response of 'Moderate' or higher (i.e., item score  $\geq 3$ ). Otherwise, the non-missing AIMS total scores is classified as 'normal'.

Item 8 of AIMS represents the global severity score. Post-Baseline AIMS global severity scores will be classified as 'worsened', 'unchanged', or 'improved', relative to a subject's Baseline response to item 8. A higher score than that of the Baseline would be classified as 'worsened'. Conversely, a lower score would be classified as 'improved'. If the score is equal to that of Baseline, the score will be classified as 'unchanged'.

AIMS is assessed at these study visits: Visit 2 and Visit 10.

The observed AIMS total score and the change from Baseline values will also be summarized descriptively by treatment group and visit. In addition, the observed AIMS total score and the change from Baseline values will be summarized descriptively by the subgroups of concomitant medication use for treatment of movement disorders.

Shift from Baseline in AIMS total score category (Normal/Abnormal) to each post-Baseline scheduled visit (Week 8/Visit 10) and to the overall post-Baseline period (including both the treatment period and the follow-up period) will be summarized descriptively by treatment group.

The observed AIMS global severity score and the change from Baseline values will be summarized descriptively by treatment group and visit. In addition, the frequency distribution of the AIMS global severity item will be summarized descriptively by treatment group and visit. Post-Baseline changes in AIMS global severity score (Worsened/Unchanged/Improved) will also be summarized descriptively by treatment group and visit.

### 17.8.3. BARNES AKATHISIA RATING SCALE (BARS)

The BARS is a rating scale geared toward assessment of neuroleptic-induced akathisia, though it can be used to measure akathisia associated with other drugs as well. The BARS consists of four items, including one item assessing objective restlessness (item 1), two items targeting subjective

| Document: | PPD |
|-----------|-----|

PROTOCOL SEP361-308 

restlessness (awareness and related distress; items 2 - 3), and one global clinical assessment of akathisia item (item 4). The objective and subjective items are anchored and utilize a 4-point scale. The global assessment item has a 6-point scale (from absence of akathisia through severe akathisia).

The BARS total score is the sum of items 1 through 3 and ranges from 0 to 9. Higher values of the BARS total score indicate higher severity of akathisia. If one or more of items 1 to 3 are missing at a visit, the BARS total score will be set to missing for that visit.

The post-Baseline BARS Global Clinical Assessment of Akathisia responses will be classified as 'worsened', 'unchanged', or 'improved', relative to a subject's Baseline response to this item. A higher score than that of the Baseline would be classified as 'worsened'. Conversely, a lower score would be classified as 'improved'. If the score is equal to that of Baseline, the score will be classified as 'unchanged'.

BARS is assessed at these study visits: Visit 2 and Visit 10.

The observed BARS total score and the change from Baseline values will also be summarized descriptively by treatment group and visit. In addition, the observed BARS total score and the change from Baseline values will be summarized descriptively by the subgroups of concomitant medication use for treatment of movement disorders.

Post-Baseline changes in BARS global clinical assessment score (Worsened/Unchanged/Improved) will be summarized descriptively by treatment group and visit.

Lastly, the observed BARS item scores and the change from Baseline values will be summarized descriptively by treatment group and visit. In addition, the frequency distribution of each BARS item will be summarized descriptively by treatment group and visit.

# 17.8.4. SIMPSON-ANGUS SCALE (SAS)

The SAS is a clinician-rated assessment of neuroleptic-induced Parkinsonism consisting of 10 items. Items are anchor-based, rated on a 5-point scale (ranging between 0 and 4), and address rigidity, gait (bradykinesia), tremor, akathisia, shoulder shaking, glabellar tap, and salivation.

SAS mean score is defined as the average of all 10 items and ranges between 0 and 4. Lower values of the SAS mean score indicate milder symptoms. If one or more of the SAS items are missing at a visit, the SAS mean score will be set to missing for that visit.

The SAS mean score at each visit will be classified as 'abnormal' if it exceeds 0.3 (Rush, et al., 2000). Otherwise, the non-missing SAS mean score will be classified as 'normal'.

SAS is assessed at these study visits: Visit 2 and Visit 10.

The observed SAS mean score and the change from Baseline values will also be summarized descriptively by treatment group and visit. In addition, the observed SAS mean score and the change from Baseline values will be summarized descriptively by the subgroups of concomitant medication use for treatment of movement disorders.

| Document: | PPD |
|-----------|-----|



Shift from Baseline in SAS mean score category (Normal/Abnormal) to each post-Baseline scheduled visit (Week 8/Visit 10) and to the overall post-Baseline period (including both the treatment period and the follow-up period) will be summarized descriptively by treatment group.

#### 17.8.5. PITTSBURGH SLEEP QUALITY INDEX

The Pittsburgh Sleep Quality Index (PSQI) consists of 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). It is used to measure the quality and patterns of sleep in adults. Only self-rated questions are included in the scoring. It differentiates "poor" from "good" sleep quality by measuring seven "component" scores, each of which has a range of 0-3 points: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction due to sleepiness over the last month.

The seven component scores are then summed to yield one global PSQI score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989).

The PSQI scoring algorithm as downloaded from the University of Pittsburgh Sleep and Chronobiology Center is inserted in APPENDIX 8. The seven component scores and the PSQI global score will be derived according to this algorithm. If one or more of the component scores are missing at a visit, the PSQI global score will be set to missing for that visit.

PSQI is assessed at these study visits: Visit 2, Visit 6 and Visit 10.

The observed PSQI global score and the change from Baseline values will be summarized descriptively by treatment group and visit.

# 17.9. SUBGROUP ANALYSIS OF SAFETY VARIABLE(S)

The subgroup analyses for AE data, vital signs data, and AIMS/BARS/SAS scales are described in their respective sections.

# 18. PHARMACOKINETIC ANALYSIS

Plasma concentrations of SEP-363856 and SEP-363854 (metabolite of SEP-363856) of all enrolled subjects will be presented in a data listing.




## 19. DATA NOT SUMMARIZED OR PRESENTED

The variables and/or domains not summarized or presented are:

- Subject initials
- Any data collected on screen failures other than disposition, basic demographics, and pre-treatment events.
- Any data collected during previously failed screening(s) for randomized subjects who were screened more than once except Adverse Events.

These domains and/or variables will not be summarized or presented but will be available in the clinical study database and SDTM datasets.

## 20. REFERENCES

- Buysse, D., Reynolds, C., Monk, T., Berman, S., & Kupfer, D. (1989). The Pittsburgh Sleep Quality Index (PSQI): A new instrument for psychiatric research and practice. *Psychiatry Research*, 28(2), 193-213.
- Hopkins, S., Ogirala, A., Loebel, A., & Koblan, K. (2018;44(3):593-602). Transformed PANSS factors intended to reduce pseudospecificity among symptom domains and enhance understanding of symptom change in antipsychotic-treated patients with schizophrenia. . *Schizophrenia Bull* .
- Hopkins, S., Ogirala, A., Loebel, A., & Koblan, K. (2020). Characterization of specific and distinct patient types in clinical trials of acute schizophrenia using an uncorrelated PANSS score matrix transform (UPSM). *Psychiatry Research*.
- Keefe, R., Philip, H., Terry, G., James, G., Trina, W., Courntey, K., & Kirsten, H. (2008). Norms and standardization of the Brief Assessment of Cognition in Schizophrenia (BACS). *Schizophrenia Reaseach*, 108-115.
- Leucht S, Crippa A, Siafis S, Patel MX, Orsini N, Davis JM. Dose-response meta-analysis of antipsychotic drugs for acute schizophrenia. American Journal of Psychiatry. 2020 Apr 1;177(4):342-53.
- Marder, S., Davis, J., & Chouinard, G. (1997;58:538–46). The effects of risperidone on the five dimensions of schizophrenia. J Clin Psychiatry.
- Rush, A., Pincus, H., First, M., Blacker, D., Endicott, J., Keith, S., . . . Zarin, D. (2000). Handbook of Psychiatric Measures. American Psychiatric Association.

| Document: | PPD |
|-----------|-----|




## APPENDIX 1. Programming Conventions for Outputs

## **IQVIA OUTPUT CONVENTIONS**

The following output conventions are to be followed:

- General presentation:
  - o The first row in the body of the table or listing should be blank
  - o Rounding should be done with the SAS function ROUND.
  - o Numbers in tables should be rounded, not truncated.
  - o The first letter of a text entry should be capitalized.
- Univariate Statistics: If the raw data has N decimal places, then the summary statistics should have the following decimal places:
  - o Minimum and maximum: N
  - o Mean, median, Q1, and Q3: N + 1
  - o SD: N + 2
  - o For lab data only, in the rare case where raw data has more than 3 decimal places, summary statistics will be presented for the scenario of N = 3. All decimals will be presented in Listings.
  - o For CGI-S score, 2 decimal places will be presented for mean, median, Q1, Q3, LS mean, LS mean difference, and 95% CI; 3 decimal places will be presented for SD and SE; 0 decimal places will be presented for min and max. 0 decimal places will be presented in listings.
  - o For UPSM scores, 3 decimal places will be presented for mean, median, Q1, Q3, LS mean, LS mean difference, and 95% CI; 4 decimal places will be presented for SD and SE; 2 decimal places will be presented for min and max. Up to 2 decimal places will be presented in Listings. No rounding will be applied in the ADaM datasets.
- Frequencies and percentages (n and %):
  - o Percentages will be reported to one decimal place, except cases where percent <100.0% but >99.9% will be presented as '>99.9%' (e.g., 99.99% is presented as >99.9%); and cases where percent < 0.1% will be presented as '<0.1%' (e.g., 0.08% is presented as <0.1%). Rounding will be applied after the <0.1% and >99.9% rule.
  - o Where counts are zero, no percentage should appear in the output.
- Confidence Intervals:

| Document: | PPD |
|-----------|-----|



- Confidence intervals and estimates are presented to one place more than the raw data, and standard errors to two places more than the raw data.
- o Boundary values of confidence intervals should be separated by a comma.
- P-values should be reported to three decimal places, except values <1.000 but >0.999 will be presented as '>0.999' (e.g., 0.9998 is presented as >0.999); and values <0.001 will be presented as '<0.001' (e.g., 0.0009 is presented as <0.001). Rounding will be applied after the <0.001 and >0.999 rule.
- Ratios should be reported to one more decimal place than the raw data.
- Missing values:
  - o A "0" should be used to indicate a zero frequency.
  - o A "-" will be used to indicate missing data in an end-of-text table or subject listing.

0

## **DATES & TIMES**

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss .

#### **SPELLING FORMAT**

English US.

## **PRESENTATION OF TREATMENT GROUPS**

For outputs, treatment groups will be represented as follows and in that order:

| Treatment Group | For Tables (Column Order) | For Listings and Graphs (Order) |
|---|---|---|
| SEP-363856 50 to 100 mg/day | SEP-363856 50 to 100 mg/day | SEP-363856 50 to 100 mg/day |

| Document: | PPD |
|-----------|-----|

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



## **LISTINGS**

All listings will be ordered by the following (unless otherwise indicated in the template):

- Enrolled subjects who did not receive any study medication will be presented at the end and labelled "Not Treated".
- Subject ID.
- Visit (where applicable)
- Original date/time (where applicable).




## APPENDIX 2. PARTIAL DATE CONVENTIONS

The actual dates as collected on the CRF will be presented in the listings. Imputed dates will not be presented in the listings unless otherwise specified.

#### **ALGORITHM FOR ADVERSE EVENTS**

As a general rule, if the start date of an AE is available and the start time of the AE is not available, the AE will be considered to have started after the study drug dose administered on the day of the AE start date.

In case of partial or missing AE start and/or end dates, impute partial or missing event start and/or end dates (if not ongoing) using the algorithm below. If an AE has some missing components in both the start and end dates, first impute the end date.

#### AE end date imputation

- If year and month (YYYY-MM) of AE end date are known, then impute the missing day to be the earlier of (last day of the month; date of last contact).
- If only year (YYYY) of AE end date is known, then impute the missing month and day to be the earlier of (31st December; date of last contact).
- If AE end date is completely missing and AE is not ongoing, then impute AE end date to be date of last contact.

## AE start date imputation

- If year and month (YYYY-MM) of AE start date are known and YYYY-MM = year and month of 361-30 study med start date, then impute AE start date to be the earlier of (361-308 study med start date; full or imputed AE end date [if non-missing]).
- If year and month (YYYY-MM) of AE start date are known and YYYY-MM ≠ year and month of 361-308 study med start date, then impute AE start date to be YYYY-MM-01.
- If only year (YYYY) of AE start date is known and YYYY = year of 361-308 study med start date, then impute AE start date to be the earlier of (361-308 study med start date; full or imputed AE end date [if non-missing]).
- If only year (YYYY) of AE start date is known and YYYY ≠ year of 361-308 study med start date, then impute AE start date to be YYYY-01-01.

| Document: | PPD |
|-----------|-----|



## PROTOCOL SEP361-308 

• If AE start date is completely missing, then impute AE start date to be the earlier of (361-308 study med start date; full or imputed AE end date [if non-missing]).

Using the full or imputed event dates, assign events into pre-treatment events vs. AE as described below.

If both event start date/time and 361-308 study med start date/time are available:

- If event start date/time < 361-308 study med start date/time, then pre-treatment event.
- If event start date/time ≥ 361-308 study med start date/time, then AE.

If (event start date is available and time is not available) and/or (361-308 study med start date is available and time is not available):

- If event start date < 361-308 study med start date, then pre-treatment event.
- If event start date ≥ 361-308 study med start date, then AE.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראח | Version Number: | 1.0 |



## **ALGORITHM FOR PRIOR / CONCOMITANT / POST-TREATMENT MEDICATIONS**

In case of partial or missing medication start and/or stop dates, impute the partial or missing dates using the algorithm below.

If a medication has some missing components in both the start and stop dates, first impute the stop date.

#### Impute stop date as latest possible date

- If only day unknown, impute to the earlier of (last day of the month; date of 361-308 last contact).
- If month and day unknown, impute to the earlier of (31st December; date of 361-308 last contact).
- If stop date is completely unknown and medication is not ongoing, impute to date of 361-308 last contact.

#### Impute start date as earliest possible date

CRF questions: 'Started prior to first dose?' = Yes; 'Started after last dose of study medication?' = No.

- If only day unknown, impute to the later of (first day of the month; date of birth [if full date is available]).
- If month and day unknown, impute to the later of (1st January; date of birth [if full date is available]).
- If start date is completely unknown, impute to the earlier of (date of informed consent\*; full or imputed medication stop date [if not missing]).

CRF questions: 'Started prior to first dose?' = No; 'Started after last dose of study medication?' = Yes.

- If only day unknown, impute to the later of (first day of the month; 361-308 study med end date + 1).
- If month and day unknown, impute to the later of (1st January; 361-308 study med end date + 1).
- If start date is completely unknown, impute to 361-308 study med end date + 1.

CRF questions: 'Started prior to first dose?' = No; 'Started after last dose of study medication?' = No.

- If only day unknown, impute to the later of (first day of the month; 361-308 study med start date).
- If month and day unknown, impute to the later of (1st January; 361-308 study med start date).
- If start date is completely unknown, impute to 361-308 study med start date.

| Document: | PPD |
|-----------|-----|



#### Then assign a medication into prior, concomitant, or post-treatment

The concept of "date" below should also include time information whenever time is available for both comparators.

- If medication stop date < 361-308 study med start date, assign as prior.
- If (medication stop date ≥ 361-308 study med start date or medication is ongoing) and medication start date ≤ 361-308 study med end date, assign
  as concomitant.
- If medication start date > 361-308 study med end date, assign as post-treatment.

#### Overriding rule

For the case where the medication start date is known and is equal to 361-308 study med end date and the medication start time is unknown, or the case where the imputed medication start date is equal to 361-308 study med end date:

- If CRF question 'Started after last dose of study medication?' = No, then assign as concomitant.
- If CRF question 'Started after last dose of study medication?' = Yes, then assign as post-treatment.




#### PARTIAL DATE IMPUTATION RULES FOR INITIAL ONSET OF SCHIZOPHRENIA

For subjects with partial onset date of schizophrenia, impute the onset date using the following rules:

- If only day unknown, impute as the earlier of: 15<sup>th</sup> of the month, or date of ICF\*.
- If both month and day unknown, impute as the earlier of: June 30<sup>th</sup> of the year, or date of ICF\*.

#### PARTIAL DATE IMPUTATION RULES FOR CURRENT ONSET OF ACUTE EXACERBATION

For subjects with partial onset date of acute exacerbation, impute the onset date using the following rules:

- If only day unknown and the known year and month is earlier than the year and month of ICF\*, impute as the later of: 15<sup>th</sup> of the month, or date of initial onset of schizophrenia (actual or imputed).
- If only day unknown and the known year and month is the same as the year and month of ICF\*, impute as the later of: earlier of (date of ICF\*, 15<sup>th</sup> of the month), or date of initial onset of schizophrenia (actual or imputed).
- If both month and day unknown and the known year is earlier than the year of ICF\*, impute as the later of: June 30<sup>th</sup> of the year, or date of initial onset of schizophrenia (actual or imputed).
- If both month and day unknown and the known year is the same as the year of ICF\*, impute as the later of: earlier of (date of ICF\*, June 30<sup>th</sup> of the year), or date of initial onset of schizophrenia (actual or imputed).

#### PARTIAL DATE IMPUTATION RULES FOR FIRST HOSPITALIZATION

For subjects with partial date of first hospitalization for treatment of schizophrenia, impute the date using the following rules:

• If only day unknown, impute as the earlier of: 15<sup>th</sup> of the month, or date of ICF\*.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראט | Version Number: | 1.0 |

<sup>\*</sup>For adolescent subjects, the later of the ICF date and IAF date should be used.

<sup>\*</sup>For adolescent subjects, the later of the ICF date and IAF date should be used.



If both month and day unknown, impute as the earlier of: June 30<sup>th</sup> of the year, or date of ICF\*.

\*For adolescent subjects, the later of the ICF date and IAF date should be used.

For subjects whose date of first hospitalization for treatment of schizophrenia is completely missing AND the number of prior hospitalizations for treatment of schizophrenia is 0, impute the date of first hospitalization to be the "Date of admission for this study hospitalization" collected on the "Psychiatric Hospitalization (HOSP)" CRF form.

#### PARTIAL DATE IMPUTATION RULES FOR FIRST ANTI-PSYCHOTIC DRUG THERAPY

For subjects with partial start date for the first anti-psychotic drug therapy of at least 2 weeks duration intended for treatment of schizophrenia, impute the start date using the following rules:

- If only day unknown, impute as the earlier of: 15<sup>th</sup> of the month, or date of ICF\*.
- If both month and day unknown, impute as the earlier of: June 30<sup>th</sup> of the year, or date of ICF\*.

#### PARTIAL DATE IMPUTATION RULES FOR ONSET OF INITIAL BEHAVIORAL DISTURBANCE

For adolescent subjects with partial onset date of initial behavioral disturbance, impute the onset date using the following rules:

- If only day unknown, impute as the earlier of: 15<sup>th</sup> of the month, or the later of (date of ICF and date of IAF).
- If both month and day unknown, impute as the earlier of: June 30<sup>th</sup> of the year, or the later of (date of ICF and date of IAF).




## **RULES FOR ASSIGNING DOSEON/DOSEA**

- In general, DOSEON/DOSEA should be the dose level immediately before the start of an AE or an assessment. In case the AE or the assessment start date/time coincides with the first dosing start date/time of the study, the DOSEON/DOSEA should be assigned to the dose level associated with that first dosing start date/time. In case the AE or the assessment start date/time coincides with a dosing start date/time other than the first dosing start date/time, the DOSEON/DOSEA should be assigned to the dose level associated with the previous dosing start date/time.
- In case of missing AE start time, missing assessment (start) time, and/or missing dosing start time, DOSEON/DOSEA should be assigned using the algorithm in the table below.

| Scenario | Data | Rules |
|---|---|---|
| Dosing start date and start time both available | Adverse Events | If AE start date is available and AE start time is missing, dose on the same day as AE start should be assigned as DOSEON. |
| | Scales/Questionnaires,<br>Vitals, Labs, ECG | If assessment start date is available and assessment start time is missing, dose on the previous day of the assessment should be assigned as DOSEA. |
| Dosing start date available but | Adverse Events | Regardless of whether AE start time is available, dose on the same day as AE start should be assigned as DOSEON. |
| start<br>time missing | Scales/Questionnaires,<br>Vitals, Labs, ECG | Regardless of whether assessment start time is available, dose on the previous day of the assessment should be assigned as DOSEA. |

In case of partial or missing AE start date, the imputed AE start date will be used for the purpose of assigning DOSEON.




## APPENDIX 3. Uncorrelated PANSS Score Matrix (UPSM)

| PANSS | UPSM-POS | UPSM-DIS | UPSM-NAA | UPSM-NDE | UPSM-HOS | UPSM-ANX | UPSM-DEP |
|---|---|---|---|---|---|---|---|
| PANSS01 | 0.5792730597 | -0.1547126840 | -0.0828932650 | 0.0071927220 | -0.0593031510 | -0.0735449620 | 0.0020484408 |
| PANSS02 | 0.0292444390 | 0.1975824582 | -0.0260173260 | -0.0234753800 | -0.0368756010 | -0.0012396240 | -0.0361645050 |
| PANSS03 | 0.2065788330 | -0.0179419820 | -0.0250663450 | -0.0133031880 | -0.0300507070 | 0.0001506005 | 0.0293001724 |
| PANSS04 | -0.0336790630 | 0.0115284348 | 0.0011652392 | -0.0723891460 | 0.1379358628 | 0.1108194656 | -0.1045224460 |
| PANSS05 | -0.0341508580 | -0.0301875430 | -0.0041019560 | -0.0233459100 | -0.0069204000 | -0.0313277060 | 0.0308288417 |
| PANSS06 | 0.3537254634 | -0.0626270750 | 0.0477329954 | 0.0012126712 | 0.0192067437 | -0.0161398140 | 0.0063264235 |
| PANSS07 | -0.0383468990 | -0.1767919370 | -0.0299340700 | 0.0314652864 | 0.5025411101 | -0.0997121200 | 0.0573604084 |
| PANSS08 | -0.0054230270 | -0.0291400280 | 0.0568702938 | 0.2474176209 | -0.0388464000 | 0.0188235393 | -0.0091524870 |
| PANSS09 | -0.0315765690 | -0.0243925850 | 0.3317907576 | -0.0228204580 | -0.0507096280 | -0.0145653830 | 0.0112689069 |
| PANSS10 | -0.0742072890 | -0.0401313020 | -0.0097485120 | 0.0161513666 | 0.0245536353 | -0.0176161520 | -0.0172218040 |
| PANSS11 | -0.0943532590 | -0.0856364190 | 0.4611503804 | -0.0286825100 | -0.0189062390 | -0.0185825180 | -0.0130433890 |
| PANSS12 | 0.0043338689 | 0.1062496353 | 0.0255910591 | -0.0301470410 | -0.0133497570 | 0.0096065791 | -0.0686802390 |
| PANSS13 | 0.0041274699 | 0.0051521898 | 0.0009558861 | 0.2576813501 | -0.0085004640 | 0.0194235006 | -0.1037459520 |
| PANSS14 | -0.0111267300 | 0.1462268689 | -0.0276416260 | 0.0023017188 | -0.0055291270 | -0.0118427800 | 0.0040128786 |
| PANSS15 | -0.0356272010 | 0.0552508287 | -0.0382627720 | 0.0110152489 | -0.0309176290 | 0.0444944076 | 0.1059845189 |
| PANSS16 | -0.0331052830 | -0.0821894470 | -0.0327376640 | -0.0533178140 | -0.0386473380 | 0.4576579818 | 0.1197800301 |
| PANSS17 | -0.0368854600 | -0.0004363100 | -0.0020681500 | -0.0407976460 | -0.0272172130 | -0.0253163640 | 0.2459654614 |
| PANSS18 | -0.0931367690 | -0.0332617600 | -0.0132943930 | 0.0231904701 | -0.0287529750 | 0.5123850161 | -0.0312522560 |
| PANSS19 | -0.0455199430 | 0.0494113554 | -0.0324174560 | 0.1026255664 | -0.0136676190 | 0.0293507269 | -0.0441735260 |
| PANSS20 | -0.0344751890 | -0.0688197670 | -0.0412738350 | 0.0381793764 | 0.0042219619 | -0.0635101090 | 0.4514426846 |
| PANSS21 | -0.0348890020 | -0.0366137810 | -0.0779782830 | 0.4409895205 | -0.0073240410 | -0.0192655290 | 0.0464131877 |
| PANSS22 | -0.0803690920 | 0.0334025939 | -0.0088488890 | -0.0200483170 | 0.2858700784 | -0.0567167860 | -0.0531076130 |
| PANSS23 | 0.1428966744 | 0.0939213700 | -0.0326143600 | -0.0367524640 | -0.0675856980 | -0.0209072840 | -0.0177890070 |
| PANSS24 | -0.0383047770 | -0.0324584080 | -0.0255393890 | -0.0180115340 | -0.0266180700 | -0.0210068530 | -0.0176029110 |
| PANSS25 | -0.1036311520 | 0.2814367260 | -0.0478918640 | 0.0029986238 | 0.0037656449 | -0.0226520240 | 0.0401351054 |
| PANSS26 | 0.0142987589 | 0.1548635741 | -0.0306089330 | -0.0331581690 | 0.0262295986 | -0.0576293550 | -0.0626180490 |
| PANSS27 | -0.0573513270 | 0.1867914227 | -0.0143489160 | 0.0581534153 | -0.0145494330 | -0.0371788310 | 0.0455412078 |
| PANSS28 | -0.0748387810 | 0.0166272025 | -0.0267498020 | -0.0031632780 | 0.2546669938 | -0.0201249190 | -0.0076420280 |
| PANSS29 | -0.0520812460 | 0.2912295497 | 0.0029775475 | -0.0324350460 | -0.0442337350 | -0.0047991290 | 0.0567191230 |

Document: PPD

Author: Version Number: 1.0

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



PROTOCOL SEP361-308 

| Document: | PPD |
|-----------|-----|



## APPENDIX 4. Internationally Agreed Order for System Organ Class

#### Internationally Agreed Order

Infections and infestations

Neoplasms benign, malignant and unspecified (incl cysts and polyps)

Blood and lymphatic system disorders

Immune system disorders

Endocrine disorders

Metabolism and nutrition disorders

Psychiatric disorders

Nervous system disorders

Eye disorders

Ear and labyrinth disorders

Cardiac disorders

Vascular disorders

Respiratory, thoracic and mediastinal disorders

Gastrointestinal disorders

Hepatobiliary disorders

Skin and subcutaneous tissue disorders

Musculoskeletal and connective tissue disorders

Renal and urinary disorders

Pregnancy, puerperium and perinatal conditions

Reproductive system and breast disorders

Congenital, familial and genetic disorders

General disorders and administration site conditions

Investigations

Injury, poisoning and procedural complications

Surgical and medical procedures

Social circumstances

Product issues

Author: PPD

Version Number: 1.0

# APPENDIX 5. Adverse Events of Potential Drug Abuse and Dependence

To ensure comprehensive and consistent selection of terminology used for analyses of drug abuse and dependence in ongoing / planned studies of SEP-363856, MedDRA preferred terms were identified from the following sources:

FDA Guidance for Industry: Assessment of Abuse Potential of Drugs (CDER, 2017; noted that the Guidance reflects MedDRA version 20.0 terminology)

MedDRA version 22.0 SMQ: Drug abuse and dependence [20000101], Broad

FDA FMQ: Study Agent Abuse Potential, Broad (released at FDA public workshop "Advancing Premarket Safety Analytics", held September 14, 2022)

## **Description:**

Preferred terms were tabulated using MedDRA version 22.0 from the sources listed above. All preferred terms (PTs) within the FDA Abuse Potential Guidance were included. All PTs listed in the MedDRA version 22.0 SMQ for Drug abuse and dependence [20000101] were included. For the FDA Study Agent Abuse Potential FMQ: No associated MedDRA PT was found for the term "Hypnogogic hallucination", and this is therefore not included. Sunovion evaluates 'Drug withdrawal' as a unique medical concept using MedDRA version 22.0 SMQ for Drug withdrawal [20000102] (Broad); any overlapping PTs from the Drug withdrawal SMQ which are listed in the FDA Study Agent Abuse Potential FMQ are not included. All other PTs listed in the FDA FMQ were included.

The table below depicts the preferred terms by source.

Table 7: Drug Abuse and Dependence Preferred Terms Using MedDRA v 22.0

| FDA Guidance 2017 | FDA Guidance 2017 | | | FDA FMQ | FDA FMQ |
|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code |
| - | - | Accidental overdose | 10000381 | Accidental overdose | 10000381 |
| - | - | - | - | Acute psychosis | 10001022 |
| Aggression | 10001488 | - | - | = | - |
| Behavioural addiction | 10081939 | - | - | - | - |
| Confusional state | 10010305 | - | - | - | - |
| - | - | - | - | Delusion of grandeur | 10012241 |
| - | - | - | - | Delusional perception | 10012258 |
| Dependence | 10012335 | Dependence | 10012335 | Dependence | 10012335 |
| - | - | - | - | Depersonalisation | 10012357 |
| - | - | - | - | Derealisation disorder | 10077810 |
| - | - | - | - | Detoxification | 10061814 |
| - | - | - | - | Disinhibition | 10013142 |
| Disorientation | 10013395 | - | - | - | - |
| - | - | Disturbance in social | 10061108 | - | - |
| | | behaviour | | | |
| Dizziness | 10013573 | - | - | - | - |
| Dopamine | 10067468 | Dopamine | 10067468 | - | - |
| dysregulation | | dysregulation | | | |
| syndrome | | syndrome | | | |




| FDA Guidance 2017 | | SMQ 20000101 | | FDA FMQ | |
|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code |
| - | - | Drug abuse | 10013654 | Drug abuse | 10013654 |
| - | - | Drug abuser | 10061111 | Drug abuser | 10061111 |
| - | - | Drug dependence | 10013663 | Drug dependence | 10013663 |
| Drug dependence, | 10013675 | Drug dependence, | 10013675 | Drug dependence, | 10013675 |
| antepartum | | antepartum | | antepartum | |
| Drug dependence, | 10013676 | Drug dependence, | 10013676 | Drug dependence, | 10013676 |
| postpartum | | postpartum | | postpartum | |
| - | - | Drug detoxification | 10052237 | Drug detoxification | 10052237 |
| - | - | Drug diversion | 10066053 | Drug diversion | 10066053 |
| - | - | Drug level above | 10061132 | - | - |
| | | therapeutic | | | |
| - | - | Drug level increased | 10013722 | - | - |
| - | - | Drug screen | 10050837 | - | - |
| - | _ | Drug screen positive | 10049177 | _ | - |
| Drug tolerance | 10052804 | Drug tolerance | 10052804 | - | _ |
| Drug tolerance | 10052805 | Drug tolerance | 10052805 | _ | _ |
| decreased | | decreased | 10032003 | | |
| Drug tolerance | 10052806 | Drug tolerance | 10052806 | _ | _ |
| increased | 10032000 | increased | 10032000 | | |
| Drug use disorder | 10079381 | Drug use disorder | 10079381 | Drug use disorder | 10079381 |
| - | - | Drug use disorder, | 10073301 | Drug use disorder, | 10073301 |
| | | antepartum | 10079382 | antepartum | 10079382 |
| - | _ | Drug use disorder, | 10073302 | Drug use disorder, | 10075302 |
| | | postpartum | 10079383 | postpartum | 10079383 |
| | _ | - postpartum | - | Energy increased | 10079383 |
| Euphoric mood | 10015535 | - | - | Euphoric mood | 10015535 |
| Feeling abnormal | 10015333 | - | - | Lupitorie mood | 10013333 |
| Feeling drunk | | - | - | Feeling drunk | 10016330 |
| reeling drunk | 10016330 | | | | 10016330 |
| | 40046353 | - | - | Feeling jittery | 10016338 |
| Feeling of relaxation | 10016352 | - | - | Feeling of relaxation | 10016352 |
| | - | - | - | Flight of ideas | 10016777 |
| Hallucination | 10019063 | - | - | Hallucination | 10019063 |
| Hallucination, | 10019070 | - | - | Hallucination, | 10019070 |
| auditory | 10010071 | | | auditory | 40046074 |
| Hallucination, | 10019071 | - | - | Hallucination, | 10019071 |
| gustatory | 400400=0 | | | gustatory | 400400=0 |
| Hallucination, | 10019072 | - | - | Hallucination, | 10019072 |
| olfactory | 10000 | | | olfactory | 10000 |
| Hallucination, | 10062824 | - | - | Hallucination, | 10062824 |
| synaesthetic | 100105- | | | synaesthetic | 10010 |
| Hallucination, tactile | 10019074 | - | - | Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 | - | - | Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 | - | - | Hallucinations, mixed | 10019079 |
| Inappropriate affect | 10021588 | - | - | Hallucination, | 10019071 |
| | | | | gustatory | |
| - | - | - | - | Hypersomnia | 10020765 |
| - | - | - | - | Hypervigilance | 10048533 |
| - | - | - | - | Hypnagogic | 10020927 |
| | | | | hallucination | 1 |

Document: PPD

Author: Version Number: 1.0



| FDA Guidance 2017 | | SMQ 20000101 | | FDA FMQ | |
|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code |
| - | - | - | - | Hypnogogic hallucination | No such code |
| - | _ | _ | _ | Hypnopompic | 10020928 |
| - | - | - | - | hallucination | 10020928 |
| - | _ | - | _ | Inappropriate affect | 10021588 |
| - | - | - | - | Infant sedation | 10082187 |
| - | - | - | - | Intentional misuse of | 10081675 |
| | | | | drug delivery system | |
| - | - | Intentional overdose | 10022523 | Intentional overdose | 10022523 |
| - | - | Intentional product | 10074903 | Intentional product | 10074903 |
| | | misuse | | misuse | |
| - | - | Intentional product | 10076308 | - | - |
| | | use issue | | | |
| - | - | - | - | Mania | 10026749 |
| - | - | Maternal use of illicit drugs | 10026938 | - | - |
| - | - | Medication overuse headache | 10072720 | - | - |
| - | - | - | - | Mixed delusion | 10076429 |
| Mood altered | 10027940 | - | - | Mood altered | 10027940 |
| Mood swings | 10027951 | - | - | - | - |
| - | - | Narcotic bowel | 10072286 | - | - |
| | | syndrome | | | |
| = | - | Needle track marks | 10028896 | - | - |
| - | - | Neonatal | 10061862 | - | - |
| | | complications of | | | |
| | | substance abuse | | | |
| - | - | - | - | Neonatal | 10050395 |
| | | | | oversedation | |
| - | - | Overdose | 10033295 | - | - |
| - | - | - | - | Paranoia | 10033864 |
| - | - | - | - | Post-injection | 10072851 |
| | | | | delirium sedation | |
| | | Dunaminti I | 40076600 | syndrome | |
| - | - | Prescription drug used without a | 10076639 | - | - |
| | | prescription | | | |
| | - | Prescription form | 10067669 | Prescription form | 10067669 |
| - | - | tampering | 1000/009 | tampering | 10007009 |
| - | _ | - | - | Psychomotor | 10037211 |
| | | | | hyperactivity | |
| Psychotic disorder | 10061920 | - | - | - | - |
| | | Reversal of opiate activity | 10039004 | - | - |
| - | - | - | - | Sedation | 10039897 |
| - | - | - | - | Sedation | 10079741 |
| | | | | complication | |
| Somnolence | 10041349 | - | - | Somnolence | 10041349 |
| - | - | - | - | Somnolence neonatal | 10041350 |

Document: PPD

Author: Version Number: 1.0



| FDA Guidance 2017 | | SMQ 20000101 | SMQ 20000101 | | |
|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code |
| - | - | - | - | Stupor | 10042264 |
| - | - | Substance abuse | 10066169 | Substance abuse | 10066169 |
| - | - | Substance abuser | 10067688 | Substance abuser | 10067688 |
| - | - | Substance dependence | 10076595 | Substance dependence | 10076595 |
| - | - | Substance use | 10070964 | - | - |
| Substance use disorder | 10079384 | Substance use disorder | 10079384 | Substance use disorder | 10079384 |
| - | - | Substance-induced mood disorder | 10072387 | Substance-induced mood disorder | 10072387 |
| - | - | Substance-induced psychotic disorder | 10072388 | Substance-induced psychotic disorder | 10072388 |
| - | - | - | - | Suspected product tampering | 10079404 |
| Thinking abnormal | 10043431 | - | - | - | - |
| - | - | Toxicity to various agents | 10070863 | - | - |
| - | - | - | - | Transient psychosis | 10056326 |
| - | - | - | - | Withdrawal<br>hypertension | 10048007 |

Document: PPD

Author: PPD




## APPENDIX 6. EXTRAPYRAMIDAL ADVERSE EVENTS

To ensure comprehensive and consistent selection of terminology used for analyses of extrapyramidal signs and symptoms in ongoing / planned studies of SEP-363856, MedDRA preferred terms were identified from the following source:

MedDRA version 22.0 SMQ: Extrapyramidal syndrome [20000095], Broad, including all 4 sub-SMQs (Akathisia [20000096], Dyskinesia [20000097], Dystonia [20000098], and Parkinson-like events [20000099])

#### **Description:**

All preferred terms listed in the MedDRA version 22.0 SMQ for Extrapyramidal syndrome [20000095] were included. The table below depicts the preferred terms by sub-SMQ.

Table 8: Extrapyramidal Syndrome SMQ Using MedDRA v 22.0

| Akathisia | | Dyskinesia | | Dystonia | | Parkinson-like | |
|---|---|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code | PT | Code |
| Akathisia | 10001540 | - | - | - | - | - | - |
| - | - | - | - | - | - | Akinesia | 10001541 |
| - | - | Athetosis | 10003620 | - | - | - | - |
| - | - | Ballismus | 10058504 | - | - | - | - |
| - | - | - | - | - | - | Bradykinesia | 10006100 |
| - | - | Buccoglossal syndrome | 10006532 | - | - | - | - |
| - | - | Chorea | 10008748 | - | - | - | - |
| - | - | Choreoathetosis | 10008754 | - | - | - | - |
| - | - | - | - | | | Cogwheel rigidity | 10009848 |
| - | - | Dopamine<br>dysregulation<br>syndrome | 10067468 | - | - | - | - |
| - | - | - | - | Dopa-<br>responsive<br>dystonia | 10080034 | - | - |
| - | - | Dyskinesia | 10013916 | - | - | - | - |
| - | - | Dyskinesia<br>neonatal | 10013922 | - | - | - | - |
| - | - | Dyskinesia<br>oesophageal | 10013924 | - | - | - | - |
| - | - | | | Dystonia | 10013983 | | |
| - | - | | | Dystonic tremor | 10073210 | | |
| - | - | - | - | Early onset primary dystonia | 10076668 | - | - |
| - | - | - | - | Emprosthotonus | 10014566 | - | - |
| - | - | - | - | - | - | Freezing phenomenon | 10060904 |
| - | - | Grimacing | 10061991 | - | - | - | - |
| - | - | - | - | - | - | Hypertonia | 10020852 |

Author: PPD

Author: Version Number: 1.0



| Akathisia | | Dyskinesia | | Dystonia | | Parkinson-like | |
|---|---|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code | PT | Code |
| - | - | - | - | - | - | Hypertonia | |
| | | | | | | neonatal | 10048615 |
| - | - | - | - | - | - | Hypokinetic | |
| | | | | | | dysarthria | 10082243 |
| _ | - | - | - | Meige's | 10027138 | | |
| | | | | syndrome | | | |
| - | - | - | - | - | - | Muscle rigidity | 10028330 |
| - | - | Oculogyric crisis | 10030071 | Oculogyric crisis | 10030071 | , | |
| - | - | - | - | - | - | On and off | 10030312 |
| | | | | | | phenomenon | |
| - | - | - | - | Opisthotonus | 10030899 | - | - |
| - | - | | | Oromandibular | 10067954 | - | - |
| | | | | dystonia | | | |
| - | - | - | - | - | - | Parkinsonian | 10048868 |
| | | | | | | crisis | |
| - | - | - | - | - | - | Parkinsonian | 10056242 |
| | | | | | | gait | |
| - | - | - | - | - | - | Parkinsonian | 10056437 |
| | | | | | | rest tremor | |
| - | - | - | - | - | - | Parkinsonism | 10034010 |
| - | - | - | - | - | - | Parkinsonism | 10071243 |
| | | | | | | hyperpyrexia | |
| | | | | | | syndrome | |
| - | - | - | - | - | - | Parkinson's | 10061536 |
| | | | | | | disease | |
| - | - | - | - | - | - | Parkinson's | 10074835 |
| | | | | | | disease | |
| | | | | | | psychosis | |
| - | - | Pharyngeal | 10070912 | - | - | - | - |
| | | dyskinesia | | | | | |
| - | - | - | - | Pharyngeal | 10081226 | - | - |
| | | | | dystonia | | | |
| - | - | - | - | Pleurothotonus | 10035628 | - | - |
| - | - | - | - | | | Propulsive gait | 10082328 |
| - | - | Protrusion | 10037076 | - | - | - | - |
| | | tongue | | | | | |
| - | - | Rabbit | 10068395 | - | - | - | - |
| | | syndrome | | | | | |
| - | - | Respiratory | 10057570 | - | - | - | - |
| | | dyskinesia | | | | | |
| - | - | - | - | - | - | Resting tremor | 10071390 |
| - | - | - | - | Spasmodic | 10067672 | - | - |
| | | | | dysphonia | | | |
| - | - | Tardive | 10043118 | - | - | - | - |
| | | dyskinesia | | | | | |
| - | - | - | - | Torticollis | 10044074 | - | - |
| - | - | - | - | Trismus | 10044684 | - | - |
| - | - | - | - | Writer's cramp | 10072249 | - | - |




| Akathisia | | Dyskinesia | | Dystonia | | Parkinson-like | |
|---|---|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code | PT | Code |
| - | - | Abnormal involuntary movement scale | 10075002 | - | - | - | - |
| = | - | = | - | = | - | Action tremor | 10072413 |
| - | - | - | - | Blepharospasm | 10005159 | | |
| - | - | - | - | - | - | Bradyphrenia | 10050012 |
| - | - | Chronic tic disorder | 10076661 | Chronic tic disorder | 10076661 | - | - |
| - | - | Complex tic | 10076663 | Complex tic | 10076663 | - | - |
| - | - | Drooling | 10013642 | Drooling | 10013642 | Drooling | 10013642 |
| - | - | - | - | - | - | Dysphonia | 10013952 |
| Extrapyramidal disorder | 10015832 | Extrapyramidal disorder | 10015832 | Extrapyramidal disorder | 10015832 | Extrapyramidal disorder | 10015832 |
| - | - | - | - | Facial spasm | 10063006 | - | - |
| - | - | - | - | - | - | Fine motor skill dysfunction | 10076288 |
| - | - | - | - | - | - | Gait<br>disturbance | 10017577 |
| - | - | - | - | Gait inability | 10017581 | - | - |
| Hyperkinesia | 10020651 | - | - | - | - | - | - |
| Hyperkinesia<br>neonatal | 10020652 | - | - | - | - | - | - |
| - | - | - | - | - | - | Hypokinesia | 10021021 |
| - | - | - | - | - | - | Hypokinesia<br>neonatal | 10021022 |
| - | - | - | - | - | - | Laryngeal<br>tremor | 10078751 |
| - | - | - | - | Laryngospasm | 10023891 | - | - |
| - | - | - | - | - | - | Micrographia | 10057333 |
| - | - | - | - | - | - | Mobility<br>decreased | 10048334 |
| Motor | 10061296 | Motor | 10061296 | Motor | 10061296 | Motor | 10061296 |
| dysfunction | | dysfunction | | dysfunction | | dysfunction | |
| Movement disorder | 10028035 | Movement disorder | 10028035 | Movement disorder | 10028035 | Movement disorder | 10028035 |
| - | - | Muscle<br>twitching | 10028347 | - | - | - | - |
| - | - | - | - | Muscle<br>contractions<br>involuntary | 10028293 | - | - |
| - | - | - | - | Muscle spasms | 10028334 | - | - |
| - | - | - | - | Muscle<br>spasticity | 10028335 | - | - |
| - | - | - | - | Muscle<br>tightness | 10049816 | - | - |
| - | - | - | - | Muscle tone<br>disorder | 10072889 | Muscle tone disorder | 10072889 |
| - | - | - | - | Muscle<br>twitching | 10028347 | - | - |

Document: PPD

Author: Version Number: 1.0 Version Date: 06MAY2024



| Akathisia | | Dyskinesia | | Dystonia | | Parkinson-like | |
|---|---|---|---|---|---|---|---|
| PT | Code | PT | Code | PT | Code | PT | Code |
| - | - | - | - | Musculoskeletal stiffness | 10052904 | Musculoskeletal stiffness | 10052904 |
| - | - | - | - | Oesophageal spasm | 10030184 | - | - |
| - | - | - | - | Oropharyngeal spasm | 10031111 | - | - |
| - | - | - | - | Posture<br>abnormal | 10036436 | - | - |
| - | - | - | - | - | - | Postural reflex impairment | 10067206 |
| - | - | - | - | - | - | Postural tremor | 10073211 |
| - | - | | | Posturing | 10036437 | - | - |
| - | - | Provisional tic disorder | 10076694 | Provisional tic disorder | 10076694 | - | - |
| Psychomotor hyperactivity | 10037211 | - | - | - | - | - | - |
| | | - | - | - | - | Reduced facial expression | 10078576 |
| Restlessness | 10038743 | - | - | - | - | - | - |
| - | - | - | - | Risus sardonicus | 10039198 | - | - |
| - | - | Secondary tic | 10076702 | Secondary tic | 10076702 | - | - |
| - | - | Tic | 10043833 | Tic | 10043833 | = | - |
| - | - | - | - | Tongue spasm | 10043981 | = | - |
| - | - | - | - | Torticollis psychogenic | 10044076 | - | - |
| - | - | - | - | - | - | Tremor | 10044565 |
| - | - | - | - | - | - | Tremor<br>neonatal | 10044575 |
| - | - | - | - | Uvular spasm | 10050908 | - | - |
| - | - | - | - | - | - | - | - |
| - | - | - | - | - | - | Walking<br>disability | 10053204 |

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ררט | Version Number: | 1.0 |



# APPENDIX 7. Predefined Potentially Clinically Significant (PCS) Criteria in SI Units

## STANDARD PCS CRITERIA FOR LABORATORY PARAMETERS - SI UNITS

| Category | | |
|---|---|---|
| Parameter Name | PCS Low | PCS High |
| Age/Sex Restriction, if any | | |
| HEMATOLOGY | | |
| WBC | ≤ 2.8 × 10 <sup>9</sup> /L | ≥ 16 × 10 <sup>9</sup> /L |
| Neutrophils (abs) | < 0.5 × 10 <sup>9</sup> /L | > 13.5 × 10 <sup>9</sup> /L |
| Lymphocytes (abs) | N/A | > 12 × 10 <sup>9</sup> /L |
| Monocytes (abs) | N/A | > 2.5 × 10 <sup>9</sup> /L |
| Eosinophils (abs) | N/A | > 1.6 × 10 <sup>9</sup> /L |
| Basophils (abs) | N/A | > 1.6 × 10 <sup>9</sup> /L |
| Neutrophils (relative) | ≤ 0.15 | > 0.85 |
| Lymphocytes (relative) | N/A | ≥ 0.75 |
| Monocytes (relative) | N/A | ≥ 0.15 |
| Eosinophils (relative) | N/A | ≥ 0.10 |
| Basophils (relative) | N/A | ≥ 0.10 |
| Hemoglobin | | |
| Male | ≤ 115 g/L | ≥ 190 g/L |
| Female | ≤ 95 g/L | ≥ 175 g/L |
| Hematocrit | | |
| Male | ≤ 0.37 | ≥ 0.60 |
| Female | ≤ 0.32 | ≥ 0.54 |
| RBC | ≤ 3.5 × 10 <sup>12</sup> /L | ≥ 6.4 × 10 <sup>12</sup> /L |
| Platelet Count | ≤ 75 × 10 <sup>9</sup> /L | ≥ 700 × 10 <sup>9</sup> /L |
| SERUM CHEMISTRY | | |
| Sodium | < 130 mmol/L | > 150 mmol/L |
| Potassium | < 3 mmol/L | > 5.5 mmol/L |
| Chloride | ≤ 90 mmol/L | ≥ 118 mmol/L |
| Calcium | < 1.75 mmol/L | ≥ 3.1 mmol/L |
| Phosphate | < 0.65 mmol/L | > 1.65 mmol/L |
| Bicarbonate | < 15.1 mmol/L | > 34.9 mmol/L |
| Magnesium | < 0.4 mmol/L | > 1.23 mmol/L |
| AST | N/A | ≥ 3 × ULN |
| ALT | N/A | ≥ 3 × ULN |
| Alkaline Phosphatase | N/A | ≥ 1.5 × ULN |
| CK | N/A | > 2.5 × ULN |
| Creatinine | N/A | ≥ 177 umol/L |
| BUN | N/A | ≥ 10.7 mmol/L |
| Total bilirubin | N/A | ≥ 34.2 umol/L OR > 2 × ULN |
| Total protein | ≤ 45 g/L | ≥ 100 g/L |
| Albumin | ≤ 25 g/L | N/A |
| Total Cholesterol | N/A | > 7.76 mmol/L |
| HDL-Cholesterol | < 0.78 mmol/L | N/A |
| LDL-Cholesterol | N/A | > 4.9 mmol/L |
| Triglycerides | N/A | > 3.42 mmol/L |

| Document: | PPD |
|-----------|-----|



| Uric acid | | |
|------------|---------------|---------------|
| Male | N/A | > 595 umol/L |
| Female | N/A | > 476 umol/L |
| Glucose | < 2.78 mmol/L | > 13.9 mmol/L |
| HbA1c | N/A | ≥ 0.075 |
| Prolactin | N/A | ≥ 5 × ULN |
| URINALYSIS | | |
| RBC | N/A | > 25 hpf |
| WBC | N/A | > 25 hpf |

Document: PPD

Author: Version Number: 1.0



## APPENDIX 8. **PSQI Scoring Sheet**

PSQI scoring reference as defined by BUYSSE is provided in following website:

https://www.sleep.pitt.edu/instruments/#psqi

Author: PPD


#### Pittsburgh Sleep Quality Index (PSQI)

#### Form Administration Instructions, References, and Scoring

#### **Form Administration Instructions**

The range of values for questions 5 through 10 are all 0 to 3.

Questions 1 through 9 are not allowed to be missing except as noted below. If these questions are missing then any scores calculated using missing questions are also missing. Thus it is important to make sure that all questions 1 through 9 have been answered.

In the event that a range is given for an answer (for example, '30 to 60' is written as the answer to Q2, minutes to fall asleep), split the difference and enter 45.

#### Reference

Buysse DJ, Reynolds CF, Monk TH, Berman SR, Kupfer DJ: The Pittsburgh Sleep Quality Index: A new instrument for psychiatric practice and research. *Psychiatry Research* 28:193-213, 1989.

## Scores - reportable in publications

On May 20, 2005, on the instruction of Dr. Daniel J. Buysse, the scoring of the PSQI was changed to set the score for Q5J to 0 if either the comment or the value was missing. This may reduce the DISTB score by 1 point and the PSQI Total Score by 1 point.

#### PSQIDURAT DURATION OF SLEEP

IF Q4 > 7, THEN set value to 0

IF Q4 < 7 and  $\geq$  6, THEN set value to 1 IF Q4 < 6 and > 5, THEN set value to 2

IF Q4 < 5, THEN set value to 3

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQIDISTB SLEEP DISTURBANCE

IF Q5b + Q5c + Q5d + Q5e + Q5f + Q5g + Q5h + Q5i + Q5j (IF Q5JCOM is null or Q5j is null, set the value of Q5j to 0) = 0, THEN set value to 0

IF Q5b + Q5c + Q5d + Q5e + Q5f + Q5g + Q5h + Q5i + Q5j (IF Q5JCOM is null or Q5j is null, set the value of Q5j to 0) > 1 and < 9, THEN set value to 1

IF Q5b + Q5c + Q5d + Q5e + Q5f + Q5g + Q5h + Q5i + Q5j (IF Q5JCOM is null or Q5i is null, set the value of Q5i to 0) > 9 and < 18, THEN set value to 2

IF Q5b + Q5c + Q5d + Q5e + Q5f + Q5g + Q5h + Q5i + Q5j (IF Q5JCOM is null or Q5j is null, set the value of Q5j to 0) > 18, THEN set value to 3

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQILATEN SLEEP LATENCY

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראח | Version Number: | 1.0 |

First, recode Q2 into Q2new thusly:

IF Q2  $\geq$  0 and  $\leq$  15, THEN set value of Q2new to 0 IF Q2 > 15 and  $\leq$  30, THEN set value of Q2new to 1 IF Q2 > 30 and  $\leq$  60, THEN set value of Q2new to 2

IF Q2 > 60, THEN set value of Q2new to 3

Next

IF Q5a + Q2new = 0. THEN set value to 0

IF Q5a + Q2new  $\geq$  1 and  $\leq$  2, THEN set value to 1 IF Q5a + Q2new  $\geq$  3 and  $\leq$  4, THEN set value to 2

IF Q5a + Q2new  $\geq$  5 and  $\leq$  6, THEN set value to 3

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQIDAYDYS DAY DYSFUNCTION DUE TO SLEEPINESS

IF Q8 + Q9 = 0, THEN set value to 0

IF Q8 + Q9  $\geq$  1 and  $\leq$  2, THEN set value to 1 IF Q8 + Q9  $\geq$  3 and  $\leq$  4, THEN set value to 2 IF Q8 + Q9  $\geq$  5 and  $\leq$  6, THEN set value to 3

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQIHSE SLEEP EFFICIENCY

Diffsec = Difference in seconds between day and time of day Q1 and day Q3

Diffhour = Absolute value of diffsec / 3600

newtib =IF diffhour > 24, then newtib = diffhour - 24
IF diffhour < 24, THEN newtib = diffhour

(NOTE, THE ABOVE JUST CALCULATES THE HOURS BETWEEN GNT (Q1)

AND GMT (Q3))

tmphse = (Q4 / newtib) \* 100

IF tmphse ≥ 85, THEN set value to 0

IF tmphse < 85 and  $\geq$  75, THEN set value to 1 IF tmphse < 75 and  $\geq$  65, THEN set value to 2

IF tmphse < 65, THEN set value to 3

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQISLPQUAL OVERALL SLEEP QUALITY

Q6

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQIMEDS NEED MEDS TO SLEEP

Q7

Minimum Score = 0 (better); Maximum Score = 3 (worse)

#### PSQI TOTAL

DURAT + DISTB + LATEN + DAYDYS + HSE + SLPQUAL + MEDS

Minimum Score = 0 (better); Maximum Score = 21 (worse)
Interpretation: TOTAL ≤ 5 associated with good sleep quality
TOTAL > 5 associated with poor sleep quality

Author: PPD


## APPENDIX 9. CLASSIFICATION OF PATIENT Type FROM UPSM FACTOR SCORES

Guided machine learning via linear support vector machine (L-SVM) algorithm in MATLAB will be used to classify subjects into 5 patient types based on UPSM factor scores. There are 5 distinct patient types described in the table below.

| TYPE | PATIENT TYPE |
|------|--------------------------|
| 1 | Prominently Disorganized |
| 2 | Prominently Negative |
| 3 | Prominently Hostile |
| 4 | Prominently Positive |
| 5 | Prominently Affective |

The classification will occur in two steps:

- Step 1: Train L-SVM in MATLAB to classify subjects into 1 of 5 patient types using 7 columns of UPSM data. Training dataset is given in the table below.
- Step 2: Use the now trained classifier function in MATLAB to classify subjects into 1 of 5 patient types using 7 columns of UPSM data.

**Table 9: Training Dataset** 

| UPSM-HOS | UPSM-DIS | UPSM-POS | UPSM-NAA | UPSM-ANX | UPSM-NDE | UPSM-DEP | TYPE |
|---|---|---|---|---|---|---|---|
| 0.110138 | 1.960813 | 0.478927 | 3.298293 | 1.382828 | 2.114771 | 0.391504 | 1 |
| 1.431769 | 1.616874 | 3.310726 | 2.225812 | 0.541127 | 1.542821 | 0.22721 | 4 |
| 0.537462 | 2.293898 | 3.358519 | 2.713077 | 2.582309 | 1.584137 | 2.762624 | 5 |
| 1.458801 | 0.51371 | 3.162632 | 4.179415 | 2.367169 | 0.687056 | 2.014098 | 5 |
| 0.491282 | 1.47429 | 0.583566 | 2.633944 | 4.227873 | 1.12837 | 3.735909 | 5 |
| 2.124307 | 2.621508 | 2.553096 | 1.81619 | 1.463642 | 0.857061 | 1.801388 | 3 |
| 0.229749 | 4.356682 | 3.900132 | 2.980611 | 1.59104 | 2.825456 | 2.487569 | 1 |
| 0.65872 | 1.492003 | 3.98728 | 1.558729 | 1.721153 | 1.716735 | 2.567419 | 4 |
| 4.311785 | 3.13258 | 3.26397 | -0.53456 | 3.583895 | 0.246863 | 3.063737 | 3 |
| 1.673673 | 2.982224 | 2.381804 | 0.168301 | 2.017634 | 2.223616 | 2.420761 | 3 |
| -0.28911 | 1.117716 | 3.325504 | 4.394722 | 0.710643 | 2.619891 | 1.77449 | 4 |
| -0.40258 | 1.164411 | 3.68884 | 2.699136 | 3.395212 | 2.032147 | 2.131544 | 5 |
| 0.120462 | 2.660464 | 3.395254 | 2.078197 | 2.900268 | 0.261296 | 2.725002 | 4 |
| 1.361992 | 3.411795 | 4.64508 | 0.18819 | 1.223746 | 2.532468 | 1.366811 | 4 |
| 3.667904 | 3.136446 | 2.321715 | 2.125103 | 3.409371 | 1.537432 | -0.2218 | 3 |
| 4.879887 | 3.475862 | 2.076838 | -0.59349 | 1.113849 | 1.688076 | 0.123996 | 3 |
| -0.02164 | 2.41729 | 2.779121 | 3.079331 | 2.108443 | 1.951256 | 1.676715 | 1 |
| -0.3092 | 2.157215 | 2.674034 | 2.803489 | 1.084307 | 0.996332 | 1.994321 | 4 |
| 0.196083 | 2.475004 | 2.878793 | 1.351682 | 1.201559 | 0.816825 | 2.181635 | 4 |
| 0.030238 | 3.526967 | 4.532129 | 0.380547 | 0.326149 | 1.986222 | 1.517082 | 4 |
| 2.275873 | 2.640193 | 3.251667 | 0.839343 | 2.051567 | 0.58417 | 2.170745 | 3 |
| 0.664909 | 2.042059 | 2.76595 | 2.366495 | 1.440192 | 0.733822 | 2.402925 | 5 |
| 1.243306 | 1.337145 | 4.074218 | 2.793057 | 2.698381 | 2.51747 | 3.318289 | 5 |
| 3.22947 | 2.860181 | 3.577492 | 3.502082 | 2.628584 | 0.298051 | 3.390157 | 5 |
| 0.901195 | 1.663412 | 2.142304 | 3.688469 | 1.330552 | 2.56257 | 2.640387 | 5 |
| 2.593164 | 3.648882 | 3.709823 | 3.206283 | 1.011247 | 1.094186 | 3.558644 | 3 |
| -0.51118 | 2.448093 | 2.437806 | 1.15006 | 2.797663 | 3.063268 | 2.065887 | 1 |
| -0.11226 | 1.666885 | 2.743509 | 1.415346 | 0.850013 | 2.305111 | 1.401516 | 4 |
| 0.461343 | 2.627467 | 4.224476 | 0.273361 | 1.87481 | 0.626399 | 1.981483 | 4 |
| 2.984818 | 3.119943 | 1.817018 | 0.766638 | 2.093436 | 1.529787 | 0.320228 | 3 |
| 3.77918 | 4.634406 | 1.565869 | 3.283619 | 0.239241 | 1.954698 | 0.044583 | 2 |

Document: PPD

Author: Version Number: 1.0



| 2.144653 | 2.782737 | 3.498727 | 0.538967 | 1.545457 | 0.710868 | 0.792113 | 3 |
|---|---|---|---|---|---|---|---|
| 0.894321 | 4.51713 | 0.328192 | 4.038478 | 0.461848 | 4.202648 | 0.153093 | 2 |
| -0.36753 | 4.43122 | 3.945508 | 3.314841 | 3.447207 | 2.09228 | 1.277813 | 1 |
| -0.54075 | 4.778543 | 0.863248 | 4.518782 | 2.584591 | 3.675675 | 1.102248 | 1 |
| 0.567503 | 3.24148 | 3.050335 | 3.616151 | 2.485309 | 1.23559 | 1.194027 | 1 |
| -0.14361 | 3.811718 | 1.934878 | 4.106673 | 2.496619 | 1.883645 | 1.255909 | 1 |
| 2.074899 | 4.309083 | 3.67494 | 2.931829 | 2.158336 | 1.564656 | 0.532635 | 2 |
| -0.19755 | 3.56726 | 2.443049 | 2.469007 | 2.522924 | 2.551866 | 4.876176 | 1 |
| 1.77413 | 1.53753 | 2.847139 | 1.882985 | 0.272108 | 1.812518 | 3.542881 | 5 |
| 1.620442 | 2.629055 | 2.66762 | -0.09426 | 2.112038 | 0.781558 | 3.528088 | 3 |
| 0.284396 | 1.770956 | 2.033619 | 2.009207 | 3.469858 | 0.528655 | 2.227344 | <u>5</u> |
| 3.932854 | 4.528324 | 2.861762 | 1.430475 | 2.837778 | 1.200249 | 2.254885 | 3 |
| -0.56969 | 0.692111 | 4.179689 | 2.437995 | 1.95239 | 1.874127 | 3.146663 | 5 |
| 4.750689 | 2.427282 | 4.856594 | 3.187711 | 1.452157 | -0.41915 | 0.793141 | 3 |
| 3.405697 | 1.355663 | 3.002656 | 3.832785 | 3.044058 | 1.05007 | 2.012123 | 5 |
| 3.246586 | 1.094777 | 3.274349 | 3.670523 | 2.797322 | 0.536438 | 3.19334 | 5 |
| -0.73954 | 2.073529 | 3.517236 | 4.06399 | 3.114689 | 3.682423 | 3.860445 | 5 |
| -0.52019 | 1.761008 | 4.510467 | 2.327021 | 2.304678 | 3.148164 | 2.974405 | 4 |
| 2.014756 | 2.407895 | 2.295336 | 2.006102 | 1.24862 | 3.567501 | 2.040139 | 2 |
| 0.617758 | 2.661608 | 1.536687 | 3.738151 | 1.672221 | 2.392486 | -0.23323 | 2 |
| 2.207155 | 1.517604 | 2.625454 | 1.804154 | 0.763335 | 0.901574 | 1.873668 | 3 |
| 1.23422 | 2.210916 | 2.561197 | 2.528093 | 1.527851 | 1.183324 | 0.255261 | 4 |
| 0.021092 | 1.402188 | 2.331655 | 1.812051 | 2.72359 | 0.272525 | 2.258971 | 5 |
| -0.954 | 5.328812 | 2.839309 | 3.194626 | 2.923765 | 1.602491 | 3.133907 | 1 |
| 3.167057 | 3.125152 | 1.146554 | 4.533739 | 1.648505 | 1.456163 | 2.409444 | 2 |
| 0.076614 | 2.337764 | 1.24781 | 1.632617 | 2.307237 | 1.494694 | 0.092505 | 1 |
| 1.769865 | 3.050355 | 3.584774 | 3.050455 | 0.435454 | 0.965985 | 1.414732 | 4 |
| -0.14345 | 2.274485 | 3.363205 | 2.516223 | 1.298419 | 0.84683 | 0.939489 | 4 |
| 0.73008 | 2.109659 | 1.353254 | 2.267853 | 1.683644 | 1.547878 | 2.385081 | 1 |
| 1.99611 | 2.845866 | 2.776477 | 2.253987 | 2.519993 | 1.293208 | 0.830398 | 3 |
| 0.070748 | 2.973237 | 2.458206 | 2.670777 | 0.933532 | 0.498741 | 0.68469 | 4 |
| 0.876838 | 1.702267 | 2.500296 | 1.205238 | 1.988358 | 1.73428 | 1.88312 | 5 |
| 2.539879 | 1.866446 | 1.194986 | 2.380642 | 1.503776 | 2.970662 | 0.607604 | 2 |
| 1.394134 | 3.329297 | 3.029867 | 2.34767 | 2.089692 | 0.610036 | 3.175958 | 5 |
| 1.370158 | 3.673851 | 0.853038 | 2.542066 | 2.93799 | 2.377451 | 1.666476 | 1 |
| 1.873059 | 1.656544 | 2.282509 | 0.870666 | 2.632208 | 0.4312 | 1.362965 | 3 |
| 2.587309 | 1.766566 | 1.972871 | 2.451865 | 2.200703 | 1.026357 | 0.802177 | 3 |
| 3.83788 | 1.83301 | 2.241711 | 3.814479 | 1.270124 | 0.82664 | 0.010026 | 3 |
| 1.139727 | 1.009246 | 2.171023 | 2.861618 | 1.94202 | 1.469105 | 2.310987 | <u>5</u> |
| 0.399375 | 1.269958 | 3.185143 | 3.451366 | 2.536612 | 1.873559 | 3.891391 | 5 |
| | 0.720076 | | | 1.676011 | | 1.931072 | 5 |
| 1.155282 | | 1.978406<br>2.176408 | 2.550957 | | 2.227286 | | |
| 1.344237 | 1.329165 | | 2.522749 | 2.36858 | 1.113254 | 1.862452 | 5 |
| 1.884397 | 0.811162 | 2.366897 | 3.193561 | 1.903167 | 0.529586 | 3.039549 | 5 |
| 0.857138 | 1.991846 | 4.143588 | 3.203741 | 2.567467 | 1.723389 | 2.662205 | 5 |
| 0.316037 | 0.913369 | 3.265191 | 3.908459 | 2.02769 | 2.805904 | 3.226179 | 5 |
| 0.941557 | 1.611534 | 3.550319 | 2.397795 | 2.465604 | 1.637112 | 2.268425 | 5 |
| 1.001373 | 0.053415 | 2.59386 | 3.243315 | 2.765545 | 1.745535 | 1.070277 | 5 |
| 0.503857 | 0.731232 | 2.859462 | 3.221411 | 1.999709 | 0.617281 | 0.785101 | 4 |
| 0.606582 | 1.644987 | 2.617478 | 3.87998 | 1.79895 | 0.52075 | 1.931541 | 5 |
| 0.028959 | 0.051636 | 2.679662 | 3.743596 | 1.258786 | 0.796158 | 2.684655 | 5 |
| 1.346641 | 0.874823 | 2.367707 | 3.081821 | 1.922213 | 0.204586 | 1.535142 | 5 |
| 1.860828 | 2.605349 | 3.667323 | 4.365784 | -0.09249 | 1.265363 | 1.238416 | 2 |
| 3.841476 | 0.719424 | 2.257701 | 4.478491 | 1.331765 | 0.100831 | 1.896058 | 5 |
| 1.661837 | 1.572432 | 2.894384 | 4.184757 | 1.296394 | 0.92299 | 2.19499 | 5 |
| 1.639518 | 1.463103 | 2.652642 | 1.584517 | 2.156156 | 1.371609 | 1.96164 | 5 |
| 0.422721 | 1.235118 | 2.915662 | 1.806378 | 1.774961 | 1.461898 | 1.782514 | 5 |
| 1.706561 | 2.255214 | 2.013119 | 3.335592 | 1.432492 | 1.106246 | 0.37835 | 2 |
| 1.400759 | 1.11035 | 3.176518 | 2.727226 | 1.683432 | 1.484354 | 2.072159 | 5 |
| 0.261743 | 1.846856 | 2.95069 | 1.604365 | 1.313196 | 2.201688 | 2.045153 | 4 |

Document: PPD

Author: Version Number: 1.0 Version Date: 06MAY2024



| 0.50000 | 4 00040 | | 0.447404 | 4 005000 | 4.00000= | 0.000004 | |
|---|---|---|---|---|---|---|---|
| 0.589363 | 1.63248 | 2.607093 | 3.117401 | 1.985862 | 1.962965 | 2.226981 | 5 |
| -0.25198 | 1.221123 | 3.025169 | 3.361783 | 1.767464 | 1.630335 | 2.390124 | 5 |
| 2.291071 | 0.293838 | 3.270165 | 3.243712 | 2.442306 | -0.00452 | 2.387481 | 5 |
| 1.537487 | 0.068818 | 3.108614 | 1.546074 | 2.023246 | 1.696579 | 2.706242 | 5 |
| 0.582496 | 1.908653 | 2.366867 | 2.51433 | 1.475041 | 0.41553 | 1.263473 | 4 |
| 2.181457 | 1.917974 | 2.429864 | 2.922081 | 1.514385 | -0.21779 | 1.973444 | 3 |
| 2.263951 | 0.29547 | 3.331314 | 1.415383 | 2.346612 | 1.031364 | 2.892756 | 5 |
| 2.009356 | 1.113335 | 3.138889 | 3.341652 | 1.883817 | 0.109166 | 1.958678 | 5 |
| 0.172439 | 1.489999 | 3.292475 | 2.720522 | 1.176231 | 1.605558 | 2.641559 | 5 |
| -0.17314 | 1.356652 | 4.442061 | 3.10633 | 2.049317 | 0.791991 | 1.912506 | 4 |
| 1.388335 | 1.095188 | 3.220865 | 1.628662 | 1.732311 | 1.352052 | 2.405447 | 5 |
| 1.205138 | 2.024409 | 3.791492 | 2.398941 | 3.006668 | 1.787416 | 2.920256 | 5 |
| 0.464397 | 1.684218 | 3.40262 | 2.726862 | 3.013933 | 1.189662 | 3.61535 | 5 |
| 1.628768 | 1.308049 | 2.95217 | 2.745054 | 1.327077 | 2.028925 | 3.357957 | 5 |
| 0.586597 | 2.536766 | 2.916748 | 3.252801 | 2.392646 | 2.207333 | 3.37449 | 5 |
| 0.668672 | 0.21496 | 3.401807 | 3.499059 | 2.747658 | 2.264928 | 3.708938 | 5 |
| 1.85842 | 1.032293 | 3.81473 | 3.017692 | 2.560804 | 1.060393 | 2.687179 | 5 |
| 0.421477 | 1.193203 | 3.072718 | 3.197042 | 2.410182 | 2.327653 | 3.342285 | 5 |
| 0.705007 | 2.094874 | 1.758942 | 2.993589 | 1.631168 | 1.769052 | 2.175233 | 1 |
| 1.341319 | 2.511154 | 2.487053 | 0.737579 | 1.309727 | 1.172314 | 2.21039 | 3 |
| -0.10475 | 3.201991 | 2.494132 | 3.312053 | 0.911785 | 2.561984 | 0.543735 | 2 |
| 1.26418 | 1.34083 | 2.50963 | 3.164473 | 0.66512 | 1.883488 | 1.486237 | 2 |
| 2.135516 | 2.140969 | 2.155306 | 4.111724 | 2.433874 | 1.272746 | 2.910099 | 5 |
| 0.11181 | 3.029033 | 2.241817 | 4.074078 | 2.229162 | 1.485626 | 1.801666 | 1 |
| 0.57075 | 4.309476 | 3.042631 | 3.640668 | 1.121444 | 1.676763 | 0.985236 | 2 |
| 2.368828 | 2.078152 | 1.757995 | 3.68918 | 2.238158 | 0.832056 | 3.202517 | 5 |
| 0.460592 | 3.343601 | 1.369653 | 3.591892 | 3.052149 | 1.590111 | 1.853283 | 1 |
| 1.039519 | 2.73413 | 2.797452 | 4.794559 | 3.188477 | 1.32171 | 2.069804 | 1 |
| -0.10856 | 3.283553 | 2.221476 | 2.861392 | 2.916771 | 1.670176 | 1.495856 | 1 |
| 1.635721 | 1.670994 | 2.776531 | 3.481021 | 3.648923 | 1.09168 | 3.517521 | 5 |
| -0.28728 | 1.550428 | 3.027047 | 1.569179 | 3.495302 | 1.675143 | 3.72542 | 5 |
| 0.629977 | 1.356138 | 4.076404 | 1.705047 | 2.22813 | 1.423955 | 2.063269 | 4 |
| 2.307646 | 2.236448 | 2.680489 | 0.969736 | 2.569013 | -0.08536 | 2.277701 | 3 |
| 2.477069 | 3.263651 | 2.163565 | 2.139497 | 1.721061 | -0.00358 | 0.65799 | 3 |
| 1.243638 | 2.913075 | 4.107979 | 2.66461 | 0.995093 | -0.14437 | 1.22687 | 4 |
| 0.527388 | 1.958446 | 1.279965 | 3.081775 | 0.643036 | 1.853639 | 2.172642 | 1 |
| 0.424628 | 2.137735 | 2.088917 | 1.156878 | 1.766872 | 1.219234 | 1.53977 | 1 |
| 2.527044 | 0.76957 | 4.013747 | 2.360512 | 3.03441 | -0.3789 | 4.007144 | 5 |
| -0.19304 | 1.261063 | 2.340497 | 2.776243 | 2.052291 | 1.922053 | 3.962693 | 5 |
| 0.533501 | 1.87061 | 4.417346 | 2.075672 | 3.323951 | -0.27006 | 4.225107 | 5 |
| 2.411661 | 1.882853 | 4.355587 | 1.036112 | 1.98607 | 0.055844 | 1.311082 | 3 |
| -0.48578 | 1.752793 | 4.45535 | 3.947321 | 1.094441 | 2.902358 | 2.033406 | 4 |
| 0.464869 | 3.413253 | 2.635796 | 2.121825 | 2.8906 | 1.996746 | 3.22642 | 1 |
| 4.132441 | 0.401081 | 2.381923 | 3.456109 | 0.953315 | 3.096096 | 0.555434 | 2 |
| 0.218247 | 3.435941 | 1.849422 | 1.196065 | 2.511003 | 1.363478 | 0.35237 | 1 |
| -0.32981 | 4.544489 | 1.360392 | 3.024887 | 1.106194 | 2.727317 | 0.572736 | 1 |
| 0.544813 | 4.282196 | 2.116876 | 2.290366 | 2.541964 | 1.369559 | 1.818978 | 1 |
| -0.47234 | 4.088985 | 0.577244 | 2.967936 | 2.63388 | 2.877609 | 2.381399 | 1 |
| -0.55527 | 4.84008 | 1.960686 | 2.982342 | 2.094423 | 1.626178 | 1.184506 | 1 |
| 0.263513 | 3.736018 | 1.959549 | 1.758239 | 1.640343 | 1.004376 | 1.472666 | 1 |
| 0.705893 | 3.718196 | 2.301378 | 0.926439 | 1.774488 | 0.994932 | 1.79793 | 1 |
| 0.069405 | 3.026261 | 2.43983 | 3.17107 | 3.19792 | 2.883761 | 1.97275 | 1 |
| -0.32695 | 0.330879 | 2.510527 | 3.441654 | 2.057765 | 2.304866 | 2.878307 | 5 |
| 2.690017 | 0.693133 | 1.730133 | 3.88509 | 2.562458 | 1.455035 | 1.213344 | 5 |
| 0.46547 | 1.287936 | 2.939181 | 1.394492 | 3.396399 | 2.015295 | 2.080734 | 5 |
| 1.394982 | 1.559578 | 2.471032 | 3.161232 | 2.57522 | 0.992441 | 2.406263 | 5 |
| 0.672309 | 2.393359 | 1.896502 | 2.598218 | 0.993053 | 3.154678 | 1.696235 | 1 |
| 4 000740 | 1.325886 | 0.880014 | 5.37448 | 1.164323 | 3.653433 | 2.895248 | 5 |
| 1.693716<br>1.356159 | 2.406733 | 2.037301 | 2.919935 | 1.869511 | 3.465406 | 1.13788 | 2 |

Document: PPD

Author: Version Number:




| T | 1 | | | 1 | | 1 | |
|---|---|---|---|---|---|---|---|
| 1.027015 | 1.062603 | 0.659294 | 4.357499 | 2.82001 | 3.266347 | 4.132878 | 5 |
| 1.436698 | -0.58649 | 1.964863 | 3.95011 | 3.191804 | 0.377813 | 4.488555 | 5 |
| 4.058956 | -0.66886 | 1.317517 | 4.606702 | 1.160914 | 2.731827 | 3.099033 | 5 |
| 1.416783 | 1.490505 | 2.933091 | 1.730763 | 3.560499 | 0.430518 | 2.821162 | 5 |
| 0.824231 | -0.19387 | 4.748215 | 0.202208 | 2.896445 | 0.69977 | 4.873985 | 5 |
| -0.36924 | 2.678109 | 3.163096 | 1.596358 | 0.59506 | 3.346233 | 1.61617 | 4 |
| 2.327808 | 1.715927 | 3.390249 | 3.327197 | -0.07099 | 1.647033 | 1.876406 | 2 |
| 1.146957 | 1.732186 | 2.467294 | 4.312694 | 0.967439 | 3.606223 | 2.364763 | 2 |
| -0.08434 | 2.371234 | 1.923559 | 2.551661 | 2.780099 | -0.41496 | 2.607441 | 5 |
| 2.330935 | 1.249285 | 1.977942 | -0.29365 | 1.750854 | 1.887952 | 3.34313 | 5 |
| -0.29097 | 2.579936 | 4.03501 | 2.453226 | 1.223345 | 1.756084 | 1.578965 | 4 |
| 2.433418 | 1.586402 | 2.744031 | 2.943148 | 2.595221 | -0.15045 | 4.456784 | 5 |
| 1.686219 | 2.133575 | 3.063004 | 2.625084 | 1.837615 | 0.138859 | 2.505072 | 5 |
| 2.182811 | 2.480894 | 3.512331 | 2.528045 | 3.359501 | 1.174893 | 2.358992 | 5 |
| 1.726701 | 2.611469 | 3.08875 | 2.914048 | 3.581237 | 1.05601 | 1.522262 | 1 |
| 0.604793 | 3.12306 | 2.124151 | 2.637198 | 2.7244 | 2.472494 | 1.200589 | 1 |
| 3.236433 | 3.290153 | 2.702033 | 2.314023 | 3.316992 | 0.3816 | 1.895082 | 3 |
| 1.425043 | 3.692046 | 3.472158 | 4.057196 | 2.405972 | 0.434079 | 2.869765 | 1 |
| 2.201707 | 3.084578 | 2.151076 | 4.021647 | 2.182574 | 2.301893 | 1.407549 | 2 |
| 1.815693 | 2.134869 | 4.303099 | 4.369005 | 1.882038 | 0.949098 | 1.847457 | 4 |
| 1.20209 | 3.064755 | 4.217095 | 3.649783 | 2.915971 | 0.357701 | 1.225159 | 4 |
| 0.046373 | 2.916968 | 4.455808 | 2.885248 | 3.107358 | 0.426352 | 2.008252 | 4 |
| -0.01844 | 3.893585 | 3.026784 | 1.817709 | 0.913144 | 3.254477 | 2.670709 | 1 |
| 0.15412 | 3.328443 | 1.620771 | 1.879719 | 2.673819 | 2.668971 | 2.431268 | 1 |
| -0.07332 | 4.359244 | 3.52468 | 1.723178 | 0.553973 | 1.862672 | 0.970363 | 4 |
| 0.708979 | 3.65687 | 2.295132 | 2.084227 | 1.178033 | 3.673556 | 0.603624 | 2 |
| 1.454947 | 3.430231 | 2.232895 | 2.447069 | 2.309456 | 2.631151 | 2.32591 | 1 |
| 0.583852 | 3.473869 | 2.416568 | 2.141427 | 0.479351 | 2.977283 | 1.947473 | 2 |
| 0.284904 | 3.74932 | 2.086627 | 3.204144 | -0.07831 | 2.28367 | 1.519997 | 2 |
| 0.882449 | 3.863615 | 3.044836 | 2.195771 | -0.10572 | 1.730727 | 0.181928 | 2 |
| 0.180445 | 1.883516 | 1.562047 | 2.663036 | 2.63216 | 2.250718 | 2.436309 | 1 |
| 0.378782 | 2.931791 | 1.708711 | 2.980852 | 2.771396 | 2.111069 | 0.610343 | 1 |
| 0.352732 | 1.89972 | 2.265854 | 3.230448 | 1.11399 | 1.21381 | 2.019503 | 5 |
| -0.07905 | 1.7187 | 0.81324 | 3.213864 | 2.58132 | 2.072825 | 1.596053 | 1 |
| -0.04268 | 2.161476 | 1.854841 | 2.9067 | 2.572292 | 2.05655 | 3.250114 | 1 |
| 0.532978 | 3.478254 | 2.049047 | 1.952408 | 2.807302 | 1.696268 | 1.824182 | 1 |
| 0.155656 | 3.999629 | 3.146047 | 1.349007 | 2.792547 | 1.478153 | 1.4613 | 1 |
| 0.796148 | 2.634837 | 3.132603 | 3.222581 | 2.680883 | 1.854805 | 2.030157 | 1 |
| 0.86594 | 2.609557 | 2.546813 | 1.751367 | 1.740951 | 1.533923 | 2.228512 | <u>-</u> |
| 1.01185 | 2.816307 | 2.912837 | 1.669116 | 2.542537 | 1.330716 | 1.168323 | 1 |
| 1.350645 | 1.989788 | 1.74757 | 3.198019 | 2.213117 | 0.804664 | 1.34773 | 1 |
| 0.349145 | 2.756305 | 1.716076 | 2.68973 | 2.739907 | 1.656974 | 1.623306 | 1 |
| 0.342705 | 1.679803 | 1.833402 | 2.032994 | 2.960676 | 1.663841 | 2.120364 | 1 |
| 1.484201 | 1.539412 | 1.50688 | 2.924464 | 2.475359 | 1.705127 | 1.683536 | 5 |
| 1.562951 | 3.030532 | 1.644437 | 2.014339 | 1.595521 | 1.644179 | 1.164406 | 1 |
| 3.029619 | 2.819386 | 1.874296 | 2.742982 | 1.788343 | 2.269874 | 1.542436 | 2 |
| 0.78352 | 1.877238 | 2.074483 | 2.627216 | 2.240644 | 2.194709 | 2.377748 | 5 |
| 0.710665 | 2.849776 | 2.364681 | 1.919057 | 2.747839 | 1.648826 | 1.233827 | <u></u> |
| 0.798178 | 2.933791 | 3.35471 | 2.705446 | 0.796685 | 3.192393 | 0.488374 | 2 |
| 1.905889 | 4.839237 | 3.456346 | 0.724097 | 2.164524 | 0.999083 | 1.83366 | 3 |
| -0.42893 | 2.354318 | 2.48451 | 3.358162 | 0.714569 | 2.794577 | 2.607276 | <u>3</u> 1 |
| 2.197681 | 2.953134 | 3.844426 | 1.086876 | 0.80736 | -0.01227 | 2.050991 | 3 |
| 1.175299 | 4.850591 | 4.181569 | 1.539452 | 1.490182 | 0.734061 | 1.239397 | 4 |
| -0.50935 | 3.131051 | 2.46547 | 2.550862 | 1.514948 | 3.740844 | 1.942203 | <u>4</u> 1 |
| -0.47872 | 2.432521 | 2.46547 | 3.345092 | 1.896522 | 3.066479 | 3.392814 | 1 |
| 1.647404 | | 0.922094 | | 2.766181 | | | 1 |
| | 2.212889 | 3.626749 | 2.565279 | | 2.737955 | 1.599062 | 5 |
| 2.466112 | 2.010557 | | 3.847344 | 2.514457 | 1.560699 | 3.442844 | |
| 3.004502<br>1.241437 | 2.637176 | 2.798804 | 3.711184 | 2.463544 | 1.57843 | 2.123784 | 3 |
| 1 /4143/ | 2.778655 | 1.589605 | 2.563038 | 2.012834 | 1.91169 | 3.491985 | 1 |

Document: PPD

Author: PPD

Version Number: Version Date:

06MAY2024

1.0

1.0

06MAY2024



Statistical Analysis Plan

| 1.486578 3.128626 2.487837 1.743571 2.003073 1.737516 1.3 2.586535 2.877124 2.287801 2.632841 1.387282 2.363598 2.4 1.66655 2.838318 2.35911 1.973314 1.859279 2.225311 2.9 1.589938 3.65255 2.956482 2.565466 0.975133 1.615948 0.4 | 144007 | $\overline{}$ |
|---|---|---|
| 2.586535 2.877124 2.287801 2.632841 1.387282 2.363598 2.4 1.66655 2.838318 2.35911 1.973314 1.859279 2.225311 2.9 1.589938 3.65255 2.956482 2.565466 0.975133 1.615948 0.4 | 941087 | 3 |
| 2.586535 2.877124 2.287801 2.632841 1.387282 2.363598 2.4 1.66655 2.838318 2.35911 1.973314 1.859279 2.225311 2.9 1.589938 3.65255 2.956482 2.565466 0.975133 1.615948 0.4 | 329548 | 1 |
| 1.66655 2.838318 2.35911 1.973314 1.859279 2.225311 2.9 1.589938 3.65255 2.956482 2.565466 0.975133 1.615948 0.4 | 153764 | 2 |
| 1.589938 3.65255 2.956482 2.565466 0.975133 1.615948 0.4 | 15387 | 1 |
| | 199501 | 2 |
| 1 1945018 1 3 050839 1 2 514292 1 3 234802 1 2 203473 1 1822279 1 1 | | |
| | .99805 | 1 |
| | 758004 | 4 |
| | 160136 | 3 |
| | .89525 | 3 |
| | 91725 | 2 |
| 1.244654 1.73021 1.827923 2.489334 1.383575 2.073081 1.3 | 360675 | 1 |
| | 276463 | 4 |
| | 737043 | 1 |
| | .87712 | 5 |
| | 968036 | 5 |
| | 79216 | 5 |
| | 325316 | 5 |
| | 330153 | 4 |
| | 87518 | 5 |
| | .51607 | 1 |
| | 302135 | 1 |
| | )22366 | 1 |
| | 2.6483 | 1 |
| 1.148024 4.715529 1.712537 1.143191 1.448075 0.735696 1.2 | 255713 | 1 |
| 0.17321 2.714301 3.093773 2.731845 3.555077 0.30472 1.9 | 964692 | 1 |
| | 062154 | 5 |
| | 221664 | 5 |
| | .45575 | 1 |
| | .09806 | 5 |
| | 642933 | 4 |
| | 183245 | 5 |
| | 797111 | |
| | | 5 |
| | 322844 | 5 |
| | 003566 | 4 |
| | 924363 | 1 |
| 1.322036 1.215882 3.921602 3.003509 2.284119 -0.24933 1.8 | 306291 | 5 |
| | .65026 | |
| | | 5 |
| | 83754 | |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 | | 5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. | 83754 | 5<br>1<br>1 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 | .76725<br>.330049 | 5<br>1<br>1<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 | .76725<br>.330049<br>.420509 | 5<br>1<br>1<br>5<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 | .76725<br>.330049<br>.20509<br>.069859 | 5<br>1<br>1<br>5<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 | 583754<br>.76725<br>330049<br>420509<br>069859<br>717352 | 5<br>1<br>1<br>5<br>5<br>1<br>2 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 | 583754<br>.76725<br>330049<br>420509<br>069859<br>717352<br>779611 | 5<br>1<br>1<br>5<br>5<br>1<br>2 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 | 583754<br>.76725<br>.330049<br>.20509<br>.69859<br>.717352<br>.779611<br>.851252 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 | 583754<br>76725<br>330049<br>120509<br>169859<br>717352<br>779611<br>351252<br>110001 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 | 583754<br>576725<br>5330049<br>120509<br>120509<br>169859<br>177352<br>1779611<br>1851252<br>100001<br>1005764 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 083754<br>076725<br>030049<br>020509<br>069859<br>077352<br>079611<br>051252<br>010001<br>005764<br>020828 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 883754<br>.76725<br>.830049<br>.820509<br>.869859<br>.717352<br>.779611<br>.851252<br>.010001<br>.005764<br>.220828<br>.796499 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 083754<br>076725<br>030049<br>020509<br>069859<br>077352<br>079611<br>05764<br>020828<br>0796499<br>014239 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 883754<br>.76725<br>.830049<br>.820509<br>.869859<br>.717352<br>.779611<br>.851252<br>.010001<br>.005764<br>.220828<br>.796499 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 083754<br>076725<br>030049<br>020509<br>069859<br>077352<br>079611<br>05764<br>020828<br>0796499<br>014239 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 883754<br>.76725<br>.830049<br>.820509<br>.869859<br>.77352<br>.779611<br>.851252<br>.010001<br>.005764<br>.220828<br>.796499<br>.114239<br>.156116 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 583754<br>.76725<br>330049<br>120509<br>120609 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 583754<br>.76725<br>330049<br>120509 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 583754<br>.76725<br>.330049<br>120509<br>169859<br>717352<br>779611<br>.351252<br>.110001<br>.105764<br>.220828<br>.796499<br>.114239<br>.156116<br>.1662573<br>.359132<br>.380617<br>.147056 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 583754<br>.76725<br>.330049<br>120509<br>169859<br>717352<br>779611<br>.351252<br>.10001<br>.005764<br>.220828<br>.796499<br>.14239<br>.156116<br>.662573<br>.359132<br>.380617<br>.447056<br>.88581 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 883754<br>.76725<br>.30049<br>120509<br>169859<br>717352<br>779611<br>.351252<br>.110001<br>.105764<br>.220828<br>.796499<br>.114239<br>.156116<br>.162573<br>.359132<br>.380617<br>.147056<br>.88581<br>.83891 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5<br>5<br>5<br>5<br>5<br>7<br>5 |
| 0.59895 3.329155 2.836852 2.202842 1.497784 1.607472 2.5 0.565399 5.191211 2.58232 2.271006 2.778369 1.798438 0. 1.891514 1.030671 2.378489 2.521739 2.470474 1.713408 1.8 2.251343 1.964833 2.782653 2.173102 2.552897 0.928943 2.4 0.827273 1.676045 1.79413 2.599383 2.936736 2.290989 1.0 0.933062 4.872175 1.858903 3.41357 1.483246 3.481183 0.7 1.319798 3.170397 2.467164 3.559172 3.259405 2.329196 0.7 1.159981 2.887268 2.048998 1.864787 1.714485 1.964015 0.8 2.594349 4.47202 1.935226 2.39397 0.807125 1.443819 1.0 2.259674 2.817409 2.241478 3.232779 1.265977 2.904775 1.0 3.853234 3.442007 3.483622 | 583754<br>.76725<br>.330049<br>120509<br>169859<br>717352<br>779611<br>.351252<br>.10001<br>.005764<br>.220828<br>.796499<br>.14239<br>.156116<br>.662573<br>.359132<br>.380617<br>.447056<br>.88581 | 5<br>1<br>1<br>5<br>5<br>1<br>2<br>1<br>1<br>2<br>2<br>3<br>1<br>2<br>5<br>5<br>5<br>5<br>1<br>2<br>5 |

PPD Document:

Author: שא Version Number: Version Date:

The contents of this document are confidential and proprietary to Sunovion Pharmaceuticals Inc. Unauthorized use, disclosure or reproduction is strictly prohibited.



| 1.725945 | 3.009119 | 2.694312 | 0.112874 | 3.046849 | 1.046677 | 2.597689 | 3 |
|---|---|---|---|---|---|---|---|
| 0.631709 | 2.429373 | 2.904648 | 1.845756 | 1.753777 | 3.513261 | 1.93335 | 1 |
| -0.23163 | 3.002049 | 3.345794 | 2.547498 | 3.554414 | 1.593511 | 3.265845 | 1 |
| -0.21477 | 2.923092 | 2.388016 | 3.395137 | 2.936315 | 2.417217 | 2.608649 | 1 |
| 2.292153 | 2.412309 | 2.891003 | 2.297742 | 1.884942 | 0.821511 | 1.938632 | 3 |
| 1.826434 | 3.195578 | 1.861429 | 3.285702 | 2.60437 | 0.337541 | 1.982752 | 1 |
| 1.081747 | 2.024036 | 3.051124 | 2.759296 | 2.689623 | 2.411139 | 3.523435 | 5 |
| 1.726368 | 2.23849 | 3.132346 | 2.316369 | 2.459357 | 2.194413 | 2.921579 | 5 |
| 0.273047 | 2.916457 | 1.761402 | 3.342903 | 1.357142 | 2.447486 | 1.642088 | 1 |
| 2.061364 | 2.246574 | 2.274476 | 2.84223 | 2.513461 | 1.435599 | 1.663619 | 5 |
| -0.44394 | 1.990884 | 2.120804 | 2.786634 | 1.973897 | 3.156599 | 3.453843 | 1 |
| 0.965206 | 1.901004 | 1.431642 | 3.042105 | 2.183742 | 2.33692 | 2.365446 | 1 |
| 1.658993 | 1.392341 | 3.179016 | 2.725544 | 1.270456 | 1.609023 | 2.18851 | 5 |
| 1.841815 | 2.190828 | 2.24286 | 3.811443 | 2.195616 | 0.758591 | 2.922796 | 5 |
| 1.22653 | 1.421029 | 2.261803 | 2.765931 | 2.425561 | 1.732311 | 3.372288 | 5 |
| -0.23487 | 2.062772 | 2.559663 | 2.79011 | 1.445805 | 2.657801 | 2.760422 | 1 |
| 0.245227 | 2.689176 | 1.443797 | 1.973458 | 2.887213 | 1.25989 | 2.374189 | 1 |
| 2.215864 | 1.754762 | 2.859705 | 4.169328 | 2.445922 | 1.18503 | 2.197257 | 5 |
| 2.827656 | 1.672037 | 1.272949 | 2.704282 | 2.616846 | 2.725432 | 3.720687 | 5 |
| 3.199189 | 1.422016 | 2.654105 | 4.302128 | 3.544407 | 1.718565 | 4.051834 | 5 |
| 2.403098 | 2.968469 | 4.036389 | 2.438671 | 1.294979 | 0.563823 | 1.703829 | 3 |
| 2.45239 | 3.234068 | 2.759748 | 1.024698 | 1.562684 | 1.112423 | 2.375853 | 3 |
| 1.502019 | 2.281229 | 1.340381 | 1.610793 | 2.423306 | 1.047639 | 1.624365 | 1 |
| 1.77479 | 1.921922 | 3.237566 | 1.352774 | 2.492678 | 1.049467 | 2.512043 | 5 |
| 1.663432 | 3.019771 | 1.897049 | 0.759906 | 3.501306 | 1.569326 | 1.914466 | 1 |
| 2.94352 | 2.35016 | 2.281449 | 0.951598 | 2.511059 | 1.019162 | 1.526363 | 3 |
| 1.68009 | 2.045579 | 1.887194 | 2.357748 | 1.978092 | 1.635593 | 2.811834 | 5 |
| 0.808124 | -0.13738 | 2.953735 | 3.906694 | 1.947323 | 1.380431 | 2.901026 | 5 |
| 1.209549 | -0.67634 | 4.084019 | 3.428157 | 1.289318 | 1.264035 | 2.480664 | 5 |
| 1.733745 | -0.34144 | 2.996359 | 2.729753 | 1.784482 | -0.03631 | 2.462543 | 5 |
| 1.619052 | 0.150902 | 4.359022 | 2.334887 | 2.914195 | -0.11285 | 1.33825 | 5 |
| -0.13043 | 0.923062 | 2.34262 | 2.347549 | 0.138352 | 3.16152 | 1.597485 | 4 |
| 1.32315 | 0.012205 | 4.865486 | 0.779994 | 1.714469 | 0.367159 | 2.011743 | 4 |
| 2.650652 | 1.224055 | 2.722871 | 2.274911 | 1.37163 | 1.630707 | 1.845764 | 3 |
| 1.607415 | 2.287416 | 2.580634 | 1.22177 | 2.238811 | 1.518263 | 0.841124 | 3 |
| 0.407971 | 0.974984 | 2.534841 | 2.228252 | 3.585527 | 2.013955 | 3.485656 | 5 |
| 1.576527 | 1.697772 | 2.575915 | 3.470199 | 2.282271 | 1.37511 | 2.962369 | 5 |
| 1.956178 | -0.46028 | 4.546977 | 2.448721 | 1.334782 | 1.148109 | 3.918205 | 5 |
| 0.18701 | 2.273386 | 4.282304 | 2.119968 | 2.185045 | 2.674903 | 1.84133 | 4 |
| 0.354561 | 1.314933 | 4.056158 | 2.91016 | 1.719733 | 1.791516 | -0.16259 | 4 |
| 0.797993 | 0.857493 | 3.688851 | 3.229713 | 3.474734 | 2.372434 | 1.533996 | 5 |
| 1.856804 | 2.053879 | 1.920647 | 2.220341 | 2.898173 | 0.918768 | 1.764507 | 5 |
| -0.13872 | 3.299856 | 3.489781 | 2.220536 | 1.711955 | 1.704413 | 3.085852 | 1 |
| 0.72802 | 2.655034 | 3.106166 | 2.872185 | 1.647015 | 1.176479 | 0.846061 | 4 |
| 0.225626 | 1.874406 | 1.825989 | 3.058365 | 2.868861 | 3.509008 | 2.042135 | 1 |
| 2.051621 | 1.818373 | 4.017949 | 2.104391 | 1.201151 | 0.575975 | 1.724579 | 3 |
| 0.59504 | 1.95428 | 5.204595 | 1.783968 | 1.497278 | 1.731733 | 1.678559 | 4 |
| 1.584827 | 0.935282 | 3.327166 | 1.94125 | 2.179968 | 0.358369 | 3.245291 | 5 |
| 0.928618 | 0.658035 | 3.076131 | 3.113168 | 2.172916 | 1.004145 | 3.430131 | 5 |
| 2.201803 | 1.135876 | 4.001561 | 1.791912 | 1.757235 | 0.255488 | 2.840382 | 5 |
| 3.807773 | 3.594538 | 1.889844 | 0.931891 | 1.714179 | -0.22761 | 0.176671 | 3 |
| 0.242025 | 1.84378 | 3.468098 | 2.711658 | 2.422419 | 0.129613 | 1.804384 | 4 |
| 2.001564 | 1.682021 | 3.01414 | 2.000518 | 1.811704 | 0.298292 | 1.451765 | 3 |
| 1.563126 | 0.95651 | 2.505286 | 2.57955 | 1.915208 | 0.43884 | 3.595415 | 5 |
| 0.166357 | 2.392899 | 3.069375 | 2.770552 | 1.708797 | 3.004771 | 0.534774 | 1 |
| 0.537015 | 2.481759 | 5.567584 | 0.735376 | 1.212872 | 0.596699 | 1.804847 | 4 |
| 1.419943 | 3.311596 | 2.146657 | 1.1977 | 1.445532 | 1.588575 | 0.49374 | 3 |
| 1.6282 | 2.717846 | 3.449848 | 2.08389 | 0.548107 | 3.320778 | 3.109258 | 2 |
| 0.74564 | 4.329717 | 3.465316 | 2.586558 | 0.874382 | 2.331343 | 0.952736 | 2 |
| 0.74504 | 4.528111 | 3.400310 | 2.300000 | 0.074302 | 2.331343 | 0.302130 | |

Document: PPD

Author: PPD


06MAY2024

1.0



| | | | | | | 1 | |
|---|---|---|---|---|---|---|---|
| -0.53777 | 2.184301 | 1.465823 | 2.443865 | 3.215783 | 3.614718 | 3.522195 | 1 |
| 0.517961 | 4.639776 | 1.693983 | 2.760274 | 1.535191 | 2.33917 | 2.777603 | 11 |
| 3.464622 | 3.305747 | 3.148404 | 1.874921 | 1.356197 | 0.483571 | 0.587682 | 3 |
| 1.831054 | 3.21794 | 1.980434 | 1.148194 | 2.693122 | 0.351515 | 2.311651 | 3 |
| 1.334201 | 2.45268 | 3.196957 | 1.766991 | 1.617076 | 0.218062 | 2.178214 | 4 |
| 1.925363 | 1.20103 | 1.434322 | 1.670427 | 2.831532 | 1.924301 | 2.443715 | 5 |
| 2.379776 | 1.265335 | 2.872741 | 2.090623 | 3.297923 | 2.679207 | 2.677931 | 5 |
| -0.50069 | 3.784005 | 2.725673 | 3.553338 | 0.042037 | 2.158042 | 2.048815 | 2 |
| 0.315685 | 2.035559 | 1.810852 | 3.164387 | 0.491681 | 3.110445 | 2.98571 | 1 |
| 1.791176 | 1.005473 | 2.139767 | 2.53269 | 1.78994 | 2.214137 | 2.723798 | 5 |
| 1.979567 | 1.748545 | 1.776153 | 2.846214 | 2.002051 | 1.003302 | 2.429969 | 5 |
| 1.853418 | 3.53585 | 3.835734 | 0.856978 | 1.400599 | 3.712702 | 2.91704 | 1 |
| 1.63315 | 1.316722 | 2.619318 | 2.937318 | 1.916679 | 1.496701 | 3.180816 | 5 |
| 1.884768 | 1.551881 | 2.123122 | 4.401792 | 3.459827 | 1.945 | 2.269949 | 5 |
| 3.020426 | 2.411129 | 2.633178 | 2.075542 | 1.667037 | 2.194526 | 2.91346 | 3 |
| 1.449371 | 3.431235 | 3.018328 | 1.125531 | 3.259058 | 1.10168 | 1.764484 | 3 |
| 0.84953 | 1.932868 | 3.02034 | 1.862252 | 3.688928 | 2.444511 | 1.698493 | 1 |
| 2.228413 | 1.91244 | 2.305406 | 2.513044 | 2.202764 | 1.670849 | 3.270545 | 5 |
| 1.208468 | 2.707595 | 4.269007 | 2.566786 | 2.451727 | 1.520423 | 1.423032 | 4 |
| 2.061931 | 1.903822 | 2.856964 | 2.327123 | 1.620568 | 0.117391 | 1.840711 | 3 |
| 0.262233 | 3.43046 | 3.196516 | 2.788729 | 2.266742 | 1.759309 | -0.00986 | 1 |
| 1.357973 | 0.780838 | 2.722596 | 2.246043 | 2.321431 | 1.691787 | 2.072079 | 5 |
| 0.114807 | 2.509803 | 2.692398 | 3.128366 | 1.181392 | 2.545597 | 1.148067 | 1 |
| 1.28309 | 0.90347 | 3.001318 | 4.109714 | 0.083325 | 2.33898 | 1.950549 | 2 |
| 0.506534 | 1.782591 | 2.399148 | 2.907124 | 2.313644 | 1.898565 | 1.305203 | 1 |
| 1.213072 | 0.529087 | 4.048949 | 2.688219 | 1.612988 | 2.403943 | 1.783422 | 5 |
| 1.313982 | 1.203218 | 2.354178 | 3.867624 | 1.752954 | 2.803632 | 0.720678 | 2 |
| 1.872386 | 0.357258 | 3.278948 | 2.103521 | 0.673257 | 2.418421 | 2.767138 | 5 |
| 0.721409 | 1.36012 | 2.099485 | 2.777914 | 1.511871 | 1.263105 | 3.078166 | 5 |
| 1.803057 | 1.579713 | 2.093822 | 2.916097 | 2.61537 | 2.381333 | 1.975054 | 5 |
| 1.511414 | 2.714801 | 2.477878 | 2.356489 | 1.608225 | 2.422306 | 1.576296 | 1 |
| 3.784065 | 1.862054 | 1.713389 | 0.213838 | 2.933285 | 1.556042 | 1.609158 | 3 |
| 1.205779 | 3.309772 | 2.478432 | 0.880979 | 1.048996 | 1.852513 | 1.572679 | 1 |
| 3.810057 | 2.116697 | 2.3975 | -0.04406 | 3.077084 | 1.416204 | 1.145462 | 3 |
| 2.507306 | 2.291566 | 2.189901 | 3.038778 | 1.571151 | 1.557165 | 1.056906 | 3 |
| 0.103926 | 2.725501 | 3.826067 | 2.194335 | 1.86495 | 2.26395 | 1.177269 | 4 |
| 0.809178 | 1.040189 | 1.730576 | 2.894496 | 3.211068 | 2.478951 | 1.698509 | 5 |
| 0.838928 | 1.784799 | 2.841608 | 0.794042 | 1.844635 | 1.75334 | 1.732254 | 4 |
| 2.569555 | 0.4746 | 3.345086 | 1.136888 | 2.120048 | 1.299826 | 1.999741 | 5 |
| 1.322061 | -0.11907 | 2.775271 | 1.95979 | 2.899401 | 1.783886 | 3.379287 | 5 |
| -0.76506 | 4.724631 | 2.893808 | 2.774245 | 2.50157 | 3.237441 | 2.484975 | 1 |
| 2.804131 | 1.719649 | 1.570869 | 1.93659 | 2.742195 | 1.139427 | 2.036416 | 3 |
| 1.205436 | 1.512286 | 3.53046 | 1.379409 | 2.993918 | 0.657272 | 2.418126 | 5 |
| 0.051672 | 0.879804 | 2.650317 | 2.384895 | 3.283675 | 1.39516 | 3.257062 | 5 |
| -0.39607 | 1.190186 | 2.649046 | 2.575062 | 2.076664 | 2.576419 | 3.426286 | 5 |
| -0.40315 | 0.425886 | 3.815744 | 3.942569 | 2.3952 | 1.989152 | 2.833274 | 5 |
| -0.07924 | 2.622817 | 4.052617 | 1.266456 | 1.17043 | 1.867025 | 1.448149 | 4 |
| -0.13567 | 2.362155 | 4.004661 | 2.462405 | 1.297833 | 2.140488 | 0.681625 | 4 |
| 0.477195 | 1.17295 | 2.913251 | 2.483704 | 2.848027 | 2.056686 | 1.758322 | 5 |
| 0.56271 | 1.616479 | 1.830526 | 2.923669 | 3.684984 | 0.849889 | 3.423473 | 5 |
| 1.579464 | 2.173769 | 2.527411 | 3.219991 | 1.767273 | 2.623521 | 2.888911 | 5 |
| 2.700568 | 1.320227 | 1.239929 | 2.207632 | 2.038575 | 1.646896 | 1.555653 | 3 |
| 2.151782 | 1.974439 | 4.213681 | 2.612496 | 2.459162 | 0.91177 | 1.399608 | 3 |
| 1.576249 | 1.452704 | 4.058938 | 2.575511 | 2.394314 | 1.063594 | 2.603736 | 5 |
| 3.780426 | 1.734454 | 3.849178 | 2.897637 | 2.083926 | 1.825276 | 1.092608 | 3 |
| 1.390327 | 2.075764 | 4.243 | 3.125061 | 1.273445 | 2.840671 | 1.859468 | 4 |
| 1.607157 | 2.968483 | 3.24849 | 2.076404 | 2.62992 | 2.696016 | 2.195731 | 1 |
| 2.569179<br>3.757162 | 2.272447 | 4.441177 | 2.249513 | 1.372362 | 2.432124 | 0.511077 | 3 |
| 3./3/102 | 1.90669 | 4.023394 | 2.056548 | 2.092316 | 0.702579 | 2.357687 | 3 |

Document: PPD

Author: Version Number:

Version Number: 1.0 Version Date: 06MAY2024



| 3.200396 | 1.822515 | 4.443242 | 2.109396 | 2.22672 | 1.391675 | 1.539029 | 3 |
|---|---|---|---|---|---|---|---|
| 2.250052 | 3.01667 | 3.066849 | 1.523405 | 2.086696 | 1.93857 | 1.362553 | 3 |
| 3.564286 | 1.622048 | 4.393762 | 2.323449 | 1.023309 | 0.742946 | 1.799375 | 3 |
| 1.820917 | 1.750117 | 4.53634 | 2.28264 | 1.228009 | 2.070476 | 1.366165 | 4 |
| 3.837824 | 3.469015 | 3.399461 | 1.508111 | 2.106133 | 0.646965 | 1.877185 | 3 |
| 3.086287 | 3.311494 | 3.384577 | 1.007094 | 2.34214 | 0.704304 | 1.716368 | 3 |
| 0.735348 | 2.431545 | 4.265286 | 3.135617 | 1.18764 | 1.246144 | 1.800427 | 4 |
| 1.061379 | 3.511977 | 3.233219 | 1.598488 | 1.538965 | 1.701663 | 1.133595 | 4 |
| 1.481552 | 3.995962 | 3.090677 | 1.705871 | 2.747919 | 0.002467 | 1.188856 | 3 |
| -0.00182 | 3.260239 | 3.669034 | 1.489115 | 1.660088 | 3.071547 | 1.895616 | 1 |
| 2.364332 | 3.423769 | 3.730801 | 0.464028 | 1.449773 | 0.034636 | 0.491184 | 3 |
| 1.790911 | 3.020807 | 2.397504 | 2.504064 | 3.159573 | 2.110374 | 2.839354 | 1 |
| 1.845525 | 2.336941 | 3.108308 | 2.925869 | 1.398286 | 1.004538 | 1.277946 | 3 |
| 3.774452 | 3.283662 | 2.601613 | 1.319941 | 3.095036 | 0.246845 | 0.737773 | 3 |
| 1.505742 | 3.82593 | 3.401152 | 2.344606 | 1.070413 | 1.189597 | 1.387092 | 4 |
| 1.612573 | 2.40045 | 3.297188 | 2.902049 | 2.074842 | 2.284885 | 2.024605 | 1 |
| 1.088512 | 2.784298 | 3.62959 | 2.500349 | 2.343832 | 3.113105 | 2.404938 | 1 |
| 1.42413 | 2.253803 | 3.343379 | 2.051898 | 2.425804 | 0.579324 | 1.473222 | 3 |
| 0.905829 | 3.986124 | 2.764364 | 2.658993 | 1.428778 | 2.003098 | 0.431219 | 2 |
| 1.778831 | 2.523333 | 3.375314 | 2.030899 | 0.692378 | 2.061231 | 0.704335 | 2 |
| 1.765234 | 2.818131 | 2.887796 | 3.433211 | 1.183735 | 2.435894 | 2.171128 | |
| 1.960731 | 4.06999 | | | | | 1.270132 | 2 |
| | 3.897983 | 4.008457<br>3.379027 | 3.39411<br>3.055913 | 0.026767<br>0.426009 | 1.542573<br>3.234069 | | |
| 0.764445 | | | | | | 0.929019 | 2 |
| 3.687367 | 1.522458 | 4.258232 | 2.500019 | 0.945134 | 1.624383 | 0.883844 | 3 |
| 2.64934 | 2.323337 | 3.874644 | 2.744603 | 1.575332 | 0.305109 | 0.525865 | 3 |
| 1.789778 | 3.038155 | 3.024023 | 3.769444 | 0.323103 | 2.528426 | 1.142301 | 2 |
| 4.672162 | 3.069382 | 3.688413 | 2.440952 | 1.405466 | 0.020889 | 1.708298 | 3 |
| 2.340334 | 2.50208 | 3.653272 | 2.672299 | 1.360596 | 1.219283 | 1.643292 | 3 |
| 1.89812 | 3.145009 | 2.649546 | 3.571723 | 1.739567 | 2.162005 | 2.432012 | 11 |
| 2.405691 | 2.557828 | 2.234228 | 3.77717 | 0.918691 | 2.055871 | 1.870516 | 2 |
| 1.991084 | 3.045781 | 3.097603 | 3.246524 | 0.560414 | 3.354772 | 2.362809 | 2 |
| 2.652284 | 2.692073 | 2.782371 | 1.637233 | 2.017997 | 0.278823 | 1.12878 | 3 |
| 2.078746 | 2.558682 | 3.375823 | 2.666212 | 0.672835 | 2.323415 | 1.714464 | 2 |
| 2.272887 | 3.299781 | 2.934946 | 3.415632 | 1.601629 | 2.553767 | 1.538921 | 2 |
| 2.174742 | 2.020834 | 3.200357 | 3.304615 | 1.962247 | 1.781806 | 1.57773 | 5 |
| 1.554845 | 3.411567 | 3.696475 | 1.814908 | 2.144365 | 0.424043 | 1.026569 | 3 |
| 2.601653 | 2.277123 | 4.083702 | 3.772831 | -0.42827 | 1.541241 | 1.480311 | 2 |
| 1.853866 | 4.368635 | 2.087155 | 1.677374 | 1.142678 | 1.287609 | 1.80835 | 3 |
| 2.681699 | 3.558978 | 3.406055 | 1.417839 | 1.343321 | 0.426572 | 0.474613 | 3 |
| 2.24989 | 0.822324 | 3.131529 | 2.802165 | 1.135157 | 0.648374 | 2.308554 | 5 |
| 2.111609 | 1.90889 | 2.584371 | 2.77702 | 1.595925 | 0.485008 | 2.907262 | 5 |
| 0.173858 | 1.347144 | 2.399445 | 2.292993 | 2.871639 | 2.099188 | 3.231836 | 5 |
| 1.546568 | 2.585044 | 3.272659 | 0.477661 | 1.807298 | 0.726058 | 1.899376 | 3 |
| 1.156342 | 1.765744 | 2.866667 | 1.718082 | 2.954764 | 1.113488 | 2.110821 | 5 |
| 1.494649 | 1.806517 | 2.856774 | 1.354115 | 2.009178 | 1.117367 | 2.192055 | 5 |
| 1.364551 | 1.615682 | 2.777178 | 1.997047 | 1.850187 | 1.154867 | 1.975221 | 5 |
| 1.412895 | 1.93883 | 2.560225 | 1.571869 | 1.177979 | 1.037155 | 1.555193 | 3 |
| 2.205521 | 1.692739 | 2.633795 | 2.812203 | 1.770763 | 1.12824 | 3.014037 | 5 |
| 0.745193 | 1.490097 | 3.379798 | 2.22975 | 2.245205 | 1.51202 | 1.55745 | 4 |
| 1.378298 | 2.662703 | 1.85831 | 1.981788 | 1.283554 | 1.282433 | 1.512774 | 1 |
| 1.884125 | 2.075508 | 2.16487 | 1.55485 | 2.294037 | 1.421776 | 2.021908 | 3 |
| 0.985738 | 2.323031 | 3.344249 | 2.186234 | 1.046613 | 1.139703 | 2.08681 | 4 |
| 1.339493 | 2.323031 | 2.640416 | 1.643363 | 1.890265 | 0.862075 | 2.452216 | 5 |
| 1.411204 | 1.768375 | 2.509155 | 2.071366 | 1.069819 | 1.270294 | | <u>5</u> |
| | | | | | | 2.138543 | |
| 1.603957 | 2.393124 | 4.600104 | 1.479665 | 0.3686 | 1.257599 | 1.671143 | 4 |
| 1.593894 | 1.808995 | 1.276598 | 2.542793 | 2.668689 | 1.234447 | 3.011351 | 5 |
| 0.437205 | 2.05325 | 2.233585 | 2.342777 | 2.863301 | 0.989024 | 3.132892 | 5 |
| 1.796248 | 1.921808 | 4.253712 | 0.987076 | 2.703099 | 0.264328 | 0.99685 | 3 |
| 1.637491 | 2.60536 | 2.78299 | 3.176663 | 3.185908 | 0.945942 | 1.681183 | 1 |

Document: PPD

Author: PPD


06MAY2024

1.0


| 0.007000 | 4 00=004 | 4.04040 | 0.407000 | 0.504000 | 4 == 4000 | 0.000004 | |
|---|---|---|---|---|---|---|---|
| 2.397302<br>2.328269 | 1.887024 | 1.91816 | 2.197268 | 2.581808<br>0.099046 | 1.771002 | 2.369984 | 5<br>2 |
| | 2.27798 | 2.125474 | 3.005204 | | 1.713398 | 1.026657 | 4 |
| 0.11416 | 2.396599 | 2.853036 | 3.178833 | 1.031306 | 1.899937 | 0.55292 | 4 |
| 0.646272 | 2.409414 | 3.949841 | 1.627033 | 1.13211 | 1.385222 | 1.246331 | |
| 1.819873 | 2.572002<br>1.199162 | 1.843449<br>2.164442 | 1.60919<br>2.545358 | 3.013846<br>2.839459 | 0.301808<br>1.856562 | 1.919204<br>2.979892 | 3 |
| 2.893933<br>1.657387 | -0.04104 | 2.817115 | | 2.252117 | 2.258384 | 3.244889 | 5<br>5 |
| 3.223918 | 1.104266 | 2.818893 | 2.885721<br>1.829432 | 1.385741 | 2.256364 | 3.350843 | 5 |
| 1.567883 | 1.69097 | 2.678636 | 3.576635 | 1.69927 | 2.373808 | 1.665361 | 5 |
| 1.444466 | 2.164448 | 3.129106 | 2.105301 | 1.025459 | 3.286115 | 2.679373 | 5 |
| 0.789237 | 2.751414 | 4.503448 | 2.279741 | 0.594937 | 1.47052 | 1.258745 | 4 |
| 1.32103 | 1.739759 | 2.91269 | 1.970637 | 1.670966 | 2.325363 | 1.734543 | 5 |
| 1.417863 | 1.565313 | 2.942052 | 2.716931 | 2.031696 | 2.665588 | 1.504992 | 5 |
| 0.105744 | 2.701506 | 3.935611 | 3.081274 | 0.140042 | 2.612532 | 1.21387 | 4 |
| 0.093926 | 1.328851 | 3.657152 | 2.021215 | 2.748042 | 1.799659 | 2.503177 | 5 |
| 2.058253 | 1.409092 | 3.385514 | 1.720862 | 1.359984 | 2.940476 | 2.368557 | 5 |
| 0.610951 | 2.617612 | 2.618744 | 2.959006 | 1.079474 | 1.703607 | 0.602328 | 2 |
| 1.620419 | 1.452286 | 3.220025 | 2.04852 | 1.620619 | 2.70717 | 2.011157 | 5 |
| 1.26425 | 2.492492 | 2.254208 | 3.149003 | 0.20461 | 2.680442 | 0.963521 | 2 |
| 0.931603 | 0.778784 | 3.816232 | 2.411449 | 1.588901 | 1.749691 | 2.903384 | 5 |
| 1.883671 | 1.958262 | 2.662179 | 2.06722 | 1.593241 | 2.260557 | 1.932458 | 5 |
| 1.616866 | 1.148898 | 3.165864 | 2.700711 | 2.133769 | 2.779107 | 2.060409 | 5 |
| 1.96896 | 1.173538 | 3.408077 | 1.916709 | 1.627131 | 2.562472 | 2.227437 | 5 |
| 0.775019 | 3.539821 | 1.948109 | 1.474039 | 1.512137 | 2.192336 | 0.356982 | 1 |
| -0.48434 | 2.801792 | 3.341801 | 1.253899 | 2.23096 | 2.792869 | 3.211511 | 1 |
| 1.735924 | 3.692729 | 4.176931 | 0.871424 | 2.20432 | -0.09871 | 1.803309 | 3 |
| 2.436967 | 2.242692 | 2.95653 | 2.42781 | 1.861757 | 1.764807 | 2.614867 | 5 |
| 1.658166 | 2.250213 | 2.272366 | 3.709927 | 2.741535 | 2.928559 | 1.376769 | 1 |
| 1.333809 | 3.28714 | 1.923658 | 2.704404 | 1.874826 | 2.942094 | 1.95615 | 1 |
| 0.304445 | 2.431619 | 3.242846 | 1.164343 | 2.616041 | 2.179615 | 2.512263 | 1 |
| 1.093769 | 2.70846 | 3.188444 | 1.452049 | 2.704276 | 2.837869 | 3.558715 | 1 |
| 0.979075 | 2.932777 | 2.236762 | 1.834613 | 3.024493 | 1.92344 | 3.156133 | 1 |
| 1.504879 | 2.118966 | 1.74156 | 1.487179 | 3.392883 | 2.680421 | 2.117358 | 1 |
| 0.235742 | 1.514871 | 2.640203 | 4.244476 | 1.9561 | 1.274938 | 3.144923 | 5 |
| 0.721346 | 2.624908 | 2.503404 | 1.783081 | 2.070988 | 2.354757 | 2.050832 | 1 |
| 1.511873 | 1.611845 | 2.686757 | 2.24819 | 2.398428 | 0.857729 | 2.340673 | 5 |
| 1.483817 | 1.742122 | 2.38017 | 2.115277 | 2.46686 | 0.885315 | 2.411145 | 5 |
| 1.412824 | 2.023799 | 2.394205 | 2.244071 | 2.566338 | 1.066282 | 1.957895 | 5 |
| 0.96656 | 1.956889 | 2.503954 | 1.889427 | 2.584678 | 0.635303 | 2.486109 | 5 |
| 1.445583 | 1.659629 | 2.820313 | 2.291001 | 1.995405 | 1.615854 | 2.326673 | 5 |
| 1.264227 | 1.559251 | 2.530892 | 2.351941 | 2.005204 | 1.908408 | 2.08316 | 5 |
| 1.300572 | 1.506208 | 2.456656 | 2.476265 | 1.930084 | 1.826288 | 2.238183 | 5 |
| 1.395494 | 2.681821 | 2.399638 | 1.861954 | 1.670527 | 2.336857 | 1.348026 | 1 |
| 1.071372 | 1.64587 | 2.335144 | 2.049403 | 2.134302 | 1.103433 | 2.192995 | 5 |
| 0.972549 | 2.213103 | 2.453235 | 1.965736 | 1.820293 | 1.210596 | 1.269824 | 1 |
| 1.492335 | 1.795098 | 2.306659 | 1.928596 | 2.03471 | 1.206811 | 2.336041 | 5 |
| 0.290952 | 2.170553 | 2.27139 | 3.121171 | 1.858355 | 1.795948 | 1.144805 | 1 |
| 1.575429 | 2.032213 | 2.465815 | 3.19347 | 1.550548 | 2.006904 | 0.837601 | 2 |
| -0.28365 | 2.768528 | 2.892846 | 2.010788 | 3.199715 | 1.111858 | 1.784 | 1 |
| 1.699107 | 1.726334 | 2.98967 | 2.659644 | 1.172693 | 1.45147 | 1.176434 | 4 |
| 2.310326 | 1.084356 | 3.212852 | 0.991361 | 2.383933 | 1.0178 | 3.223335 | 5 |
| 0.538985 | 0.684544 | 2.87213 | 3.319863 | 0.471048 | 1.146485 | 3.037455 | 5 |
| 1.320483 | 0.370392 | 2.959414 | 2.893502 | 3.208969 | 0.487022 | 2.159851 | 5 |
| 0.632746 | 0.962392 | 3.786251 | 3.674781 | 1.636723 | 0.976119 | 0.43589 | 4 |
| 1.260572 | 1.114517 | 3.471529 | 3.147704 | 2.509499 | 0.784426 | 0.739571 | 4 |
| 1.81431 | 0.908937 | 3.437827 | 3.115334 | 1.089183 | 0.8543 | 1.536967 | 5 |
| 0.480491 | 1.603937 | 3.497161 | 3.171849 | 2.858567 | 1.045461 | 0.796103 | 4 |
| 2.448276 | 0.9507 | 3.11357 | 2.242604 | 2.513886 | 1.092078 | 1.001218 | 3 |
| 1.667621 | 0.720564 | 3.065787 | 2.789554 | 2.601914 | 1.00463 | 1.646084 | 5 |

Author: PPD


06MAY2024



| 4.00540 | 0.474004 | 0.070400 | 0.00000 | 0.040400 | 0.000004 | 0.077004 | |
|---|---|---|---|---|---|---|---|
| 1.36549 | 0.471031 | 3.670106 | 2.32908 | 2.812428 | 0.692981 | 2.377931 | 5 |
| 1.782831 | 0.668699 | 4.303075 | 2.950578 | 1.196954 | 1.473613 | 2.410163 | 5 |
| 1.779422 | 1.804898 | 2.372978 | 2.236031 | 1.796164 | 1.101095 | 2.408556 | 5 |
| 0.752197 | 1.221928 | 3.601867 | 1.913002 | 2.917384 | 0.485048 | 2.184378 | 5 |
| 1.090207 | 0.371767 | 3.657906 | 3.103313 | 2.695586 | 1.088557 | 2.130409 | 5 |
| 1.449626 | 1.446819 | 4.565353 | 2.201232 | 1.589811 | 1.28579 | 1.45593 | 4 |
| 1.538993 | 0.432944 | 3.880188 | 2.973588 | 2.369882 | 1.22025 | 3.079243 | 5 |
| 1.267368 | 0.956728 | 3.771335 | 2.573059 | 2.060642 | 1.354038 | 2.111837 | 5 |
| 0.812903 | 2.100727 | 2.003404 | 2.841437 | 1.176845 | 4.042103 | 2.308406 | 11 |
| -0.12421 | 2.607063 | 2.9329 | 2.202843 | 1.640928 | 2.10373 | 2.387402 | 11 |
| 0.542068 | 2.551937 | 3.744826 | 2.376175 | 0.753738 | 3.505419 | 2.13489 | 4 |
| 0.372456 | 3.354352 | 3.712648 | 1.479283 | 0.715589 | 1.445332 | 0.635211 | 4 |
| 0.305215 | 2.289783 | 4.46517 | 2.340381 | 1.999469 | 2.164077 | 1.869376 | 4 |
| 2.755486 | 3.573517 | 3.853695 | 1.941299 | 2.051228 | 1.450862 | 2.118203 | 3 |
| 1.626729 | 2.778755 | 1.826495 | 3.451388 | 1.873129 | 3.158793 | 0.826211 | 2 |
| 0.076946 | 1.646119 | 2.222775 | 2.737351 | 1.203729 | 2.5871 | 4.468302 | 5 |
| 1.013232 | 2.162299 | 3.088201 | 2.495127 | 1.321445 | 0.938687 | 1.910282 | 4 |
| 1.20519 | -0.07545 | 2.885382 | 1.956822 | 2.266986 | 2.416183 | 3.019212 | 5 |
| 1.39817 | 1.852987 | 3.197305 | 2.136321 | 1.394049 | 0.442642 | 2.051922 | 4 |
| 0.873249 | 2.555248 | 2.54208 | 2.041056 | 2.167741 | 0.808359 | 1.213751 | 1 |
| 0.806786 | 1.256641 | 3.512638 | 2.772089 | 1.439192 | 2.428634 | 3.160887 | 5 |
| 0.026556 | 1.299047 | 2.254734 | 2.758667 | 2.102032 | 2.059072 | 2.925602 | 5 |
| -0.37456 | 1.577272 | 2.356102 | 3.532591 | 1.521418 | 2.161338 | 1.712706 | 1 |
| 0.294225 | 1.883966 | 2.915752 | 2.171537 | 1.986679 | 0.595522 | 1.150333 | 4 |
| 1.332085 | 0.698822 | 2.722347 | 3.810148 | 1.240012 | 1.953593 | 2.289551 | 5 |
| 1.531207 | 1.639334 | 2.208954 | 2.580159 | 1.424991 | 1.388167 | 2.864206 | 5 |
| 0.649526 | 1.983378 | 3.004372 | 2.763197 | 0.644957 | 1.465754 | 1.641154 | 4 |
| 1.062165 | 1.703427 | 4.137153 | 3.523577 | -0.25471 | 0.274785 | 2.414101 | 4 |
| 1.613615 | 1.567968 | 2.01006 | 2.909649 | 1.084012 | 1.64672 | 3.082602 | 5 |
| 2.611317 | 1.360381 | 2.572052 | 3.842697 | 2.318571 | 1.267588 | 1.442266 | 5 |
| 0.244814 | 0.983054 | 2.619721 | 3.328562 | 3.670014 | 1.220171 | 3.959349 | 5 |
| 0.212633 | 1.470245 | 3.736618 | 2.26854 | 3.534922 | 1.163535 | 2.752749 | 5 |
| 0.210494 | 2.000189 | 3.356024 | 2.1878 | 2.134824 | 1.09907 | 3.104368 | 5 |
| 1.926494 | 2.720868 | 1.743791 | 1.398287 | 2.173038 | 3.352568 | 2.561924 | 1 |
| 1.072198 | 3.31218 | 4.423606 | 0.480775 | 1.247225 | 1.562622 | 3.173473 | 4 |
| 1.357499 | 2.189561 | 2.255633 | 3.35382 | 1.874947 | 3.258765 | 3.437023 | 5 |
| 1.497423 | 1.962183 | 2.210324 | 1.454927 | 2.617754 | 2.249815 | 2.748368 | 5 |
| 1.704547 | 1.358564 | 2.589937 | 2.18018 | 2.343222 | 1.467078 | 3.609101 | 5 |
| 1.339563 | 2.526236 | 2.490679 | 1.016699 | 2.780961 | 2.661584 | 2.361953 | 1 |
| 2.328581 | 2.394616 | 2.552002 | 1.14282 | 2.842293 | 0.484683 | 4.308226 | 5 |
| 1.85317 | 1.934251 | 3.869415 | 0.499016 | 2.363052 | 1.674276 | 1.029997 | 3 |
| 1.45469 | 2.190708 | 3.760847 | 1.722148 | 1.768372 | 3.116628 | 3.478788 | 5 |
| 3.470967 | 3.439438 | 3.360445 | 0.721942 | -0.20575 | -0.06164 | 0.009922 | 3 |
| 1.296298 | 2.090994 | 1.963986 | 3.324418 | 1.359161 | 1.950194 | 4.18974 | 5 |
| 0.814951 | 2.698575 | 2.986318 | 0.932067 | 2.782515 | 1.42676 | 0.998865 | 1 |
| 0.701812 | 2.816236 | 4.503632 | 3.118434 | 1.809571 | 2.136325 | 1.220668 | <u> </u> |
| -0.10962 | 4.748057 | 1.311358 | 3.02705 | 1.085849 | 3.705541 | 2.662043 | 1 |
| 1.458165 | 3.619007 | 2.461477 | 1.602822 | 1.411744 | 2.264779 | 2.547659 | 1 |
| 0.800917 | 4.262438 | 2.544643 | 2.894222 | 0.613533 | 3.956862 | 1.671726 | 2 |
| 0.717591 | 4.02109 | 1.879332 | 2.441721 | 1.49057 | 2.877834 | 0.429284 | 2 |
| 0.643691 | 3.855714 | 1.005858 | 3.175629 | 0.103246 | 3.558945 | 0.795806 | 2 |
| 0.460533 | 3.698006 | 2.572437 | 2.387381 | 2.850441 | 2.808884 | 3.094858 | 1 |
| 4.04329 | 2.578201 | 0.799226 | 1.244423 | 1.632081 | 1.311067 | 1.735986 | 3 |
| 1.774165 | 4.058947 | 4.405546 | 1.785724 | 2.283782 | 0.758058 | 0.79129 | 3 |
| 2.724334 | 4.789961 | 1.917886 | 3.663023 | 0.860011 | 2.905804 | -0.22034 | 2 |
| 1.890045 | 3.070056 | 2.121002 | 2.630324 | 1.471761 | 1.45338 | 1.399154 | 2 |
| | | | | 2.39835 | 0.483349 | | |
| 1.179053 | 2.241616 | 2.464325 | 1.743874 | | 0.483349 | 2.739105 | 5 |
| 0.910327 | 1.109921 | 3.392557 | 1.840023 | 3.649984 | | 2.727363 | 5 |
| -0.76467 | 2.630535 | 4.08284 | 1.372603 | 1.512798 | 2.614801 | 1.87896 | 4 |

Author: Version Number:

Version Number: 1.0 Version Date: 06MAY2024



| 0.018361 | 2.910309 | 2.608297 | 1.602254 | 2.228515 | -0.1038 | 2.327382 | 4 |
|---|---|---|---|---|---|---|---|
| 2.31223 | 2.140411 | 3.730239 | 2.46278 | 1.824992 | 1.428426 | 2.476548 | 3 |
| 2.000375 | 2.189982 | 3.724534 | 2.161509 | 1.635054 | 1.57342 | 0.200782 | 3 |
| 3.566437 | 0.913912 | 4.240227 | 1.9238 | 2.017575 | 2.399885 | 0.391107 | 3 |
| 1.62852 | 1.018615 | 3.425307 | 2.069394 | 2.752738 | 2.893608 | 1.471069 | 5 |
| 2.456128 | 1.924375 | 4.611679 | 1.543373 | 2.675139 | 1.215867 | 0.819487 | 3 |
| 2.955322 | 1.138264 | 3.747873 | 1.707216 | 2.573102 | 0.483788 | 0.805569 | 3 |
| 2.62885 | 1.755127 | 3.044607 | 2.3257 | 3.162495 | 2.415337 | 1.155672 | 3 |
| 2.310367 | 1.524535 | 3.543808 | 2.150572 | 2.369389 | 2.057397 | 0.899822 | 3 |
| 2.827557 | 1.951977 | 3.069947 | 1.919696 | 2.682531 | 1.73087 | 1.301477 | 3 |
| 2.354338 | 1.852527 | 4.186875 | 2.762147 | 2.727398 | 1.526546 | 1.348267 | 3 |
| 3.133866 | 1.126868 | 3.578091 | 2.250377 | 2.22218 | 0.989612 | 2.052883 | 3 |
| 3.902417 | 1.344091 | 2.9635 | 2.392058 | 2.238225 | 1.139263 | 1.925944 | 3 |
| 4.044799 | 2.560889 | 2.663006 | 2.169593 | 0.901192 | 1.77012 | 1.96679 | 3 |
| 4.155056 | 3.609037 | 2.424906 | 2.437343 | 0.670008 | 2.751403 | 1.023351 | 2 |
| 3.229569 | 3.060956 | 1.07279 | 2.674057 | 0.661189 | 2.715768 | 2.115442 | 2 |
| 2.921269 | 3.279488 | 2.066332 | 2.23657 | 1.842327 | 2.123827 | 1.809801 | 3 |
| 3.044779 | 4.07456 | 3.89887 | 1.460329 | 1.288036 | 0.384507 | 1.178261 | 3 |
| 2.740083 | 1.644629 | 2.55435 | 3.62446 | 1.955832 | 2.066756 | 0.815177 | 2 |
| 3.672096 | 3.42332 | 1.365735 | 3.932623 | 0.190274 | 3.855517 | 0.758265 | 2 |
| 3.179953 | 3.568001 | 2.620359 | 2.696917 | -0.87467 | 3.369777 | 0.541363 | 2 |
| 2.519518 | 3.268074 | 3.607177 | 2.930387 | 1.07823 | 3.237732 | 2.437606 | 2 |
| 2.225039 | 3.775535 | 1.123748 | 3.689868 | 1.819697 | 3.939923 | 2.586388 | 2 |
| 3.709609 | 3.536046 | 2.146801 | 3.13129 | 1.525033 | 3.051844 | 1.077151 | 2 |
| 3.922836 | 3.537094 | 2.352621 | 3.817752 | 0.344085 | 3.99746 | 1.601192 | 2 |
| 2.559641 | 4.363924 | 3.081225 | 3.940225 | 1.04974 | 4.147581 | 1.955423 | 2 |
| 2.506535 | 3.511332 | 2.686218 | 2.671171 | 0.351229 | 3.135231 | 1.534423 | 2 |
| | 4.140873 | 2.759899 | 3.567679 | 0.327898 | 3.496142 | 1.915584 | 2 |
| 3.611068 | 4.030347 | 2.759699 | 1.898102 | 0.623562 | | 0.318056 | |
| 5.041109 | | 2.811553 | | 0.623562 | 2.481326<br>2.530565 | 0.318056 | <u>3</u> |
| 3.987555<br>3.206587 | 3.862457<br>3.376827 | | 2.815862<br>3.04708 | 0.253199 | 3.026795 | 1.442369 | 2 |
| 2.687183 | | 1.547706 | | | | | |
| | 3.33638 | 2.737193 | 3.16023 | 0.407868 | 1.803257 | 1.018576 | 2 |
| 4.22479 | 4.024705 | 2.715407 | 2.974781 | 0.622469 | 2.100873 | 0.07855 | 2 |
| 3.485571 | 4.124516 | 1.799485 | 1.550554 | 0.865302 | 2.835845 | 0.512219 | 2 |
| 3.689093 | 2.992012 | 2.750544 | 2.126705 | 0.951029 | 1.841686 | 1.154485 | 3 |
| 1.507022 | 1.700048 | 3.643006 | 1.920586 | 1.721019 | 1.670477 | 0.88364 | 4 |
| 2.276998 | 1.872161 | 3.071937 | 1.551547 | 1.758093 | 1.456656 | 3.036033 | 5 |
| 1.722543 | 1.742988 | 3.195897 | 1.77644 | 1.623838 | 1.707611 | 1.691541 | 3 |
| 2.065441 | 1.855082 | 2.560649 | 1.429018 | 1.677676 | 1.63554 | 1.462513 | 3 |
| 1.74568 | 2.356083 | 3.455882 | 1.940336 | 1.498636 | 1.462326 | 1.919923 | 3 |
| 0.158772 | 2.513544 | 4.247838 | 2.551583 | 1.045512 | 1.299605 | 1.587535 | 4 |
| 1.80119 | 2.071641 | 4.041234 | 1.902576 | 1.296598 | 1.057213 | 0.731661 | 4 |
| 2.215429 | 2.553712 | 3.092798 | 1.870086 | 2.016486 | 1.713556 | 1.211197 | 3 |
| 2.561767 | 1.359762 | 3.215666 | 1.723347 | 2.649111 | 1.506876 | 1.212116 | 3 |
| 2.008407 | 2.326931 | 2.699744 | 1.797094 | 2.059043 | 1.621615 | 1.595778 | 3 |
| 2.063938 | 2.29876 | 3.576087 | 1.683763 | 1.536197 | 1.5092 | 1.604547 | 3 |
| 1.870314 | 3.05033 | 2.832324 | 1.120539 | 1.534361 | 0.937647 | 1.53327 | 3 |
| 1.545386 | 2.699153 | 2.90158 | 1.987278 | 1.572393 | 0.979358 | 2.326712 | 3 |
| 1.459833 | 2.793298 | 2.536495 | 1.525111 | 1.671519 | 1.382715 | 1.130589 | 3 |
| 2.883239 | 1.229672 | 3.978406 | 2.649253 | 1.311891 | 0.28695 | 1.875801 | 3 |
| 3.555512 | 0.756289 | 4.859439 | 2.591224 | -0.00136 | 1.007842 | 1.233879 | 3 |
| 0.508175 | 3.178791 | 4.788698 | 1.290105 | -0.27008 | 1.16648 | 1.256636 | 4 |
| -0.43375 | 2.490532 | 4.749263 | 2.352686 | -0.37615 | 2.187117 | 0.105813 | 4 |
| 3.964904 | 4.089137 | 4.415442 | 3.244999 | -1.16908 | 1.236213 | -0.05455 | 2 |
| 2.359152 | 2.995853 | 2.391476 | 2.378635 | 0.185879 | 0.813561 | 0.190325 | 2 |
| 1.015333 | 3.244709 | 3.91884 | 1.170988 | -0.83935 | 0.70902 | 1.389022 | 4 |
| -0.1317 | 3.371376 | 2.410057 | 3.437201 | 0.297436 | 2.487018 | 0.199548 | 2 |
| | | | | | 2.158269 | 1.332632 | 4 |
| 1.47955 | 1.064245 | 4.922544 | 1.301369 | 0.974274 | 2.130209 | 1.332032 | 4 |

Author: PPD


06MAY2024



| 1.978596 | 2.050605 | 4.222893 | 1.545038 | 2.620691 | 1.180971 | 2.380491 | 3 |
|---|---|---|---|---|---|---|---|
| 1.621695 | 1.681869 | 2.94142 | 2.467838 | -0.34802 | 1.869441 | 0.368981 | 2 |
| 1.218523 | 1.811689 | 4.994002 | 2.11 | -0.69899 | 2.880036 | 1.550563 | 4 |
| 2.064395 | 1.173791 | 3.932134 | 2.708803 | 1.250605 | 1.115845 | 0.557882 | 4 |
| 0.532071 | 1.356335 | 3.948873 | 2.254287 | 2.468433 | 1.466865 | 1.992075 | 4 |
| 1.429912 | 3.253482 | 2.093267 | 3.097008 | 2.026439 | 2.325492 | 1.059837 | 1 |
| 1.462999 | 2.915668 | 2.516664 | 3.674496 | 3.004662 | 1.589824 | 0.748062 | 1 |
| 0.733537 | 2.892451 | 2.643295 | 3.09355 | 3.151582 | 1.65196 | 1.337782 | 1 |
| 0.791875 | 2.884693 | 2.779237 | 3.413417 | 2.44907 | 2.601256 | 1.424172 | 1 |
| -0.10517 | 3.040316 | 3.360112 | 2.855718 | 2.873678 | 1.188593 | 0.322964 | 1 |
| 0.875719 | 2.924053 | 3.610616 | 2.741726 | 2.132826 | 1.585964 | 0.493479 | 4 |
| 2.176518 | 4.067647 | 1.934115 | 2.559868 | 2.254118 | 2.083677 | 1.380008 | 1 |
| -0.17358 | 3.503438 | 2.423085 | 3.051185 | 2.147663 | 1.953754 | 2.706169 | 1 |
| 1.679471 | 2.53749 | 2.705387 | 2.011349 | 3.219434 | 1.704823 | 2.592947 | 5 |
| -0.62134 | 3.307752 | 3.073545 | 2.275577 | 1.186566 | 2.329074 | 1.121935 | 1 |
| -0.58953 | 4.10793 | 2.459029 | 3.07827 | 1.627415 | 1.960017 | 0.474559 | 1 |
| -0.4566 | 3.748106 | 2.48163 | 1.703436 | 2.031344 | 2.439934 | 2.085523 | 1 |
| -0.40305 | 4.629888 | 1.803605 | 2.719529 | 0.109098 | 2.449213 | 0.376085 | 2 |
| -0.13362 | 3.298538 | 2.094871 | 2.657361 | 2.068097 | 2.119957 | 1.46328 | 1 |
| 1.051681 | 3.044125 | 1.860595 | 2.414682 | 1.750706 | 2.127842 | 0.624443 | 1 |
| -0.46756 | 3.672684 | 2.609306 | 2.798242 | 2.727397 | 2.08414 | 1.927971 | 1 |
| -0.22257 | 3.403974 | 3.992026 | 1.594233 | 0.951226 | 1.79945 | 1.564202 | 4 |
| 0.879599 | 2.559537 | 2.682985 | 2.436528 | 1.732751 | 1.685048 | 0.478358 | 1 |
| 2.068797 | 4.083433 | 2.641366 | 3.421411 | 2.299622 | 2.077696 | 0.331541 | 2 |
| 3.216228 | 3.0991 | 2.141928 | 3.095791 | 1.858518 | 2.550298 | 0.088065 | 2 |
| 3.29187 | 3.301854 | 1.867055 | 2.807832 | 2.601268 | 1.726811 | 0.402809 | 3 |
| 3.144054 | 3.6932 | 1.424622 | 1.494059 | 2.486708 | 2.370872 | 0.574533 | 3 |
| 2.457114 | 2.686718 | 2.077536 | 2.537355 | 2.735416 | 1.764817 | 0.329161 | 3 |
| 1.390182 | 3.449505 | 1.922259 | 2.738923 | 2.591671 | 0.9854 | 1.00846 | 1 |
| 2.120156 | 2.579095 | 2.882224 | 2.725341 | 2.006488 | 1.055209 | 0.117931 | 3 |
| 1.970891 | 3.700663 | 1.468186 | 1.396667 | 1.40279 | 2.8171 | 2.009906 | 1 |
| 2.336216 | 3.764322 | 2.473572 | 2.329863 | 2.576363 | 1.084098 | 1.365232 | 3 |
| -0.10381 | 3.389959 | 2.547536 | 3.543453 | 2.283116 | 2.61914 | 1.589867 | 1 |
| 1.530012 | 3.427078 | 3.194501 | 2.701941 | 1.67882 | 0.968439 | 1.025129 | 4 |
| 0.857718 | 3.392356 | 0.472536 | 3.279675 | 2.230862 | 2.233642 | 1.218844 | 1 |
| 1.505968 | 2.621823 | 1.743091 | 2.215408 | 1.95822 | 2.639966 | 2.912557 | 1 |
| 0.725015 | 3.984839 | 1.182635 | 3.701695 | 1.594431 | 2.084002 | 1.741048 | 1 |
| 1.473229 | 3.459439 | 1.638031 | 3.406329 | 1.333691 | 1.702277 | 0.560334 | 2 |
| 1.060838 | 4.181436 | 2.247993 | 3.323963 | 1.172574 | 1.898132 | 0.339313 | 2 |
| 2.990401 | 2.281804 | 3.070215 | 3.687298 | -0.31184 | 1.27937 | 0.285347 | 2 |
| 0.769166 | 3.840194 | 2.731756 | 3.841705 | 1.747542 | 2.137993 | 1.252245 | 1 |
| 0.75415 | 3.558579 | 3.263125 | 2.647108 | 1.429326 | 2.333785 | 1.492619 | 1 |
| 1.303379 | 3.795161 | 1.530871 | 3.377136 | 2.072449 | 1.99248 | 1.083788 | 1 |
| 0.524407 | 3.859915 | 0.853766 | 3.074975 | 2.435645 | 3.317072 | 2.826819 | 1 |
| 0.12645 | 3.785307 | 2.629406 | 3.674972 | 1.265829 | 3.524083 | 1.271341 | 2 |
| 0.343963 | 3.983414 | 2.502811 | 1.906588 | 1.645706 | 0.417935 | 0.845107 | 1 |
| 1.710316 | 3.076969 | 2.060937 | 1.610017 | 1.059669 | 2.128205 | 0.703361 | 2 |
| 0.417446 | 3.648473 | 1.424328 | 3.711073 | 2.197958 | 3.114104 | 3.181453 | 1 |
| 2.04927 | 3.750571 | 1.462268 | 2.262071 | 2.189925 | 2.108657 | 0.792803 | 1 |
| 0.69803 | 2.205002 | 2.111445 | 2.568238 | 1.649992 | 2.488567 | 2.237445 | 1 |
| 0.951935 | 2.583197 | 3.095091 | 1.735256 | 2.707042 | 2.199157 | 0.645377 | 1 |
| 1.068594 | 2.818606 | 1.152625 | 2.573538 | 1.774493 | 3.034217 | 1.334008 | 1 |
| 1.308397 | 2.569901 | 3.080408 | 2.525086 | 2.007064 | 1.700561 | 0.976378 | 1 |
| 1.712708 | 2.433669 | 2.691373 | 2.580652 | 1.52399 | 1.378826 | 1.194658 | 3 |
| 0.91916 | 2.37196 | 2.775352 | 2.330603 | 1.599222 | 2.702074 | 0.89072 | 1 |
| 0.817149 | 3.12306 | 2.784622 | 2.661203 | 1.768797 | 1.560057 | 1.036902 | 1 |
| 0.791967 | 2.595179 | 1.847499 | 3.263682 | 2.414274 | 2.375985 | 1.818882 | 1 |
| 0.849967 | 2.071186 | 2.320527 | 2.101878 | 1.589166 | 3.016033 | 2.319835 | 1 |
| 1.60647 | 1.993996 | 2.891402 | 2.562998 | 2.438122 | 2.625546 | 1.083263 | 1 |
| | | - | | | | | |

Author: PPD


06MAY2024



| 0.040000 | 0.075000 | 0.000004 | 0.700400 | 4.040004 | 0.400050 | 0.400400 | |
|---|---|---|---|---|---|---|---|
| 0.942826 | 2.975032 | 2.008094 | 2.730432 | 1.613834 | 2.493358 | 0.169133 | 2 |
| 1.07511 | 2.919006 | 2.379194 | 3.328983 | 1.773508 | 2.139629 | 0.766729 | 2 |
| 1.325045 | 2.690406 | 2.595724 | 1.726559 | 2.106144 | 2.474342 | 0.974182 | 1 |
| 1.411178 | 2.448139 | 2.713626 | 1.825376 | 2.091093 | 2.512333 | 0.987373 | 1 |
| 1.433908 | 3.131516 | 2.788815 | 2.250392 | 0.990708 | 2.570261 | 0.605752 | 2 |
| 0.880346 | 2.425598 | 2.678058 | 1.88785 | 2.024216 | 2.640519 | 1.366953 | 1 |
| 0.260364 | 2.906487 | 2.683074 | 2.969851 | 2.87145 | 1.602331 | 0.491496 | 1 |
| 0.423654 | 3.974504 | 2.400218 | 2.156817 | 1.89691 | 1.267873 | 0.473422 | 11 |
| 0.427651 | 3.447316 | 3.1171 | 2.700789 | 0.708482 | 1.333679 | 0.149171 | 4 |
| 0.579635 | 3.585689 | 2.21721 | 2.667774 | 2.940801 | 2.46273 | 0.537045 | 1 |
| -0.02029 | 3.840243 | 2.522009 | 2.530284 | 1.500204 | 2.86294 | 0.081363 | 1 |
| -0.06372 | 4.230166 | 3.597157 | 1.843047 | 0.983072 | 1.515249 | -0.07676 | 4 |
| -0.26029 | 3.873231 | 3.083164 | 2.437457 | 1.954143 | 1.404252 | 0.414916 | 1 |
| -0.09942 | 2.776442 | 2.750918 | 2.707537 | 3.145203 | 1.570567 | 0.377695 | 1 |
| 0.275255 | 2.768954 | 4.02854 | 3.181462 | 2.991128 | 2.109993 | 1.402953 | 1 |
| 0.113402 | 2.605435 | 3.763227 | 2.119889 | 2.826393 | 0.865589 | 0.907433 | 4 |
| 0.149213 | 2.508363 | 3.846134 | 2.298856 | 2.899768 | 0.618085 | 1.543748 | 4 |
| 0.340557 | 2.541882 | 3.976928 | 2.681444 | 2.89268 | 1.145417 | 2.776941 | 5 |
| -0.22202 | 2.844312 | 3.663467 | 3.049983 | 2.78542 | 0.617824 | 1.919961 | 4 |
| -0.42178 | 2.192275 | 3.690923 | 2.891726 | 2.728776 | 1.202586 | 1.759638 | 4 |
| 0.457553 | 2.492178 | 3.576297 | 2.309842 | 2.744103 | 1.488316 | 0.765272 | 4 |
| -0.07661 | 2.609934 | 2.688168 | 3.119072 | 3.314492 | 1.011728 | 2.009197 | 1 |
| -0.30624 | 2.770384 | 3.647785 | 2.925661 | 2.651414 | 1.323014 | 1.751405 | 4 |
| 0.140752 | 2.594201 | 3.258795 | 3.069871 | 3.47017 | 0.903461 | 0.651931 | 1 |
| 1.494952 | 2.999964 | 2.300849 | 1.995311 | 1.425531 | 2.775196 | 1.773108 | 1 |
| 1.41039 | 2.949323 | 2.387595 | 1.69254 | 2.185164 | 2.487053 | 1.731274 | 1 |
| 1.118924 | 2.488969 | 3.415318 | 2.801899 | 2.178712 | 2.20894 | 1.709332 | 1 |
| 0.680572 | 3.258869 | 2.936039 | 1.918446 | 2.464094 | 2.07186 | 1.309618 | 1 |
| 1.141929 | 3.06936 | 2.624611 | 2.402971 | 2.363638 | 2.640456 | 1.426466 | 1 |
| 0.746483 | 3.534708 | 3.054122 | 2.286824 | 2.79205 | 2.205442 | 1.267024 | 1 |
| 1.011091 | 3.031657 | 2.571288 | 2.223547 | 2.575557 | 2.478644 | 1.656454 | 1 |
| 1.40917 | 2.33553 | 2.061849 | 1.689985 | 1.99935 | 1.701782 | 1.404149 | 1 |
| 0.768691 | 3.058953 | 2.917657 | 1.717871 | 2.803346 | 1.933463 | 1.826406 | 1 |
| 0.623259 | 3.10424 | 3.355942 | 1.998985 | 2.639103 | 2.307023 | 1.329493 | 1 |
| 1.357966 | 3.236041 | 1.628006 | 1.779124 | 2.009948 | 2.126546 | 2.923375 | 1 |
| 2.07341 | 2.95349 | 2.752977 | 0.969581 | 1.431418 | 1.74605 | 0.802422 | 3 |
| 0.792031 | 2.649246 | 3.21402 | 2.835091 | 2.391127 | 1.799076 | 1.483771 | 1 |
| 0.858457 | 3.130532 | | 2.654074 | 2.640759 | 1.527418 | 0.322885 | 1 |
| 0.80738 | 2.732501 | 3.015193<br>1.65259 | 2.665072 | 1.627335 | 2.728416 | 2.013305 | <u> </u> |
| | 3.110723 | | 2.698361 | 2.430201 | 1.879455 | 2.229385 | 1 |
| 2.121461<br>1.359222 | 3.174655 | 1.16904<br>1.435069 | 2.530789 | 2.244504 | 2.450394 | 2.229365 | <u> </u> |
| | | 2.997585 | 3.838252 | 1.685823 | 1.335476 | 0.356832 | 2 |
| 0.801118 | 3.074178 | | | | | | |
| 0.080879 | 2.361793 | 4.274073 | 3.686526 | 2.221517 | 1.268115 | 0.479096 | 4 |
| -0.17235 | 2.88178 | 4.48302 | 3.728202 | 1.719875 | 1.135475 | 0.350021 | 4 |
| 1.761006 | 2.297744 | 2.459649 | 3.053792 | 1.618949 | 1.878463 | 0.104232 | 2 |
| 0.216599 | 2.173008 | 3.770535 | 2.930397 | 2.304761 | 1.358994 | 0.372433 | 4 |
| 0.269085 | 2.048156 | 4.424645 | 2.43455 | 2.333657 | 0.970885 | 0.469465 | 4 |
| 0.065369 | 2.640117 | 2.597345 | 2.581476 | 2.209659 | 2.753815 | 1.558239 | 1 |
| 0.345163 | 2.569093 | 3.249664 | 3.07534 | 2.493951 | 1.078831 | 0.499263 | 4 |
| 0.052513 | 2.518404 | 3.110811 | 3.134081 | 3.319594 | 0.871954 | 0.68042 | 1 |
| 0.30771 | 3.104776 | 3.560694 | 3.132041 | 2.383767 | 0.800719 | 0.482138 | 4 |
| 1.154284 | 3.557102 | 1.593781 | 2.129454 | 2.591031 | 2.608611 | 1.732789 | 1 |
| 3.548581 | 3.065902 | 3.364989 | 2.870269 | -0.19792 | 0.576981 | 0.807048 | 3 |
| 1.265666 | 2.865337 | 3.30641 | 1.610438 | 0.737536 | 0.923749 | 1.090937 | 4 |
| 1.399631 | 3.450565 | 3.602698 | 2.993068 | 1.321121 | 3.436824 | 2.859307 | 2 |
| 2.071889 | 4.124985 | 2.273219 | 3.721401 | 1.332661 | 2.351524 | 0.687626 | 2 |
| 0.876012 | 3.10726 | 5.157052 | 2.502289 | 1.431415 | 0.674595 | 1.330972 | 4 |
| 2.349308 | 2.583863 | 1.776008 | 3.662912 | 2.041628 | 1.749898 | 2.531925 | 5 |
| 2.0.0000 | | | | | | | 3 |

Document: PPD

Author: PPD


06MAY2024

| 0.007407 | 0.050500 | 0.404470 | 0.407007 | 4.000040 | 0.755400 | 4.050005 | 0 |
|---|---|---|---|---|---|---|---|
| 2.987487 | 2.852596 | 2.434173 | 2.467237 | 1.838249 | 2.755136 | 1.358205 | 2 |
| 0.81905 | 1.825397 | 3.348165 | 4.522798 | 1.350309 | 1.59561 | 1.848665 | 5 |
| 1.774038 | 2.862877 | 2.685874 | 2.435596 | 2.107649 | 1.280506 | 0.910797 | 3 |
| 2.471096 | 2.604342 | 2.691034 | 2.817636 | 1.91936 | 2.006992 | 1.160133 | 3 |
| 3.060003 | 2.389687 | 3.987338 | 3.677606 | 1.309749 | 0.365417 | 0.614433 | 3 |
| 3.262966 | 3.396536 | 4.41932 | 0.726091 | 2.244941 | 0.726714 | 0.128801 | 3 |
| 2.494411 | 3.012345 | 4.550361 | 1.22457 | 1.950454 | 1.090167 | 0.322092 | 3 |
| 2.079433 | 2.14239 | 3.469334 | 1.070271 | 2.489137 | 1.932302 | 0.438562 | 3 |
| 2.268403 | 1.873654 | 4.282994 | 1.313821 | 1.418581 | 2.464574 | 0.276199 | 3 |
| 3.08802 | 1.748826 | 4.565023 | -0.33519 | 2.055988 | 2.092309 | 0.217988 | 3 |
| 2.777448 | 1.078595 | 4.10723 | 2.455113 | 1.397793 | 2.134951 | 0.741937 | 3 |
| 3.102757 | 1.592921 | 3.055213 | 1.054164 | 2.005069 | 1.878598 | 0.214148 | 3 |
| 3.479759 | 1.33687 | 3.174094 | 1.2196 | 2.175686 | 2.51985 | -0.06827 | 3 |
| 0.623457 | 2.841408 | 1.295385 | 3.855206 | 2.838636 | 3.356909 | 2.354045 | 1 |
| 1.847572 | 3.354191 | 3.861348 | 3.103105 | 0.405502 | 2.467452 | 1.557334 | 2 |
| 2.32006 | 2.266582 | 2.220428 | 2.264085 | 0.940936 | 1.327739 | 1.041959 | 3 |
| 2.959903 | 2.952272 | 3.331057 | 3.012319 | 0.19202 | 1.653348 | 0.098445 | 2 |
| 1.703666 | 4.825642 | 2.81377 | -0.18771 | 1.279538 | 0.122421 | 0.405711 | 3 |
| 0.475181 | 2.03538 | 3.124756 | 3.793217 | 2.522743 | 3.14862 | 3.03574 | 5 |
| 2.204704 | 4.680761 | 3.398592 | -0.06387 | 1.459862 | 0.056371 | 0.729264 | 3 |
| 2.002607 | 2.755353 | 3.376209 | 0.036351 | 1.407113 | 0.555023 | 2.247859 | 3 |
| 0.907119 | 1.708706 | 4.912416 | 2.140988 | 1.922985 | 2.28953 | 1.116472 | 4 |
| 1.825809 | 2.128214 | 4.741464 | 0.159796 | 1.636236 | 2.063124 | 0.352333 | 3 |
| 0.153648 | 2.889437 | 2.800667 | 0.352795 | 2.08095 | 2.082555 | 1.234468 | 1 |
| 0.587994 | 3.861874 | 2.269366 | 1.68284 | 1.605637 | 1.89417 | 0.802835 | 1 |
| 1.024508 | 3.664618 | 2.874202 | 0.661802 | 1.556209 | 1.204374 | 0.130695 | 3 |
| 0.283041 | 3.817617 | 2.288075 | 1.913851 | 1.877978 | 1.808863 | 1.815715 | 1 |
| 0.311823 | 3.273917 | 2.51415 | 3.816218 | 1.458316 | 2.762033 | 2.043699 | 1 |
| 0.718942 | 4.25634 | 4.459668 | 2.072599 | 1.638075 | 0.100716 | 1.716839 | 4 |
| 0.008545 | 2.195237 | 3.234108 | 2.99666 | 2.548574 | 1.681762 | 2.171549 | 1 |
| -0.47133 | 4.246083 | 1.528641 | 2.336485 | 0.732913 | 3.646783 | -0.41321 | 2 |
| 1.077048 | 4.530622 | 3.141172 | 1.851634 | 0.845131 | 1.322201 | -0.08585 | 2 |
| 1.705065 | 3.239689 | 4.050878 | 1.401745 | 0.04819 | 0.238856 | 0.758254 | 4 |
| 2.025447 | 3.033307 | 2.675933 | 2.113983 | 1.52901 | 0.942658 | 2.129124 | 3 |
| 0.244751 | 4.092002 | 3.424906 | 1.330836 | 2.236125 | 0.876376 | 0.474374 | 4 |
| 0.151119 | 2.98758 | 3.568751 | 1.451563 | 1.656526 | 1.805595 | 1.468168 | 4 |
| -0.24368 | 2.750309 | 3.5265 | 1.860395 | 1.715834 | 0.987104 | 1.895436 | 4 |
| 2.648074 | 3.621529 | 3.486606 | 2.933279 | 0.373718 | 2.709986 | -0.22809 | 2 |
| 2.066586 | 3.066316 | 3.580333 | 2.246909 | 1.180946 | 1.055538 | 0.656804 | 3 |
| 1.944425 | 1.998555 | 3.567294 | 2.594938 | 1.536046 | 2.975502 | 0.613735 | 2 |
| 1.121274 | 2.724664 | 2.638417 | 2.486761 | 2.431015 | 2.384841 | 1.565011 | 1 |
| 2.850815 | 1.654452 | 3.992092 | 2.263066 | 2.418238 | 1.276869 | 1.221492 | 3 |
| 0.684173 | 2.59755 | 4.093945 | 1.046064 | 3.083327 | 0.362483 | 1.38296 | 4 |
| 0.174206 | 3.493588 | 3.316332 | 1.816635 | 2.951768 | 0.969128 | 0.733653 | 1 |
| 1.860815 | 1.680196 | 2.476973 | 1.941281 | 1.753742 | 1.344025 | 1.426395 | 3 |
| 1.752092 | 2.024168 | 2.66644 | 1.898802 | 1.6596 | 1.209577 | 1.477241 | 3 |
| 1.321311 | 2.063387 | 2.163432 | 2.908879 | 1.330973 | 1.88362 | 2.361532 | 5 |
| 1.647948 | 2.270076 | 1.86041 | 1.867999 | 1.454386 | 1.969179 | 2.568774 | 5 |
| 1.325019 | 2.361829 | 1.478412 | 2.266887 | 1.764518 | 2.642484 | 1.702186 | 1 |
| 1.088055 | 2.85659 | 2.246922 | 2.880238 | 1.555623 | 1.051089 | 1.817443 | 1 |
| 1.062752 | 2.864692 | 2.06805 | 2.854408 | 1.648133 | 1.414439 | 1.940907 | 1 |
| 1.898748 | 2.937805 | 2.14582 | 2.108399 | 1.533958 | 0.926171 | 1.734107 | 3 |
| 1.164505 | 3.039528 | 2.132053 | 2.855484 | 1.416871 | 1.0435 | 2.152127 | 1 |
| 1.217726 | 2.459069 | 2.369937 | 2.894859 | 1.596448 | 1.29165 | 1.294127 | 1 |
| 1.205169 | 2.99523 | 2.238958 | 2.69529 | 1.1099 | 1.645469 | 0.920897 | 2 |
| 2.247636 | 1.559871 | 2.359851 | 2.345988 | 0.75245 | 2.326831 | 2.011774 | 2 |
| 0.515809 | 3.209018 | 2.974778 | 0.088037 | 0.354395 | 2.184264 | 0.377669 | 4 |
| 2.664913 | 2.258446 | 2.453266 | 2.835131 | 0.94236 | 1.093029 | 1.450462 | 3 |
| 2.332702 | 2.904314 | 2.102263 | 3.80914 | 4.423846 | 2.545838 | 2.19781 | 1 |
| 2.002102 | 2.004014 | ۷. ۱۷۷۷۷ | 5.00314 | 7.720040 | 2.040000 | 2.18101 | I |

Document: PPD

Author: PPD

Version Number: Version Date: 1.0 06MAY2024



| 0.858277 | 2.789032 | 2.675953 | 3.975471 | 2.940192 | 3.199923 | 1.756495 | 1 |
|---|---|---|---|---|---|---|---|
| 0.135326 | 3.130819 | 1.787072 | 3.322858 | 3.569177 | 3.067827 | 1.901571 | 1 |
| 0.210271 | 2.715819 | 3.337833 | 3.945324 | 2.118081 | 3.089931 | 2.290278 | 1 |
| -0.10692 | 3.305084 | 3.883783 | 3.738765 | 2.271649 | 1.095572 | 2.372052 | 4 |
| 2.940514 | 2.045527 | 1.655645 | 3.337987 | 2.325931 | 1.995342 | 2.523698 | 5 |
| 0.017031 | 3.471114 | 2.781549 | 3.449273 | 3.063424 | 1.982684 | 2.810396 | 1 |
| 0.217045 | 3.102494 | 2.257095 | 3.712236 | 3.227408 | 2.424947 | 2.706707 | 1 |
| 1.168394 | 3.158382 | 2.397039 | 2.875788 | 3.195214 | 1.667232 | 2.237079 | 1 |
| 2.166365 | 2.328856 | 3.406558 | 3.882285 | 2.341709 | 1.610299 | 1.985158 | 5 |
| 1.207266 | 3.701287 | 3.536277 | 2.471503 | 2.445392 | 1.455107 | 1.94385 | 1 |
| 0.350961 | 3.216452 | 3.756608 | 3.369897 | 2.633468 | 1.71541 | 1.968044 | 1 |
| 2.142924 | 3.021736 | 4.265552 | 2.12064 | 0.265916 | 2.962148 | 1.455148 | 2 |
| 0.33667 | 1.944071 | 2.455792 | 1.119593 | 2.806737 | 2.954146 | 1.19752 | 1 |
| -0.37456 | 4.684672 | 1.857995 | 2.673432 | 2.43409 | 1.675507 | 0.615034 | 1 |
| -0.45765 | 2.951242 | 3.57413 | 2.673064 | 2.310049 | 1.494068 | 1.204785 | 4 |
| 2.241543 | 3.295219 | 1.761795 | -0.46674 | 2.062207 | 0.658954 | 3.085202 | 3 |
| 2.274352 | 3.904877 | | 1.090103 | | 1.008027 | 1.615303 | 3 |
| | | 0.965383 | | 2.177539 | | | |
| 0.542086 | 1.246405 | 4.771957 | 2.932708 | 1.626256 | 0.35913 | 2.19558 | 4 |
| 1.405164 | 4.017422 | 2.502021 | 2.645762 | 2.199201 | 0.974838 | 1.105484 | 1 |
| 1.596445 | 2.820486 | 2.350912 | 1.453811 | 3.042025 | 1.647329 | 1.921859 | 1 |
| -0.10552 | 2.818759 | 2.971996 | 3.080708 | 1.907297 | 0.083147 | 0.823936 | 4 |
| -0.32487 | 3.260904 | 3.534991 | 2.253789 | 0.849691 | 0.516675 | 1.967281 | 4 |
| -0.1682 | 2.358753 | 3.087227 | 0.986124 | 3.435746 | 2.779199 | 2.729604 | 1 |
| 2.247645 | 4.286214 | 0.019446 | 3.584856 | 2.068911 | 1.866873 | 0.807345 | 2 |
| 0.47302 | 1.446077 | 0.663542 | 3.750715 | 1.414859 | 3.605458 | 1.93925 | 1 |
| -0.59701 | 1.675585 | 3.925224 | 1.716529 | 2.459564 | 3.219338 | 0.880136 | 4 |
| 0.861698 | 3.040857 | 2.553108 | 1.336346 | 1.43595 | 1.136466 | 0.604058 | 4 |
| 0.957117 | 2.787028 | 3.658154 | 0.801289 | -0.61602 | 1.330431 | 0.835537 | 4 |
| 0.124301 | 2.421105 | 2.705534 | 2.460809 | 1.797187 | 2.180488 | 1.753949 | 1 |
| 1.006473 | 1.997175 | 1.029746 | 2.796541 | 2.776268 | 0.984417 | 2.779216 | 5 |
| 0.366053 | 2.322168 | 4.060788 | 1.559525 | 1.519204 | 0.253499 | 2.169938 | 4 |
| 1.583427 | 3.27796 | 2.562148 | 1.507864 | 2.014645 | 0.852825 | 2.43981 | 3 |
| 0.751172 | 3.492416 | 4.487172 | 2.507872 | 1.848005 | 0.476099 | 2.176782 | 4 |
| 0.859564 | 2.121968 | 3.57061 | 2.07186 | 1.694885 | 2.381739 | 1.771004 | 4 |
| 1.150281 | 2.229375 | 3.993247 | 1.538726 | 1.713609 | 1.263208 | 2.984529 | 4 |
| 1.009329 | 2.523104 | 3.632711 | 1.751953 | 2.49709 | 0.747835 | 1.973844 | 4 |
| 0.800092 | 2.313618 | 1.947549 | 2.129778 | 2.779523 | 2.736547 | 1.287074 | 1 |
| 0.507842 | 2.126182 | 3.709382 | 2.025182 | 2.014483 | 2.499448 | 1.949562 | 4 |
| 1.707627 | 1.784648 | 3.412401 | 2.081609 | 1.543876 | 1.982379 | 2.252024 | 5 |
| 1.520279 | 2.053032 | 3.102355 | 2.341057 | 1.547812 | 1.045763 | 2.045449 | 5 |
| 2.051176 | 1.709775 | 3.481137 | 1.391418 | 1.709236 | 1.635493 | 3.759327 | 5 |
| | 1.734922 | | | 2.121027 | 3.065789 | 1.925379 | 1 |
| 0.911119 | | 3.484695 | 1.986006 | | | | 5 |
| 1.401215 | 1.524107 | 2.979994 | 1.938822 | 2.037472 | 0.806494 | 2.666591 | |
| 1.082589 | 1.594227 | 3.461005 | 1.861188 | 2.047426 | 1.824083 | 2.205309 | 5 |
| 0.782273 | 1.504928 | 3.980124 | 1.198786 | 2.167906 | 1.904642 | 2.458123 | 4 |
| 1.130089 | 1.618194 | 3.558431 | 1.84232 | 1.224004 | 2.513945 | 1.961609 | 4 |
| 0.777959 | 2.330444 | 4.134831 | 2.302482 | 1.573921 | 1.895572 | 1.789862 | 4 |
| 1.708766 | 1.298943 | 2.563442 | 2.053514 | 2.096883 | 1.721538 | 2.927518 | 5 |
| 1.154063 | 2.688875 | 2.425242 | 2.718147 | 2.253345 | 1.159137 | 1.198447 | 1 |
| 0.809999 | 1.599301 | 2.619081 | 2.243507 | 1.198234 | 2.379065 | 3.111126 | 5 |
| 1.98482 | 1.356919 | 3.401547 | 2.87027 | 2.888688 | 0.917695 | 1.559026 | 5 |
| 2.623055 | 0.067936 | 2.551413 | 1.795425 | 2.420002 | 0.685113 | 3.023309 | 5 |
| 0.104503 | 0.941991 | 2.736113 | 4.900371 | 2.223849 | 2.112671 | 1.511158 | 5 |
| 1.397307 | 0.341324 | 2.840602 | 2.29184 | 2.505188 | 0.169115 | 3.259495 | 5 |
| 1.270621 | 0.496461 | 2.746452 | 2.312243 | 3.044293 | 0.303743 | 3.174375 | 5 |
| 2.274565 | 0.005369 | 2.76484 | 2.662452 | 2.414838 | 0.887809 | 2.310469 | 5 |
| 0.086942 | 2.180963 | 2.659627 | 3.723745 | -0.4808 | 2.794365 | 2.358254 | 2 |
| 2.554201 | 2.382038 | 2.613128 | 2.197507 | 2.622773 | 0.417857 | 2.937588 | 5 |
| 0.665437 | -0.15309 | 3.013491 | 3.591409 | 2.397752 | 0.910813 | 3.196063 | 5 |
| 0.005457 | -0.10008 | 0.010431 | 5.531403 | 2.031102 | 0.310013 | 5.180003 | J |

Document: PPD

Author: PPD


06MAY2024



| 0.219131 | 0.988948 | 2.949241 | 2.832939 | 2.812933 | 1.931909 | 2.337423 | 5 |
|---|---|---|---|---|---|---|---|
| 0.08191 | 1.904748 | 2.697057 | 2.395814 | 2.909281 | 0.849056 | 1.816543 | 11 |
| -0.5757 | 2.364009 | 3.812397 | 1.903619 | 2.952605 | 1.246934 | 2.699965 | 4 |
| 0.281395 | 2.412998 | 4.491506 | 1.717264 | 1.527465 | 0.20048 | 1.743169 | 4 |
| -0.37792 | 0.853802 | 3.500635 | 4.447944 | 1.770293 | 2.376319 | 2.945239 | 5 |
| 1.43101 | 1.729342 | 2.285234 | 3.594539 | 2.158406 | 1.41163 | 2.35083 | 5 |
| 2.242448 | 0.452776 | 2.03011 | 2.175292 | 2.960922 | 0.892266 | 3.490946 | 5 |
| 0.772287 | 1.044562 | 4.099495 | 2.099755 | 2.303216 | -0.07957 | 3.408013 | 5 |
| 1.687683 | 0.705034 | 3.483106 | 3.50241 | 0.084663 | 1.296573 | 1.360677 | 4 |
| 0.08152 | 2.497989 | 2.633608 | 2.102286 | 1.992036 | 2.405288 | 2.854927 | 1 |
| 0.564148 | 0.290457 | 1.858481 | 3.457962 | 2.040157 | 2.621054 | 4.093532 | 5 |
| 1.432265 | 2.214134 | 2.28557 | 2.447828 | 3.114609 | 1.697488 | 0.560871 | 1 |
| 1.22986 | 4.209676 | 4.152368 | 1.648818 | 2.4148 | 1.380472 | 3.982964 | 1 |
| 1.798733 | 2.321707 | 1.944999 | 2.484884 | 2.09713 | 2.497045 | 3.945049 | 5 |
| 1.548915 | 2.98621 | 2.419907 | 4.166224 | 1.884883 | 3.007174 | 1.354243 | 2 |
| 1.736698 | 2.102224 | 2.781879 | 2.624937 | 1.287076 | 1.154947 | 2.066471 | 5 |
| 1.841468 | 2.779364 | 2.014616 | 1.952026 | 1.864021 | 0.832871 | 2.831117 | 5 |
| 1.850788 | 3.557185 | 1.247119 | 2.762191 | 2.367131 | 2.073187 | 2.334656 | 1 |
| 1.988117 | 1.848378 | 1.617975 | 3.235807 | 3.561746 | 0.849005 | 3.282251 | 5 |
| 2.963195 | 1.875433 | 2.294584 | 2.090209 | 1.373802 | 0.773446 | 1.733781 | 3 |
| 1.280458 | 3.577684 | 3.18186 | 2.344035 | 3.374431 | 2.15427 | 2.751256 | 1 |
| 0.884161 | 5.784644 | 3.534264 | 1.819497 | 2.386301 | 3.77747 | 0.141682 | <del>- i</del> |
| 0.074259 | 3.574523 | 1.619785 | 2.533091 | 0.988846 | 2.903029 | 2.823716 | <del>- </del> |
| 3.04004 | 2.314318 | 2.13163 | 1.6602 | 1.868691 | 0.651936 | 2.527277 | 3 |
| 2.717961 | 1.981777 | 1.938336 | 2.53088 | 2.20996 | 0.031930 | 1.92194 | 3 |
| 1.469363 | 2.818761 | 1.884582 | 2.648021 | 2.089939 | 2.410461 | 1.996118 | 1 |
| 2.709623 | 2.493832 | 1.025723 | 2.408424 | 3.062117 | 3.46406 | 1.106719 | 1 |
| 2.161146 | 1.174376 | 2.314965 | 2.254531 | 3.234909 | 1.291243 | 2.520153 | 5 |
| 2.287607 | 1.838934 | 1.818019 | 2.927362 | 2.361122 | 0.866097 | 2.034928 | 5 |
| 3.353594 | 3.559703 | 2.04658 | 2.406643 | -0.54042 | 0.195315 | 0.023831 | 3 |
| 1.392493 | 2.078828 | 2.6005 | 1.897844 | 2.84124 | 0.383242 | 0.947499 | 3 |
| 1.725897 | 3.336555 | 1.507295 | 1.7479 | 3.54761 | 2.859758 | 2.606246 | 1 |
| 1.2252 | 3.287465 | 2.245327 | 2.208732 | 1.496208 | 2.975495 | 2.753529 | 1 |
| 1.518102 | 2.010543 | 2.173446 | 2.299928 | 2.45509 | 2.839368 | 2.859943 | 5 |
| 1.289588 | 3.386302 | 4.211413 | 2.154531 | 1.303094 | 0.481756 | 2.964039 | 4 |
| 1.012439 | 4.384014 | 3.35423 | 2.879892 | 0.911968 | 4.236695 | 1.938896 | 2 |
| -0.18313 | 2.332953 | 2.817455 | 2.991674 | 1.413407 | 2.469997 | 1.751645 | 1 |
| -0.50824 | 2.851968 | 3.078299 | 3.017893 | 1.511157 | 3.204069 | 1.452336 | 1 |
| 2.015306 | 1.892684 | 3.122085 | 2.005002 | 1.28295 | 1.431305 | 2.252795 | 3 |
| 1.810405 | 2.313179 | 2.719985 | 2.289299 | 1.433045 | 1.995691 | 2.279748 | 5 |
| -0.36417 | 2.441534 | 4.741204 | 2.029903 | 2.179041 | 1.560313 | 1.344052 | 4 |
| 1.612228 | 3.39865 | 3.771511 | 2.523235 | 1.798751 | 1.338797 | 1.638589 | 4 |
| 0.498329 | 2.028352 | 3.80679 | 2.242893 | 1.021459 | 2.388737 | 1.175935 | 4 |
| -0.18434 | 2.373169 | 3.690509 | 2.559589 | 2.106675 | 1.890076 | 2.149593 | 4 |
| 1.521238 | 2.119707 | 2.963294 | 1.800389 | 1.566119 | 1.958181 | 0.758386 | 3 |
| 3.747659 | 1.227065 | 2.861703 | 2.434098 | 1.443798 | 2.781314 | 2.597393 | 5 |
| -0.4823 | 1.90793 | 3.373967 | 2.878178 | 2.004723 | 3.40478 | 2.332985 | 1 |
| 0.899904 | 4.377078 | 2.276759 | 2.487403 | 0.184471 | 1.761139 | 0.685288 | 2 |
| 1.801516 | 3.019131 | 3.060307 | 2.431625 | 1.409738 | 1.490599 | 0.428911 | 2 |
| 0.524149 | 2.633798 | 3.796815 | 1.644169 | 0.667038 | 1.265146 | 1.836087 | 4 |
| 2.832446 | 3.170785 | 1.759903 | 1.961723 | 1.444286 | 1.823112 | 1.105778 | 3 |
| -0.07634 | 2.224685 | 3.774898 | 3.031975 | -0.1915 | 1.917331 | 1.714644 | 4 |
| -0.00896 | 3.683818 | 3.356392 | 2.308612 | 1.307789 | 3.677818 | 0.323892 | 2 |
| 1.756645 | 2.94947 | 3.107809 | 2.888338 | 0.822709 | 3.959166 | 1.271949 | 2 |
| 2.132132 | 2.038671 | 2.938456 | 2.077305 | 1.016538 | 1.692268 | 1.867374 | 3 |
| 2.027801 | 2.090666 | 3.044967 | 2.391921 | 1.466157 | 2.999378 | 1.451428 | 2 |
| 2.365434 | 0.881948 | 2.909211 | 2.874983 | 1.970898 | 2.364969 | 2.719813 | 5 |
| 1.951106<br>1.155816 | 1.417047<br>1.648827 | 3.499015 | 3.274452 | 1.057297 | 1.360355 | 2.54604 | <u>5</u><br>5 |
| | 1 6/1887/ | 3.136144 | 3.231095 | 1.479935 | 2.61277 | 2.369647 | 5 |

Document: PPD

Author: PPD


06MAY2024

| | | 1 | - | | 1 | | |
|---|---|---|---|---|---|---|---|
| 1.771195 | 1.978266 | 2.468392 | 2.849778 | 1.952468 | 2.637186 | 2.539566 | 5 |
| 2.175577 | 0.957878 | 1.749733 | 4.318935 | 2.408992 | 2.347051 | 3.083741 | 5 |
| 1.730574 | 1.460436 | 2.355927 | 2.801036 | 2.458172 | 2.805657 | 3.037723 | 5 |
| 1.625811 | 1.123879 | 2.555173 | 2.98834 | 1.932035 | 2.598875 | 3.107223 | 5 |
| 1.300338 | 1.27347 | 2.863889 | 2.670251 | 2.788495 | 2.009867 | 4.144211 | 5 |
| 1.058618 | 1.640886 | 3.14455 | 3.155436 | 1.597802 | 1.754571 | 2.858831 | 5 |
| 1.714292 | 1.198592 | 2.361832 | 3.655121 | 2.911294 | 2.190251 | 2.968629 | 5 |
| 1.240011 | 1.509991 | 2.984057 | 1.286569 | 2.708608 | 1.855332 | 3.967645 | 5 |
| 1.152672 | 1.764461 | 2.576472 | 2.889279 | 2.721701 | 1.695326 | 2.606245 | 5 |
| 1.255709 | 1.355849 | 2.521385 | 2.856854 | 2.597104 | 1.876426 | 3.207666 | 5 |
| 0.74156 | 1.575887 | 3.573962 | 3.438606 | 3.075308 | 2.406598 | 2.848083 | 5 |
| 1.487389 | 2.083264 | 1.877643 | 2.610233 | 2.580977 | 2.734694 | 3.221042 | 5 |
| 1.02402 | 0.666849 | 3.200515 | 3.967067 | 2.679366 | 2.374665 | 3.865079 | 5 |
| 0.904672 | 0.738232 | 2.490656 | 2.403095 | 2.3109 | 1.981781 | 2.503543 | 5 |
| 1.97023 | 1.764496 | 2.422681 | 3.936467 | 1.939548 | 2.512576 | 3.901476 | 5 |
| 2.676331 | 1.08356 | 3.41355 | 3.33541 | 0.698102 | 2.519931 | 3.287986 | 5 |
| 2.614462 | 4.775062 | 3.793557 | -0.19917 | -0.981 | 0.09312 | 1.252973 | 3 |
| 0.092529 | 2.213861 | 1.666891 | 3.141264 | 2.591698 | 3.012315 | 1.884515 | 1 |
| 0.62021 | 3.504931 | 2.630801 | 1.965301 | 1.737083 | 2.335864 | 1.035281 | 1 |
| -0.10889 | 2.970387 | 2.077207 | 2.483217 | 2.67454 | 2.810844 | 2.125511 | 1 |
| -0.28494 | 2.862408 | 4.948831 | 1.475156 | 1.273039 | 0.024325 | 2.188301 | 4 |
| 0.141229 | 1.826175 | 2.57906 | 3.825405 | 2.331338 | 2.178282 | 3.733651 | 5 |
| -0.27393 | 1.798164 | 2.281096 | 1.096077 | 3.405163 | 2.22112 | 2.368599 | 1 |
| 1.889118 | 2.197416 | 2.662556 | 0.938291 | 1.45778 | 1.768633 | 1.850104 | 3 |
| | | | | | | | 3 |
| 2.026809 | 1.43333 | 2.852578 | 2.062381 | 2.494402 | 2.510134 | 1.003418 | |
| 0.4547 | 1.822873 | 1.642994 | 1.648994 | 2.465097 | 2.307406 | 2.260072 | 1 |
| 1.180574 | 1.979456 | 2.190599 | 0.638097 | 1.822171 | 1.684538 | 1.976499 | 1 |
| -0.15376 | 2.113963 | 2.755861 | 2.31101 | 2.417009 | 2.151042 | 2.155638 | 1 |
| 2.937327 | 0.559019 | 3.293035 | 1.705683 | 1.755515 | 1.537882 | 2.362831 | 5 |
| 0.356661 | 2.212595 | 2.084012 | 1.942391 | 2.012923 | 1.77337 | 1.492639 | 1 |
| 1.257337 | 1.708001 | 1.806124 | 1.843787 | 2.280795 | 1.967791 | 2.486759 | 5 |
| 1.302175 | 2.292117 | 3.27532 | 2.309357 | 0.828285 | 1.952833 | 1.783675 | 4 |
| 1.714566 | 2.866174 | 2.614927 | 1.165569 | 2.346443 | -0.46207 | 1.580056 | 3 |
| 2.336772 | 1.820066 | 2.107818 | 2.778122 | 2.028988 | 1.729201 | 2.644071 | 5 |
| -0.531 | 1.905626 | 2.663749 | 4.288357 | 2.308736 | 3.089625 | 4.707173 | 5 |
| 1.955097 | 2.75595 | 1.720104 | 1.485425 | 2.439215 | 0.383829 | 2.150109 | 3 |
| 0.424371 | 2.775628 | 2.618747 | 3.105367 | 1.291942 | 1.385739 | 1.814535 | 1 |
| 2.682818 | 1.975018 | 3.091693 | 2.359624 | 2.077224 | 1.058987 | 2.189526 | 3 |
| 1.640291 | 2.201269 | 3.686279 | 2.493968 | 3.027828 | 0.383334 | 1.950114 | 5 |
| 1.962298 | 2.543239 | 1.478078 | 2.839681 | 0.880412 | 1.964117 | 2.524755 | 2 |
| 1.518659 | 3.192809 | 2.697412 | 1.905137 | 2.597932 | -0.15954 | 2.23207 | 3 |
| 1.834275 | 1.687792 | 3.803747 | 2.399916 | 1.433644 | 0.562578 | 1.025609 | 4 |
| 1.540272 | 1.983626 | 2.956717 | 3.394021 | 1.800051 | 1.677738 | 0.662117 | 2 |
| 1.509981 | 2.642669 | 3.116794 | 1.549859 | 1.938711 | 1.855646 | 1.954819 | 3 |
| 2.134296 | 1.907773 | 2.690553 | 3.23495 | 1.495158 | 0.775124 | 1.619342 | 3 |
| 0.427512 | 2.987253 | 2.561937 | 2.27099 | 1.3845 | 2.114721 | 0.565118 | 1 |
| 1.466702 | 2.301835 | 2.37308 | 2.599048 | 2.254712 | 1.407731 | 1.813743 | <u> </u> |
| 1.027552 | 1.923318 | 3.15668 | 3.298839 | 1.721175 | 1.344687 | 1.461926 | 4 |
| 2.925279 | 2.151205 | 3.252401 | 2.148987 | 1.787043 | 1.139834 | 1.406604 | 3 |
| 1.803615 | 0.897055 | 2.381724 | 4.027319 | 0.612286 | 2.102622 | 0.497539 | 2 |
| 0.501035 | 1.594727 | 3.748318 | 3.202126 | 2.717837 | 1.217422 | 2.0056 | 5 |
| 1.135913 | 2.46013 | 2.699918 | 2.040346 | 1.05604 | 2.40855 | 1.437545 | 2 |
| 1.47729 | 1.576555 | 2.766053 | 2.486893 | 3.088382 | 0.238345 | 2.288514 | 5 |
| 2.322109 | 1.8903 | 1.856853 | 3.043669 | 1.448824 | 1.854425 | 2.292022 | 5 |
| 0.943979 | 2.865445 | 2.334755 | 2.361299 | 1.84453 | 1.57974 | 1.455633 | 1 |
| 1.09441 | 2.61972 | 2.570202 | 2.266813 | 0.822919 | 1.006511 | 1.137528 | 4 |
| 1.446558 | 2.894173 | 3.720822 | 2.312959 | 2.573729 | 1.242164 | 1.410237 | 4 |
| 0.736881 | 2.07327 | 3.906554 | 3.063998 | 1.881051 | 1.369881 | 0.160261 | 4 |
| 0.665234 | 2.183043 | 2.941374 | 2.995214 | 1.14126 | 3.139709 | 0.670783 | 2 |

Document: PPD

Author: Version Number:

Version Number: 1.0 Version Date: 06MAY2024

| | | , | | | | | |
|---|---|---|---|---|---|---|---|
| 1.431209 | 2.102447 | 2.877089 | 3.272383 | 1.528063 | 1.667444 | 0.597345 | 2 |
| 0.48805 | 2.199462 | 2.791748 | 3.053477 | 1.218693 | 3.241743 | 0.81835 | 2 |
| 1.729035 | 2.60887 | 2.382874 | 2.946179 | 1.154216 | 2.539631 | 0.705188 | 2 |
| 0.923982 | 2.09841 | 3.134973 | 3.049035 | 1.577602 | 2.226752 | 0.562968 | 2 |
| 0.473393 | 1.823634 | 2.603832 | 3.244876 | 2.472785 | 2.388323 | 0.70335 | 1 |
| 0.643718 | 3.162341 | 2.628687 | 3.124583 | 0.697315 | 3.489079 | 0.444281 | 2 |
| 1.231598 | 1.489925 | 2.575601 | 2.956323 | 1.393692 | 3.056498 | 2.419777 | 5 |
| 0.885313 | 3.604693 | 2.334157 | 2.907145 | 1.783189 | 2.383189 | 0.473879 | 2 |
| 1.486663 | 2.382557 | 2.521454 | 3.405304 | 0.122165 | 2.458242 | 1.897779 | 2 |
| 1.305746 | 2.536706 | 2.503103 | 2.726279 | 1.370371 | 2.271897 | 0.760181 | 2 |
| -0.12128 | 2.931554 | 2.985789 | 3.448854 | 2.373757 | 3.0748 | 0.750214 | 1 |
| -0.3651 | 3.29011 | 2.870149 | 3.014172 | 0.790517 | 3.231845 | 1.216384 | 1 |
| 1.310901 | 2.905656 | 3.206514 | 2.745517 | 2.308938 | 2.328841 | 1.60868 | 1 |
| 0.8192 | 2.058696 | 3.311621 | 2.910875 | 2.063997 | 2.20247 | 1.529922 | 1 |
| 1.579844 | 2.31691 | 1.764519 | 2.700399 | 1.475303 | 3.338388 | 1.799588 | 2 |
| 1.650651 | 1.172353 | 2.25335 | 2.336537 | 1.40992 | 2.091142 | 1.840565 | 5 |
| 2.400323 | 0.610945 | 2.145213 | 1.814261 | 2.156261 | 2.594137 | 1.989301 | 5 |
| 1.337072 | 1.787411 | 2.435036 | 2.180727 | 1.476423 | 1.703351 | 2.390161 | 5 |
| 1.334314 | 3.493188 | 3.203095 | 0.739232 | 2.752471 | 1.577154 | 1.506409 | 3 |
| 2.395664 | 1.784892 | 2.990832 | 1.597801 | 3.454405 | 1.431834 | 2.221238 | 5 |
| 2.834376 | 1.372208 | 2.467716 | 1.487558 | 2.422688 | 2.178153 | 2.292664 | 5 |
| 1.271013 | 2.190323 | 2.02582 | 1.854061 | 2.466391 | 2.423069 | 2.725961 | 1 |
| 0.129491 | 1.944993 | 3.627968 | 1.689957 | 1.382203 | 2.063105 | 2.376668 | 4 |
| 0.915972 | 2.036587 | 2.390177 | 2.812893 | 1.865705 | 1.996444 | 1.482858 | 1 |
| -0.29183 | 2.254987 | 2.829684 | 2.300647 | 0.747438 | 3.259114 | 1.744497 | 1 |
| 0.234823 | 3.984334 | 2.709338 | 3.583035 | 0.06296 | 3.288988 | 0.717452 | 2 |
| -0.03279 | 1.956234 | 3.73337 | 2.42477 | 1.51287 | 1.496175 | 2.24365 | 4 |
| -0.22374 | 3.954465 | 4.147648 | 3.000342 | 2.095893 | 1.375367 | 0.174058 | 4 |
| 4.446452 | 3.112146 | 3.834213 | -0.56448 | 2.322335 | 0.081094 | 0.815274 | 3 |
| 0.254195 | 2.219487 | 2.347961 | 1.5985 | 2.939996 | 1.619148 | 2.003347 | 1 |
| 0.722066 | 1.84351 | 3.439109 | 3.028911 | 0.858413 | 2.820346 | 2.055325 | 4 |
| -0.27786 | 1.621398 | 3.810628 | 3.493549 | 1.61931 | 2.388291 | 1.959439 | 4 |
| 1.95763 | 2.243665 | 2.419941 | 1.550256 | 2.339185 | 1.526504 | 0.87867 | 3 |
| -0.17712 | 3.679931 | 2.027275 | 3.438949 | 1.227549 | 4.346655 | 0.565953 | 2 |
| -0.52016 | 2.644474 | 4.985067 | 2.777575 | 2.129857 | 1.603163 | 1.322 | 4 |
| 0.139093 | 3.077551 | 3.155317 | 1.84699 | 1.544916 | 0.909727 | 2.255974 | 4 |
| -0.29745 | 3.924371 | 3.427086 | 2.814315 | -0.34252 | 2.52275 | -0.12371 | 2 |
| 1.197751 | 1.139765 | 2.959802 | 3.724448 | 2.00368 | 1.870335 | 3.248781 | 5 |
| -0.55263 | 2.850451 | 3.603637 | 2.159742 | 1.61182 | 3.131141 | 2.21753 | <u></u> |
| -0.09923 | 3.147932 | 3.515215 | 1.300025 | 2.023952 | 0.341102 | 1.147187 | 4 |
| 1.482171 | 0.598118 | 4.524763 | 2.495524 | 1.920755 | 1.016522 | 1.752847 | 4 |
| 0.435803 | 0.030049 | 2.99525 | 5.212456 | 3.600696 | 2.278578 | 3.051625 | 5 |
| 0.896986 | 2.123555 | 1.956048 | 3.483763 | 3.273525 | 1.450855 | 1.995661 | <u>5</u> 1 |
| 1.727307 | 1.314198 | 3.995778 | 4.880579 | 3.273323 | 2.337371 | 2.479633 | 5 |
| 1.007479 | 1.779471 | 4.011855 | 3.485044 | 1.019926 | 0.992437 | 0.427342 | 4 |
| 1.133501 | 3.612282 | 3.371249 | 4.166631 | 0.783912 | 2.980189 | 0.390786 | 2 |
| 0.447813 | 1.584168 | 4.595198 | 4.146647 | 1.49147 | 1.118816 | 2.154007 | 4 |
| 1.36141 | | | 4.615451 | | | | |
| | 0.164857 | 4.184602 | | 0.680796<br>1.538351 | 2.828915 | 2.215485 | <u>5</u><br>4 |
| 0.237311 | 1.661926 | 4.718851 | 3.915297 | | 2.461316 | 0.972878 | |
| 1.675214 | 2.703634 | 3.664126 | 1.781546 | 1.381758 | 1.584137 | 2.177306 | 4 |
| -0.0933 | 4.003946 | 3.094488 | 2.609247 | -0.45808 | 3.497689 | 1.265117 | 2 |
| 1.115991 | 1.93992 | 2.449696 | 2.209266 | 1.989389 | 2.600533 | 1.638723 | 1 |
| 0.565087 | 1.267156 | 1.971504 | 1.821961 | 2.941994 | 2.362466 | 1.948297 | 5 |
| 0.2899 | 2.425688 | 2.527741 | 1.688038 | 2.859624 | 1.102273 | 1.363903 | 1 |
| 0.012578 | 2.713523 | 2.772004 | 1.695502 | 2.556442 | 1.490683 | 1.172728 | 1 |
| 0.457526 | 2.242863 | 2.640553 | 1.38489 | 2.9747 | 1.112302 | 1.723175 | 1 |
| 0.269487 | 1.856392 | 2.378915 | 2.310383 | 2.23644 | 1.466357 | 2.292227 | 5 |
| -0.30298 | 2.039958 | 2.487779 | 2.484312 | 2.889577 | 1.778061 | 2.620527 | 1 |
| -0.059 | 2.329745 | 2.661882 | 1.800231 | 2.943895 | 0.849261 | 2.4205 | 1 |

Document: PPD

Author: PPD


06MAY2024

1.0

06MAY2024



#### Statistical Analysis Plan

| 3.234036 | 3.172942 | 2.152633 | 1.247851 | 1.830191 | 0.741028 | 1.367281 | 3 |
|---|---|---|---|---|---|---|---|
| -0.14962 | 3.212166 | 2.838131 | 2.052148 | 0.76686 | 2.904901 | 0.926416 | 11 |
| 1.008297 | 3.605593 | 1.552424 | 2.545575 | 1.459873 | 2.458237 | 1.063863 | 11 |
| 0.069645 | 3.442147 | 2.503456 | 2.854764 | 2.551114 | 2.401892 | 1.840573 | 11 |
| -0.19621 | 2.856654 | 2.546963 | 3.078251 | 1.409379 | 1.312913 | 2.43579 | 11 |
| 0.922144 | 3.392091 | 3.413087 | 1.786973 | 0.876997 | 1.979531 | 0.815435 | 4 |
| 0.439565 | 3.695894 | 3.233887 | 3.19461 | -0.65113 | 2.981872 | 0.096498 | 2 |
| 0.463794 | 3.118323 | 2.945531 | 2.132446 | 0.692042 | 1.676786 | 1.832364 | 4 |
| 2.046115 | 1.860467 | 4.503206 | 1.44212 | 0.944814 | 0.960159 | 1.702708 | 4 |
| 0.822082 | 1.752166 | 3.96031 | 3.670542 | 0.432142 | 2.094926 | 1.835506 | 4 |
| 1.384499 | 1.676338 | 3.335121 | 2.344334 | 1.708029 | 1.973757 | 3.015226 | 5 |
| 2.913171 | 2.251743 | 3.828942 | 2.862465 | 3.506109 | 2.288636 | 0.682411 | 3 |
| 2.838667 | 1.587802 | 3.139398 | 2.455651 | 1.986433 | 1.559845 | 2.010168 | 3 |
| 1.984939 | 1.226032 | 3.974135 | 2.871381 | 1.764569 | 2.52817 | 2.269736 | 5 |
| 1.882535 | 0.965832 | 3.62802 | 2.424984 | 3.088003 | 2.571588 | 1.442444 | 5 |
| 2.834767 | 2.291731 | 2.914424 | 1.828595 | 2.676055 | 2.190016 | 0.904297 | 3 |
| 2.406044 | 2.421871 | 3.677239 | 1.100186 | 2.528083 | 1.850513 | 0.909268 | 3 |
| 3.333304 | 1.738452 | 3.145411 | 1.694157 | 2.436078 | 0.861111 | 2.058184 | 3 |
| 2.809199 | 2.201564 | 3.268227 | 2.439596 | 2.217548 | 2.20399 | 0.443276 | 3 |
| 3.232019 | 2.695417 | 3.21763 | 1.39774 | 1.641224 | 1.386497 | 0.029767 | 3 |
| 2.562955 | 1.649742 | 4.191257 | 1.75234 | 3.416616 | 0.008248 | 0.947485 | 3 |
| 2.653311 | 2.213077 | 2.654112 | 1.964367 | 0.998636 | 3.271016 | 3.047206 | 5 |
| 4.088227 | 3.519633 | 1.458443 | 1.578193 | 0.700923 | 2.177483 | 3.025567 | 3 |
| 1.621409 | 1.437943 | 3.781382 | 2.457539 | 0.583088 | 1.380606 | 1.395895 | 4 |
| 2.902669 | 2.219219 | 2.532083 | 1.780608 | 1.705037 | 1.497211<br>0.680305 | 1.210752<br>0.244186 | 3 |
| 3.005859 | 2.263617 | 5.64921 | 1.245774 | -0.42109 | | | 3 |
| 2.362506 | 1.144091<br>2.06235 | 2.361297<br>2.689261 | 2.453162<br>2.022982 | 2.143155<br>2.280881 | 1.79232<br>1.219565 | 2.288028<br>1.887121 | <u>5</u><br>5 |
| 1.667598<br>1.808149 | 1.78866 | 4.051322 | 1.885426 | 2.260661 | 0.817292 | 1.620497 | 3 |
| 0.687603 | 3.206993 | 4.031322 | 3.315963 | -0.20797 | 1.946517 | 1.362868 | 4 |
| 2.862084 | 2.377349 | 2.555443 | 3.876989 | 0.702746 | 2.024126 | 1.165072 | 2 |
| 0.710643 | 1.936612 | 2.900109 | 3.781125 | 2.51583 | 1.740071 | 2.016443 | 5 |
| 2.057296 | 3.589327 | 2.526465 | 2.853584 | -0.28298 | 1.54849 | 0.178033 | 2 |
| 1.717724 | 3.312208 | 3.219567 | 3.832021 | 0.433151 | 1.332947 | 0.398813 | 2 |
| 1.784393 | 3.483958 | 1.901055 | 2.434483 | 0.562683 | 3.044089 | 0.828156 | 2 |
| 2.365971 | 2.201863 | 3.519977 | 1.583483 | 1.150986 | 1.335765 | 0.655795 | 3 |
| 4.319165 | 1.590442 | 3.087611 | 1.69606 | 0.770118 | 0.599462 | 1.282893 | 3 |
| 3.346217 | 1.09885 | 4.812988 | 1.455227 | 0.212139 | 1.128825 | 1.865715 | 3 |
| 3.530807 | 1.567584 | 4.504891 | 1.8653 | 0.940612 | 0.82131 | 0.77248 | 3 |
| 2.891285 | 1.89644 | 4.433179 | 2.19465 | 1.006817 | 1.09154 | 0.498398 | 3 |
| 1.928594 | 2.236547 | 4.683135 | 1.988054 | 0.544993 | 1.246763 | 0.558855 | 4 |
| 2.285322 | 2.125545 | 4.559235 | 2.288247 | 0.666203 | 1.084367 | 0.472938 | 4 |
| 1.89005 | 1.011516 | 5.266577 | 2.797959 | 0.412246 | 0.880222 | 0.483154 | 4 |
| 0.418664 | 1.731204 | 5.061108 | 3.2518 | 0.698308 | 3.020168 | 0.715598 | 4 |
| 1.367057 | 2.925187 | 4.655244 | 3.350586 | -0.01201 | 3.470676 | 0.821254 | 2 |
| 2.309585 | 1.804595 | 2.978303 | 3.676435 | 0.676995 | 2.935604 | 1.066488 | 2 |
| 1.8683 | 1.609789 | 3.585674 | 3.410347 | 1.090116 | 2.76966 | 0.538212 | 2 |
| 1.582343 | 1.893786 | 4.194117 | 3.161633 | 1.008141 | 2.783293 | 0.669849 | 2 |
| 2.150257 | 2.572329 | 2.223382 | 1.867505 | 2.895349 | 1.994313 | 3.149671 | 5 |
| 2.438346 | 4.148842 | 2.612882 | 3.155902 | 0.171949 | 1.607915 | 2.041156 | 2 |
| 2.643976 | 3.492028 | 2.734121 | 3.093574 | 0.779863 | 2.711358 | 1.925412 | 2 |
| 2.855769 | 2.880836 | 1.739848 | 1.828785 | 2.194659 | 2.847119 | 1.926847 | 3 |
| 3.399597 | 3.245786 | 2.023543 | 2.512159 | 1.595768 | 2.089901 | 1.455838 | 3 |
| 2.737046 | 3.037004 | 0.67967 | 3.566229 | 1.882432 | 3.613259 | 1.022656 | 2 |
| 2.989004 | 3.050118 | 1.218374 | 2.338301 | 1.72523 | 2.930881 | 2.004095 | 2 |
| 3.730418 | 3.135985 | 1.6401 | 2.053811 | 1.028681 | 2.857294 | 2.173015 | 2 |
| 2.463663 | 0.859639 | 5.162668 | 0.886539 | 1.554102 | 0.509594 | 2.314751 | 3 |
| 2.946992 | 0.400476 | 4.639125 | 3.18962 | 1.353431 | 1.528145 | 2.900802 | 5 |
| 3.042424 | 4.105682 | 3.575925 | 0.706032 | -0.75609 | -0.13641 | 0.230446 | 3 |

PPD Document:

Author: שא Version Number: Version Date:

| 2.253494 | 0.88575 | 4.05183 | 1.474706 | 3.073917 | 0.406476 | 3.763321 | 5 |
|---|---|---|---|---|---|---|---|
| 1.675898 | 2.724666 | 4.647242 | 2.097785 | 0.23467 | 0.574127 | 0.663669 | 4 |
| 2.582725 | 2.741702 | 4.9941 | 1.059533 | 1.35462 | 1.077715 | 1.16564 | 3 |
| 1.050035 | 2.210001 | 5.021932 | 3.464061 | 1.364692 | 0.340931 | 1.686686 | 4 |
| 1.561219 | 0.545155 | 4.069079 | 1.690497 | 3.179686 | 0.016492 | 3.553318 | 5 |
| 1.265462 | 3.092702 | 3.594905 | 2.829159 | 0.750077 | 3.152979 | 1.644279 | 2 |
| 1.074474 | 3.037171 | 4.680648 | 3.823089 | 0.788346 | 0.936433 | 0.868559 | 4 |
| 1.091429 | 3.677598 | 3.423406 | 2.745653 | 1.001984 | 2.498806 | 1.66485 | 2 |
| 2.720772 | 2.102133 | 3.405409 | 2.797069 | 0.364539 | 1.46441 | 1.087318 | 3 |
| 3.226577 | 1.922205 | 2.953435 | 1.647369 | 0.593546 | 2.083638 | 0.851123 | 3 |
| 2.96997 | 2.214062 | 3.505646 | 2.499191 | 0.846053 | 0.964966 | 1.384221 | 3 |
| 3.651752 | 1.742185 | 4.164508 | 2.691835 | 0.553888 | 1.162542 | 1.663439 | 3 |
| 1.774319 | 2.621301 | 3.839708 | 2.941738 | 1.179815 | 1.918955 | 1.74463 | 4 |
| 3.320918 | 1.48185 | 3.289602 | 2.379944 | 0.653762 | 1.801415 | 1.466398 | 3 |
| 2.604631 | 2.198748 | 3.566384 | 3.787496 | 0.095679 | 1.115488 | 1.241199 | 2 |
| 3.833065 | 2.359699 | 3.028004 | 2.96456 | 0.979526 | 1.33778 | 1.312105 | 3 |
| 3.004658 | 1.994467 | 3.340586 | 3.123453 | 0.168374 | 1.183954 | 1.303827 | 3 |
| 3.557233 | 1.908423 | 3.907425 | 3.378859 | 0.393898 | 1.68292 | 1.077381 | 3 |
| 2.411464 | 2.16817 | 3.985166 | 2.790466 | 1.111273 | 1.797105 | 1.584131 | 3 |
| 1.491612 | 2.692824 | 3.446391 | 1.610859 | 2.136308 | 1.597012 | 0.673667 | 3 |
| 1.570925 | 1.579912 | 3.93983 | 2.736112 | 1.868873 | 0.511005 | 2.476103 | 5 |
| 1.74664 | 1.266399 | 2.752911 | 3.290547 | 2.346396 | 2.387008 | 4.022284 | 5 |
| 1.154398 | 2.149252 | 1.965355 | 2.992882 | 1.978235 | 3.127639 | 0.860784 | 1 |
| 0.688774 | 2.974488 | 1.694827 | 3.193321 | 2.122084 | 3.338055 | 1.028929 | 1 |
| 1.131356 | 2.409504 | 3.316011 | 4.297027 | -0.46325 | 1.780486 | 0.505052 | 2 |
| 2.478426 | 4.047283 | 2.050103 | 4.226233 | -0.2782 | 3.394542 | -0.23253 | 2 |
| 2.083689 | 3.657652 | 2.921747 | 3.583169 | -0.01864 | 2.614121 | -0.05174 | 2 |
| 0.436883 | 4.775917 | 2.633991 | 3.694657 | -0.60229 | 3.109147 | 0.170619 | 2 |
| 4.010344 | 4.141069 | 2.630313 | 3.047465 | -0.95245 | 2.075121 | -0.17676 | 2 |
| -0.12992 | 3.393718 | 5.397824 | 0.854292 | 2.35004 | 0.100554 | 2.472098 | 4 |
| 1.590358 | 2.277793 | 1.279885 | 3.553163 | 2.987285 | 1.843279 | 1.926848 | 1 |
| 0.723736 | 3.291846 | 0.950193 | 3.990674 | 0.001098 | 3.059685 | 0.568444 | 2 |
| 2.182197 | 3.841742 | 3.585516 | 1.894945 | -0.17265 | 1.744152 | 0.364155 | 2 |
| 3.352942 | 2.882326 | 3.866515 | 1.546324 | 0.773397 | 0.696639 | 1.2335 | 3 |
| 2.389582 | 2.199895 | 5.216224 | 1.660491 | 0.991467 | 0.364649 | 1.546675 | 4 |
| 1.212857 | 3.882324 | 5.050131 | 1.263146 | -0.44613 | 1.522973 | 1.118274 | 4 |
| 0.472468 | 3.753695 | 4.995122 | 2.815492 | 0.027114 | 1.436463 | 0.056062 | 4 |
| 0.938919 | 3.164955 | 5.159946 | 0.67008 | 1.569086 | 0.043587 | 1.313561 | 4 |
| 1.298786 | 3.083568 | 1.830169 | 2.236362 | 2.000518 | 3.179449 | 1.594717 | 1 |
| 0.366913 | 2.044937 | 2.617066 | 3.038203 | 3.593626 | 1.970333 | 0.407605 | 1 |
| -0.20437 | 3.531738 | 2.182952 | 2.036282 | 1.892294 | 2.801329 | 1.66814 | 1 |
| 0.28563 | 2.587021 | 2.643787 | 2.445734 | 3.925445 | 0.792276 | 0.350427 | 1 |
| 0.996504 | 3.106436 | 2.692807 | 1.902592 | 3.575833 | 1.568171 | -0.2585 | 1 |
| 2.260508 | 3.017908 | 2.137207 | 1.674803 | 1.196457 | 2.873861 | 1.848838 | 2 |
| -0.03506 | 3.609465 | 2.625299 | 2.368762 | 1.671222 | 3.0121 | 1.916716 | 1 |
| 0.854331 | 1.998625 | 3.000042 | 3.004479 | 3.726537 | 1.246325 | 0.524352 | 1 |
| 0.262891 | 2.741493 | 2.465511 | 3.593546 | 2.739738 | 1.530374 | 0.298851 | 1 |
| 2.270781 | 2.561758 | 2.539467 | 0.271137 | 3.602786 | 0.407443 | 0.328955 | 3 |
| 1.318672 | 2.621613 | 2.430487 | 2.202098 | 3.112685 | 0.926337 | 0.382588 | 1 |
| 1.473336 | 3.617204 | 2.026884 | 3.569903 | 3.190754 | 1.528451 | 0.754648 | 1 |
| 3.029609 | 3.419414 | 0.786625 | 4.327039 | 3.598551 | 1.734834 | 0.51481 | 1 |
| 1.792849 | 2.884772 | 2.081495 | 3.645535 | 2.82959 | 1.953796 | 0.623779 | 1 |
| 1.334464 | 2.874837 | 2.544076 | 3.153225 | 2.856396 | 1.395013 | 0.581578 | 1 |
| 1.368727 | 3.383985 | 2.730762 | 3.125914 | 3.853141 | 1.181855 | 0.793415 | 1 |
| 1.158614 | 2.646456 | 2.146818 | 2.3928 | 2.766568 | 2.142429 | 1.291993 | 1 |
| 0.880486 | 3.031536 | 2.821478 | 1.423451 | 0.733423 | 2.545687 | 1.142586 | 2 |
| 1.174285 | 2.721081 | 2.441791 | 2.207948 | 1.827167 | 2.157325 | 0.964771 | 1 |
| 0.870188 | 3.398999 | 2.271434 | 2.450359 | 2.154208 | 1.686502 | 0.205592 | 1 |
| 1.653495 | 3.671909 | 1.899133 | 3.211423 | 3.15191 | 1.735527 | 0.69995 | 1 |

Document: PPD

Author: PPD


06MAY2024

| 0.682774 | 4.503063 | 1.489453 | 2.222444 | 1.302957 | 2.698368 | 1.259985 | 11 |
|---|---|---|---|---|---|---|---|
| 2.663757 | 3.054066 | 3.250958 | 2.184488 | 2.114672 | 1.565751 | 0.71493 | 3 |
| -0.03549 | 2.627792 | 3.353033 | 2.490402 | 1.333189 | 3.449527 | 2.01461 | 1 |
| 0.176902 | 3.363572 | 1.788922 | 2.632445 | 2.046902 | 1.661218 | 1.862941 | 1 |
| 1.665005 | 3.096207 | 1.841999 | 2.76653 | 2.242893 | 2.006812 | 0.692106 | 1 |
| 0.434799 | 3.054804 | 2.514313 | 1.468836 | 0.715913 | 1.864575 | 0.778837 | 4 |
| 2.414456 | 2.360334 | 2.306623 | 2.052518 | 1.905444 | 2.084339 | 1.41141 | 3 |
| 1.548719 | 2.645218 | 2.647588 | 3.017119 | 1.307344 | 2.603688 | 1.402963 | 2 |
| 1.043513 | 2.563992 | 0.768526 | 3.563116 | 1.338746 | 4.07294 | 0.737781 | 2 |
| 2.75563 | 2.346252 | 3.231356 | 2.059784 | 2.305691 | 0.999648 | 2.35069 | 3 |
| 1.618229 | 1.55903 | 2.663824 | 2.071062 | 1.269606 | 2.184555 | 2.946364 | 5 |
| 1.927056 | 2.062933 | 2.708249 | 2.422282 | 0.670938 | 1.652872 | 0.78742 | 2 |
| 1.888032 | 1.739451 | 3.022219 | 0.731892 | 0.901051 | 1.484288 | 2.493283 | 3 |
| 1.373058 | 3.726288 | 2.173993 | 1.611522 | 1.419764 | 1.355206 | 1.332446 | 1 |
| 1.587711 | 4.845681 | 1.633788 | 2.276364 | 0.613327 | 2.951609 | 0.774923 | 2 |
| 1.107882 | 4.1896 | 0.662106 | 3.017648 | 2.54298 | 3.18947 | 1.811624 | 1 |
| 0.80748 | 4.128602 | 3.05368 | 0.753182 | 1.523971 | 2.218486 | 1.551826 | 1 |
| 1.792069 | 5.297029 | -1.4584 | 4.517665 | 0.420555 | 3.75568 | -0.2235 | 2 |
| 0.29681 | 2.154562 | 4.291881 | -0.71309 | 3.192156 | 4.1492 | 2.884095 | 1 |
| 2.641933 | 4.808604 | 1.697382 | 3.192166 | 0.262471 | 2.395388 | 1.412021 | 2 |
| 1.862043 | 3.096722 | 2.942964 | 1.87311 | 2.463407 | 1.027912 | 2.61095 | 3 |
| 2.842538 | 4.881212 | 0.084864 | 3.656311 | 1.139249 | 2.492176 | 1.855205 | 2 |
| -0.56891 | 4.003578 | 3.196236 | 3.384194 | 0.419863 | 2.238542 | 0.05731 | 2 |
| 2.881629 | 2.605602 | 4.146121 | 2.6831 | -0.69501 | 1.296744 | 1.351407 | 2 |
| 1.066547 | 2.269026 | 3.176295 | 3.933355 | 0.905649 | 3.788415 | 2.012815 | 2 |
| -0.27702 | 5.214505 | 3.964305 | -0.42548 | 3.649732 | 1.399817 | 2.064414 | 1 |
| 3.247233 | 1.250798 | 1.933796 | 3.519258 | 1.290077 | 3.216229 | 3.350252 | 5 |
| 5.269156 | 3.595336 | 1.57854 | 4.563517 | 3.322321 | 2.0089 | 2.253221 | 3 |
| 0.402385 | 3.988677 | 1.888783 | 3.045963 | 2.415748 | 2.16155 | 2.283636 | 11 |
| 1.305141 | 3.669467 | 2.596833 | 3.356985 | 1.244654 | 1.832795 | 2.358681 | 1 |
| 1.198453 | 3.482618 | 2.315618 | 2.959246 | 0.01394 | 2.162574 | 0.785387 | 2 |
| 2.34431 | 4.126819 | 2.223733 | 1.390981 | 1.353677 | 1.772295 | 1.929 | 3 |
| 1.125582 | 2.252314 | 3.475507 | 3.005104 | 1.493761 | 0.598888 | 1.6825 | 4 |
| 0.540524 | 2.337962 | 4.474714 | 1.180037 | 1.137322 | 1.401177 | 1.350397 | 4 |
| 0.605022 | 2.493479 | 3.007678 | 3.416692 | 1.835619 | 3.153643 | 1.208213 | 1 |
| 1.70579 | 2.90063 | 2.763136 | 3.22817 | 2.736035 | 1.453346 | 1.065606 | 1 |
| 1.774505 | 2.964929 | 4.050098 | 0.483415 | 1.620176 | 2.106961 | 1.469905 | 3 |
| 0.37949 | 3.798105 | 3.253912 | 2.618223 | 2.893426 | 1.931221 | 1.662662 | 1 |
| 4.088323 | 4.086708 | 1.203542 | 3.401486 | 1.006494 | 1.889707 | 1.626608 | 2 |
| 1.119508 | 1.699654 | 3.586956 | 2.997562 | 1.258626 | 1.989826 | 0.903255 | 4 |
| 0.613604 | 3.759827 | 3.856952 | 2.125737 | 1.154775 | 0.907478 | 1.761888 | 4 |
| 0.907833 | 2.530289 | 2.395073 | 2.958473 | 0.736132 | 1.751963 | 0.549846 | 2 |
| 3.173489 | 3.591836 | 4.33018 | 2.384611 | 3.189142 | 3.388148 | 1.267663 | 3 |
| 0.198984 | 2.664969 | 2.869373 | 4.610011 | 0.313022 | 2.824204 | 0.625394 | 2 |
| 0.630253 | 2.095562 | 4.612635 | 3.10251 | 0.403171 | 0.586135 | 1.524354 | 4 |
| 1.172078 | 3.404195 | 2.258 | 4.688623 | 0.018005 | 3.749981 | 0.113934 | 2 |
| 4.007734 | 4.416939 | 3.65958 | 2.156696 | 1.668164 | 2.136666 | -0.46751 | 3 |
| 1.868898 | 3.149336 | 2.275342 | 3.520585 | 0.30994 | 2.832434 | 1.386088 | 2 |
| 0.780472 | 3.074664 | 2.209664 | 2.923805 | 1.234535 | 3.130313 | 0.715847 | 2 |
| 4.848926 | 2.952455 | 3.823995 | 0.591641 | 1.587537 | 2.18594 | -0.83412 | 3 |
| 1.211911 | 3.276599 | 1.160352 | 3.7608 | 0.172588 | 3.302692 | 0.900316 | 2 |
| 1.345695 | 4.407982 | 2.247066 | 3.577123 | 1.592001 | 1.564087 | 2.094433 | 1 |
| 1.224475 | 3.147634 | 2.941942 | 3.798999 | 1.535248 | 2.344394 | 1.478652 | 2 |
| 3.814597 | 3.334847 | 3.097241 | 4.383301 | 1.594088 | 3.575003 | 2.193627 | 2 |
| 2.618453 | 3.317255 | 1.941214 | 3.630248 | 2.69847 | 3.52205 | 2.648051 | 1 |
| 1.294275 | 1.56371 | 3.043611 | 2.412047 | 2.498057 | 1.647309 | 1.693621 | 5 |
| 0.789672 | 3.383044 | 3.337881 | 3.451955 | 2.680502 | 1.791768 | -0.33461 | 1 |
| | | | | 3.165442 | | | |
| 5.565368<br>0.669129 | 3.181652 | 3.711348 | 1.365467 | | 0.633596 | 1.577293 | 3 |
| U 009179 | 2.118351 | 2.117884 | 2.709941 | 1.785749 | 2.353919 | 1.396308 | 1 |

Document: PPD

Author: PPD


06MAY2024



| 0.400074 | 0.070500 | 4.000400 | 0.044000 | 4 404000 | 0.054004 | 4.040047 | 0 |
|---|---|---|---|---|---|---|---|
| 2.122874 | 2.370528 | 4.039168 | 0.044906 | 1.404239 | 0.054061 | 1.210217 | 3 |
| -0.31367 | 1.429249 | 3.608487 | 3.153238 | 3.435385 | 2.595252 | 1.562 | 1 |
| 2.998431 | 3.071495 | 3.935008 | -0.03663 | 1.493068 | -0.0469 | 0.969036 | 3 |
| 1.208636 | 1.198679 | 3.797957 | 1.94229 | 3.154749 | 1.181498 | 1.587801 | 5 |
| 1.238483 | 2.984314 | 4.102558 | 1.020331 | 1.746735 | 0.210602 | 0.596202 | 4 |
| 0.721211 | 2.570974 | 4.789879 | 1.510915 | 0.470652 | 0.495575 | 0.773934 | 4 |
| 2.182478 | 2.318548 | 4.180739 | 2.217635 | 1.400813 | 1.181345 | 1.366411 | 3 |
| 4.973196 | 1.25845 | 3.181555 | 1.930606 | 1.754247 | 0.502145 | 0.808431 | 3 |
| 1.299859 | 3.358898 | 2.963783 | 2.996693 | 1.210242 | 2.837687 | 2.661287 | 1 |
| 1.721604 | 4.747844 | 2.938984 | 3.246941 | 0.280358 | 1.577821 | -0.18553 | 2 |
| 2.151246 | 2.475189 | 2.327683 | 1.99312 | 0.50071 | 1.478181 | 2.367488 | 3 |
| -0.52803 | 2.946022 | 3.74577 | 3.453622 | 1.366665 | 1.530891 | 2.898386 | 4 |
| 2.520474 | 2.840891 | 4.605005 | 2.492233 | 1.505935 | 0.933693 | 1.547949 | 3 |
| 1.953568 | 4.710961 | 2.059415 | 3.21843 | 0.404182 | 2.072298 | -0.48158 | 2 |
| 0.67322 | 2.059827 | 3.378463 | 3.263051 | 1.593942 | 1.411997 | 3.478853 | 5 |
| 0.482849 | 1.669846 | 5.337114 | 3.92286 | 0.857681 | 2.098765 | 1.276031 | 4 |
| 1.436908 | 3.006341 | 2.111445 | 3.63576 | 1.17833 | 2.696489 | -0.03468 | 2 |
| -0.16469 | 3.037464 | 2.593747 | 2.19126 | 1.150814 | 1.183965 | 2.885273 | 1 |
| 3.098244 | 2.591925 | 4.55368 | 2.771836 | 0.409717 | 4.100465 | 1.1617 | 2 |
| 0.287138 | 2.638836 | 3.863141 | 2.410391 | 1.952481 | 0.480413 | 3.121472 | 4 |
| 0.88184 | 3.625722 | 4.892386 | 0.792852 | -0.38779 | 0.599907 | 0.319505 | 4 |
| 2.150267 | 2.531001 | 1.798742 | 1.734505 | 2.569138 | 1.474977 | 1.943503 | 3 |
| 0.080232 | 1.944229 | 2.89941 | 3.091852 | 1.297553 | 1.130481 | 1.479588 | 4 |
| 1.307558 | 3.242025 | 3.928579 | 0.550179 | 0.489302 | -0.2167 | 1.569607 | 4 |
| -0.23345 | 2.508582 | 4.13559 | 3.019692 | 1.012514 | 0.803014 | 2.163831 | 4 |
| 0.452287 | 4.095796 | 2.938024 | 2.755959 | 1.197267 | 1.736364 | 1.48946 | 1 |
| 0.333146 | 3.491975 | 2.998474 | 2.348185 | 2.863105 | 2.005441 | 1.99996 | 1 |
| -0.2021 | 2.38004 | 4.119341 | 2.26864 | 1.40722 | 0.247862 | 1.495971 | 4 |
| 1.27648 | 2.71056 | 3.416199 | 3.573639 | 1.124956 | 2.475951 | 1.110492 | 2 |
| 1.071622 | 0.058392 | 4.1753 | 3.035761 | 3.147516 | 0.463041 | 3.434267 | 5 |
| 0.767058 | 2.902141 | 2.81539 | 1.046366 | 3.481824 | 2.314722 | 3.456745 | 1 |
| 3.199205 | 1.794078 | 3.094138 | 0.666184 | 2.680831 | 0.969656 | 3.012809 | 3 |
| 0.381606 | 1.855712 | 2.180899 | 2.28543 | 2.69681 | 2.129198 | 3.061778 | 5 |
| 1.199252 | 1.771864 | 3.210781 | 2.048203 | 2.117378 | 1.37389 | 2.377955 | 5 |
| 0.91132 | 1.981741 | 2.199601 | 2.419341 | 2.215353 | 2.0596 | 2.989397 | 5 |
| 1.465285 | 2.997421 | 3.137443 | 1.03661 | 2.101259 | 0.412757 | 0.556006 | 3 |
| 1.445957 | 2.331573 | 1.916218 | 2.899514 | 1.818489 | 2.843057 | 2.654736 | 1 |
| 2.190434 | 2.781964 | 2.697725 | 2.215768 | 1.935821 | 3.086303 | 2.382583 | 1 |
| 3.060515 | 2.893715 | 3.843192 | 1.274351 | 2.77693 | 1.999967 | 1.625444 | 3 |
| 3.43918 | 4.685975 | 2.511207 | 0.606142 | 2.48964 | 0.899216 | 2.126643 | 3 |
| 2.248858 | 3.078349 | 2.536622 | 1.289691 | 2.240462 | 3.084218 | 2.519339 | 1 |
| 3.37998 | 3.32946 | 4.457823 | 2.144631 | 1.21309 | 0.40427 | 0.75011 | 3 |
| 1.485575 | 0.653133 | 3.573337 | 1.804786 | 2.614735 | 1.700206 | 2.294768 | 5 |
| -0.11639 | 1.697496 | 3.894954 | 1.163997 | 2.803677 | 1.62084 | 3.170209 | 5 |
| 0.265337 | 0.794674 | 3.483188 | 3.196532 | 2.270673 | 0.733305 | 3.105335 | 5 |
| 0.487467 | 2.134018 | 3.509739 | 2.158815 | 1.670326 | 3.086941 | 1.766996 | 1 |
| 1.785974 | 2.325783 | 3.97547 | 1.09789 | 1.533602 | 0.00662 | 0.661087 | 3 |
| 2.199662 | 1.043731 | 3.230455 | 1.471481 | 1.594108 | 0.196087 | 1.699968 | 3 |
| 0.432774 | 0.473242 | 3.749216 | 2.000787 | 2.260527 | 2.0028 | 2.936089 | 5 |
| -0.03225 | 1.823518 | 3.460935 | 2.026709 | 2.073493 | 1.822957 | 2.199521 | 4 |
| 2.922641 | 1.912792 | 2.869191 | 1.92473 | 2.23171 | 1.463312 | 1.771086 | 3 |
| 1.95851 | 2.620691 | 3.209711 | 2.40885 | 2.167502 | 1.410435 | 0.780651 | 3 |
| 1.673373 | 3.1535 | 3.384783 | 2.665686 | 2.386609 | 3.045046 | 1.306632 | 1 |
| 2.052142 | 2.801713 | 3.616672 | 2.376778 | 2.198514 | 2.571284 | 2.109671 | 1 |
| 2.398755 | 2.656117 | 3.599123 | 2.113145 | 1.85368 | 1.955369 | 1.029531 | 3 |
| 1.600749 | 2.772373 | 2.97559 | 2.356207 | 2.179088 | 2.727056 | 2.963031 | 1 |
| 2.407436 | 2.876793 | 3.588069 | 2.349736 | 2.603454 | 1.472847 | 1.481762 | 3 |
| 1.477092 | 2.367975 | 3.279323 | 3.706314 | 2.496294 | 1.970748 | 2.027569 | 5 |
| 2.117032 | 3.129461 | 3.33882 | 2.353723 | 1.303854 | 3.213898 | 2.046513 | 2 |
| | | | , | , , , , , , | | | <del></del> |

Document: PPD

Author: Version Number:


| 2 222252 | 4 =0=004 | 4 000==0 | 0.000004 | 4 =00=04 | 4 = 0 = 0 0 | 0.040040 | |
|---|---|---|---|---|---|---|---|
| 0.862852 | 1.787891 | 4.693773 | 3.920364 | 1.536504 | 1.598562 | 0.812846 | 4 |
| 2.124976 | 2.522997 | 2.142115 | 2.017715 | 1.329319 | 1.353485 | 2.01721 | 3 |
| 2.053942 | 1.282666 | 2.60817 | 2.173067 | 1.883355 | 1.446771 | 1.932743 | 5 |
| 1.051968 | 1.351924 | 2.743535 | 2.133289 | 2.15663 | 1.277404 | 1.947453 | 5 |
| 1.711215 | 1.470019 | 2.419263 | 1.720749 | 1.882597 | 1.273467 | 2.368535 | 5 |
| 2.929092 | 1.337477 | 2.249875 | 2.137536 | 0.784348 | 1.365049 | 2.001452 | 3 |
| 1.158983 | 1.4628 | 2.915975 | 1.823459 | 1.509886 | 0.551248 | 2.793893 | 5 |
| 2.091268 | 1.750324 | 3.37735 | 1.24898 | 0.459163 | 1.414763 | 2.315137 | 3 |
| 2.076045 | 1.774582 | 2.512304 | 2.256736 | 1.866886 | 1.14936 | 2.611307 | 5 |
| 0.888772 | 2.398703 | 2.96251 | 3.053851 | 0.409217 | 0.752585 | 2.749108 | 4 |
| 1.385868 | 2.726663 | 4.786969 | 1.926702 | -0.29151 | 1.447619 | 0.300511 | 4 |
| 1.573504 | 1.385677 | 2.765509 | 1.797339 | 2.803497 | 0.70662 | 1.886113 | 5 |
| 1.36709 | 2.250416 | 2.120969 | 3.156059 | 0.953453 | 0.834286 | 0.332707 | 2 |
| 1.83963 | 1.020248 | 2.261243 | 3.005754 | 1.931713 | 0.376005 | 1.855818 | 5 |
| 1.601561 | 1.25261 | 2.891928 | 2.486944 | 1.195034 | 1.634183 | 1.888287 | 5 |
| -0.02354 | 3.287441 | 3.06615 | 1.477316 | 0.788567 | 1.769741 | 0.388055 | 4 |
| 1.218747 | 0.968508 | 2.310128 | 1.840931 | 3.599996 | 2.546517 | 2.353331 | 5 |
| 2.273433 | 1.691484 | 4.048696 | 2.607554 | 3.589263 | 1.255111 | 0.435131 | 3 |
| 2.088968 | 1.147388 | 2.211211 | 2.663832 | 2.513624 | 1.159295 | 2.510907 | 5 |
| 1.671819 | 1.377036 | 3.442522 | 3.119088 | 2.535569 | 0.140997 | 2.209565 | 5 |
| 0.655599 | 2.044898 | 3.029 | 2.970167 | 1.316146 | 2.118602 | 2.10233 | 4 |
| 1.85728 | 0.119835 | 2.531109 | 2.346743 | 1.542376 | 2.049295 | 3.632266 | 5 |
| 0.810013 | 0.519835 | 2.208672 | 2.690966 | 1.793883 | 2.252788 | 3.340709 | 5 |
| -0.53672 | 1.90413 | 3.751989 | 2.896342 | 2.684364 | 0.736452 | 2.240227 | 4 |
| 0.912099 | 0.843401 | 3.863282 | 1.466242 | 1.900905 | 1.511621 | 3.068371 | 5 |
| 0.717642 | 1.816272 | 2.257425 | 3.060543 | 1.17801 | 1.755652 | 3.457668 | 5 |
| -0.58683 | 3.081178 | 4.155074 | 3.340262 | -0.52844 | 2.870146 | 1.44833 | 4 |
| 0.948814 | 1.329927 | 2.309509 | 2.638619 | 2.425392 | 2.050609 | 2.055008 | 5 |
| 1.405381 | 2.577678 | 4.286141 | 1.980834 | 2.432689 | -0.09613 | 1.148452 | 4 |
| 1.567328 | 2.933253 | 3.513708 | 2.585126 | 1.043179 | -0.13341 | 2.420696 | 4 |
| 0.654842 | 2.497284 | 3.603089 | 3.237035 | 1.70472 | 1.099211 | 1.797649 | 4 |
| 1.512999 | 0.611854 | 2.683634 | 2.169291 | 2.81694 | 1.732635 | 3.711279 | 5 |
| 1.750541 | 0.9083 | 3.874494 | 4.076287 | -0.0004 | 3.253308 | 1.558526 | 2 |
| 3.554138 | 3.798572 | 3.92936 | 3.171349 | 1.134508 | -0.27824 | 2.674967 | 3 |
| 1.843493 | 2.035074 | 1.975868 | 1.991719 | 2.417606 | 0.563503 | 2.469965 | 5 |
| 1.717436 | 2.392262 | 3.051026 | 2.060343 | 2.753362 | 1.495397 | 3.641729 | 5 |
| -0.42161 | 4.174919 | 2.381554 | 3.388356 | 0.438055 | 3.444924 | 1.033751 | 2 |
| 1.763247 | 1.821026 | 3.455334 | 0.63166 | 3.032002 | 1.410237 | 2.909767 | 5 |
| 1.676444 | 2.552671 | 2.604784 | 0.875316 | 1.878914 | -0.17302 | 2.688803 | 3 |
| 2.421358 | 0.897852 | 1.757336 | 1.945325 | 2.978777 | 0.589719 | 2.963783 | 5 |
| 1.091983 | 1.664438 | 3.094837 | 2.810642 | 2.668531 | 3.176472 | 3.365537 | 5 |
| 0.95825 | 2.322112 | 2.79394 | 1.357469 | 2.849933 | 1.464401 | 1.685897 | 11 |
| 1.686879 | 1.209325 | 2.357908 | 1.591704 | 2.3949 | 2.815835 | 3.473977 | 5 |
| 0.679991 | 0.490045 | 3.649338 | 3.121814 | 3.233997 | 1.803668 | 3.433076 | 5 |
| 0.576465 | 1.683357 | 3.679851 | 3.021204 | 2.972976 | 2.905107 | 2.180476 | 5 |
| 0.136986 | 3.709519 | 2.895228 | 2.006352 | 2.08725 | 0.559701 | 0.559701 | 4 |
| 1.992158 | 1.887124 | 2.751854 | 4.05701 | 2.787676 | 3.611463 | 1.616108 | 11 |
| 2.188311 | 1.67236 | 3.624552 | 2.120629 | 2.385157 | -0.40732 | 2.290743 | 3 |
| 1.103505 | 3.213246 | 3.56517 | 1.335934 | 2.322979 | 2.073316 | 2.533389 | 1 |
| 1.172266 | 1.179647 | 3.3055 | 0.938081 | 2.639 | 3.333973 | 2.398904 | 5 |
| 0.946777 | 1.12983 | 3.224024 | 2.29541 | 2.958102 | 2.775739 | 1.638153 | 5 |
| 1.180773 | 2.20079 | 3.909757 | 0.784649 | 2.537993 | 1.654572 | 2.353767 | 4 |
| -0.29837 | 2.708103 | 4.010237 | 3.212327 | 2.782713 | 2.544077 | 2.617483 | 1 |
| 0.999984 | 1.601736 | 3.175787 | 1.809006 | 2.008332 | 2.584361 | 2.924514 | 5 |
| 1.191219 | 1.61463 | 2.640179 | 2.097072 | 2.463071 | 2.923712 | 2.126753 | 5 |
| 0.81584 | 1.766591 | 1.901241 | 3.201082 | 3.089132 | 1.507481 | 2.906519 | 5 |
| -0.52005 | -0.21152 | 3.877069 | 3.117811 | 2.445868 | 1.942376 | 3.528102 | 5 |
| 0.698561 | 1.581811 | 3.206016 | 2.966686 | 2.174549 | 2.628289 | 3.4346 | 5 |
| 0.294319 | 1.243359 | 3.264264 | 2.504067 | 2.125595 | 1.764063 | 2.399821 | 5 |

Document: PPD

Author: Version Num


1.0

06MAY2024



#### Statistical Analysis Plan

| 0.550500 | 4.04400 | 0.000707 | 0.050400 | 4.000004 | 4.004744 | 0.040400 | 4 |
|---|---|---|---|---|---|---|---|
| 0.552522 | 1.94189 | 3.663707 | 2.656138 | 1.682984 | 1.361744 | 2.218496 | 4 |
| 3.133129 | -0.27546 | 2.912236 | 2.424335 | 1.345903 | 0.670599 | 2.517861 | 5 |
| -0.24638 | 0.480544 | 3.246561 | 3.188092 | 2.920533 | 2.712854 | 0.739785 | 5 |
| 1.14412 | 0.149335 | 2.163497 | 1.884293 | 2.33313 | 3.013641 | 3.065498 | 5 |
| 1.106268 | 1.42373 | 4.030908 | 3.058467 | 1.784729 | 1.151248 | 3.145549 | 5 |
| 1.747898 | 2.289926 | 3.193032 | 2.342344 | 1.836667 | 2.341647 | 2.572253 | 5 |
| 1.249783<br>1.369205 | 1.366357 | 1.891003 | 3.500575 | 2.873969 | 2.428008 | 3.977269 | 5 |
| | 1.426718 | 3.489257 | 2.725576 | 2.382661 | 1.919912 | 3.088201 | 5 |
| 2.047065 | 0.823226 | 2.345861 | 3.062785 | 1.533924 | 2.751118 | 4.369498 | 5 |
| 1.665568 | 1.758852 | 2.102023 | 2.36764 | 1.985868 | 2.164683 | 2.997736 | 5 |
| 1.235974 | 1.308576 | 2.981051 | 2.429463 | 1.928441 | 2.464002 | 2.952178 | 5 |
| 1.8261 | 1.512971 | 3.123711 | 2.497745 | 2.373443 | 2.094497 | 3.044643 | 5 |
| 2.84051 | 1.175393 | 2.586929 | 3.28986 | 2.33567 | 2.090763 | 3.742619 | 5 |
| 0.279548 | 1.895825 | 5.388341 | 2.120073 | 2.247174 | 0.868701 | 1.081032 | 4 |
| 0.99619 | 1.012696 | 1.960564 | 3.89922 | 2.166986 | 3.011827 | 2.011537 | 5 |
| 0.40928<br>0.215144 | 3.185794<br>2.091797 | 2.623647 | 1.940549<br>2.320654 | 1.825407<br>3.369494 | 1.698621<br>3.191467 | 1.568015<br>1.64836 | 1<br>1 |
| 2.510542 | 2.017149 | 4.171211<br>2.234838 | 3.722974 | 3.594265 | 1.538423 | 4.527227 | 5 |
| 2.191789 | 2.27999 | 0.75166 | 3.750002 | 2.901422 | 1.686636 | 2.481703 | 5 |
| 3.326313 | 2.528328 | 3.928792 | 3.121216 | 1.453615 | 1.682897 | 1.617506 | 3 |
| 1.664394 | 3.09397 | 1.78878 | 1.884236 | 2.924941 | 1.515557 | 2.520133 | <u> </u> |
| 3.639972 | 2.296478 | 1.151978 | 4.058536 | 3.114612 | 3.240043 | 1.390437 | 2 |
| 0.449924 | 1.48284 | 0.97592 | 2.929817 | 3.717695 | 4.493118 | 4.460917 | 5 |
| 2.003783 | 1.617244 | 1.483172 | 3.165291 | 2.814826 | 1.544825 | 3.40854 | 5 |
| 1.642709 | 2.599317 | 2.743092 | 2.478182 | 1.216038 | 1.569686 | 2.955092 | 5 |
| 2.020474 | 3.031131 | 1.458374 | 1.963512 | 2.002057 | 0.863468 | 1.791431 | 3 |
| 1.588088 | 1.83981 | 1.621011 | 2.296312 | 2.576374 | 1.595488 | 3.050562 | 5 |
| -0.03704 | 2.618573 | 2.73468 | 3.523944 | 1.728803 | 3.092423 | 1.011341 | 1 |
| 1.507168 | 2.289949 | 2.907394 | 2.494175 | 0.342619 | 2.955806 | 2.238876 | 2 |
| 0.65722 | 1.948092 | 3.384632 | 3.591149 | 1.093019 | 1.948022 | 2.226399 | 4 |
| 0.906972 | 2.341611 | 3.474023 | 3.766265 | 1.319244 | 2.054854 | 0.849818 | 2 |
| 1.099988 | 2.333797 | 3.238913 | 2.937232 | 0.493977 | 1.700426 | 1.402933 | 4 |
| 1.280015 | 2.513557 | 2.225763 | 1.868445 | 1.739776 | 1.374607 | 1.782267 | 1 |
| -0.11139 | 2.095035 | 2.947376 | 3.142256 | 3.032293 | 1.639643 | 0.480099 | 1 |
| 1.551912 | 1.887402 | 2.344782 | 3.686308 | 2.768613 | 2.681956 | 1.157552 | 1 |
| -0.08866 | 3.745314 | 2.220336 | 3.071661 | 2.849671 | 1.862011 | 1.695552 | 1 |
| -0.14035 | 2.459132 | 2.989569 | 2.991661 | 2.682929 | 2.55258 | 1.272708 | 1 |
| 0.863472 | 1.802155 | 2.07836 | 2.793182 | 3.686965 | 2.535373 | 3.223135 | 5 |
| 1.939982 | 1.028043 | 2.661535 | 3.283031 | 2.849478 | 1.791159 | 2.935827 | 5 |
| 0.202088 | 2.772472 | 3.860564 | 2.418321 | 1.221271 | 2.686473 | 3.045804 | 4 |
| 1.536423 | 3.963189 | 3.539271 | 3.213546 | 2.934773 | 0.878772 | 1.750439 | 1 |
| 0.716654 | 3.769872 | 2.337558 | 3.21909 | 3.257411 | 3.09655 | 1.200753 | 1 |
| 0.002053 | 2.579149 | 1.708619 | 1.826842 | 2.902119 | 2.69227 | 1.846354 | 1 |
| 1.878384 | 1.367029 | 2.529927 | 2.219242 | 3.170144 | 1.372932 | 2.595525 | 5 |
| 1.113165 | 4.083788 | 2.197008 | 2.347144 | 2.640993 | 3.571014 | 1.565829 | 1 |
| -0.55411 | 3.677333 | 2.607452 | 2.868568 | 1.895632 | 1.742989 | 1.350166 | 1 |
| 0.728818 | 5.38512 | 1.999552 | 1.995521 | 1.688124 | 1.794364 | 1.567654 | 11 |
| 2.000957 | 2.156025 | 2.529648 | 2.916682 | 2.007876 | 1.796838 | 1.507756 | 3 |
| 1.464876 | 4.794305 | 2.399407 | 2.661065 | 2.77422 | 2.379961 | 2.595127 | 1 |
| 1.639087 | 2.011963 | 1.930406 | 2.611254 | 3.568298 | 2.516589 | 2.812242 | 5 |
| 1.446411 | 3.638014 | 2.57226 | 2.162072 | 2.791145 | 2.57307 | 1.488721 | 1 |
| 1.167265 | 2.626558 | 2.203502 | 2.296486 | 1.842762 | 2.90644 | 1.855448 | 1 |
| 2.792874 | 1.787912 | 2.792314 | 2.672087 | 2.421138 | 2.292698 | 1.817582 | 3 |
| 1.661313 | 1.518343 | 3.330552 | 2.900845 | 1.686547 | 3.210328 | 0.977498 | 2 |
| 1.818558 | 1.962483 | 3.011182 | 2.984796 | 2.464553 | 2.212576 | 2.227476 | 5 |
| 2.368946 | 1.765466 | 2.807844 | 3.021599 | 1.988137 | 2.766653 | 1.264226 | 2 |
| 1.519612 | 1.349884 | 2.745033 | 2.585421 | 1.414565 | 2.762992 | 0.696093 | 2 |
| 2.525452 | 1.940259 | 3.229155 | 2.42824 | 1.51069 | 1.699371 | 0.8384 | 3 |
| 1.470027 | 2.213906 | 2.174315 | 2.641719 | 2.62319 | 2.124632 | 1.701656 | 1 |

Document: PPD

Author: Version Number: Version Date:



| 4 400=4 | 4 0 4 4 4 7 0 | 4.004040 | 0.00000 | 0.00=0=0 | 4 = 2 2 2 2 2 | 0.040=00 | |
|---|---|---|---|---|---|---|---|
| 1.40074 | 1.014476 | 4.221012 | 2.082268 | 2.397258 | 1.566852 | 2.246523 | 5 |
| 3.364591 | 1.251376 | 3.290845 | 2.500423 | 2.222562 | 2.499598 | 1.64981 | 3 |
| 2.129269 | 2.710131 | 2.313439 | 3.013249 | 3.038706 | 2.468915 | 1.469671 | 1 |
| 3.640786 | 2.112478 | 2.740796 | 2.354109 | 1.865754 | 1.397937 | 0.737311 | 3 |
| 1.421128 | 1.717524 | 3.14217 | 3.412806 | 1.643833 | 2.767619 | 1.014461 | 2 |
| 3.634259 | 3.829661 | 2.455371 | 1.544377 | 1.340034 | 3.256891 | 2.485461 | 3 |
| 2.697317 | 2.840325 | 2.636191 | 2.10339 | 1.209549 | 2.466469 | 1.862657 | 3 |
| 2.125605 | 1.718318 | 2.887255 | 2.48321 | 2.397532 | 1.066204 | 2.379777 | 5 |
| 3.792892 | 2.650793 | 2.764114 | 1.400925 | 1.851319 | 2.681576 | 2.986922 | 3 |
| 2.072001 | 3.045846 | 3.962105 | 2.177186 | 2.573999 | 0.25015 | 0.832666 | 3 |
| 3.47285 | 2.593043 | 2.890262 | 3.791422 | 0.974418 | 0.107865 | 1.905316 | 3 |
| 3.442853 | 2.49001 | 3.917911 | 2.182262 | 1.331236 | 0.624292 | 0.56678 | 3 |
| 2.219969 | 2.735774 | 2.653031 | 1.323758 | 1.209602 | 2.197175 | 1.866327 | 3 |
| 3.544702 | 2.323891 | 2.279193 | 1.803041 | 1.570909 | 2.167078 | 2.118647 | 3 |
| 3.420414 | 1.926201 | 3.185597 | 0.632802 | 0.632656 | 1.50262 | 1.384866 | 3 |
| 3.209916 | 2.705199 | 3.627112 | 1.981629 | 2.297275 | 1.142996 | 1.049544 | 3 |
| 3.048556 | 2.6651 | 3.121058 | 2.043578 | 1.409733 | 1.083988 | 0.612292 | 3 |
| 2.713898 | 2.765805 | 2.622923 | 3.012792 | 2.375676 | 2.068843 | 1.575362 | 3 |
| 2.443942 | 2.666966 | 2.428546 | 0.891082 | 0.771637 | 2.603498 | 1.684131 | 3 |
| 2.905297 | 3.397697 | 2.938849 | 1.225181 | 1.163792 | 1.690736 | 1.431206 | 3 |
| 3.593219 | 4.593676 | 2.85064 | 2.031216 | 0.486013 | 2.463427 | 1.85159 | 2 |
| 2.102827 | 2.396113 | 2.513477 | 3.23259 | 0.053848 | 0.624753 | 1.872851 | 2 |
| 1.064304 | 1.898978 | 2.016754 | 3.140289 | 0.964322 | 2.533744 | 1.1192 | 2 |
| 2.444071 | 2.783835 | 4.013843 | 2.538264 | -0.99133 | 1.913701 | 1.514094 | 2 |
| 0.597051 | 2.841435 | 3.260321 | 2.331223 | 2.770425 | 1.762876 | 1.657292 | 1 |
| 1.277791 | 1.224479 | 4.027602 | 2.223094 | 1.528438 | 1.553553 | 1.985067 | 4 |
| 2.544969 | 1.139785 | 3.265251 | 2.26823 | -0.46458 | 2.591822 | 0.882637 | 2 |
| 1.825547 | 1.669443 | 3.223452 | 3.179786 | -0.42529 | 1.875906 | 1.452051 | 2 |
| 2.962217 | 3.600508 | 5.143498 | 1.353762 | 0.671814 | 0.235175 | 0.560646 | 3 |
| 1.456116 | 2.008452 | 4.33278 | 2.854759 | 0.605656 | 0.405156 | 2.166573 | 4 |
| 0.626556 | 3.945301 | 3.324774 | 2.371494 | -0.03127 | 1.118954 | 0.265501 | 4 |
| -0.31383 | 2.113856 | 2.59672 | 1.908942 | 1.667484 | 2.524643 | 2.408832 | 1 |
| 1.228335 | 1.387955 | 5.154633 | 1.452413 | 1.155377 | 0.786883 | 1.862063 | 4 |
| 1.25387 | 2.254079 | 4.47892 | 1.999785 | 1.359129 | 0.771985 | 2.204713 | 4 |
| 2.077432 | 1.663845 | 5.072246 | 2.79507 | -0.51169 | 0.56814 | 0.610627 | 4 |
| 0.599443 | 1.280542 | 4.815207 | 2.746904 | 1.803925 | 0.649366 | 2.415114 | 4 |
| 0.598819 | 1.589002 | 4.750287 | 3.058779 | 1.458149 | 1.533219 | 1.688224 | 4 |
| 0.931227 | 2.847927 | 4.160636 | 2.13367 | 0.982232 | 1.452196 | 1.729529 | 4 |
| 0.316014 | 1.483445 | 5.063682 | 1.620782 | 1.363688 | 0.744981 | 2.184789 | 4 |
| 1.805851 | 0.751263 | 4.905275 | 2.126935 | 0.927103 | 0.411213 | 1.870546 | 4 |
| 1.817658 | 1.874295 | 3.402797 | 2.738788 | 0.632739 | 3.089684 | 0.283125 | 2 |
| 2.080507 | 1.479588 | 3.698097 | 2.018675 | 1.102444 | 3.123037 | 0.499457 | 2 |
| 2.155577 | 1.737956 | 3.83843 | 2.286946 | 1.14978 | 2.696318 | 0.43201 | 2 |
| 1.608477 | 1.801606 | 3.90294 | 2.616016 | 0.307342 | 3.013917 | 0.867098 | 2 |
| 2.281242 | 0.685045 | 2.986646 | 2.985925 | 1.546753 | 3.087632 | 0.720522 | 2 |
| 2.214117 | 0.65798 | 3.986178 | 2.320973 | 1.01724 | 3.012481 | 0.405324 | 2 |
| 0.781439 | 0.915361 | 4.091384 | 2.741706 | 1.203266 | 2.853794 | 0.715125 | 4 |
| 1.727043 | 2.106237 | 3.150811 | 3.001749 | 0.701208 | 2.788492 | 0.486409 | 2 |
| 1.728331 | 1.779813 | 3.270322 | 2.618096 | 0.884794 | 3.065053 | 0.971797 | 2 |
| 1.749562 | 1.403262 | 3.229064 | 3.006373 | 1.472604 | 2.900566 | 0.640564 | 2 |
| 0.679291 | 1.950655 | 4.747832 | 2.835375 | 0.382722 | 2.499583 | 0.591783 | 4 |
| 1.147152 | 1.826271 | 4.035526 | 2.320126 | -0.02238 | 3.159645 | 0.731292 | 2 |
| 1.941818 | 2.082537 | 2.989712 | 2.260192 | -0.00818 | 2.787371 | 1.151937 | 2 |
| 1.249031 | 1.527114 | 4.299129 | 2.535885 | -0.5818 | 2.879486 | 0.525447 | 2 |
| 1.19344 | 1.077144 | 4.43854 | 2.214834 | 1.010501 | 3.005332 | 0.498575 | 4 |
| 1.38946 | 2.086965 | 3.925157 | 2.506738 | 0.61587 | 2.518739 | 0.56424 | 4 |
| 1.877671 | 2.377552 | 3.591046 | 2.443115 | -0.60871 | 2.798473 | 0.648804 | 2 |
| 2.957277 | 2.94879 | 2.629078 | 2.712291 | 2.437214 | 2.745738 | 2.306572 | 3 |
| 2.992108 | 2.599115 | 2.293851 | 3.124804 | 2.015908 | 3.133204 | 2.268303 | 2 |

Document: PPD

Author: Version Number:

Version Number: 1.0 Version Date: 06MAY2024

| 1.728135 3 0.89866 3 0.108157 3 0.949288 3 1.685074 3 2.355394 2 1.392201 2 4.06007 1 2.515136 3 2.353872 3 3.092874 2 2.985002 3 2.991006 2 2.991006 2 2.992435 3 3.732834 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 3 2.089671 2 2.089671 2 2.088354 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 3.011791<br>3.382881<br>3.708311<br>3.70854<br>3.908633<br>3.335918<br>2.924333<br>2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.3356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 1.363058 2.602387 3.08077 4.751098 4.21671 4.22883 3.329398 3.262224 3.365211 4.366534 3.164015 3.277328 3.090189 3.149261 3.128822 3.712698 3.266269 4.925664 4.289369 4.52097 4.555364 3.980479 3.628399 4.51504 6.417695 5.504821 6.131995 6.237579 | 2.752717 3.073562 2.230172 2.833147 2.584499 2.169423 1.851904 3.078521 2.991789 2.666384 2.511792 3.030188 3.004494 2.913923 2.930944 3.228355 3.874878 2.483556 5.662817 0.52877 2.821781 1.786325 3.051233 3.199279 0.828802 0.619534 0.715511 | 2.051352<br>1.122538<br>1.323137<br>1.226326<br>1.12431<br>1.972558<br>1.452708<br>1.380314<br>1.430271<br>0.004945<br>0.303662<br>0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449<br>1.160781 | 2.988232<br>2.970503<br>1.21315<br>1.494066<br>2.357137<br>2.209607<br>1.768292<br>2.171287<br>1.604211<br>2.058869<br>2.456513<br>1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393<br>1.224874 | 2.550854<br>0.769473<br>0.775188<br>0.657168<br>1.324043<br>1.534274<br>1.320825<br>1.551109<br>1.31471<br>1.022499<br>1.106662<br>1.083689<br>0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979<br>0.05934 | 2<br>4<br>4<br>4<br>4<br>3<br>2<br>3<br>3<br>2<br>2<br>2<br>2 |
|---|---|---|---|---|---|---|---|
| 0.89866 3 0.108157 3 0.949288 3 1.685074 3 2.355394 2 1.392201 2 4.06007 1 2.515136 3 2.353872 3 3.092874 2 2.991006 2.498692 2.932435 3 3.732834 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 1.288354 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 3.708311<br>3.703654<br>3.908633<br>3.335918<br>2.924333<br>2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.143928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.08077<br>4.751098<br>4.21671<br>4.22883<br>3.329398<br>3.262224<br>3.365211<br>4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.230172 2.833147 2.584499 2.169423 1.851904 3.078521 2.991789 2.666384 2.511792 3.030188 3.004494 2.913923 2.930944 3.228355 3.874878 2.483556 5.662817 0.52877 2.821781 1.786325 3.051233 3.199279 0.828802 0.619534 | 1.323137 1.226326 1.12431 1.972558 1.452708 1.380314 1.430271 0.004945 0.303662 0.686356 0.234085 0.221522 0.71372 0.051874 1.708321 -0.84478 1.16513 1.356926 -0.36831 -0.66089 -1.17422 -0.98896 1.741449 | 1.21315 1.494066 2.357137 2.209607 1.768292 2.171287 1.604211 2.058869 2.456513 1.732787 1.989451 2.037312 1.97819 2.453515 0.299856 1.269878 2.814028 0.340221 1.590714 0.481637 0.352569 1.381106 0.852393 | 0.775188 0.657168 1.324043 1.534274 1.320825 1.551109 1.31471 1.022499 1.106662 1.083689 0.991129 0.911563 0.9461 0.868749 2.488879 -0.24187 1.745695 0.917349 0.438113 0.032882 0.381981 0.015064 0.681979 | 4<br>4<br>4<br>4<br>3<br>2<br>3<br>3<br>2<br>2<br>2<br>2 |
| 0.108157 3 0.949288 3 1.685074 3 2.355394 2 1.392201 2 1.872292 2 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.98354 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 3.703654<br>3.908633<br>3.335918<br>2.924333<br>2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.143928<br>1.765644<br>4.3356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.751098<br>4.21671<br>4.22883<br>3.329398<br>3.262224<br>3.365211<br>4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.833147 2.584499 2.169423 1.851904 3.078521 2.991789 2.666384 2.511792 3.030188 3.004494 2.913923 2.930944 3.228355 3.874878 2.483556 5.662817 0.52877 2.821781 1.786325 3.051233 3.199279 0.828802 0.619534 | 1.226326 1.12431 1.972558 1.452708 1.380314 1.430271 0.004945 0.303662 0.686356 0.234085 0.221522 0.71372 0.051874 1.708321 -0.84478 1.16513 1.356926 -0.36831 -0.66089 -1.17422 -0.98896 1.741449 | 1.494066 2.357137 2.209607 1.768292 2.171287 1.604211 2.058869 2.456513 1.732787 1.989451 2.037312 1.97819 2.453515 0.299856 1.269878 2.814028 0.340221 1.590714 0.481637 0.352569 1.381106 0.852393 | 0.657168 1.324043 1.534274 1.320825 1.551109 1.31471 1.022499 1.106662 1.083689 0.991129 0.911563 0.9461 0.868749 2.488879 -0.24187 1.745695 0.917349 0.438113 0.032882 0.381981 0.015064 0.6681979 | 4<br>4<br>4<br>4<br>3<br>2<br>3<br>3<br>2<br>2<br>2<br>2 |
| 0.949288 3 1.685074 3 2.355394 2 1.392201 2 1.872292 2 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 2.089671 2 2.872695 2 2.089671 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 3.908633<br>3.335918<br>2.924333<br>2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.21671<br>4.22883<br>3.329398<br>3.262224<br>3.365211<br>4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.584499 2.169423 1.851904 3.078521 2.991789 2.666384 2.511792 3.030188 3.004494 2.913923 2.930944 3.228355 3.874878 2.483556 5.662817 0.52877 2.821781 1.786325 3.051233 3.199279 0.828802 0.619534 | 1.12431 1.972558 1.452708 1.380314 1.430271 0.004945 0.303662 0.686356 0.234085 0.221522 0.71372 0.051874 1.708321 -0.84478 1.16513 1.356926 -0.36831 -0.66089 -1.17422 -0.98896 1.741449 | 2.357137<br>2.209607<br>1.768292<br>2.171287<br>1.604211<br>2.058869<br>2.456513<br>1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.324043<br>1.534274<br>1.320825<br>1.551109<br>1.31471<br>1.022499<br>1.106662<br>1.083689<br>0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 4<br>4<br>3<br>2<br>2<br>3<br>2<br>3<br>3<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>2<br>2<br>3<br>2 |
| 1.685074 3 2.355394 2 1.392201 2 1.872292 2 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 2.089671 2 2.872695 2 2.089671 2 2.872695 3 2.089671 2 2.872695 3 2.089671 2 2.872695 3 2.089671 2 2.872695 3 2.089671 2 1.288354 2 1.624061 3 2.445324 3 1.445021 2 | 3.335918<br>2.924333<br>2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.22883 3.329398 3.262224 3.365211 4.366534 3.164015 3.277328 3.090189 3.149261 3.128822 3.712698 3.26629 4.925664 4.289369 4.52097 4.555364 3.980479 3.628399 4.51504 6.417695 5.504821 6.131995 | 2.169423<br>1.851904<br>3.078521<br>2.991789<br>2.666384<br>2.511792<br>3.030188<br>3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 1.972558<br>1.452708<br>1.380314<br>1.430271<br>0.004945<br>0.303662<br>0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.209607<br>1.768292<br>2.171287<br>1.604211<br>2.058869<br>2.456513<br>1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.534274 1.320825 1.551109 1.31471 1.022499 1.106662 1.083689 0.991129 0.911563 0.9461 0.868749 2.48879 -0.24187 1.745695 0.917349 0.438113 0.032882 0.381981 0.015064 0.681979 | 4<br>3<br>2<br>2<br>3<br>2<br>3<br>3<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>2<br>3<br>2<br>2<br>2<br>4<br>3<br>2<br>2<br>2<br>4<br>3<br>2<br>2<br>2<br>4<br>3<br>2<br>2<br>2<br>2 |
| 2.355394 2 1.392201 2 1.872292 2 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 2.088221 2 1.624061 3 2.445324 3 1.445021 2 | 2.924333<br>2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>1.765644<br>4.3356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.329398<br>3.262224<br>3.365211<br>4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 1.851904<br>3.078521<br>2.991789<br>2.666384<br>2.511792<br>3.030188<br>3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 1.452708<br>1.380314<br>1.430271<br>0.004945<br>0.303662<br>0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 1.768292 2.171287 1.604211 2.058869 2.456513 1.732787 1.989451 2.037312 1.97819 2.453515 0.299856 1.269878 2.814028 0.340221 1.590714 0.481637 0.352569 1.381106 0.852393 | 1.320825 1.551109 1.31471 1.022499 1.106662 1.083689 0.991129 0.911563 0.9461 0.868749 2.488879 -0.24187 1.745695 0.917349 0.438113 0.032882 0.381981 0.015064 0.681979 | 3<br>2<br>2<br>3<br>2<br>3<br>3<br>2<br>2<br>2<br>3<br>3<br>2<br>2<br>2<br>2<br>2<br>2<br>3<br>3<br>2<br>2<br>3<br>3<br>2<br>2<br>2<br>3<br>2<br>2<br>2<br>3<br>2<br>3<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>2<br>3<br>2<br>2<br>2<br>3<br>2<br>2<br>2<br>2<br>3<br>2<br>2<br>2<br>2<br>3<br>2 |
| 1.392201 2 1.872292 2 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 2.646019<br>2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>1.765644<br>4.3356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.262224<br>3.365211<br>4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.078521<br>2.991789<br>2.666384<br>2.511792<br>3.030188<br>3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 1.380314<br>1.430271<br>0.004945<br>0.303662<br>0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.171287<br>1.604211<br>2.058869<br>2.456513<br>1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.551109<br>1.31471<br>1.022499<br>1.106662<br>1.083689<br>0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>3<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>2<br>2<br>2 |
| 1.872292 2 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.932435 3 3.732834 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 2.088221 2 1.624061 3 2.445324 3 1.445021 2 | 2.807496<br>1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.3356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.365211<br>4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.991789 2.666384 2.511792 3.030188 3.004494 2.913923 2.930944 3.228355 3.874878 2.483556 5.662817 0.52877 2.821781 1.786325 3.051233 3.199279 0.828802 0.619534 | 1.430271 0.004945 0.303662 0.686356 0.234085 0.221522 0.71372 0.051874 1.708321 -0.84478 1.16513 1.356926 -0.36831 -0.66089 -1.17422 -0.98896 1.741449 | 1.604211 2.058869 2.456513 1.732787 1.989451 2.037312 1.97819 2.453515 0.299856 1.269878 2.814028 0.340221 1.590714 0.481637 0.352569 1.381106 0.852393 | 1.31471<br>1.022499<br>1.106662<br>1.083689<br>0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>3<br>2<br>2<br>2<br>2<br>2<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>2<br>4<br>4<br>4<br>4 |
| 4.06007 1 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.932435 3 3.732834 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.089671 2 1.288354 2 1.624061 3 2.445324 3 1.445021 2 | 1.952389<br>3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.366534<br>3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.666384<br>2.511792<br>3.030188<br>3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.004945<br>0.303662<br>0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.058869<br>2.456513<br>1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.022499 1.106662 1.083689 0.991129 0.911563 0.9461 0.868749 2.488879 -0.24187 1.745695 0.917349 0.438113 0.032882 0.381981 0.015064 0.681979 | 3<br>2<br>2<br>2<br>2<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>2<br>2<br>4 |
| 2.515136 3 2.353872 3.092874 2 2.985002 3 2.991006 2.498692 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 2.089671 2 1.288354 2 1.624061 3 2.445324 3 1.445021 2 | 3.582175<br>2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.164015<br>3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.511792<br>3.030188<br>3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.303662<br>0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.456513<br>1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.106662<br>1.083689<br>0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>2<br>2<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>4 |
| 2.353872<br>3.092874<br>2.985002<br>3.991006<br>2.498692<br>3.732834<br>3.732834<br>3.732834<br>2.764755<br>1.3089919<br>2.476432<br>2.910139<br>4.3135612<br>2.872695<br>2.089671<br>1.288354<br>2.068221<br>1.624061<br>3.445324<br>3.1445021<br>2.945002<br>3.156002<br>3.1 | 2.84456<br>2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.277328<br>3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.030188<br>3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.686356<br>0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 1.732787<br>1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.083689<br>0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>2<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>4 |
| 3.092874 2 2.985002 3 2.991006 2.498692 3 3.732834 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.878354 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 2.935414<br>3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.090189<br>3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.004494<br>2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.234085<br>0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 1.989451<br>2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.991129<br>0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>2<br>4 |
| 2.985002 3 2.991006 2.498692 3 2.932435 3 3.732834 3 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 2.872695 2 1.288354 2 1.624061 3 2.445324 3 1.445021 2 | 3.046288<br>3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.149261<br>3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.913923<br>2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.221522<br>0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.037312<br>1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.911563<br>0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>2<br>3<br>2<br>2<br>3<br>2<br>3<br>2<br>3<br>2<br>2<br>3<br>2<br>4 |
| 2.991006<br>2.498692<br>3.732834<br>3.732834<br>3.732834<br>3.089919<br>3.476432<br>2.910139<br>4.3135612<br>2.872695<br>2.089671<br>1.288354<br>2.068221<br>2.624061<br>3.445324<br>3.445324<br>3.445324<br>3.445321<br>2.445324<br>3.49692<br>3.49692<br>3.49692<br>3.49692<br>4.49692<br>4 | 3.1423<br>3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.128822<br>3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.930944<br>3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.71372<br>0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 1.97819<br>2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.9461<br>0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>3<br>2<br>2<br>3<br>2<br>3<br>2<br>2<br>3<br>2 |
| 2.498692 3<br>2.932435 3<br>3.732834 3<br>2.764755 1<br>3.089919 3<br>2.476432 2<br>2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 3.030364<br>3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.712698<br>3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.228355<br>3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.868749<br>2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>3<br>2<br>2<br>3<br>2<br>3<br>2<br>2<br>4 |
| 2.932435 3<br>3.732834 3<br>2.764755 1<br>3.089919 3<br>2.476432 2<br>2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 0.051874<br>1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.453515<br>0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 3<br>2<br>2<br>3<br>2<br>3<br>2<br>2<br>4 |
| 2.932435 3<br>3.732834 3<br>2.764755 1<br>3.089919 3<br>2.476432 2<br>2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 3.234334<br>3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.266269<br>4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.874878<br>2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 1.708321<br>-0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 0.299856<br>1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 2.488879<br>-0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 3<br>2<br>2<br>3<br>2<br>3<br>2<br>2<br>4 |
| 3.732834 3<br>2.764755 1<br>3.089919 3<br>2.476432 2<br>2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 3.443928<br>1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.925664<br>4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.483556<br>5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | -0.84478<br>1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 1.269878<br>2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | -0.24187<br>1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>2<br>3<br>2<br>3<br>2<br>2<br>2<br>4 |
| 2.764755 1 3.089919 3 2.476432 2 2.910139 4 3.135612 4 2.872695 3 2.089671 2 1.288354 2 2.068221 2 1.624061 3 2.445324 3 1.445021 2 | 1.765644<br>3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.289369<br>4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 5.662817<br>0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 1.16513<br>1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 2.814028<br>0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 1.745695<br>0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>3<br>2<br>3<br>2<br>2<br>4 |
| 3.089919 3<br>2.476432 2<br>2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 3.356786<br>2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.52097<br>4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 0.52877<br>2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | 1.356926<br>-0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 0.340221<br>1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.917349<br>0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 3<br>2<br>3<br>2<br>2<br>4 |
| 2.476432 2<br>2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 2.565019<br>4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.555364<br>3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 2.821781<br>1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | -0.36831<br>-0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 1.590714<br>0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.438113<br>0.032882<br>0.381981<br>0.015064<br>0.681979 | 2<br>3<br>2<br>2<br>4 |
| 2.910139 4<br>3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 4.087892<br>4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.980479<br>3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 1.786325<br>3.051233<br>3.199279<br>0.828802<br>0.619534 | -0.66089<br>-1.17422<br>-0.98896<br>1.741449 | 0.481637<br>0.352569<br>1.381106<br>0.852393 | 0.032882<br>0.381981<br>0.015064<br>0.681979 | 3<br>2<br>2<br>4 |
| 3.135612 4<br>2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 4.630961<br>3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 3.628399<br>4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.051233<br>3.199279<br>0.828802<br>0.619534 | -1.17422<br>-0.98896<br>1.741449 | 0.352569<br>1.381106<br>0.852393 | 0.381981<br>0.015064<br>0.681979 | 2<br>2<br>4 |
| 2.872695 3<br>2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 3.720954<br>2.377447<br>2.713286<br>2.422813<br>3.815175 | 4.51504<br>6.417695<br>5.504821<br>6.131995 | 3.199279<br>0.828802<br>0.619534 | -0.98896<br>1.741449 | 1.381106<br>0.852393 | 0.015064<br>0.681979 | 2<br>4 |
| 2.089671 2<br>1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 2.377447<br>2.713286<br>2.422813<br>3.815175 | 6.417695<br>5.504821<br>6.131995 | 0.828802<br>0.619534 | 1.741449 | 0.852393 | 0.681979 | 4 |
| 1.288354 2<br>2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 2.713286<br>2.422813<br>3.815175 | 5.504821<br>6.131995 | 0.619534 | | | | |
| 2.068221 2<br>1.624061 3<br>2.445324 3<br>1.445021 2 | 2.422813<br>3.815175 | 6.131995 | | 1.160781 | 1 224874 | 0.05934 I | |
| 1.624061 3<br>2.445324 3<br>1.445021 2 | 3.815175 | | ∩ 715511 I | | | | 4 |
| 2.445324 3<br>1.445021 2 | | 6 227570 | | 2.167848 | 1.25567 | 0.822885 | 4 |
| 1.445021 2 | | | 2.066145 | -1.00305 | 2.208537 | 0.277069 | 4 |
| | 3.714635 | 5.837543 | 0.946298 | -0.31739 | 1.034344 | 0.393447 | 4 |
| | 2.958948 | 2.395126 | 3.098661 | 2.870223 | 0.928077 | 0.090669 | 1 |
| 2.375642 | 2.68096 | 2.183977 | 3.157854 | 2.235614 | 1.306861 | 0.393268 | 3 |
| 1.505374 2 | 2.723895 | 3.330147 | 2.767737 | 3.015288 | 0.696092 | 0.640706 | 3 |
| 1.567687 2 | 2.888448 | 2.295104 | 3.176463 | 3.193394 | 1.005992 | 0.495985 | 1 |
| 2.912557 2 | 2.523757 | 1.949625 | 3.107942 | 2.987511 | 1.188252 | 0.531214 | 3 |
| 1.851181 3 | 3.069879 | 2.227234 | 3.15 | 2.626483 | 1.087311 | 0.423944 | 1 |
| | 2.854885 | 1.961183 | 2.925096 | 3.283892 | 1.388586 | 1.156093 | 3 |
| | 2.694963 | 3.178889 | 2.979329 | 2.500077 | 1.289893 | 1.388323 | 1 |
| | 2.35197 | 2.874528 | 3.014931 | 2.432711 | 1.772328 | 0.987868 | 1 |
| | 2.431548 | 2.221421 | 3.091684 | 2.478228 | 1.352556 | 0.871416 | 3 |
| | 4.262361 | 1.874516 | 2.474586 | 2.511507 | 2.529192 | 0.508671 | 2 |
| | 3.696322 | 1.49651 | 3.046902 | 2.934443 | 2.880074 | 0.135186 | 2 |
| | 3.55922 | 2.511403 | 2.548477 | 2.859269 | 2.493715 | | 3 |
| | | | | | | 0.459517 | |
| | 3.580969 | 1.643502 | 2.802134 | 2.574489 | 1.719936 | 0.253408 | 3 |
| | 3.415299 | 2.264899 | 2.677293 | 2.42812 | 2.083265 | 0.589096 | 3 |
| | 3.61867 | 2.115313 | 3.326557 | 3.243235 | 1.954775 | 0.300382 | 3 |
| | 3.585996 | 2.497658 | 3.382737 | 2.407784 | 1.805826 | 0.848883 | 2 |
| | 3.158151 | 2.642835 | 2.811435 | 3.556004 | 2.073591 | 0.192526 | 3 |
| | 3.29477 | 2.061836 | 3.531687 | 2.321305 | 2.139039 | 0.260408 | 2 |
| 2.866981 3 | 3.461092 | 2.503888 | 3.076605 | 2.320136 | 2.322889 | 0.164261 | 2 |
| 3.02909 3 | 3.796378 | 1.622972 | 3.100696 | 2.428454 | 2.112373 | 0.302758 | 2 |
| 1.832561 3 | 3.035723 | 2.92606 | 3.152572 | 1.969182 | 1.66836 | 2.027277 | 1 |
| | 3.724756 | 1.959737 | 2.563242 | 2.126821 | 1.498965 | 0.513307 | 1 |
| | 3.205037 | 1.664459 | 3.411925 | 1.951163 | 2.136093 | 1.881294 | 1 |
| | 3.496502 | 1.921167 | 2.296864 | 2.092613 | 1.947697 | 1.894757 | 1 |
| | 3.535061 | 3.032781 | 1.687279 | 2.179816 | 1.986136 | 3.189025 | <del>:</del><br>1 |
| | 3.098997 | 2.935675 | 2.583162 | 0.79795 | 1.274482 | 1.279583 | 4 |
| | 3.729742 | 3.438625 | 3.315709 | 1.270037 | 1.351169 | 0.323621 | 4 |
| | 2.878876 | 2.439134 | 3.205687 | 2.056859 | 1.26008 | 0.245724 | 2 |
| | 3.260611 | 1.669527 | 2.611259 | 2.802661 | 1.975953 | 1.996848 | 1 |

Document: PPD

Author: PPD


06MAY2024



| 0.929042 | 4.229001 | 0.958476 | 1.837791 | 2.345441 | 0.85991 | 0.266006 | 1 |
|---|---|---|---|---|---|---|---|
| 0.835028 | 4.094564 | 1.624835 | 3.745215 | 0.676649 | 1.596787 | 0.633265 | 2 |
| 0.518017 | 3.482631 | 0.026971 | 3.232487 | 2.585949 | 1.714216 | 1.247258 | 11 |
| 2.142077 | 2.763266 | 1.717985 | 2.132657 | 1.981876 | 1.682524 | 1.359786 | 3 |
| 1.163136 | 2.278781 | 2.040656 | 1.66038 | 2.28934 | 2.245927 | 2.48422 | 1 |
| 1.773945 | 1.815762 | 2.296841 | 2.241036 | 2.003111 | 2.440107 | 2.329185 | 5 |
| 0.370864 | 1.828904 | 3.135938 | 1.977168 | 1.213476 | 1.233708 | 2.011518 | 4 |
| 1.286832 | 2.260544 | 3.247904 | 2.244789 | 1.087078 | 2.409808 | 1.666524 | 4 |
| 0.665569 | 2.919365 | 2.218953 | 2.267884 | 1.69468 | 1.892542 | 1.390264 | 1 |
| 0.499638 | 1.950232 | 2.077153 | 2.111414 | 2.362764 | 2.243769 | 2.65479 | 1 |
| 1.813017 | 3.779611 | 3.381505 | 1.889955 | 2.499938 | 1.561516 | 0.468737 | 3 |
| 0.397136 | 4.680782 | 2.396155 | 3.188569 | 3.35778 | 3.188256 | 1.316963 | 1 |
| 1.019573 | 2.844814 | 3.271878 | 1.693419 | 1.576868 | 2.980728 | 1.484369 | 1 |
| -0.12102 | 2.640397 | 1.937596 | 2.509998 | 2.081944 | 2.465172 | 1.921706 | 1 |
| 0.52094 | 4.365047 | 0.079631 | 3.39627 | 0.649761 | 3.180026 | 0.097283 | 2 |
| 2.731117 | 3.182713 | 2.077638 | 3.00734 | 2.583772 | 1.26684 | 0.103849 | 3 |
| 1.771354 | 3.13086 | 2.349316 | 1.061821 | 2.445899 | 2.343069 | 1.002997 | 1 |
| 2.059941 | 3.055221 | 2.663597 | 1.88279 | 2.215695 | 1.325664 | 0.702866 | 3 |
| 1.303168 | 2.959174 | 2.820694 | 2.397158 | 2.033969 | 1.579769 | 2.122712 | 1 |
| 2.429935 | 2.785714 | 1.96915 | 1.688699 | 2.165227 | 2.253247 | 1.325774 | 3 |
| 0.891107 | 2.804571 | 3.191638 | 2.048713 | 1.508145 | 1.19412 | 1.88979 | 4 |
| 1.907596 | 2.544843 | 1.657253 | 2.422589 | 1.154796 | 1.183471 | 1.661215 | 3 |
| 2.385735 | 3.027558 | 1.489701 | 1.884331 | 0.99354 | 1.180347 | 1.127258 | 3 |
| 1.251581 | 3.68027 | 2.711777 | 2.1435 | 1.619374 | 1.509578 | 0.333364 | 2 |
| 0.798065 | 3.178204 | 1.337118 | 2.323722 | 1.813707 | 1.180386 | 0.886322 | 1 |
| 2.252769 | 3.452674 | 2.544877 | 4.622918 | -0.07422 | 2.354946 | 0.115854 | 2 |
| 0.583991 | 1.996347 | 3.522147 | 2.550794 | 2.507082 | 2.036728 | 2.388671 | 5 |
| -0.13509 | 2.898338 | 2.444281 | 2.521597 | 1.825635 | 2.888208 | 1.921385 | 1 |
| -0.36838 | 2.995744 | 3.441612 | 2.97643 | 1.572292 | 2.68975 | 1.238128 | 1 |
| -0.30352 | 3.100945 | 3.418419 | 1.915066 | 2.18415 | 2.148555 | 2.157188 | 1 |
| 1.244294 | 3.111563 | 2.930995 | 1.059978 | 0.847236 | 1.804209 | 0.909519 | 4 |
| -0.14236 | 1.646401 | 3.496471 | 1.485099 | 1.650087 | 0.930843 | 2.037234 | 4 |
| 1.19828 | 2.207907 | 2.349218 | 1.552053 | 1.722359 | 1.499779 | 1.598663 | 11 |
| 0.38149 | 3.928541 | 1.372957 | 2.687336 | 1.838206 | 2.154214 | 0.524778 | 1 |
| 2.481611 | 3.481827 | 2.197603 | 2.130881 | 1.476809 | 2.260437 | 1.234254 | 2 |
| 0.481608 | 2.39286 | 2.337152 | 1.8301 | 3.06498 | 1.393734 | 2.654131 | 1 |
| 2.037414 | 2.085096 | 1.496653 | 2.455538 | 3.879859 | 1.623686 | 2.888888 | 5 |
| 1.550216 | 3.153218 | 1.742108 | 1.904519 | 1.712383 | 1.807038 | 1.351736 | 11 |
| 1.648021 | 2.673175 | 1.638725 | 3.046737 | 1.692765 | 2.351428 | 1.857887 | 1 |
| 1.374126 | 2.435089 | 2.234815 | 2.18588 | 1.898093 | 2.19479 | 0.889646 | 11 |
| 1.019342 | 2.647679 | 2.648263 | 2.498198 | 1.115062 | 0.804325 | 2.647109 | 4 |
| 2.736435 | 0.551078 | 3.752571 | 1.417281 | 1.549031 | 0.691697 | 3.033024 | 5 |
| 1.076616 | 4.06708 | 2.069281 | 1.842046 | 1.935288 | 1.900541 | 2.868004 | 1 |
| 1.33195<br>2.77427 | 2.484582<br>3.355737 | 2.416758<br>2.304729 | 2.379112<br>1.78513 | 1.760003<br>0.741504 | 3.692732<br>2.762615 | 0.736447 | 2 |
| | | | | | 0.850391 | 1.853789 | 4 |
| 1.110734 | 3.632882 | 3.21394 | 1.776796 | 1.612268 | | 0.641557 | |
| 2.389185 | 2.881695 | 1.795131 | 3.20699 | 0.41942 | 3.494308 | 1.27316 | 2 |
| 0.730482 | 2.662928 | 2.413819 | 2.880268 | 1.47977 | 2.413753 | 1.470869 | 1 |
| 1.544426 | 3.943903 | 2.727814 | 1.735903 | 0.3283 | 1.153388 | 0.127138 | 2 |
| 1.279774 | 1.859157 | 2.630356 | 2.828011 | 0.364033 | 1.515973 | 1.979112<br>1.325387 | 4 |
| 1.793325 | 3.012943 | 1.797364 | 3.337012 | 0.706964 | 2.779247 | | 2 |
| 2.238936 | 3.999729 | 2.426756 | 1.92557 | 2.32772 | 3.174616 | 1.094697 | 2 |
| 1.328915 | 2.584895 | 2.436472 | 2.695512 | 0.404388 | 2.423566 | 0.966932 | 2 |
| 0.949881 | 2.271697 | 2.870003 | 1.331377 | 3.139382 | 1.581926 | 2.831327 | 5 |
| 1.447089 | 4.561358 | 2.758321 | 1.890039 | 1.155236 | 2.090646 | -0.24765 | 2 |
| 1.559906 | 3.743831 | 2.957692 | 2.926744 | 0.70788 | 3.029807 | 1.492514 | 2 |
| 0.037952 | 2.623521 | 2.977699 | 2.60586 | 1.7889 | 1.516554 | 1.752384 | 1 |
| 0.544136 | 2.470642 | 3.054143 | 1.796674 | 2.630448 | 1.995703 | 1.006744 | 1 |
| 1.103825 | 2.393463 | 3.065722 | 1.774394 | 2.428612 | 1.982995 | 0.895501 | 1 |

Document: PPD

Author: PPD


06MAY2024

| 1.399663 | 2.370678 | 3.102827 | 1.824285 | 1.496074 | 2.043118 | 0.86195 | 4 |
|---|---|---|---|---|---|---|---|
| 0.897121 | 2.54747 | 3.141174 | 1.854219 | 1.595786 | 2.011652 | 0.804589 | 4 |
| 1.201974 | 2.640957 | 2.332992 | 2.627714 | 2.533396 | 2.930975 | 1.314934 | 1 |
| 1.363306 | 2.722 | 2.897964 | 1.712665 | 1.587274 | 2.16176 | 0.545037 | 2 |
| 0.723609 | 3.782392 | 3.074652 | 2.64536 | 2.840634 | 1.366008 | 0.711355 | 1 |
| 0.719305 | 3.75657 | 2.379346 | 3.293745 | 1.618362 | 3.079174 | 0.353328 | 2 |
| 0.328069 | 3.287281 | 2.131284 | 2.691661 | 1.991577 | 1.488309 | 0.506056 | 1 |
| -0.64046 | 2.981621 | 2.625653 | 2.987986 | 1.415446 | 2.682281 | 2.372283 | 1 |
| 0.787829 | 3.43195 | 2.429392 | 3.333081 | 1.33786 | 2.979558 | 0.795472 | 2 |
| 0.227007 | 3.521006 | 2.724771 | 3.137629 | 0.03393 | 2.165901 | 0.06169 | 2 |
| -0.40163 | 3.609939 | 2.626096 | 3.870232 | -0.36079 | 2.958831 | 0.209338 | 2 |
| 1.965187 | 3.49462 | 2.311837 | 3.878262 | -0.49392 | 1.852627 | -0.02262 | 2 |
| 1.791554 | 2.700887 | 2.96369 | 2.574842 | 1.361732 | 1.22905 | 0.905313 | 3 |
| 0.592842 | 2.498902 | 3.325384 | 1.998149 | 2.970382 | 1.484991 | 2.433574 | 1 |
| 0.93449 | 3.04107 | 3.092865 | 3.005954 | 3.044192 | 1.088331 | 1.023012 | 1 |
| 0.003281 | 2.687613 | 3.929499 | 2.543304 | 2.892851 | 2.191037 | 3.148313 | 1 |
| 1.068601 | 3.440496 | 2.803361 | 2.066853 | 2.684096 | 1.392016 | 0.972695 | 1 |
| 0.253151 | 3.366974 | 3.134181 | 2.849601 | 1.98879 | 1.665742 | 1.794241 | 1 |
| 0.568625 | 2.599822 | 3.489269 | 2.403426 | 2.2514 | 1.457632 | 1.842686 | 4 |
| | 2.891183 | | 2.837727 | 2.056235 | | 1.521558 | 1 |
| 0.00812<br>0.032748 | 2.470632 | 3.527231<br>2.393383 | 2.837727 | 2.050235 | 2.082804<br>2.522461 | 3.323862 | 1 |
| | | | 1.648248 | | | | 1 |
| 0.542252<br>0.489436 | 2.924785<br>2.782794 | 2.188542<br>2.799251 | 2.348694 | 1.714741<br>2.562243 | 2.188392<br>2.045669 | 2.210163<br>2.597358 | 1 |
| 0.598497 | 3.537035 | 2.270759 | 1.885296 | 2.640754 | 1.931446 | 1.9822 | 11 |
| 2.684479 | 4.627392 | 1.323444 | 2.104489 | 3.085864 | 1.524276 | 4.186668 | 11 |
| 0.655399 | 2.42486 | 2.702211 | 1.692073 | 2.686051 | 2.115035 | 1.992235 | 1 |
| 1.00012 | 2.63573 | 1.946578 | 1.927783 | 2.474008 | 2.149825 | 2.785688 | 1 |
| 0.803679 | 2.576829 | 1.90842 | 2.733659 | 2.142713 | 2.062206 | 2.425543 | 1 |
| 1.362799 | 2.747179 | 1.705736 | 1.951721 | 2.795911 | 2.423492 | 1.966459 | 1 |
| 0.963135 | 3.36129 | 1.576244 | 2.275032 | 2.391988 | 1.914535 | 2.548146 | 1 |
| 0.957478 | 3.325917 | 2.675156 | 2.401962 | 0.999558 | 1.423449 | 0.931414 | 2 |
| 0.847499 | 2.932603 | 2.498088 | 1.810525 | 2.707284 | 2.590633 | 2.0517 | 1 |
| 1.234055 | 2.177802 | 2.697905 | 2.809799 | 2.466852 | 1.403281 | 2.495561 | 5 |
| 2.015017 | 3.586158 | 1.209095 | 0.797506 | 1.692396 | 1.815927 | 1.146375 | 3 |
| 1.555804 | 2.938869 | 1.394756 | 0.825921 | 2.281687 | 1.885865 | 1.503032 | 11 |
| 1.919184 | 2.652597 | 2.006072 | 1.579702 | 1.47809 | 1.927411 | 1.892786 | 3 |
| 1.164025 | 3.354408 | 1.683151 | 2.741454 | 2.56621 | 1.453452 | 2.74602 | 1 |
| 0.86959 | 2.681597 | 1.65861 | 2.77981 | 2.819379 | 1.416855 | 2.724348 | 1 |
| 1.043517 | 2.337804 | 1.855299 | 2.055885 | 2.697255 | 1.476669 | 2.311822 | 11 |
| 2.083676 | 4.361556 | 1.724352 | 2.17223 | 2.581234 | 2.50454 | 1.35888 | 1 |
| 2.615128 | 3.571862 | 0.682013 | 3.528703 | 2.241834 | 3.449389 | 2.821293 | 1 |
| 2.085683 | 3.602037 | 1.088369 | 2.923386 | 2.205792 | 2.28507 | 2.979874 | 1 |
| 1.898764 | 3.276854 | 1.77007 | 2.506758 | 1.517037 | 2.607894 | 1.089812 | 2 |
| 2.5278 | 2.059308 | 1.713481 | 3.124673 | 1.225085 | 3.026174 | 3.025545 | 5 |
| 2.864402 | 3.013686 | 1.637174 | 1.573196 | 2.441859 | 1.623372 | 1.120725 | 3 |
| 2.072019 | 3.282316 | 0.870472 | 2.358488 | 2.208217 | 2.802844 | 1.730093 | 1 |
| 1.63954 | 3.096221 | 2.814322 | 2.561726 | 2.063223 | 1.377709 | 1.451547 | 1 |
| 2.309299 | 3.454196 | 1.661915 | 2.559652 | 1.830277 | 1.966368 | 0.014157 | 2 |
| 0.72982 | 2.395892 | 2.585869 | 2.750007 | 2.132678 | 2.026769 | 1.971763 | 1 |
| 2.549466 | 3.574283 | 2.038015 | 3.583879 | 1.986217 | 2.118853 | 0.140961 | 2 |
| 2.083922 | 3.433225 | 1.320953 | 2.441424 | 2.589508 | 2.780382 | 1.209729 | 1 |
| 1.293829 | 3.273937 | 1.462928 | 2.817106 | 1.721652 | 3.104604 | 2.554968 | 1 |
| 1.195288 | 3.769418 | 1.210908 | 2.98681 | 1.044027 | 2.749903 | 0.60132 | 2 |
| 2.061813 | 2.704437 | 2.316068 | 2.554463 | 2.553281 | 3.014762 | 2.00189 | 1 |
| 2.468648 | 2.98751 | 2.060243 | 3.21991 | 1.330698 | 2.781815 | 2.311667 | 2 |
| 0.936901 | 2.780699 | 1.501068 | 3.119347 | 1.893182 | 1.345022 | 1.445776 | 1 |
| 2.096261 | 3.729782 | 2.528279 | 2.942293 | 2.272058 | 1.668373 | 0.184038 | 2 |
| -0.06866 | 2.323305 | 2.466225 | 3.008179 | 2.310103 | 1.806849 | 1.758138 | 1 |
| 2.600323 | 1.57889 | 2.767321 | 2.701491 | 1.678983 | 0.431804 | 0.746914 | 3 |
| 2.000020 | 1.07000 | 2.101021 | 2.101701 | 1.070000 | 0101004 | 0.7 700 17 | <u> </u> |

Document: PPD

Author: PPD


06MAY2024

| | | | | | 1 | | |
|---|---|---|---|---|---|---|---|
| 1.904414 | 1.941858 | 2.790823 | 1.733361 | 1.862784 | 0.627279 | 1.648438 | 3 |
| 1.596553 | 2.69657 | 2.367887 | 2.664833 | 1.633339 | 1.978123 | 0.121749 | 2 |
| 1.07667 | 1.205244 | 2.672278 | 1.959053 | 2.384767 | 1.783993 | 3.279252 | 5 |
| 1.595228 | 3.077974 | 2.380944 | 2.815531 | 1.774421 | 1.243553 | 0.373183 | 2 |
| 3.05165 | 1.742192 | 3.165878 | 2.403648 | 1.464842 | 0.801114 | 0.72373 | 3 |
| 2.207574 | 2.570317 | 1.919201 | 3.671462 | -0.20097 | 2.181307 | 0.583058 | 2 |
| 1.136287 | 2.834087 | 3.186852 | 2.882391 | 1.934227 | 0.932035 | 1.06899 | 4 |
| 3.138606 | 1.675005 | 3.392111 | 2.846753 | 0.800305 | 1.366669 | 0.36267 | 3 |
| 3.006056 | 1.788769 | 2.430313 | 2.210938 | 2.343229 | 0.8086 | 1.471998 | 3 |
| 3.301842 | 2.534269 | 2.727616 | 1.645315 | 2.297743 | 1.398658 | 0.504945 | 3 |
| 1.045698 | 3.34271 | 2.926759 | 2.671772 | -0.54325 | 3.05828 | 1.151877 | 2 |
| 1.474318 | 3.49987 | 3.358005 | 2.668088 | -0.34163 | 0.727697 | 0.198376 | 2 |
| 1.418577 | 3.540259 | 1.859501 | 1.848117 | 0.758087 | 1.62029 | 1.178268 | 2 |
| 1.792042 | 3.571176 | 2.781245 | 2.623082 | 2.059251 | 2.687523 | 0.663873 | 2 |
| 2.246787 | 3.973687 | 2.288619 | 2.616655 | 0.964431 | 2.932953 | 0.383798 | 2 |
| 2.557149 | 3.009742 | 3.015698 | 2.63141 | 1.263235 | 2.701192 | 0.65265 | 2 |
| 2.406639 | 2.86216 | 2.747641 | 2.887785 | 2.069158 | 2.148691 | 0.371257 | 2 |
| 2.144278 | 3.008093 | 3.211825 | 4.019281 | 0.030605 | 2.866497 | 0.860084 | 2 |
| 2.555363 | 2.579017 | 3.075949 | 2.0346 | 2.256304 | 2.102979 | 0.446911 | 3 |
| 2.53739 | 3.435742 | 2.628374 | 3.319847 | 1.749244 | 2.053878 | 1.172975 | 2 |
| 2.645764 | 3.632515 | 2.547884 | 2.116629 | 2.961363 | 2.525557 | 0.751793 | 3 |
| 2.167688 | 3.177878 | 2.822987 | 2.693744 | 2.104781 | 2.348668 | 0.571723 | 2 |
| 1.225418 | 2.761464 | 2.284974 | 2.906629 | 1.555919 | 2.234763 | 1.344509 | 1 |
| 2.549378 | 1.883245 | 4.847159 | -0.38613 | 2.328991 | 0.399031 | 0.899669 | 3 |
| 0.835491 | 3.410214 | 3.238864 | 2.174315 | 1.569618 | 3.313993 | 1.048845 | 1 |
| 0.197072 | 3.720005 | 3.210243 | 1.462301 | 1.715089 | 3.289458 | 0.349891 | 11 |
| 0.956348 | 1.634326 | 4.496375 | 2.859105 | 1.713968 | 2.541391 | 0.572134 | 4 |
| 2.710831 | 2.895985 | 4.542081 | 1.117162 | 1.602833 | 0.638402 | 1.605333 | 3 |
| 0.468519 | 2.775847 | 4.793864 | 1.572114 | 2.577669 | 2.142251 | 0.374559 | 4 |
| 0.801185 | 3.856247 | 4.476053 | 1.102946 | 1.665504 | 2.180561 | 1.051688 | 4 |
| 1.396774 | 2.38184 | 3.159023 | 2.272422 | 1.642917 | 2.218226 | 0.494604 | 2 |
| 1.029972 | 1.815946 | 3.624451 | 2.805185 | 1.766394 | 1.950249 | 0.557906 | 4 |
| 2.351785 | 2.454701 | 1.492669 | 4.377274 | 1.452214 | 3.421769 | 1.610619 | 2 |
| 2.32405 | 3.466859 | 1.816886 | 2.125494 | 2.298043 | 2.802006 | 1.772149 | 1 |
| 1.22715 | 2.873227 | 2.457041 | 2.742809 | 1.886899 | 1.460491 | 1.371267 | 1 |
| 1.281567 | 3.046454 | 2.498313 | 1.471574 | 2.914418 | 2.038731 | 1.977465 | 1 |
| 0.288136 | 1.74727 | 3.931425 | 2.686452 | 2.618377 | 2.564444 | 2.479821 | 5 |
| 2.522687 | 2.759939 | 1.745555 | 1.6985 | 2.060347 | 0.322064 | 1.304326 | 3 |
| 0.543637 | 2.544981 | 3.348045 | 1.906861 | 2.258307 | 1.031273 | 1.44175 | 4 |
| 1.620347 | 3.401088 | 2.574342 | -0.41533 | 2.252736 | 0.219513 | 1.438078 | 3 |
| 1.842942 | 3.37822 | 2.328411 | 1.420737 | 2.466913 | 0.174455 | 2.317012 | 3 |
| 0.948361 | 3.600731 | 3.023847 | 2.142095 | 2.757594 | 0.861544 | 1.1149 | 1 |
| 1.868794 | 3.629237 | 1.867504 | 3.675692 | 1.405051 | 3.091689 | 0.902801 | 2 |
| 0.109365 | 3.572819 | 2.384525 | 2.616362 | 1.429333 | 1.794456 | 1.190442 | 1 |
| | | | | 2.02835 | | 2.584236 | |
| 2.186493 | 1.83317 | 2.188746 | 1.631281 | | 1.133724 | | 5 |
| -0.19669 | 3.080497 | 2.427698 | 1.772721 | 1.871182 | 2.58294 | 1.963527 | 1 |
| 1.045365 | 3.084264 | 2.502615 | 1.233211 | 2.190984 | 1.398955 | 2.304011 | 11 |
| 0.498219 | 3.184056 | 3.006726 | 1.873029 | 1.272331 | 2.277158 | 2.527363 | 1 |
| 0.064184 | 3.279553 | 2.142248 | 1.683496 | 2.028901 | 1.967967 | 2.81393 | 1 |
| 1.294706 | 3.528197 | 2.401889 | 2.620905 | 1.628489 | 2.505685 | 1.915161 | 1 |
| 1.237893 | 4.214992 | 3.247795 | 1.255129 | 1.727378 | 1.922664 | 1.535637 | 1 |
| 0.895371 | 2.295853 | 2.195042 | 3.304022 | 1.494507 | 2.228977 | 1.607169 | 11 |
| -0.15976 | 2.294287 | 3.693329 | 1.853443 | 2.346265 | 2.371389 | 1.889254 | 4 |
| 0.765196 | 3.619231 | 3.406026 | 2.56884 | 1.039612 | 2.176356 | 1.173186 | 2 |
| 0.040116 | 2.078193 | 3.350767 | 1.54803 | 2.515734 | 2.492502 | 1.961021 | 1 |
| -0.01981 | 2.391736 | 2.677275 | 2.01822 | 2.822933 | 2.111246 | 2.320911 | 1 |
| | 3.088558 | 2.695161 | 1.66284 | 2.394352 | 1.829432 | 2.164855 | 3 |
| 2.137868 | 3.000330 | 2.033101 | 1.0020- | | | | |
| 2.137868<br>2.081211 | 1.547291 | 3.061405 | 1.85112 | 1.647561 | 2.145304 | 1.606017 | 3 |

Document: PPD

Author: PPD


06MAY2024



| 1.758938 | 3.006452 | 2.01326 | 0.699399 | 3.04425 | 1.384979 | 0.665989 | 3 |
|---|---|---|---|---|---|---|---|
| 1.237003 | 2.523978 | 2.330382 | 2.049435 | 1.997275 | 1.271707 | 0.498445 | 1 |
| 0.667497 | 2.718609 | 2.958894 | 1.611983 | 2.782766 | 2.031715 | 2.059987 | 1 |
| 2.0786 | 2.254637 | 2.013767 | 2.860412 | 1.253703 | 2.580455 | 1.367255 | 2 |
| 1.137981 | 2.2767 | 2.173088 | 2.474196 | 1.543822 | 2.78904 | 1.474368 | 1 |
| 0.83508 | 2.375671 | 2.923106 | 2.319775 | 1.112637 | 1.568078 | 1.782344 | 4 |
| 1.532628 | 2.452578 | 4.199479 | 2.184313 | 1.28271 | 1.39555 | 1.30231 | 4 |
| 2.832667 | 3.229237 | 2.248558 | 5.046877 | -0.14981 | 3.168044 | 0.514728 | 2 |
| 2.804329 | 3.544024 | 3.281753 | 1.443864 | 0.979548 | 1.515588 | 2.244697 | 3 |
| 4.176895 | 3.853278 | 3.442913 | 3.436163 | -0.20598 | 1.787425 | 0.697663 | 2 |
| 1.447793 | 1.661014 | 4.651958 | 1.638069 | 0.705343 | 1.763816 | 0.192127 | 4 |
| 0.837814 | 3.230974 | 2.320599 | 3.009408 | 0.461031 | 2.905844 | 1.343623 | 2 |
| 1.802944 | 1.716569 | 3.558995 | 2.552908 | 0.4513 | 2.238213 | -0.50813 | 2 |
| 0.957177 | 1.475594 | 3.511604 | 2.462799 | 0.950496 | 1.55846 | 1.053852 | 4 |
| 1.767879 | 2.111048 | 3.558412 | 1.886744 | -0.32273 | 1.971333 | -0.18521 | 2 |
| 0.567263 | 0.795808 | 2.30941 | 2.196065 | 2.747347 | 1.982559 | 2.3133 | 5 |
| 1.47234 | 2.608456 | 2.826792 | 2.398996 | 1.022706 | 2.533647 | 0.7236 | 2 |
| 1.025226 | 2.719732 | 2.423171 | 2.797212 | 2.343007 | 2.681939 | 1.803731 | 1 |
| 1.665459 | 0.517428 | 3.510286 | 1.925527 | 2.679155 | 2.339655 | 2.32634 | 5 |
| 0.626203 | 3.278759 | 4.570286 | 1.802226 | 1.454045 | 0.984405 | 1.873493 | 4 |
| 0.989795 | 3.025333 | 2.064807 | 1.322011 | 2.195479 | 2.639946 | 1.743527 | 1 |
| 0.748755 | 2.27195 | 2.717904 | 3.103542 | 2.114782 | 3.677446 | 1.694106 | 1 |
| -0.54808 | 3.454881 | 2.794786 | 0.243503 | 2.598806 | 2.136147 | 2.934898 | 1 |
| 1.73608 | 2.049779 | 2.363716 | 2.801236 | 2.019415 | 1.639227 | 1.9725 | 5 |
| 2.540272 | 3.227549 | 3.596597 | 2.319795 | 1.413479 | 2.179313 | 0.192601 | 2 |
| 4.283287 | 3.240125 | 2.663105 | 2.760057 | 0.818601 | 1.64212 | 1.574151 | 3 |
| 1.391141 | 2.810916 | 2.450279 | 2.953166 | 2.210613 | 2.323273 | 1.154374 | 1 |

Document: PPD

Author: PPD


# APPENDIX 10. Marder PANSS Negative Symptoms (MPNS)

#### **HETEROGENEITY INDEX METHOD**

Subject-level PANSS item scores between two assessments (e.g., Screening and Baseline) are encoded in a variance-covariance difference (VCD) vector. The VCD vector captures the intra-item variance, between-item covariance, and between-item differences of PANSS items between two assessment time points from a single subject.

Briefly, for each subject h, a variance-covariance matrix of the 30 PANSS items is defined as

$$V = \begin{bmatrix} \sigma_{s_1}^2 & \cdots & \sigma_{s_{1,30}} \\ \vdots & \ddots & \vdots \\ \sigma_{s_{30,1}} & \cdots & \sigma_{s_{30}}^2 \end{bmatrix},$$

where

$$\sigma_{s_j}^2 = \sum_{t=1}^2 (s_t^j - \bar{s^j})^2,$$

is the unbiased estimator of the variance of  $s^{j}$  (score of PANSS item j), j=1,2,...,30, and

$$\sigma_{s_{i,j}} = \sum_{t=1}^{2} (s_t^i - \overline{s^I})(s_t^j - \overline{s^J}),$$

is the unbiased estimator of the covariance of  $s^i$  and  $s^j$  (scores of PANSS items i and j), and

$$\bar{s^{I}} = \frac{\sum_{t=1}^{2} s_{t}^{j}}{2}; \ \bar{s^{I}} = \frac{\sum_{t=1}^{2} s_{t}^{i}}{2}.$$

Note that the denominators of  $\sigma_{s_i}^2$  and  $\sigma_{s_{i,i}}$  are 2 – 1 = 1, for two time points.

The unique elements of V for subject h are kept in vector  $u_{cov_h}$ , consisting of the elements of V on and below the main diagonal.

Separately, for each subject h and each timepoint t, a different matrix for the 30 PANSS items is defined as

$$D = \begin{bmatrix} d_{s_{1,1}} & \cdots & d_{s_{1,30}} \\ \vdots & \ddots & \vdots \\ d_{s_{30,1}} & \cdots & d_{s_{30,30}} \end{bmatrix},$$

where  $d_{s_{i,j}}=s^i-s^j$  for scores of items i and j. Note that the diagonal elements of D are 0.

The unique elements of D for subject h at timepoint t are kept in vector  $d_{t(h)}$ , consisting of elements of D below the main diagonal.

Together, the VCD vector of subject h for 2 timepoints (e.g., Screening and Baseline) is defined as

$$VCDV_{h(t=1,t=2)} = \begin{bmatrix} u_{cov_h} & d_{1(h)}, d_{2(h)} \end{bmatrix} \to \mathbb{R}^{1,1335},$$

and the VCD vector for N subjects is

| Document: | PPD |
|-----------|-----|

$$VCDV_{(t=1,t=2)} = \begin{bmatrix} VCDV_{h_1(t=1,t=2)} \\ VCDV_{h_2(t=1,t=2)} \\ \vdots \\ VCDV_{h_N(t=1,t=2)} \end{bmatrix} \rightarrow \mathbb{R}^{N,1335}.$$

Using the PANSS-defined VCD vector, and the 7 items of the Marder PANSS Negative Symptoms factor, a new vector of 84 elements per subject is used to define a Marder Negative Heterogeneity Index (MNHI). Table 7 lists the parameters used to derive the MNHI.

Table 10: Parameters Used to Derive the Marder Negative Heterogeneity Index (MNHI)

| $\sigma_{s_i}^2$ | Variance of PANSS item $\it i$ between Screening and Baseline for subject $\it h$ |
|---|---|
| $\Delta\sigma^2_{s_{(i.j)_t}}$ | $\sigma_{s_i}^2 - \sigma_{s_j}^2$ at visit $t$ for subject $h$ |
| $\sigma_{s_{i,j}}$ | Covariance of PANSS item $i$ and PANSS item $j$ between Screening and Baseline for subject $h$ |
| $d_{s_{i,j}}$ | Difference between PANSS item $\it i$ and PANSS item $\it j$ at a given timepoint for subject $\it h$ |
| P | Set of combinations of two Marder PANSS Negative Symptoms factor items |
| C(x) | Count of x |

The 7 items of the Marder PANSS Negative Symptoms factor are congruent based on the Marder factor model. Therefore,  $\sigma_{s_i}^2 - \sigma_{s_j}^2$  is expected to be small for all p combinations. Similarly,  $\Delta \sigma_{s(i,j)_t}^2$  is expected to be small for all p combinations, at t = Screening and t = Baseline. Furthermore,  $C\left(\sigma_{s_{i,j}}|<0\right)$  is expected to be small for all p combinations. Hence, the raw Marder Negative Heterogeneity Index (rMNHI) of subject t is defined as the sum of L1 norm of variance differences, count of negative covariance, L1 norm of between item differences at Screening and Baseline. It can be expressed as

$$rMNHI = \left\| \Delta \sigma_{s_P}^2 \right\|_1 + \sum_{p=1}^{21} C \left( \sigma_{s_p} | < 0 \right) + \left\| d_{s_P, t=1} \right\|_1 + \left\| d_{s_P, t=2} \right\|_1.$$

The min-max scaling (min = 0, max = 223) is then applied to rMNHI to derive the MNHI for subject h.

The optimal threshold to classify MPNS enriched subjects is determined by fitting the one-factor Marder Negative model through computing confirmatory factor analysis (CFA) statistics (comparative fit index [CFI], Tucker Lewis index [TLI], and root mean square error of approximation [RMSEA]) iteratively. The first iteration draws samples from the range of MNHI from the lowest to the lowest + 0.01 point. The range expands incrementally by 0.01 point for each iteration until the upper bound of the range is above the observed maximum MNHI. The smallest upper bound MNHI corresponds to the median CFI (>0.95), TFI (>0.95), and/or RMSEA (<0.08) and is identified as 0.113. It is used to classify subjects into MPNS enriched (MNHI  $\leq$  0.113) or deenriched (MNHI  $\leq$  0.113) groups.

| Document: | PPD | | |
|-----------|-----|-----------------|-----------|
| Author: | ראח | Version Number: | 1.0 |

## APPENDIX 11. SCHEDULE OF EVENTS

Table 2: Schedule of Assessments

| | Screening | | | | | | | | | | Follow-up Period |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 2 | Period | *** | Treatment Period | | | | | | | | |
| | V1 | | 100 | | | 1000 | - | | | | V11 |
| | | Pre-switch | Week | Week | Week | Week | Week | Week | Week | Week 8b | Week 9 <sup>d</sup> |
| N. A. | Screening <sup>a</sup> | Baseline | 1 | 2 | 3 | 4 | 5 | 6 | 7 TC | EOT/ET <sup>c</sup> | Follow-up |
| Study Day e | Days -21 to -1 | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>22 | Day<br>29 | Day<br>36 | Day<br>43 | Day<br>50 | Day<br>57 | 7 ± 2 days<br>after last dose |
| Informed consent | X | | , a | | | | | 2 | | | 2 |
| Informed consent for duplicate subject check | X | | | | | | | | | | |
| CCI | | | | | | | | | | | |
| Review inclusion/exclusion<br>criteria | X | X | | 2 | | | | | | S. 8 | |
| Prior/concomitant medication review | X | X | X | X | X | X | X | X | X | X | X |
| Dispensation of study drugg | | X | X | X | X | X | X | X | | 8 | |
| Study drug accountability | | | X | X | X | X | X | X | | X | |
| Demography | X | | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Psychiatric history | X | | | 7. | | | | 2 | | | |
| Nicotine use information | X | | 19 83 | | | | | 5 | | X | |
| SCID-5-CTh | X | | | | | | | | | | |
| Physical and neurological examination | X | | | | | | | | | х | X |
| Height | X | | | | | | | | | | |
| Vital signsi | X | X | X | X | X | X | X | X | | X | X |
| Weight (including BMI) <sup>j</sup> | X | X | | | | X | | | | X | |
| Waist circumference | | X | | 70 | 1 | X | | | | X | |
| 12-lead Electrocardiogram<br>(ECG) | X | X | | | | | | | | X | |
| Hematology, chemistry, and urinalysis <sup>k</sup> | х | X | | | | | | | | Х | 8 |
| Blood sample for hepatitis screening | X | | 19 | | | | | | , | | |

Author: PPD




Table 2: Schedule of Assessments (Continued)

| | Screening<br>Period | Treatment Period | | | | | | | | | Follow-up Period |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | V1<br>Screening <sup>a</sup> | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 |
| | | Pre-switch<br>Baseline | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5 | Week<br>6 | Week<br>7 TC | Week 8b<br>EOT/ET <sup>c</sup> | Week 9 <sup>d</sup><br>Follow-up |
| Study Day e | Days<br>-21 to -1 | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>22 | Day<br>29 | Day<br>36 | Day<br>43 | Day<br>50 | Day<br>57 | 7 ± 2 days<br>after last dose |
| Serum follicle stimulating<br>hormone (FSH) <sup>1</sup> | X | | | | | | | | | | |
| Serum human chorionic<br>gonadotropin (β-hCG),<br>(females) | X | | | | | | | | × | x | |
| Urine β-hCG (females) <sup>m</sup> | | X | | | | X | | | 95 | | X |
| Rapid urine β-hCG (females) <sup>m</sup> | | 100,000.0 | | | | 44.5 | | | | X | Phone |
| CI | | | | | | | | | | | |
| Blood sample for POPPK° | | X | X | | | X | | | | X | |
| Urine drug screen <sup>p</sup> | X | X | | | | X | | | 7. | X | ) |
| Rapid urine drug screen p | | | | | | | | | | X | |
| Positive and Negative<br>Syndrome Scale (PANSS) | x | X | X | X | 0 | X | | X | 30 | X | 8 |
| Clinical Global Impression –<br>Severity (CGI-S) | X | X | X | X | | X | | X | | X | |
| Clinical Global Impression –<br>Improvement (CGI-I) | | | X | X | | X | | X | | X | |
| Brief Negative Symptom<br>Scale (BNSS) | | х | | | 8 | X | | | - | X | |
| Pittsburg Sleep Quality Index<br>(PSQI) | | X | | | | X | | | - | X | |
| Columbia Suicide Severity<br>Rating Scale (C-SSRS) | х | X | X | X | X | X | X | X | X | X | X |
| Simpson-Angus Scale (SAS)q | | X | | | 2 | | | | 50 | X | 7 |
| Barnes Akathisia Rating Scale<br>(BARS) <sup>q</sup> | | х | | | | | | | | X | |





Table 2: Schedule of Assessments (Continued)

| | Screening<br>Period<br>V1<br>Screening <sup>a</sup> | Treatment Period | | | | | | | | | Follow-up Period |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11<br>Week 9 <sup>d</sup><br>Follow-up |
| | | Pre-switch<br>Baseline | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5 | Week<br>6 | Week<br>7 TC | Week 8b<br>EOT/ET <sup>c</sup> | |
| Study Day e | Days -21 to -1 | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>22 | Day<br>29 | Day<br>36 | Day<br>43 | Day<br>50 | Day<br>57 | 7 ± 2 days<br>after last dose |
| Abnormal Involuntary<br>Movement Scale (AIMS) <sup>q</sup> | | х | | | | | | | | X | |
| SF-12 | | X | | | | | | | | X | |
| Medication Satisfaction<br>Questionnaire (MSQ) | | х | | | | | | | | Х | |
| Personal and Social<br>Performance Scale (PSP) | | х | | | | | | | | Х | |
| Healthcare Resource<br>Utilization (HCRU) <sup>r</sup> | 5 | х | | × × | | | | | | X | |
| Pretreatment/Adverse events<br>(AE) monitoring <sup>5</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Duplicate Subject Check <sup>t</sup> | X | | | | | | | | | X | |
| Tokenization<br>consent (optional) <sup>f</sup> | Х | | | | | | | 0.00 | | | |

Abbreviations: AE = adverse event; BARS = Barnes Akathisia Rating Scale; β hCG = human chorionic gonadotropin; BMI = Body Mass Index; BNSS = Brief' Negative Symptom Scale; C-SSRS = Columbia Suicide Severity Rating Scale; eCRF = electronic case report form; EDC = electronic data capture; DSM-5 = Diagnostic and Statistical Manual of Mental Disorders – Fifth Edition; EOT = end of treatment; ET = early termination; FSH = Follicle stimulating hormone; MSQ = Medication Satisfaction Questionnaire; PANSS = Positive and Negative Syndrome Scale; PSP = Personal and Social Performance Scale; PK = pharmacokinetic; PSQI = Pittsburg Sleep Quality Index; SAS = Simpson-Angus Scale; SCID-5-CT = Structured Clinical Interview for DSM-5; SF-12 = Short Form Health survey; Clinical Trials Version; TC = telephone contact visit; UDS = urine drug screen.

f. Requested, but not required for study participation.



a. Subjects who screen fail can be re-screened up to 2 times after consultation with the Medical Monitor. Screening assessments may occur over multiple days. The Screening Period may be extended for up to 7 days after approval from the Medical Monitor.

b. All procedures and assessments scheduled for Week 8 will be utilized as Baseline procedures and assessments for the open-label extension study (SEP361-309).

<sup>&</sup>lt;sup>c.</sup> If a subject discontinues from the study, all Early Termination (ET) procedures should be performed at the ET visit, within 48 hours of last study dose.

d Subjects who discontinue early from the study or complete the study and do not enter the extension study (SEP361-309) will have a safety Follow-up Visit 7 (± 2) days after their last dose of study drug. While every effort should be made to complete the Follow-up Visit in the clinic, administration of C-SSRS, and collection of AEs, and concomitant medications may occur by telephone contact if the subject is unable to come to the clinic for the Follow-up Visit.

Wisit window for Day 8 is +2 days, and visit windows post Day 8 are: ± 2 days for every Visit.



- g. All study drug will be taken once daily in the evening at bedtime by mouth, without regard to food.
- h. The SCID-5-CT will be used to support the DSM-5 diagnosis and must be administered by a qualified rater with at least 2 years' experience with the population under study.
- 1 Vital signs will include respiratory rate, oral body temperature and supine and standing measurements of blood pressure and pulse rate.
- 1 BMI will be calculated and recorded in the eCRF by the clinical site at screening. For other visits, BMI will be derived in the EDC system.
- k Subjects must be fasted (no food or drink except water at least 8 hours prior to specified blood tests) at Pre-switch Baseline (Visit 2) and Week 8/EOT/ET (Visit 10). Fasting for 8 hours prior to Screening (Visit 1) is also recommended to avoid potential retests. Blood samples should be drawn in the morning followed by a snack or meal. A list of clinical laboratory tests is provided in Section 23.
- Blood samples for follicle stimulating hormone (FSH) will be collected for post-menopausal women or if menopause is suspected.
- <sup>m</sup> Positive urine drug screen (UDS) results should be discussed with the Medical Monitor.

#### CCL

- °. Blood samples for determination of plasma SEP-363856 concentrations will be collected predose (prior to administration of the first dose) on Day 1; 3 additional samples will be collected on Days 8, 29 and 57/ET. The time and date of the previous dose of study drug and the time and date of blood sampling must be recorded. The remaining plasma samples, after PK measurement is completed.
- P. Any positive urine β-hCG test should be confirmed by a serum β-hCG test.
- 4 Unscheduled SAS, BARS and AIMS scales should be administered if a subject develops extrapyramidal symptoms (EPS) requiring treatment.
- Lealthcare resource utilization questions are described in Section 11.5.8. Baseline will have 3-month lookback period. Week 8/ET will be since last assessment.
- 5. Events occurring prior to first dose of study drug are pretreatment events. Events occurring after first dose of study drug are adverse events. Determination done programmatically.
- Where local regulations allow, duplicate subject check will be performed. Following the last contact with a subject, the duplicate enrollment system should be updated, as appropriate.
